

### STATISTICAL ANALYSIS PLAN

For Interim and Primary Analyses at Week 12

### 1 TITLE PAGE

| Study Title | Vagus Nerve Stimulation Using the SetPoint System for Moderate to Severe<br>Rheumatoid Arthritis: The RESET-RA Study |
|---|---|
| Protocol Number | SPM-020 |
| ClinicalTrials.gov<br>Identifier | T04539964 |
| Investigational Device | The SetPoint System |
| Study Sponsor's Name<br>and Address | SetPoint Medical, Inc.<br>25101 Rye Canyon Loop<br>Valencia, CA 91355 |
| Biostatistics and Data<br>Analysis | SetPoint Medical, Inc. |

Statistical considerations addressing the impact of COVID-19 on the primary and key secondary endpoints are detailed in Section 10.

### CONFIDENTIALITY STATEMENT

This document is the property of SetPoint Medical, Inc. The document is highly confidential and is to be used only in connection with matters authorized by a senior representative of SetPoint Medical, and no part of it is to be disclosed to a third party without prior written permission from SetPoint Medical.




# TABLE OF CONTENTS

| 1 | TITL | E PAGE | 1 |
|---|------|----------------------------------------------------|----|
| 2 | LIST | OF ABBREVIATIONS | 6 |
| 3 | INTR | RODUCTION | 9 |
| | 3.1 | Study Objective | 9 |
| | 3.2 | Study Design | 9 |
| | 3.3 | Study Visits and Assessments | 9 |
| | 3.4 | Sample Size and Power | 10 |
| 4 | TYPI | E OF PLANNED ANALYSIS | 11 |
| | 4.1 | DMC Analysis | 11 |
| | 4.2 | Interim Analysis | 11 |
| | 4.3 | Primary Analysis | 14 |
| 5 | STAT | TISTICAL METHODS | 15 |
| | 5.1 | General Considerations for Data Analyses | 15 |
| | 5.2 | Analysis Populations | 16 |
| | 5.3 | Baseline | 16 |
| | 5.4 | Study Day Calculation | 17 |
| | 5.5 | Randomization | 17 |
| | 5.6 | Change from Baseline Calculation. | 17 |
| | 5.7 | Relative Difference Calculation | 17 |
| | 5.8 | Missing Dates | 18 |
| | 5.9 | Data Assurance. | 20 |
| | 5.10 | Consistency Across Study Centers. | 20 |
| | 5.11 | Coding Dictionaries | 20 |
| 6 | SUBJ | JECT DISPOSITION | 20 |
| | 6.1 | Subject Enrollment and Disposition | 20 |
| 7 | DEM | OGRAPHICS AND BASELINE CLINICAL CHARACTERISTICS | 21 |
| 8 | EFFI | CACY ANALYSES | 21 |
| | 8.1 | General Considerations | 21 |
| | 8.2 | Clinical Variables | 22 |
| | 8.3 | Primary Efficacy Endpoint | 24 |
| | 8.4 | Key Secondary Endpoints | 26 |
| | 8.5 | Multiplicity Adjustment of Key Secondary Endpoints | 27 |



| | 8.6 | Exploratory Secondary Endpoints | 29 |
|---|---|---|---|
| | 8.7 | Blinding Assessment | 34 |
| 9 | SAFE | ETY EVALUATION | 34 |
| | 9.1 | AE and SAEs | 34 |
| | 9.2 | Protocol Deviations | 35 |
| | 9.3 | Device Deficiencies | 35 |
| 10 | STAT | TISTICAL CONSIDERATIONS RELATED TO COVID-19 | 35 |
| | 10.1 | Impact of COVID-19 on Study Integrity | 35 |
| | 10.2 | COVID-19 Analysis Considerations | 36 |
| 11 | REFI | ERENCES | 37 |
| 12 | APPI | ENDICES | 38 |
| APPI | ENDIX | A: SCHEDULE OF ASSESSMENTS | 38 |
| APPI | ENDIX | B: TABLE MOCKUPS | 40 |
| APPI | ENDIX | C: LISTING MOCKUPS | 129 |
| | 8.7 Blinding Assessment 34 9.1 AE and SAEs 34 9.2 Protocol Deviations 35 9.3 Device Deficiencies 35 10. STATISTICAL CONSIDERATIONS RELATED TO COVID-19 35 10.1 Impact of COVID-19 on Study Integrity 35 10.2 COVID-19 Analysis Considerations 36 11 REFERENCES 37 12 APPENDICES 38 APPENDIX A: SCHEDULE OF ASSESSMENTS 38 APPENDIX B: TABLE MOCKUPS 40 APPENDIX C: LISTING MOCKUPS 129 LIST OF TABLES Fable 1: Power Calculation Based on Estimated ACR Response Rate 10 Fable 2: True Probability of Stopping after Stage 1 and Power of Study Success Based on Pooled Data 12 Fable 3: Interim Data Access Matrix 13 Fable 4: Summary of Primary and Secondary Efficacy Endpoints at Week 12 14 Fable 5: RA Disease Activity Assessments to Be Collected on the Day of Informed Consent and Used as the Baseline Assessments for Determination of the Primary and Key Secondary Efficacy Endpoints 16 Fable 6: HAQ-DI Category Scores Depending on Aids, Devices or Physical Assistance 23 | | |
| | | LIST OF TABLES | |
| Table | 1: Pow | ver Calculation Based on Estimated ACR Response Rate | 10 |
| Table | 2. True | Probability of Stopping after Stage 1 and Power of Study Success Bases | d on |
| rabic | | | |
| Table | 3: Inter | rim Data Access Matrix | 13 |
| Table | 4: Sum | nmary of Primary and Secondary Efficacy Endpoints at Week 12 | 14 |
| rabie | | | |
| | | | 16 |
| Table | 6: HA0 | Q-DI Category Scores Depending on Aids, Devices or Physical Assistance | e 23 |
| Table | 7: EIII | AR Response Criteria | 27 |
| 10010 | | | |



# **Revision History**

| Revision | Revision Date | Summary of Changes |
|----------|---------------|--------------------|
| A | 01DEC2020 | Initial release |


# SETPOINT MEDICAL

# Doc# CLP-004 Rev D, 15JUL2024

| C | 29JAN2024 | <ul> <li>Updated enrollment from "up to 250 randomized subjects" to "at least 240 and up to 250 randomized subjects" and included information for 240 subjects in power analysis (pp. 9, 10, 12 and 17)</li> <li>Updates made for consistency with current revision of CLP-001, Clinical Investigational Protocol SPM-020 (The RESET-RA Study) (pp. 9-10)</li> <li>Updates made for consistency with current version of CLP-003, Data Monitoring Committee Charter for SPM-020 (The RESET-RA Study) (pp. 11 and 13)</li> <li>Specified the Communication Plan that occurred for Interim Analysis (pp. 12-13)</li> <li>Added PTE analyses for primary outcome and key secondary outcomes (pp. 14, 16 and Appendix B pp. 9, 19-20)</li> <li>Clarified missing data approaches (pp. 14, 20, 21, 26)</li> <li>Generalized language pertaining to software requirements for statistical analysis (p. 15)</li> <li>Added additional strata for Cochran-Mantel Haenszel test and variables to the MMRM to reflect stratification factors of Stage 1 and 2 subjects (pp. 15-16, 17, table footers throughout Appendix B)</li> <li>Removed reference to collecting safety data once a subject is withdrawn from the study (p. 16)</li> <li>Added text to delineate the start of the open label/long term follow-up period for instances in which a Week 12 assessment date is missing (p. 19)</li> <li>Limited requirement to set all subsequent visits to treatment failure in the case of rescue with oral steroids considering the relatively limited half-life and averaged use between study visits. (p. 19)</li> <li>Specified corticosteroid injection rescue conditions (p. 19)</li> <li>Added detail on methods for calculating and analyzing RAMRIS scores (pp. 31-32)</li> <li>Removed information on calculation of SF-36 scores and replaced with reference to the same information which is found in the SF-36 User's Manual (p. 32)</li> <li>Clarified information on calculation of the EQ-5D-5L score (pp. 32-33, Appendix B, pp. 63-67)</li> <li>Updated description of how AEs are categorized for consistency with</li></ul> |
|---|---|---|
| D | 15JUL2024 | <ul> <li>Extended study duration by adding 6 visits as part of open-label, long-<br/>term follow-up after completion of Week 12 (pp. 9-11)</li> </ul> |




# 2 LIST OF ABBREVIATIONS

| Abbreviation | Expansion |
|----------------|--------------------------------------------------|
| ACR | American College of Rheumatology |
| AE | Adverse event |
| CARLOS | Cartilage Loss Score |
| CDAI | Clinical Disease Activity Index |
| CI | Confidence interval |
| СМН | Cochran-Mantel-Haenszel |
| СМО | Chief Medical Officer |
| CRF | Case report form |
| CSR | Clinical study report |
| DAS | Disease Activity Score |
| DMARD | Disease-modifying antirheumatic drug |
| DMC | Data monitoring committee |
| EDC | Electronic data capture |
| EGA | Evaluator's global assessment |
| eGFR | Estimated glomerular filtration rate |
| EQ-5D-5L | EuroQol 5 domains 5 levels |
| EULAR | European League Against Rheumatism |
| H <sub>0</sub> | Null hypothesis |
| Hı | Alternate hypothesis |
| HAQ-DI | Health Assessment Questionnaire Disability Index |
| hsCRP | High-sensitivity C-reactive protein |
| IL | Interleukin |
| IRB | Institutional Review Board |
| IRT | Interactive response technology |
| ITT | Intent to treat |
| JAKi | Janus kinase inhibitors |
| LDA | Low disease activity |
| LOCF | Last observation carried forward |


# Statistical Analysis Plan for Interim and Primary Analyses in SPM-020 (The RESET-RA Study)



# Doc# CLP-004 Rev D, 15JUL2024

| Abbreviation | Expansion |
|--------------|----------------------------------------------|
| MAR | Missing at random |
| MCID | Minimal clinically important difference |
| MedDRA | Medical Dictionary for Regulatory Activities |
| MMP3 | Matrix metalloproteinase 3 |
| MMRM | Mixed-effect Model Repeated Measure |
| MRI | Magnetic resonance imaging |
| NRI | Non-responder imputation |
| NRS | Numerical rating scale |
| ОС | Observed case |
| PCS | Physical component summary |
| PD | Protocol deviation |
| PF | Physical functioning |
| PMA | Premarket Approval |
| PT | Pre ferred term |
| PTE | Per-treatment evaluable |
| QC | Quality check |
| RA | Rheumatoid arthritis |
| RAMRIS | Rheumatoid Arthritis MRI Scoring System |
| RF | Rheumatoid factor |
| SAA | Serum amyloid A |
| SADE | Serious adverse device effect |
| SAE | Serious adverse event |
| SAP | Statistical analysis plan |
| SAS | Statistical Analysis Software |
| SD | Standard deviation |
| SF | Social functioning |
| SF-36 | Short Form Survey with 36 items |
| SGA | Subject's global assessment |
| SJC28 | Swollen joint count for 28 different joints |
| SOC | System organ class |

# Statistical Analysis Plan for Interim and Primary Analyses in SPM-020 (The RESET-RA Study)



# Doc# CLP-004 Rev D, 15JUL2024

| Abbreviation | Expansion |
|--------------|---------------------------------------------|
| SOP | andard operating procedure |
| TEAE | atment emergent adverse event |
| TJC28 | ender joint count for 28 different joints |
| UADE | Jnanticipated adverse device effect |
| USADE | Jnanticipated serious adverse device effect |
| WHO | World Health Organization |




### 3 INTRODUCTION

This document outlines the statistical analysis plan (SAP) for the RESET-RA study conducted by SetPoint Medical under protocol SPM-020 entitled "Vagus Nerve Stimulation Using the SetPoint System for Moderate to Severe Rheumatoid Arthritis: The RESET-RA Study." The SAP specifies the data listings, tabular summaries, and analyses to be performed for the primary, secondary and exploratory endpoints and safety evaluation using the randomized, controlled, double-blind data through Week 12 to support an application for Premarket Approval (PMA).

The data listings, tabular summaries, and analyses to be performed for the exploratory endpoints and long-term safety evaluation using the open-label follow-up data through Week 264 are detailed in a separate SAP (CLP-008). The PMA application will include supporting data on long-term safety for all subjects for whom long-term data are available at the time of application.

# 3.1 Study Objective

The overall objective of this study is to evaluate the safety and efficacy of the SetPoint System for the treatment of adult patients with active, moderate to severe RA who have had an inadequate response or intolerance to biologic or targeted synthetic DMARDs.

# 3.2 Study Design

This is an operationally seamless, 2-stage, randomized, sham-controlled, double-blind, multicenter pivotal study enrolling at least 240 and up to 250 randomized subjects at up to 45 study centers across the U.S. Enrollment will be conducted in 2 consecutive stages:

- Stage 1 with 60 randomized subjects at up to 25 study centers; and
- Stage 2 with approximately 190 randomized subjects at up to 45 study centers, including those from Stage 1.

There will be a pause in enrollment after enrollment in Stage 1 is completed. This pause in enrollment is intended to allow completion of Week 12 assessments by 60 enrolled and randomized subjects and an interim analysis (see Section 4.2). The primary analysis will occur after the last enrolled and randomized subject in Stage 2 completes Week 12 assessments, which is defined as the last subject's Week 12 visit (see Section 4.3).

After completing primary endpoint assessments at Week 12, there will be a one-way crossover of control subjects to active stimulation and a 252-week open-label follow-up with all subjects receiving active stimulation to evaluate long-term safety. Blinding will be maintained until the last enrolled and randomized subject in Stage 2 completes Week 12 assessments, and the study dataset for the primary analysis is locked.

### 3.3 Study Visits and Assessments

On the same day that written consent is obtained, each subject will undergo physical examination, RA disease activity assessments and review of prior and current RA medications to confirm their initial eligibility and baseline values for the primary and key secondary efficacy endpoints. The




remaining screening assessments, including blood work and pre-surgical clearance, will be completed prior to Implant Procedure, which shall be performed within 30 days from informed consent. Post-Surgical Clearance will be performed between 14 and 21 days from Implant Procedure. Day 0 assessments, randomization and initial device titration will be performed after completing Post-Surgical Clearance and within 14-21 days from Implant Procedure. There will be 3 additional device titration visits (Titration 1, 2, 3 at Week 1, 2 and 3, respectively), 3 follow-up RA assessment visits (Week 4, 8, 12 primary efficacy endpoint and a one-way crossover) as detailed in Schedule of Assessments (see **Appendix A**).

During open-label, long-term follow-up there will be 3 device titration visits (Titration 4, 5, 6 at Week 13, 14, 15, respectively), and 21 follow-up RA assessment visits every 12 weeks from Week 24 through Week 264 (end of study) as detailed in CLP-001.

# 3.4 Sample Size and Power

The sample size is calculated based on an estimated 60% response rate at Week 12 in the treatment group and 30% response rate at Week 12 in the control group. A sample size of 250 randomized subjects, 125 in each group, offers 96% power to detect a difference of 30% at the one-sided alpha of 0.025. If the true response rates are 50% in the treatment and 30% in the control group, the sample size of 250 subjects has 77% power to detect a difference of 20% at the one-sided alpha of 0.025. The table below provides additional power calculations for 250 subjects using estimated response rates of 20 to 40% in control and 35-70% in treatment (**Table 1**). The table also shows power if enrollment ends at 240 subjects. The decrease in power is <1% for all scenarios and most often <0.5%.

Table 1: Power Calculation Based on Estimated ACR Response Rate

| Control (%) | Treatment (%) | Difference (%) | Power<br>N = 250 | Power<br>N=240 |
|---|---|---|---|---|
| 20 | 50 | 30 | 0.967 | 0.966 |
| 20 | 45 | 25 | 0.917 | 0.916 |
| 20 | 40 | 20 | 0.812 | 0.807 |
| 20 | 35 | 15 | 0.609 | 0.601 |
| 30 | 60 | 30 | 0.959 | 0.959 |
| 30 | 55 | 25 | 0.900 | 0.898 |
| 30 | 50 | 20 | 0.773 | 0.770 |
| 30 | 45 | 15 | 0.555 | 0.549 |
| 40 | 70 | 30 | 0.959 | 0.958 |
| 40 | 65 | 25 | 0.897 | 0.893 |
| 40 | 60 | 20 | 0.762 | 0.750 |

All p-values are one-sided based on the chi-square test stratified incomplete response to JAKi and include futility stopping. Power based upon 1,000,000 simulations per scenario.




The smallest statistically significant difference that can be detected in the sample of 250 randomized subjects ranges from 11.2% to 12.8% for control rates of 20% to 40%, respectively.

### 4 TYPE OF PLANNED ANALYSIS

### 4.1 DMC Analysis

An independent Data Monitoring Committee (DMC) consisting of external, independent rheumatology, surgery and biostatistics experts will be assessing the safety and efficacy of the interventions during the trial and perform ongoing monitoring of overall study conduct. The DMC's role and responsibilities and the scope of study oversight are detailed in the DMC Charter, which defines the DMC membership, meeting logistics, and meeting frequency.

After initiation of the study, the DMC will meet regularly (i.e., after enrollment of every 15 subjects through Stage 1 and once every three months from the start of Stage 2 until the last study subject has been enrolled, and then once every six months after completing Stage 2 enrollment through Week 264. In accordance with the DMC Charter, the DMC will provide recommendations for continuing or stopping the study based on their ongoing review of cumulative safety data, including reasons for screening failure, subject disposition, AEs, SAEs, device deficiencies, protocol deviations, and concomitant medications, as well as descriptive summaries of TJC28 and SJC28. At the end of Stage 1, the DMC will review the outcomes of a formal interim analysis (see Section 4.2). Closed Sessions will occur until the study is unblinded after data lock and primary analysis.

# 4.2 Interim Analysis

One formal interim analysis is planned at the end of Stage 1 when approximately 60 randomized subjects have reached their Week 12 endpoints. The purpose of this interim analysis is to check for safety risks and a lack of efficacy prior to commencing enrollment for Stage 2. No early success stopping may possibly occur. Therefore, there is no alpha-spending as there is no possibility for early claim. As these data contribute to the overall device experience for the safety review, and no early success stopping is permissible, no Type I error inflation occurs with such interims.

# 4.2.1 Stopping rule

The DMC and FDA will review the 12-week unblinded data from Stage 1, including demographics, efficacy, safety, enrollment rates, and device implantation rates, and determine whether the following stopping rule is met:

 The observed difference between treatment and control in the proportion of subjects achieving the ACR20 response at Week 12 from baseline on the day of informed consent is less than 10%.




This stopping rule in 60 subjects balances the need to stop a trial with a projected low probability of success with a need to avoid prematurely stopping a potentially successful trial after Stage 1, given the decision is based on a dichotomous endpoint in a relatively small number of subjects.

For illustrative purposes, the table below provides stopping probabilities for 60 randomized subjects and their effect on power in 250 randomized subjects, using an estimated ACR20 response rate of 30% in the control group and a range of 35-60% in the treatment group (**Table 2**). The proposed rule has a 50% probability of stopping a study having < 30% power to meet the primary efficacy objective in 250 subjects. Type 1 error is maintained at 2.5% even without the futility stop. The last column in the table shows power if enrollment ends at 240 subjects. Again, the power decreases by < 1% in all scenarios.

Table 2: True Probability of Stopping after Stage 1 and Power of Study Success Based on Pooled Data

| Control | Treatment | Probability of Stopping | Power | Power |
|---|---|---|---|---|
| | | N = 60 (Stage 1) | N = 250 (Stage $1 + 2$ ) | N = 240 (Stage $1 + 2$ ) |
| 30% | 60% | 0.040 | 0.959 | 0.959 |
| 30% | 55% | 0.089 | 0.900 | 0.898 |
| 30% | 50% | 0.173 | 0.773 | 0.770 |
| 30% | 45% | 0.293 | 0.555 | 0.549 |
| 30% | 40% | 0.444 | 0.291 | 0.282 |
| 30% | 35% | 0.608 | 0.096 | 0.093 |
| 30% | 30% | 0.760 | 0.017 | 0.017 |

Operating characteristics calculated by simulating 1,000,000 trials per scenario using chi-square test.

### 4.2.2 Communication plan

The Stage 1 efficacy and safety data for all 60 enrolled and randomized subjects will be exported from the database and directly delivered to an independent, non-voting, biostatistician who will analyze the data and report to the DMC without any involvement from the sponsor and study biostatisticians (**Table 3**). The independent biostatistician will analyze the data by randomization group, create an interim report and submit the report with the datasets, programs and program outputs to the DMC. The interim report will be reviewed by the DMC in a Closed Session. The DMC Chairperson will convey whether or not the stopping rule is triggered to the Chief Executive Officer (CEO) of SetPoint Medical.

If the stopping rule is triggered, the CEO or designee will notify the FDA about the DMC's decision and the study will be terminated. The study will be unblinded, and all Stage 1 data analyzed. The sponsor will submit to the FDA a report with the DMC's decision together with the datasets, programs and program outputs as well as any proposals for further clinical research.

If the stopping rule is not triggered, the sponsor will initiate an IDE Supplement to the FDA to request commencement of Stage 2 enrollment, and will provide the name and contact information


# Statistical Analysis Plan for Interim and Primary Analyses in SPM-020 (The RESET-RA Study)

Doc# CLP-004 Rev D, 15JUL2024



of the statistician from whom the FDA will request the Interim Report containing unblinded data. The unblinded data will be provided directly to the FDA upon request, maintaining blinding of the sponsor. The study will advance to Stage 2 only after receiving approval from the FDA.

The DMC Chairperson may also convey to the CEO the point estimates for ACR20 response rate in the treatment and control groups, if requested by the Board of Directors or potential key investors as a contingency for financing of Stage 2. The request and response will be documented and not shared with anyone directly or indirectly involved in the management of the study. The access to and communication of the interim findings will be tightly controlled to mitigate the introduction of operational bias and documented in reports submitted by the CEO to the DMC Chairperson following the communication procedures detailed in the DMC Charter.

Table 3: Interim Data Access Matrix

| Department/Role | Blinded | Unblinded | Note |
|---|---|---|---|
| CEO | В | - | Receiving DMC's recommendations and decision as yes or no on the<br>Stage 1 stopping rule and point estimates if requested by the board or<br>investors as a contingency for financing Stage 2 |
| Clinical Operations <sup>1</sup> | В | - | Not having access to randomization assignments or DMC Closed<br>Session reports to preserve blinding of everyone involved directly or<br>indirectly in the study conduct until locking the study dataset for the<br>primary efficacy analysis at Week 12 |
| Clinical Data<br>Management | В | - | Consultants to sponsor responsible for managing EDC and IRT,<br>generating blinded data exports and not having access to randomization<br>assignments until locking the study dataset for the primary efficacy<br>analysis at Week 12 |
| Study Biostatisticians | В | - | Consultants to sponsor responsible for programming but not having access to randomization assignments until locking the study dataset for the primary efficacy analysis at Week 12 |
| Independent<br>Biostatistician | | U | Non-voting statistician reporting to DMC responsible for receiving blinded data exports, accessing randomization assignments, conducting unblinded analyses and preparing outputs for review during DMC closed sessions |
| DMC | | U | DMC chairperson, biostatistician, and clinicians participating in closed meetings |

Abbreviations: B, blinded; CMO, Chief Medical Officer; CRA, clinical research associates; DMC, data monitoring committee; EDC, electronic data capture; IRT, Interactive response technology; U, unblinded;.

<sup>1</sup>Clinical operations includes, but is not limited to, Chief Medical Officer, Vice President of Clinical Affairs, Managers of Clinical Affairs/Operations, Clinical Research Associates, Field Clinical Engineers




# 4.3 Primary Analysis

After the last enrolled and randomized subject in Stage 2 has completed all Week 12 assessments or been lost to follow-up, all outstanding data queries related to primary analysis have been resolved or determined to be unresolvable, and the data have been cleaned, finalized and locked, the study blind will be broken, and the primary analysis of the efficacy and safety data will be performed. The primary analysis at Week 12 will include all population analyses and endpoints using pooled data from all subjects enrolled and randomized in Stage 1 and 2 (**Table 4**: Summary of Primary and Secondary Efficacy Endpoints at Week 12).

Table 4: Summary of Primary and Secondary Efficacy Endpoints at Week 12

| Endpoint | Display | ITT | PTE | Sensitivity | Subgroup | Missing Data<br>Imputation |
|---|---|---|---|---|---|---|
| Primary | | | | | | |
| ACR20 response | T, L | Y | Y | Y [1] | Y | NRI |
| Key Secondary Adjusted for Multiplicity | | | | | | |
| ACR20 response from Day 0 | T, L | Y | Y | Y [1] | Y | NRI |
| DAS28-CRP good/moderate EULAR response | T, L | Y | Y | Y [2] | Y | NRI |
| DAS28-CRP response (MCID) | T, L | Y | Y | Y [2] | Y | NRI |
| HAQ-DI response (MCID) | T, L | Y | Y | Y [2] | Y | NRI |
| Exploratory Secondary [3] | | | | | | |
| ACR50/70 response | T, L | Y | | | | |
| ACR Components (TJC28, SJC28, Subject Pain, SGA, EGA, HAQ-DI, hsCRP) 20/50/70 response | T, L | Y | | - | - | - |
| Mean HAQ-DI score change at Week 12 | T, L | Y | | | | - |
| DAS28-CRP score change, LDA/remission | T, L | Y | | | | - |
| CDAI score change, LDA/remission, response | T, L | Y | | | | |
| SF-36/PCS/MCS score change | T, L | Y | | | | |
| EQ-5D-5L score change | T, L | Y | | | | |
| RAMRIS (bone erosion, osteitis, synovitis,<br>CARLOS) score change, progression (bone erosion) | T, L | Y | | - | - | - |
| Percent change in plasma biomarkers | T, L | Y | | | | |
| BI for subject's blinding assessment | T, L | Y | Y | | | |
| BI for Joint Evaluator's blinding assessment | T, L | Y | Y | | | |
| BI for Co-PI Rheumatologist's blinding assessment | T, L | Y | Y | | | |

Abbreviations: ACR, American College of Rheumatology; BI, Bang's blinding index; CARLOS, cartilage loss score; CDAI, Clinical Disease Activity Index; CRP, C-reactive protein; DAS, Disease Activity Score; EGA, evaluator's global assessment; EQ-5D-5L, EuroQol 5 domains 5 levels; EULAR, European League Against Rheumatism; HAQ-DI, Health Assessment Questionnaire Disability Index; hsCRP, high sensitivity CRP; ITT, intent to treat; L, listings; LDA, low disease activity; NRI, non-responder imputation; PTE, per treatment evaluable; RAMRIS, Rheumatoid Arthritis MRI Scoring System; SF-36, Short Form Survey with 36 items; SGA, subject's global assessment; T, tables; TJC, tender joint count; SJC, swollen joint count; Y, yes.

Note: All response rates are at Week 12 based on change from baseline, unless stated otherwise. Refer to Section 8.1 for definitions of missing data imputation strategies. Refer to Sections 8.2, 8.3, 8.4 and 8.6 for definition of response for specific endpoints. All score values are determined at all timepoints and for change from baseline.


<sup>[1]</sup> Sensitivity analyses for rescue treatments and missing data.

<sup>[2]</sup> Sensitivity analysis for timing of baseline, rescue treatments and missing data.

<sup>[3]</sup> Approaches to handling of missing data are given in Section 8.1



### 5 STATISTICAL METHODS

# 5.1 General Considerations for Data Analyses

The primary efficacy endpoint, all secondary efficacy endpoints, exploratory analyses identified here, and safety evaluations are considered *a priori* analyses because they have been prespecified in the SAP prior to locking the dataset and reviewing unblinded results. All other analyses, if any, designed subsequent to locking the dataset will be considered *post-hoc* analyses, and their results will be considered exploratory. Any *post hoc* analyses will be clearly identified in the clinical study report.

Continuous data will be summarized in terms of the mean, SD, median, minimum, maximum and number of observations, unless otherwise stated. The minimum and maximum will be reported to the same number of decimal places as the raw data recorded in the database. The mean and median will be reported to 1 more decimal place than the raw data recorded in the database. The SD will be reported to 2 more decimal places than the raw data recorded in the database. In general, the maximum number of decimal places reported shall be 4 for any summary statistic.

Categorical data will be summarized in terms of the number of subjects providing data at the relevant time point, frequency counts and percentages. If not stated otherwise, percentages will be presented with one decimal place. Percentages will not be presented for zero counts. Percentages will be calculated using n as the denominator. 100% will be presented without decimal places.

P-values greater than or equal to 0.001, in general, will be presented to 3 decimal places. P-values less than 0.001 will be presented as "< 0.001".

95% Confidence intervals (CI) will be presented to 1 more decimal place than the raw data. Unless stated otherwise, a two-sided 95% confidence level will be calculated when confidence interval is presented.

Data from the protocol-specified visits (i.e., as reported in CRF) will be used in the summary tables (**Appendix B**) and data listings (**Appendix C**). All report outputs will be produced using a software package widely recognized as acceptable for analyzing clinical data in a secure and validated environment.

The analyses for the primary and secondary efficacy endpoints are detailed below:

- The primary ACR20 response at Week 12 will be analyzed with the Cochran-Mantel-Haenszel (CMH) test. For Stage 1 subjects, stratification factors are prior inadequate response or loss of response to JAKi and RA disease severity of < 4 TJC28 or < 4 SJC28 at Day 0. For Stage 2 subjects, stratification factors are RA disease severity at Day 0 and inadequate response or loss of response to ≥ 4 biological DMARDs with ≥ 2 mechanisms of action. Other binary response endpoints at Week 12 will be analyzed similarly.</p>
- The secondary efficacy endpoints that are continuous variables (change from baseline) will be analyzed using Mixed-effect Model Repeated Measure (MMRM) statistics. The repeatedmeasures analysis will be based on the restricted maximum likelihood method assuming an unstructured covariance structure to model the within-subject errors. The model, including:




treatment group; stratification factors - inadequate response or loss of response to JAKi and RA disease severity at Day 0 (Stage 1 subjects); RA disease severity at Day 0 and inadequate response or loss of response to ≥ 4 biological DMARDs with ≥ 2 mechanisms of action (Stage 2 subjects); visit (all visits from Week 4 to Week 12); and treatment-by-visit interaction as fixed effects and baseline as a covariate, will be used to test the difference between the treatment and control group in a given efficacy endpoint change from baseline to Week 12. The data collected after receiving rescue therapy will be set to missing. Therefore, the MMRM analysis assumes a missing-at-random (MAR) mechanism for missing data due to dropout and post-rescue data.

## 5.2 Analysis Populations

Analysis population defines the subjects to be included in an analysis. The primary efficacy analyses for the primary and key secondary endpoints will be conducted on the intent-to-treat (ITT) and per-treatment-evaluable (PTE) populations. The exploratory analyses will be conducted on the ITT population as detailed in **Table 4**. All analysis populations are defined below:

- ITT population. All enrolled and randomized subjects in Stage 1 and 2.
- PTE population. Subjects from ITT population who have received the assigned treatment, who
  have no major procedural protocol deviations (see Section 9.2) and for whom follow-up data
  are available.
- Safety population. All enrolled subjects in Stage 1 and 2.

### 5.3 Baseline

Information and RA disease activity assessments collected during Screening on the day of informed consent will be used to confirm initial eligibility and as the baseline assessments for determination of the primary and key secondary efficacy endpoints (**Table 5**).

Baseline assessments for the exploratory endpoints (e.g., EQ-5D-5L, SF-36, RAMRIS, biomarkers) will be collected during Screening.

Table 5: RA Disease Activity Assessments to Be Collected on the Day of Informed Consent and Used as the Baseline Assessments for Determination of the Primary and Key Secondary Efficacy Endpoints

| Endpoint | HAQ-DI | SGA | Subject<br>Pain | TJC28 | SJC28 | EGA | hsCRP |
|---|---|---|---|---|---|---|---|
| Primary | | | | | | | |
| ACR20 response | Y | Y | Y | Y | Y | Y | Y |
| Key Secondary Adjusted for Multiplicity | | | | | | | |
| ACR20 response from Day 0 | Y | Y | Y | Y | Y | Y | Y |
| DAS28-CRP good/moderate EULAR response | | Y | | Y | Y | | Y |
| DAS28-CRP response (MCID) | | Y | | Y | Y | | Y |
| HAQ-DI response (MCID) | Y | - | | - | | - | |

Abbreviations: ACR, American College of Rheumatology; CRP, C-reactive protein; DAS, Disease Activity Score; EGA, evaluator's global assessment; EULAR, European League Against Rheumatism; HAQ-DI, Health Assessment Questionnaire Disability Index; hsCRP, high sensitivity CRP; SGA, subject's global assessment; TJC, tender joint count; SJC, swollen joint count; Y, yes.

Note: All response rates are at Week 12 based on change from baseline at the time of informed consent, unless stated otherwise.




# 5.4 Study Day Calculation

Doc# CLP-004 Rev D, 15JUL2024

Study day is calculated relative to the date of Day 0 (randomization) and will appear in the listings where applicable. If the date of event is on or after Day 0, study day will be calculated as:

Study day = date of event - date of Day 0 (randomization)

### 5.5 Randomization

After completing the protocol-required assessments at Day 0, all enrolled subjects (i.e., meeting all the inclusion and none of the exclusion criteria in whom the implant procedure was attempted) that were implanted will be assigned in a 1:1 ratio to either the treatment or the control group. The randomization scheme will be generated by the study biostatisticians and implemented centrally through Interactive Response Technology (IRT).

The randomization will be stratified to help ensure balanced distribution between treatment groups. For Stage 1 subjects, stratification factors are inadequate response or loss of response to JAKi and RA disease severity of < 4 TJC28 or < 4 SJC28 at Day 0. For Stage 2 subjects, stratification factors are RA disease severity at Day 0 and inadequate response or loss of response to  $\ge 4$  biological DMARDs with  $\ge 2$  mechanisms of action.

Enrollment will continue until at least 240 and up to 250 subjects are randomized. If there are discrepancies in stratification factor values between the IRT and EDC systems, the data recorded in the EDC will be used for analyses.

### 5.6 Change from Baseline Calculation

Percent change from baseline to any time point (e.g., Day 0, Week 4, 8 or 12) will be calculated as follows:

[Value (Post-baseline) - Value (Baseline)] / Value (Baseline) x 100

A negative value reflects a decrease in a given parameter, while a positive relative difference reflects an increase in the parameter.

### 5.7 Relative Difference Calculation

Serial Number: 8f9f5f23-bec3-4670-b6ee-899072db2597 accessed by Melissa Evangelista (MEVANGELISTA) on Thu, 28 Aug 2025 18:19:41 GMT.

Relative difference between treatment and control groups at any time point will be calculated as: [Value t – Value c] / Value x 100

A negative relative difference reflects a decrease in a given parameter on the treatment side compared to control, while a positive relative difference reflects an increase in the parameter on the treatment side compared to control.




### 5.8 Missing Dates

In analysis of AEs and medication, a complete date will be established in order to identify AEs or medication as occurring during treatment or not. For handling partially reported onset/start and outcome/end dates for AEs or medication the following algorithms are applied:

### AEs:

- Missing onset day, but month and year present:
  - If baseline visit occurred in the same month and year as the occurrence of the AE, then
    the onset day of the event is assigned to the date of baseline visit.
  - Otherwise, the onset day is set to the first day of the month (e.g., XX-Sep-2020 is considered as 01-Sep-2020).
- Missing onset day and month, but year present:
  - If baseline visit occurred in the same year as the occurrence of the AE, then the onset date of the event is assigned to the date of baseline visit.
  - Otherwise, the onset day and month is set to 01 January (e.g., XX-XXX-2020 is considered as 01-Jan-2020).
- Missing outcome day, but month and year present:
  - The day is set to the last day of the month (e.g., XX-Sep-2020 is considered as 30-Sep-2020).
- Missing outcome day and month, but year present:
  - The outcome day and month is set to 31 December (e.g., XX-XXX-2020 is considered as 31-Dec-2020).

### Medications:

- Missing start day, but month and year present:
  - If baseline visit occurred in the same month and year as the occurrence of the medication, then the start day of the medication is assigned to the date of baseline visit. Otherwise, the start day is set to the first day of the month (e.g., XX-Sep-2020 is considered as 01-Sep-2020).
- Missing start day and month, but year present:
  - If baseline visit occurred in the same month in the same year as the occurrence of the medication, then the start date of the medication is assigned to the date of baseline visit.
  - Otherwise, the start day and month is set to 01 January (e.g., XX-XXX-2020 is considered as 01-Jan-2020).
- Missing stop day, but month and year present:
  - The day is set to the last day of the month (e.g., XX-Sep-2020 is considered as 30-Sep-2020).
- Missing stop day and month, but year present:


# SETPOINT MEDICAL

### Doc# CLP-004 Rev D, 15JUL2024

- The stop day and month is set to 31 December (e.g., XX-XXX-2020 is considered as 31-Dec-2020).
- Date of RA diagnosis:
  - Missing day, but month and year present:
    - Date is set to the first day of the month (e.g., XX-Sep-2010 is considered as 01-Sep-2010).
  - Missing day and month, but year present:
    - Date is set to 01 January (e.g., XX-XXX-2010 is considered as 01-Jan-2010)
- Week 12 visit:
  - If the Week 12 visit date is missing (e.g., the subject missed the Week 12 assessment but is still participating in the study), the Week 12 visit date will be set to the date that subject's MicroRegulator was re-registered for open-label, long-term follow-up

### 5.8.1 Missing data for efficacy and safety endpoints

Missing data for each efficacy endpoint will be handled as described in Sections 8.2, 8.3, 8.4 and 8.6.

For continuous endpoints, change from baseline will be set to missing at visits with missing postbaseline values or where data were imputed to missing. Continuous efficacy endpoints will be set to missing for subjects who received rescue treatment before Week 12.

For binary endpoints, subjects with missing efficacy data, early withdrawals, or subjects who received rescue treatment before Week 12 will be imputed as non-responders and therefore treated as a failure (e.g., no ACR20/50/70 response, DAS28-CRP remission or no moderate/good EULAR response).

Additional rules for handling of missing data and rescue treatments are detailed below:

- Missing efficacy data. Visits with missing data (due to a missed visit or missing component
  of a composite endpoint) will be set to treatment failure.
- Early withdrawals. Only visits following the early withdrawal visit will be set to treatment failure.
- Prednisone equivalent >10 mg/day. The visit after a period (time from previous visit up to the
  day before the current visit) of average daily corticosteroid use exceeding 10 mg/day
  prednisone will be set to treatment failure and continuous endpoints set to missing due to
  rescue.
- Corticosteroid injection. If subject received a corticosteroid injection within 30 days prior to
  a study visit, that visit will be set to treatment failure and continuous endpoints set to missing
  due to rescue.
- b/ts/csDMARD. Subjects who receive treatment before Week 12 with biologic, targeted synthetic, or additional conventional synthetic DMARD, or increased dose of background


# Statistical Analysis Plan for Interim and Primary Analyses in SPM-020 (The RESET-RA Study)



### Doc# CLP-004 Rev D, 15JUL2024

conventional synthetic DMARD will be set to treatment failure at all subsequent visits and continuous endpoints set to missing due to rescue.

- Missing baseline value. For efficacy endpoints, a missing value at baseline will not be imputed, and the endpoint will be set to missing for all visits.
- Missing analytes/ retests. If an analyte value is missing/its concentration cannot be reliably determined (e.g., sample was lost, damaged, etc.), a retest value will be used for that analyte. If an initial value is non-missing and reliable but the analyte was retested, the value that coincides with the date of clinical assessment will be used. If neither an initial nor retest value is available, the analyte value will be set to missing.

### 5.8.2 Multiple Assessments and Visits

If a variable (e.g., MRI, TJC, SJC) has been assessed multiple times at the same visit, only the last assessment will be used.

Only completed scheduled visits will be included in summary tables (**Appendix B**). Listings will include scheduled and unscheduled visits (**Appendix C**).

### 5.9 Data Assurance

All tables, figures and data listings to be included in the report will be independently checked for consistency, integrity and in accordance with the study sponsor's SOPs.

### 5.10 Consistency Across Study Centers

The consistency of ACR 20 response rate across the study centers will be evaluated using Breslow Day test for homogeneity. Any center with < 5 subjects with ACR20 data in any treatment group will be pooled from largest to smallest until the pooled center has 5 subjects in each treatment group. If heterogeneity is found, exploratory analysis will be conducted to investigate the issue. This may include analysis adjusted for baseline characteristics that significantly differ across sites.

### 5.11 Coding Dictionaries

AEs will be coded using the Medical Dictionary for Regulatory Activities (MedDRA, version 21.0 or later). Concomitant medications will be coded using the March 2019 or later version of the WHO Drug Global dictionary.

### 6 SUBJECT DISPOSITION

### 6.1 Subject Enrollment and Disposition

A summary of subject enrollment will be provided by treatment group for each site. The summary will present the number and percentage of subjects enrolled. For each column, the denominator for the percentage calculation will be the total number of subjects analyzed for that column.


## Statistical Analysis Plan for Interim and Primary Analyses in SPM-020 (The RESET-RA Study) Doc# CLP-004 Rev D, 15JUL2024



A similar enrollment table will be provided by stratification factor stratum. The denominator for the percentage of subjects in the stratum will be the total number of enrolled subjects. If there are discrepancies in the value used for stratification assignment between the IRT and EDC systems, the value collected in the EDC will be used for the summary.

A listing of subjects with discrepancies in the value used for stratification assignment between the IRT and EDC systems at the time of data finalization will be provided.

The randomization schedule used for the study will be provided in a listing and as an appendix to CSR.

The number and percentage of subjects in whom the implant procedure was attempted and in whom it was successful will be summarized. The primary reason for subject discontinuation will be summarized. Screen failures will be reported in the data listings and the summary table. Data for subject disposition, including termination date and reason, will be listed.

### 7 DEMOGRAPHICS AND BASELINE CLINICAL CHARACTERISTICS

Demographic data (i.e., age, gender, race, ethnicity) and baseline clinical characteristics (i.e., years since RA diagnosis, treatment history with biologic, targeted synthetic and conventional synthetic DMARDs, baseline clinical variables) will be summarized per treatment group and overall using descriptive statistics for continuous variables and using number and percentage of subjects for categorical variables.

### 8 EFFICACY ANALYSES

#### 8.1 General Considerations

## 8.1.1 Missing endpoint data imputation

Below are the descriptions for the imputation methods that may be used throughout the efficacy analyses:

- Observed case (OC). Missing values remain missing. For the categorical composite endpoints, in the case that some components are missing, the composite endpoint assessment will be derived based on the non-missing components. If non-missing components are not sufficient to determine final composite endpoint, then the composite endpoint will be set as missing. For continuous composite endpoints, if any components are missing, the composite endpoints will be set as missing.
- Last observation carried forward (LOCF). Baseline and Day 0 measurements will not be carried forward to post-baseline. Only measurements post Day 0 will be LOCF for continuous and binary response measures. For the composite endpoints, the last non-missing, post-Day 0 observation will be carried forward to subsequent visits for each individual component first, and then the composite endpoints using individual components imputed by LOCF will be calculated as described above. If a subject does not have a non-missing observed record for a post-Day 0 visit, the last post-Day 0 record prior to the missed visit will be used. If the last non-missing observation prior to the missing visits cannot be determined due to multiple


# SETPOINT MEDICAL

### Doc# CLP-004 Rev D, 15JUL2024

measurements occurring at the same time or the time not available within the same day, the worst outcome will be used for LOCF. If missing components still exist after LOCF, the composite endpoints will be calculated using the same rules as described in OC.

Non-responder imputation (NRI). For all binary response measurements, starting from OC, all
missing will be set as non-responders.

If subject only had baseline measurements, LOCF and OC analyses will not include this subject. But this subject will be treated as non-responder in NRI analyses.

### 8.2 Clinical Variables

### 8.2.1 TJC28 and SJC28

The assessment for swelling is the total number of joints with a present swelling and ranges from 0 to 28 for SJC28. The assessment for tenderness is the total number of joints with a present tenderness and ranges from 0 to 28 for TJC28. The following 28 joints will be taken into account for TJC28 and SJC28: shoulder (2 joints), knee (2), elbow (2), wrist (2), fingers (PIP, MCP: 20). All joint assessments will be performed by an independent, blinded joint evaluator. Artificial, ankylosed and missing joints are excluded from swelling and tenderness assessment.

If there are missing observations for tender or swollen joints, then the remaining observations will be assessed and weighted by dividing the number presented by number of non-missing and by multiplying by 28 for the joint count. No imputations for individual joints will be done. If a joint is not evaluable at baseline, then that joint is set to missing throughout the study. If data for more than 50% of the joints are missing at the time of a given assessment, then the total count will be set to missing for that visit.

### 8.2.2 SGA

Subjects will complete a global assessment of their RA disease activity using the subject's global assessment of disease activity (SGA) item, a numerical rating scale (NRS) from "0" (inactive) to "10" (very active).

No imputations for missing data will be done.

### 8.2.3 Subject's Pain Assessment

Subjects will assess the severity of their current RA-related pain using a NRS from "0" (no pain) to "10" (worst pain imaginable).

No imputations for missing data will be done.

### 8.2.4 EGA

The joint evaluator will complete the evaluator's global assessment of disease activity item (EGA) using a NRS from "0" (inactive) to "10" (very active).




No imputations for missing data will be done.

# 8.2.5 HAQ-DI

The functional status of the subject will be assessed by means of the Health Assessment Questionnaire Disability Index (HAQ-DI). This 20-question instrument assesses the degree of difficulty a person has in accomplishing tasks in 8 functional areas:

- Dressing and grooming
- Arising
- Eating
- Walking
- Hygiene
- Reach
- Grip
- Common daily activities

Each functional area contains at least 2 questions. For each question, there is a 4-level response set that is scored from 0 (without any difficulty) to 3 (unable to do). If aids or devices or physical assistance are used for a specific functional area (**Table 6**), and the maximum response of this functional area is 0 or 1, the according value is increased to a score of 2.

Table 6: HAQ-DI Category Scores Depending on Aids, Devices or Physical Assistance

| Aid or Equipment | Will be Associated with Category Score |
|---|---|
| Walking stick/frame, crutches, wheelchair | Walking |
| Aids used for dressing | Dressing and grooming |
| Specially adapted utensils | Eating |
| Specially adapted chair | Rising |
| Raised toilet seat, bath rail, bath seat | Hygiene |
| Long-handled appliance in bathroom | Hygiene |
| Long-handled appliance for reaching | Reach |
| Jar opener | Grip |
| Other (1) | Dressing & grooming, rising, eating, walking |
| Other (2) | hygiene, reach, grip, common daily activities |

If "other" is marked as an aid or equipment, then this can be assigned to a group of four functional areas and will be handled as an aid or equipment for each of the four functional areas. Therefore,


# Statistical Analysis Plan for Interim and Primary Analyses in SPM-020 (The RESET-RA Study)



Doc# CLP-004 Rev D, 15JUL2024

if the maximum score of a functional area is 0 or 1, that value is increased to a score of 2 for each of the four functional areas.

Regarding these corrections, the highest response within each functional area determines the score of that specific functional area. If no questions within a given functional area were answered, no score will be provided for that category (even if answers on aids or equipment are available).

HAQ-DI score is only calculated if there are at least 6 functional area scores available. The average of these non-missing functional area scores defines the continuous HAQ-DI score ranging from 0 to 3. If there are less than 6 functional area scores available, no imputation will be done, and the HAQ-DI will be set to missing for the corresponding assessment.

A HAQ-DI score reduction from baseline by 0.22 represents the MCID.

### 8.2.6 hsCRP

Blood concentration of hsCRP (mg/L) for all subjects will be determined by a central laboratory.

### 8.3 Primary Efficacy Endpoint

ACR20 response at Week 12

### 8.3.1 Definition

A subject achieves ACR20 response when this subject experiences a ≥ 20% improvement from baseline on the day of informed consent to Week 12 in TJC28, SJC28, and at least 3 of the following 5 items:

- Subject's pain assessment
- SGA
- EGA
- HAQ-DI
- hsCRP

For all visits, if any of the component scores are missing, then those scores will be considered as not having met the criteria for improvement. If 3 or more of the 5 remaining ACR measures are missing, ACR20 will each be considered as "no response" in the final dataset.

For component scores with missing baseline values or a baseline value of 0, the percentage improvement cannot be calculated, and the component will be considered as not having met the criteria for improvement for all visits.

### 8.3.2 Statistical Hypothesis

The hypothesis of interest is:


Statistical Analysis Plan for Interim and Primary Analyses in SPM-020 (The RESET-RA Study) Doc# CLP-004 Rev D, 15JUL2024



$$H_0: p_t - p_c = 0$$

$$H_1: p_t - p_c > 0$$

where  $p_t$  is the response rate in the treatment group and  $p_c$  is the response rate in the control group. The study will test the null hypothesis (H<sub>0</sub>) that there is no difference between the treatment and control groups in the proportion of subjects achieving ACR20 response at Week 12 versus the alternative hypothesis (H<sub>1</sub>) that treatment group response rate exceeds the control group response rate. The study will be considered successful if there is a statistically significant improvement in the proportion of subjects with ACR20 response in favor of the SetPoint System at the one-sided alpha of 0.025.

### 8.3.3 Primary Analysis

The primary analysis of the ITT population will be the CMH test. ACR20 response is the outcome variable. Subjects who received rescue treatment before Week 12 or who had missing data at Week 12 will be considered non-responders in the primary analysis.

### 8.3.4 Sensitivity Analyses

### Sensitivity analysis for rescue intervention

Because rescue interventions can potentially confound the primary efficacy outcome, a sensitivity analysis will be performed to test the robustness of the efficacy conclusion to actual interventions given.

In this analysis, data imputations will be performed if intervention is given prior to Week 12, then ACR20 value prior to the intervention will be used in the analysis (LOCF).

### Sensitivity analysis for missing data

Subjects with missed visit, lost to follow-up or partial ACR20 will be considered as missing data. If more than 5% of the primary efficacy data are missing, the following imputation analyses will be performed to assess the sensitivity of conclusions to missing data:

- A "tipping point" analysis in which all the primary analysis will be performed with all combinations of missing data. For instance, with M<sub>C</sub> subjects with missing Week 12 data in the control group and M<sub>t</sub> subjects with missing Week 12 data in the treatment group, then all Mc × Mt possible interims are completed. Between-treatment comparisons will be performed using a chi-squared test for each possible combinations of J (from 0 to Mc) and K (from 0 to Mt). The tipping point analysis will include the following cases:
  - Impute "ACR20 responder" for all missing values in the control group and "ACR20 nonresponder" in the treatment group; this is a worst-case imputation.
  - Impute "ACR20 non-responder" for all missing values in the control group and "ACR20 responder" in the treatment group; this is a best-case imputation.


# SETPOINT MEDICAL

### Doc# CLP-004 Rev D, 15JUL2024

- If the decision about the null hypothesis using worst-case imputation agrees with the decision about the null hypothesis using best-case imputation, the tipping point analysis will include no further cases.
- In addition, an analysis will be conducted in which ACR20 responder or non-responder will be imputed based upon the last observed value (at Week 8 or Week 4) according to fully conditional specification predictive mean matching multiple imputation approach of Berglund and Heeringa (2014).

### 8.3.5 Subgroup Analyses

The primary efficacy endpoint will be examined using the following subgroups (including but not limited to the ones listed below):

- Age (< 65 vs. ≥ 65)</li>
- Gender (male vs. female)
- Race (White vs. Non-White, including Black or African American, American Indian or Alaska Native, Asian, Native Hawaiian or other Pacific Islander)
- Duration of RA (< 5 years vs. ≥ 5 to < 10 years vs. ≥ 10 years)</li>
- Number of prior biologic and targeted synthetic DMARDs (e.g., < 4 vs. ≥ 4)</li>
- Prior use of JAKi (Yes vs. No)
- RA disease activity at Screening (DAS28-CRP ≤ 5.1 vs. DAS28-CRP > 5.1)
- Moderate-to-severe RA at Day 0 (< 4 TJC28 or < 4 SJC28 vs. ≥ 4 TJC28 and ≥ 4 SJC28)</li>

## 8.4 Key Secondary Endpoints

- ACR20 response at Week 12 from Day 0
- DAS28-CRP good/moderate EULAR response at Week 12 from baseline
- DAS28-CRP response (MCID -1.2) at Week 12 from baseline
- HAQ-DI response (MCID -0.22) at Week 12 from baseline

### 8.4.1 Definitions of key secondary endpoints

# ACR20 response at Week 12 from Day 0

A subject achieves ACR20 response when this subject experiences a  $\geq$  20% improvement at Week 12 from the post-surgical baseline at Day 0 in TJC28 and SJC28 and 3 out of 5 ACR core measures and follows the same general and statistical analyses as for ACR20 response at Week 12 from baseline on the day of informed consent (see Section 8.3.1).




### DAS28-CRP good/moderate EULAR response at Week 12

DAS28-CRP EULAR response at Week 12 is defined based on the combination of the current DAS28-CRP score and its improvement relative to baseline on the day of inform consent as illustrated in **Table 7**.

Table 7: EULAR Response Criteria

| DAS28-CRP Score | DAS28-CRP Score Decrease from Baseline Value | | |
|---|---|---|---|
| Week 12 | > 1.2 | > 0.6 to ≤ 1.2 | ≤ 0.6 |
| ≤3.2 | Good response | Moderate response | No response |
| $> 3.2 \text{ to} \le 5.1$ | Moderate response | Moderate response | No response |
| > 5.1 | Moderate response | No response | No response |

A subject is considered having a moderate treatment response at Week 12 if:

- DAS28-CRP score improvement from baseline to Week 12 is > 0.6 and ≤ 1.2, and the DAS28-CRP score at Week 12 is ≤ 5.1; or
- DAS28-CRP score improvement from baseline to Week 12 is > 1.2, and the DAS28-CRP score at Week 12 is > 3.2.

A subject is considered having a good treatment response at Week 12 if:

 DAS28-CRP score improvement from baseline to Week 12 is > 1.2 and the DAS28-CRP score at Week 12 is ≤ 3.2.

If the post-baseline DAS28-CRP score is missing, then the corresponding EULAR category will be missing.

Missing DAS28-CRP values will be considered as not achieving remission.

### DAS28-CRP response (MCID -1.2) at Week 12

A DAS28-CRP score reduction by at least 1.2 from baseline on the day of inform consent to Week 12 represents the MCID response (see Section 8.6.1).

### HAQ-DI response (MCID -0.22) at Week 12

A HAQ-DI score reduction by at least 0.22 from baseline on the day of inform consent to Week 12 represents the MCID response (see Section 8.2.5).

### 8.5 Multiplicity Adjustment of Key Secondary Endpoints

This section describes the methods that will be used to control the familywise type 1 error rate (FWER) among these 4 secondary endpoints. If and only if the primary efficacy objective is met,


# SETPOINT MEDICAL

### Doc# CLP-004 Rev D, 15JUL2024

the Hochberg's step-up procedure (Hochberg 1988) will be used to control the FWER at a 1-sided significance level of 0.025 for the following 4 secondary endpoints:

ACR20 response at Week 12 from Day 0

O Test: H<sub>0</sub>: pt - pc = 0 H<sub>1</sub>: pt - pc > 0, using stratified CMH test, as detailed in Section 5.1

DAS28-CRP good/moderate EULAR response at Week 12 from baseline on the day of informed consent

• Test:  $H_0$ : pt - pc = 0  $H_1$ : pt - pc > 0, using stratified CMH test

DAS28-CRP response (MCID -1.2) at Week 12 from baseline on the day of informed consent

O Test: H<sub>0</sub>: pt - pc = 0 H<sub>1</sub>: pt - pc > 0, using stratified CMH test

HAQ-DI response (MCID -0.22) at Week 12 from baseline on the day of informed consent

Test: H<sub>0</sub>: pt - pc = 0 H<sub>1</sub>: pt - pc > 0, using stratified CMH test

The procedures rank the p-values from the above 4 tests from the least significant and examines the other p-values in a sequential manner until it reaches the most significant one, i.e., p(4) > p(3) > p(2) > p(1).

The decision rule for the Hochberg procedure is defined as follows:

- Step 1. If p(4) > 0.025, retain H(4) and go to the next step. Otherwise reject all hypotheses and stop.
- Step 2. If p(3) > 0.025/2, retain H(3) and go to the next step. Otherwise reject all hypotheses and stop.
- Steps 3. If p(2) > 0.025/3, retain H(2) and go to the next step. Otherwise reject all remaining hypotheses and stop.
- Steps 4. If p(1) > 0.025/4, retain H(1) otherwise reject it.

The adjusted p-value is calculated as detailed below:

Adjusted p(i) = p(4) for i = 4 other adjusted p(i) = minimum of [adjusted p(i+1), (5-i)\*p(i)] for i = 3, 2, 1.

If any adjusted p-value exceeds 1, it is set to 1. Using this procedure, any adjusted p-value that is < 0.025 is statistically significant and supports a claim for the corresponding endpoint, while any adjusted p-value  $\ge 0.025$  is not statistically significant. Both adjusted and unadjusted p-values will be reported.

### 8.5.1 Sensitivity analyses of key secondary endpoints

The key secondary efficacy endpoints will be evaluated using the same sensitivity analyses for rescue intervention and missing data as those used for the primary efficacy endpoint (see Section




**8.3.4**). In addition, a sensitivity analysis for timing of baseline assessment will be performed to evaluate the impact of it on the secondary efficacy conclusions.

# Sensitivity analysis for timing of baseline assessment

In this analysis, the baseline is defined as Day 0 assessments performed prior to randomization and initiation of stimulation.

### 8.5.2 Subgroup Analysis of Key Secondary Endpoints

The 4 key secondary endpoints will be summarized for the following subgroups:

- Number of prior biologic and targeted synthetic DMARDs (e.g., < 4 vs. ≥ 4)</li>
- Prior use of JAKi (Yes vs. No)
- RA disease activity at informed consent (DAS28-CRP ≤ 5.1 vs. DAS28-CRP > 5.1)
- Moderate-to-severe RA at Day 0 (< 4 TJC28 or < 4 SJC28 vs. ≥ 4 TJC28 and ≥ 4 SJC28)</li>

# 8.6 Exploratory Secondary Endpoints

The exploratory secondary endpoints through Week 12 include:

- ACR50/70 response
- Component (TJC28, SJC28, Subject Pain, SGA, HAQ-DI, EGA, hsCRP) 20/50/70 response
- DAS28-CRP score change from baseline and LDA/remission
- CDAI score change from baseline, LDA/remission and MCID response
- Mean HAQ-DI score change from baseline
- RAMRIS bone erosion, osteitis, synovitis, and CARLOS score changes from baseline
- RAMRIS bone erosion progression (> 0.5) rate from baseline
- SF-36/PCS/MCS score change from baseline
- EQ-5D-5L score change from baseline and response
- Percent change in plasma biomarker concentrations (e.g., IL-1, SAA, MMP-3)

# 8.6.1 Definitions of Exploratory Secondary Endpoints

### ACR50/70 response at Week 12

ACR50/70 response corresponds to 50% and 70% improvement at Week 12 from baseline on the day of informed consent, respectively, in TJC28 and SJC28 and 3 out of 5 ACR core measures and follows the same general and statistical analyses as for ACR20 (see Section 8.3.1).




### Component 20/50/70 response

20/50/70 response for each component (TJC28, SJC28, Subject Pain, SGA, HAQ-DI, EGA, hsCRP) corresponds to 20, 50 and 70% improvement from baseline to Week 12, respectively (see Section 8.2), and follows the same general and statistical analyses as for ACR20 (see Section 8.3.1).

# DAS28-CRP score change and LDA/remission

The Disease Activity Score (DAS) is a derived measurement of 4 components with differential weighting:

- TJC28
- SJC28
- hsCRP (mg/L)
- SGA

A total score ranges from 0 to 10 and is computed as follows:

DAS28-CRP = 0.56 \* sqrt(TJC28) + 0.28 \* sqrt(SJC28) + 0.36 \* ln(CRP+1) + 0.014 \* SGA + 0.96

If one of the components is missing at an individual assessment point, the DAS28-CRP value for that assessment will be set to missing. An alternative imputation method for missing components may be applied as described in Section 8.1.

The DAS28-CRP score corresponds to the current RA activity:

- 0 to < 2.6 Remission</li>
- 2.6 to < 3.2 Low disease activity (LDA)</li>
- 3.2 to ≤ 5.1 Moderate activity
- > 5.1 High activity

If one of the components is missing at a given assessment point, no imputations will be done, and the DAS28-CRP value for that assessment will be set to missing.

### CDAI LDA/remission and MCID response at Week 12

The Clinical Disease Activity Index (CDAI) is a composite score consisting of the sum of:

- SJC28
- TJC28
- SGA/10
- EGA/10


# SETPOINT MEDICAL

### Doc# CLP-004 Rev D, 15JUL2024

The CDAI score is calculated as follows and ranges from 0 to 76 with higher values representing higher disease activity:

CDAI = TJC28 + SJC28 + SGA + EGA

The CDAI score corresponds to the current RA activity:

- 0 to < 2.8 Remission</li>
- >2.8 to ≤ 10 Low disease activity (LDA)
- >10 to ≤ 22 Moderate activity
- > 22 High activity

The MCID varies depending on RA activity at baseline:

- -12 for high activity
- -6 for moderate activity
- 1 for low activity

If one of the components is missing at a given assessment point, no imputations will be done, and the CDAI value for that assessment will be set to missing. An imputation method for missing components may be applied as described in Section 5.8.1.

# HAQ-DI score change from baseline

Change from baseline on the day of inform consent to Week 12 in mean HAQ-DI score as determined by subjects (see Section 8.2.5).

### RAMRIS score and progression at Week 12

RAMRIS is the standardized system for RA MRI scoring of 4 different types of joint pathologies in the wrist and the hand. A total score for each pathology is generated by the summation of individual joint/bone scores as follows:

- Synovitis. 8 joints each scored on a scale from 0 = normal to 3 = severe, resulting in a total score from 0 to 24.
- Bone erosion. 25 bones each scored on a scale from 0 to 10, resulting in a total score from 0 to 250. An increase of > 0.5 from baseline to Week 12 will represent disease progression.
- Osteitis. 25 bones scored on a scale from 0 to 3, resulting in a total score from 0 to 75.
- CARLOS (cartilage loss). 25 joints each scored on a scale from 0 to 4, resulting in a total score from 0 to 100.

Subjects will undergo MRI at Screening (baseline) and Week 12, and the MRI images will be scored by independent centralized blinded readers. Scores for each bone/joint will be calculated as the average of the score provided by each of the two readers. If a RAMRIS score from one of the readers is missing, then the RAMRIS score from the other reader will be used. If the score was


# Statistical Analysis Plan for Interim and Primary Analyses in SPM-020 (The RESET-RA Study)



### Doc# CLP-004 Rev D, 15JUL2024

missing for both readers at any given time point, the average score is considered missing. An imputation method for missing components may be applied as described in Section 5.8.1. A listing will be provided that presents change in total score from baseline by subject for each of the RAMRIS pathologies. The number of observations and the total score change mean, minimum, maximum and 95% confidence interval will be presented for the treatment and control groups in a table.

The smallest detectable change (SDC) will be calculated for each of the joint pathologies to assess whether a patient experienced a change beyond measurement error. The SDC is calculated as:

 $\pm 1.96 \text{ x SD}_{\Delta(\text{CHANGE SCORES})}/(\sqrt{2} \text{ x } \sqrt{k})$ 

where CHANGE SCORE = change in RAMRIS total score between two timepoints,  $SD_{\Delta(CHANGESCORES)}$  represents the standard deviation of difference in change scores between the two readers, and k= the number of readers (Bruynesteyn et al., 2005).

In addition, subgroup analyses will be performed for subjects with and without baseline joint damage that is predictive of future progression (Gandjbakhch et al, 2014).

# SF-36/PCS/MCS score change from baseline to Week 12

Health-related quality of life will be assessed using the subject-completed Medical Outcomes Study Short-Form 36 (SF-36), which is a generic health survey that contains 36 questions covering eight domains of health. The SF-36 yields an 8-scale profile of functional health and well-being scores as well as physical and mental component health summary scores. The version 2, 4-week recall questionnaire will be used. Recoding, calculations, and standardization will be done as recommended in the User's manual for the SF-36 (Mariush, 2011). Each of the 8 domain scores is the sum of some of the overall 36 item scores.

Domain scores will only be calculated if less than half of the item scores are missing. Missing item scores will be imputed as the mean of the other item scores within the same domain. If at least half of the item scores of a domain are missing, imputation will not be performed, and the domain will be set to missing. An imputation method for missing components may be applied as described in Section 5.8.1.

# EO-5D-5L response at Week 12

A standardized instrument for measuring general health status within the following 5 dimensions:

- Mobility
- Self-care
- Usual activities
- Pain/discomfort


# Statistical Analysis Plan for Interim and Primary Analyses in SPM-020 (The RESET-RA Study)

# Doc# CLP-004 Rev D, 15JUL2024



Anxiety/depression

Each dimension is scored on 5-point scale as:

- 1 = No problems
- 2 = Slight problems
- 3 = Moderate problems
- 4 = Severe problems
- 5 = Extreme problems/Unable

General health status is scored on a VAS (0 = poor to 100 = the best). An imputation method for missing components may be applied as described in Section 5.8.1.

Reduction in the proportion of subjects with problems (moderate, severe or extreme) will represent improvement.

An EQ-5D summary index score can be derived by applying a formula that attached weights, or index values, to each of the levels in each dimension. The index is calculated by deducting the appropriate weights from the value for full health (i.e., 1). Value sets are country specific and can be obtained from the EuroQol website (EuroQol Research Foundation, 2023).

# 8.6.2 Analysis of Exploratory Secondary Endpoints

The following endpoints will be analyzed with the CMH test, as described in Section 5.1:

- ACR50/70 response at Week 12
- DAS28-CRP LDA/remission at Week 12
- CDAI response at Week 12
- HAQ-DI response at Week 12
- EQ-5D-5L response at Week 12
- RAMRIS bone erosion progression (> 0.5) at Week 12

The MMRM will be used to analyze the following endpoints, as described in Section 5.1:

- Mean CDAI score change from baseline to Week 12
- Mean HAQ-DI score change from baseline to Week 12
- Mean EQ-5D-5L score change from baseline to Week 12
- Mean SF-36/PCS/MCS score change from baseline to Week 12
- Mean RAMRIS bone erosion, osteitis, synovitis, and CARLOS score change from baseline to Week 12
- Percent change in plasma biomarkers (e.g., IL-6, SAA, MMP3)




### 8.7 Blinding Assessment

The effectiveness of blinding of subjects, joint evaluators and Co-PI Rheumatologists will be evaluated at Week 4 and Week 12 using a blinding questionnaire with the following questions:

- I strongly believe I am [or subject is] in the treatment group and receiving therapeutic stimulation
- I somewhat believe I am [or subject is] in the treatment group and receiving therapeutic stimulation
- I somewhat believe I am [or subject is] in the control group and receiving non-therapeutic stimulation
- I strongly believe I am [or subject is] in the control group and receiving non-therapeutic stimulation
- I don't know which group I am [or subject is] and which stimulation I am [or subject is] receiving

The statistical test will be Bang's blinding index (BI) and its associated 95% confidence interval (Bang 2010). The BI will be calculated for both the ITT and PTE populations.

### 9 SAFETY EVALUATION

#### 9.1 AE and SAEs

The incidence of AEs and SAEs from informed consent date to Week 12 will be tabulated. Each AE will be evaluated by clinical investigators in terms of seriousness, severity (i.e., mild, moderate, severe) and strength of relationship (i.e., not related, unlikely related, probably related, definitely related, indeterminate) to the implant procedure, implant device, stimulation, Energizer, and explant procedure. Any AE that is determined by a participating investigator to be related (definitely related or probably related) to the implant procedure, implant device, stimulation, Energizer, or explant procedure will be categorized as device related. In unblinded analyses, if the subject was assigned to the control group, but the AE indicates relationship to stimulation, the AE relationship will be updated to "not related."

For all AE tables, a subject reporting the same adverse event more than once will be counted once when calculating the number and percentage of subjects with that particular event. If a subject reports the same AE more than once or has the same AE on multiple occasions, the maximum severity grade and relationship will be presented.

The frequencies and percentages of treatment-emergent adverse events will be presented by MedDRA system organ class (SOC) and preferred term (PT). Complete subject listings of all AE will be provided. For each AE the following will be specified: start and stop dates, severity grade, MedDRA SOC and PT, relationship (not related, unlikely related, probably related, definitely related, or indeterminate) to the implant procedure, implant device, stimulation, Energizer, and explant procedure, , as well as action taken, outcome of the adverse event, and seriousness.




### 9.2 Protocol Deviations

All protocol deviations will be tabulated with reasons for deviations, reviewed by sponsor using blinded data and reported in compliance with the study protocol, IRB requirements and sponsor's SOPs.

Protocol deviations will be categorized as major procedural if a study subject:

- Undergoes any study-related procedure before signing an IRB-approved informed consent form, or
- Receives study treatment not consistent with the treatment assignment, or
- Is no longer eligible but received study treatment.

Summary tables with the number and percentage of subjects with protocol deviations will be provided by treatment group and by type of deviation (**Appendix B**). A by-subject listing of all protocol deviations will be provided (**Appendix C**).

A sensitivity analysis for protocol deviations that could impact the primary endpoint will be performed to address potential bias from minor deviations. Protocol deviations will be reviewed by the Sponsor and those identified as possibly impacting the primary endpoint will be summarized in the CSR.

### 9.3 Device Deficiencies

All device deficiencies related to the identity, quality, durability, reliability, safety or performance of the study device, including device malfunctions, use errors, and inadequate labelling will be tabulated. Summary tables with the number and percentage of device deficiencies will be provided by type (**Appendix B**). A by-subject listing of all device malfunctions will be provided (**Appendix C**).

#### 10 STATISTICAL CONSIDERATIONS RELATED TO COVID-19

The statistical considerations detailed in this section are consistent with the FDA's guidance on the conduct of clinical trials during the COVID-19 pandemic (Guidance for Industry on Statistical Considerations for Clinical Trials During the COVID-19 Public Health Emergency; Issued June 2020) and recommendations for the statistical analysis of the primary and key secondary endpoints to help ensure that the COVID-19-related changes to the RESET-RA study conduct will provide interpretable findings with correct statistical quantification of uncertainty.

### 10.1 Impact of COVID-19 on Study Integrity

Unavoidable protocol modifications may be required due to COVID-19 illness and/or COVID-19 control measures to protect subject safety and the to address its impact on the ability to collect data. The context and/or reasons for post-baseline events as they relate to COVID-19, such as discontinuation of treatment, withdrawal from the trial, use of alternative or rescue treatments, missed endpoint assessments, and the use of alternative endpoint assessment methods will be


## Statistical Analysis Plan for Interim and Primary Analyses in SPM-020 (The RESET-RA Study) Doc# CLP-004 Rev D, 15JUL2024



captured at the subject level. Information not specific to individual subjects, such as information on site closure (rheumatology or surgery) and its impact on disrupting administration of the investigational study device (i.e., implant procedure, device titration, device adjustments) will also be captured. This information at both the subject and site levels may be useful for incorporating into additional sensitivity analyses related to the impact of COVID-19.

# 10.2 COVID-19 Analysis Considerations

The impact of COVID-19 on the study integrity will be assessed and included into summaries of pooled data from Stage 1 and 2 over treatment groups, including information on missing data, protocol deviations, subject discontinuation or interruption of the investigational treatment, subject withdrawal, and changes in endpoint assessments (e.g., virtual visit).

To address adequately the impact of COVID-19 on evaluating the primary and key secondary endpoints, the following analysis strategies may be considered:

- If the study is stopped earlier than planned because of COVID-19, a smaller sample size or less follow-up time may result in loss of statistical power than was anticipated for the final analysis. A blinded power assessment will be conducted to estimate the power of the modified study. The assessment will use the actual event rates pooled over treatment group or the observed variability pooled over treatment group in the completed portion of the trial.
- Stopping the study earlier because of COVID-19 may impact the statistical inference (e.g., p-values, confidence intervals). Any modification to the study, including the original planned analyses, should not be based on data that reveal information on the treatment effect.
- If the study is stopped earlier because of COVID-19, the planned interim analysis may be
  appropriate for the statistical interference. Modifications can be considered to maintain control
  over Type 1 error. The actual results may be less statistically significant or have a wider
  confidence interval than the trial was designed for because of reduced information (e.g., fewer
  endpoint events).
- Extending the protocol-defined windows and using alternative remote methods for assessment
  of the primary and secondary efficacy endpoints may be warranted to address the impact of
  COVID-19. The data from these late or modified assessments can be leveraged based on
  scientifically based rationale and clinical judgement.
- Any differences in the assessment methods between treatment groups or among subjects with different baseline characteristics may be explored though sensitivity analyses stratified by the method and timing of the endpoint assessment. Additional sensitivity analyses will examine differences in baseline characteristics and post-baseline events (including endpoints and AEs) between the originally enrolled subjects and those with missing endpoint assessments or interrupted investigational treatment because of COVID-19.
- The available data at baseline and post-baseline, including COVID-19-related information will
  be leveraged using the prespecified methods for handling missing data in Section 5.8. The
  analysis will take into consideration the actual event rates pooled over treatment groups or the
  observed variability pooled over treatment groups in the completed portion of the study.

Statistical Analysis Plan for Interim and Primary Analyses in SPM-020 (The RESET-RA Study) Doc# CLP-004 Rev D, 15JUL2024



#### 11 REFERENCES

Bang H, Flaherty S, Kolahi J, Park J. Blinding assessment in clinical trials: A review of statistical methods and a proposal of blinding assessment protocol. Clin Res Reg Affairs. 2010;27:42-51.

Berglund P, Heeringa SG. Multiple imputation of missing data using SAS. SAS Institute Inc. Cary NC. 2014.

Bruynesteyn K, Boers M, Kostense P, van der Linden S, van der Heijde D. Deciding on progression of joint damage in paired films of individual patients: smallest detectable difference or change. Ann Rheum Dis. 2005;64:179-182.

EuroQol Research Foundation. EQ-5D-5L. Online Available: https://euroqol.org/eq-5d-instruments/eq-5d-5l-about/. 2023.

FDA Guidance for Industry on Statistical Considerations for Clinical Trials During the COVID-19 Public Health Emergency. June 2020.

FDA Guidance for Industry, Investigators, and Institutional Review Boards on Conduct of Clinical Trials of Medical Products During COVID-19 Public Health Emergency. 2020; updated September 21, 2020.

Gandjbakhch F, et al. Determining a magnetic resonance imaging inflammatory activity acceptable state without subsequent radiographic progression in rheumatoid arthritis: results from a followup MRI study of 254 patients in clinical remission or low disease activity. J Rheumatol. 2014 Feb;41(2):398-406.Hochberg Y. A sharper Bonferroni procedure for multiple tests of significance. Biometrika. 1988;75:800-2.

Maruish M. (Ed.). User's manual for the SF-36v2 Health Survey (3rd ed.). Lincoln, RI: QualityMetric Incorporated. 2011.




#### 12 APPENDICES

#### Appendix A: Schedule of Assessments

| Assessment | Informed Consent & Screening (Baseline) | Enrollment & Implant Procedure (≤ 30d post-Informed Consent) | Post-Surgical Clearance (14-21d post- Implant Procedure) | Day 0 (Randomization & Initiation of Stimulation) (14-21d post- | Titration 1 $(7 \pm 2d2)$ | Titration 2<br>(14 ± 2d2) | Titration 3 $(21 \pm 2d2)$ | Week 4<br>(28 ± 3d2) | Week 8<br>(56 ± 5d2) | Week 12<br>(Primary<br>Endpoint & One-<br>way Crossover)<br>(84 ± 7d2) |
|---|---|---|---|---|---|---|---|---|---|---|
| Informed consent | X* | | | ** | | | | | | ** |
| Vital signs | X* | | | X | | | | | | X |
| Physical exam and medical history | X* | | | | | | | | | |
| Pregnancy test (childbearing female) | X* | X | X | X | X | X | X | X | X | X |
| RA disease activity assessments <sup>1</sup> | X* | | | X | | | | X | X | X |
| RA prior and current medication | X* | | | | | | | | | |
| Energizer fit test | X* | | | | | | | | | |
| SF-36 & EQ-5D-5L questionnaires | X | | | X | | | | X | X | X |
| Blood collection (RF, ACPA, eGFR) | X | | | | | | | | | |
| Blood collection (CBC, biomarkers) | X | | | X | | | | X | X | X |
| Hand MRI | X | | | | | | | | | X |
| 12-lead ECG | X | | | | | | | | | X |
| X-ray cervical spine | X | | | | | | | | | |
| Surgical clearance | X | | X | | | | | | | |
| Implant procedure in operating room | | X | | | | | | | | |
| Randomization | | | | X | | | | | | |
| Subject training on the use of Energizer | | | | X | | | | | | |
| Device check & dose titration | | | | X | X | X | X | | | $X^3$ |
| Device check & dose adjustment if needed | | | | | | | | X | X | |
| Blinding assessment 4 | | | | | | | | X | | X |
| Treatment decision for long-term follow-up | | | | | | | | | | X |
| Device deficiency reporting | | X | X | X | X | X | X | X | X | X |
| Adverse event reporting | X | X | X | X | X | X | X | X | X | X |
| Concomitant medication | X | X | X | X | X | X | X | X | X | X |

Abbreviations: ACPA, anti-citrullinated protein antibodies; CBC, complete blood count; d, day; EGA, evaluator's global assessment; eGFR: estimated glomerular filtration rate; HAQ-DI, Health Assessment Questionnaire Disability Index; hsCRP, high-sensitivity C-reactive protein; MRI, magnetic resonance imaging; RA, rheumatoid arthritis; RF, rheumatoid factor; SGA, subject's global assessment; SJC, swollen joint count; TJC, tender joint count


<sup>\*</sup> Screening assessments that must be conducted on the day of informed consent to determine subject's initial eligibility and baseline values for the primary and key secondary efficacy endpoints.



#### Doc# CLP-004 Rev D, 15JUL2024

- RA disease activity assessments include: HAQ-DI, SGA, subject's pain assessment, TJC28, SJC28, EGA, and hsCRP. Subjects must have ≥ 4TJC28 and ≥ 4SJC28 at consent to be eligible.
- <sup>2</sup> From Day 0 (randomization).
- 3 Dose titration is not performed if subject and Co-PI Rheumatologist decide that subject should not receive active stimulation in open-label, long-term follow-up period.
- 4 Blinding assessments are completed by the subject, Joint Evaluator and Co-PI Rheumatologist.


#### Statistical Analysis Plan for Interim and Primary Analyses in SPM-020 (The RESET-RA Study) Doc# CLP-004 Rev D, 15JUL2024



### Appendix B: Table Mockups

| Table 14.1.1.1 | Subject Disposition (All Subjects) | 42 |
|---|---|---|
| Table 14.1.1.2 | Demographic and Baseline Characteristics (ITT Population) | 43 |
| Table 14.1.2.1 | ACR20 Response (ITT Population) | 47 |
| Table 14.1.2.1.0 | ACR20 Response (PTE Population) | 48 |
| Table 14.1.2.1.1 | Sensitivity Analysis of ACR20 Response: Rescue Treatment (ITT Population) | 49 |
| Table 14.1.2.1.2 | Sensitivity Analysis of ACR20 Response: Missing Data (ITT Population) | 50 |
| Table 14.1.2.1.3 | Sensitivity Analysis of ACR20 Response: Impact of COVID-19 (ITT Population) | 51 |
| Table 14.1.2.1.3.1 | Descriptive Analysis of Diagnosis of COVID-19 (ITT Population) | 52 |
| Table 14.1.2.1.4 | Subgroup Analysis of ACR20 Response: Age (ITT Population) | 53 |
| Table 14.1.2.1.5 St | abgroup Analysis of ACR20 Response: Gender (ITT Population) | 54 |
| Table 14.1.2.1.6 | Subgroup Analysis of ACR20 Response: Race (ITT Population) | 54 |
| Table 14.1.2.1.7 | Subgroup Analysis of ACR20 Response: RA Duration (ITT Population) | 54 |
| Table 14.1.2.1.8 | Subgroup Analysis of ACR20 Response: Prior b/tsDMARDs (ITT Population) | 54 |
| Table 14.1.2.1.9 | Subgroup Analysis of ACR20 Response: Prior JAKi (ITT Population) | 54 |
| Table 14.1.2.1.10 | Subgroup Analysis of ACR20 Response: RA Disease Activity at Screening (ITT Population) | |
| Table 14.1.2.1.11 | Subgroup Analysis of ACR20 Response: Moderate-to-severe RA at Day 0 (ITT Population) | |
| Table 14.1.2.2 | Key Secondary Endpoints Adjusted for Multiplicity (ITT Population) | 57 |
| Table 14.1.2.2.1 | Key Secondary Endpoints (PTE Population) | 58 |
| Table 14.1.2.2.2 | Sensitivity Analysis of Key Secondary Endpoints: Timing of Baseline (ITT Population) | |
| Table 14.1.2.2.3 | Sensitivity Analysis of Key Secondary Endpoints: Rescue Treatments (ITT Population) | |
| Table 14.1.2.2.4 | Sensitivity Analysis of Key Secondary Endpoints: Missing Values (ITT Population) | 63 |
| Table 14.1.2.2.5 | Subgroup Analysis of Key Secondary Endpoints: Prior b/tsDMARDs (ITT Population) | |
| Table 14.1.2.2.6 | Subgroup Analysis of Key Secondary Endpoints: Prior JAKi (ITT Population) | 66 |
| Table 14.1.2.2.7 | Subgroup Analysis of Key Secondary Endpoints: RA Disease Activity at Screening (ITT Population) | 66 |
| Table 14.1.2.2.8 | Subgroup Analysis of Key Secondary Endpoints: Moderate-to-severe RA a<br>Day 0 (ITT Population) | 66 |
| Table 14.1.2.3 | ACR50/70 (ITT Population) | 67 |
| Table 14.1.2.4 | TJC28 (ITT Population) | |
| Table 14.1.2.5 | SJC28 (ITT Population) | 71 |




#### Doc# CLP-004 Rev D, 15JUL2024

| Table 14.1.2.6 | Subject's Assessment of Pain (ITT Population) | 74 |
|---|---|---|
| Table 14.1.2.7 | SGA (ITT Population) | 77 |
| Table 14.1.2.8 | EGA (ITT Population) | 80 |
| Table 14.1.2.9 | hsCRP (ITT Population) | 83 |
| Table 14.1.2.10 | HAQ-DI (ITT Population) | 86 |
| Table 14.1.2.11 | DAS28-CRP (ITT Population) | 91 |
| Table 14.1.2.12 | CDAI (ITT Population) | 95 |
| Table 14.1.2.13 | RAMRIS (ITT Population) | 99 |
| Table 14.1.2.14 | EQ-5D-5L (ITT Population) | 102 |
| Table 14.1.2.15 | SF-36 (ITT Population) | 107 |
| Table 14.1.2.16 | Subject's Blinding Assessment (ITT Population) | 110 |
| Table 14.1.2.16.1 | Subject's Blinding Assessment (PTE Population) | 110 |
| Table 14.1.2.17 | Joint Evaluator's Blinding Assessment (ITT Population) | 111 |
| Table 14.1.2.17.1 | Evaluator's Blinding Assessment (PTE Population) | 111 |
| Table 14.1.2.18 | Co-PI Rheumatologist's Blinding Assessment (ITT Population) | 112 |
| Table 14.1.2.18.1 | Co-PI Rheumatologist's Blinding Assessment (PTE Population) | 112 |
| Table 14.1.2.19 | Inflammatory Biomarkers (ITT Population) | 113 |
| Table 14.1.2.20 | RA Rescue Treatments and Follow-up Interventions (ITT Population) | 115 |
| Table 14.1.2.22 | Implant Performance (ITT Population) | 117 |
| Table 14.1.3.1 | Adverse Events (Safety Population) | 118 |
| Table 14.1.3.2 | Adverse Events by SOC and Maximum Severity: All Events Safety Population | 120 |
| Table 14.1.3.3 | Implant Procedure-Related Adverse Events by SOC and Maximum Severity: All Events (Safety Population) | |
| Table 14.1.3.4 | Implant Device-Related Adverse Events by SOC and Maximum Severi<br>All Events (Safety Population) | - |
| Table 14.1.3.5 | Stimulation-Related Adverse Events by SOC and Maximum Severity: A Events (Safety Population) | |
| Table 14.1.3.6 | Explant Procedure-Related Adverse Events by SOC and Maximum Severity: All Events (Safety Population) | 126 |
| Table 14.1.3.7 | Energizer-Related Adverse Events by SOC and Maximum Severity: All Events (Safety Population) | |
| Table 14.1.3.8 | Device Deficiency (Safety Population) | 127 |
| Table 14 1 3 9 | Protocol Deviations (ITT Population) | 128 |




Table 14.1.1.1 Subject Disposition (All Subjects)

| | Treatment | Control | All |
|---|---|---|---|
| Number of subjects: | | | |
| Consented | _ | _ | xxx |
| Screen failure | _ | _ | xxx |
| Enrolled | XXX | xxx | xxx |
| Implanted | xxx | xxx | xxx |
| Randomized | xxx | xxx | xxx |
| ITT population [1] | xxx | xxx | xxx |
| PTE population [2] | xxx | XXX | xxx |
| Safety population [3] | xxx | XXX | XXX |
| Withdrawn | XXX | XXX | XXX |
| Completed study through Week 12 | xxx | XXX | XXX |
| Primary reason for withdrawal [4]: | | | |
| Subject decision to withdraw consent | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| Investigator decision or medical judgement | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| Lost to follow-up | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| Device malfunction | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| Adverse event | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| Subject no longer eligible | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| Death | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| Study terminated | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| Sponsor or IRB decision | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| Other | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |

Abbreviations: ITT, intent to treat; PTE, per-treatment-evaluable.

Reference: Listing 16.x.x.x

SOURCE: xxxxx SAS 9.4 {program location} {run date/time}


<sup>[1]</sup> ITT population comprises all enrolled and randomized subjects in Stage 1 and 2.

<sup>[2]</sup> PTE population comprises subjects from the ITT population who have received the assigned treatment, have no major procedural protocol deviations, and for whom follow-up data are available.

<sup>[3]</sup> Safety population comprises all enrolled subjects in Stage 1 and 2.

<sup>[4]</sup> Percentage calculated based on ITT population.



Table 14.1.1.2 Demographic and Baseline Characteristics (ITT Population)

| | (11 1 Topulation) | | |
|---|---|---|---|
| | Treatment | Control | All |
| | (N=xxx) | (N=xxx) | (N=xxx) |
| N | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| Age (years) | | | |
| N | XXX | xxx | xxx |
| Mean (SD) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) |
| Median | xx.xx | xx.xx | xx.xx |
| Min-Max | xx.x - xx.x | xx.x - xx.x | xx.x - xx.x |
| Gender [1] | | | |
| Male | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| Female | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| Ethnicity [1] | | | |
| Hispanic or Latino | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| Not Hispanic or Latino | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| Not disclosed | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| Race [1][2] | | | |
| American Indian or Alaska Native | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| Asian | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| Black or African American | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| Native Hawaiian or other Pacific Islander | xxx (xx.x%) | xxx (xx.x%) | xxx (xx,x%) |
| White | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| Other | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| RA duration (years) | | | |
| N | xxx | xxx | XXX |
| Mean (SD) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) |
| Median | xx.xx | xx.xx | XX,XX |
| Min-Max | xx.x - xx.x | xx.x - xx.x | xx.x - xx.x |
| BMI (kg/m²) | | | |
| N | XX | xx | XX |
| Mean (SD) | xxx.x (xxx.xx) | xxx.x (xxx.xx) | xxx.x (xxx.xx) |


## SETPOINT MEDICAL

#### Doc# CLP-004 Rev D, 15JUL2024

| | Treatment | Control | All |
|---|---|---|---|
| | (N=xxx) | (N=xxx) | (N=xxx) |
| Median | xxx.xx | xxx.xx | XXX,XX |
| Min-Max | xxx.x-xxx.x | xxx.x - xxx.x | xxx.x - xxx.x |
| RF [1] | | | |
| Positive | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| ACPA [1] | | | |
| Positive | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Positive serology (RF and/or ACPA positive) [1] | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| hsCRP (mg/L) | | | |
| N | xx | xx | XX |
| Mean (SD) | xxx.x (xxx.xx) | xxx.x (xxx.xx) | xxx.x (xxx.xx) |
| Median | xxx.xx | xxx.xx | xxx.xx |
| Min-Max | xxx.x - xxx.x | xxx.x - xxx.x | xxx.x - xxx.x |
| TJC28 | | | |
| N | xx | XX | XX |
| Mean (SD) | xxx.x (xxx.xx) | xxx.x (xxx.xx) | xxx.x (xxx.xx) |
| Median | xxx,xx | xxx.xx | xxx.xx |
| Min-Max | xxx.x - xxx.x | xxx.x - xxx.x | xxx.x - xxx.x |
| SJC28 | | | |
| N | xx | XX | XX |
| Mean (SD) | xxx.x (xxx.xx) | xxx.x (xxx.xx) | xxx.x (xxx.xx) |
| Median | xxx.xx | xxx.xx | xxx.xx |
| Min-Max | xxx.x - xxx.x | xxx.x - xxx.x | xxx.x - xxx.x |
| CDAI score | | | |
| N | xx | XX | XX |
| Mean (SD) | xxx.x (xxx.xx) | xxx.x (xxx.xx) | xxx.x (xxx.xx) |
| Weatt (SD) | | xxx.xx | xxx.xx |
| Median | XXX,XX | AAA, AA | AAA.AA |


Doc# CLP-004 Rev D, 15JUL2024

| | Treatment | Control | All |
|----------------|----------------|----------------|----------------|
| | (N=xxx) | (N=xxx) | (N=xxx) |
| N | XX | xx | XX |
| Mean (SD) | xxx.x (xxx.xx) | xxx.x (xxx.xx) | xxx.x (xxx.xx) |
| Median | xxx.xx | xxx.xx | XXX,XX |
| Min-Max | xxx.x - xxx.x | xxx.x - xxx.x | xxx.x - xxx.x |
| HAQ-DI score | | | |
| N | XX | XX | XX |
| Mean (SD) | xxx.x (xxx.xx) | xxx.x (xxx.xx) | xxx.x (xxx.xx) |
| Median | xxx.xx | xxx.xx | XXX.XX |
| Min-Max | xxx.x - xxx.x | xxx.x - xxx.x | xxx.x - xxx.x |
| EQ-5D-5L Index | | | |
| N | XX | XX | XX |
| Mean (SD) | xxx.x (xxx.xx) | xxx.x (xxx.xx) | xxx.x (xxx.xx) |
| Median | xxx.xx | xxx.xx | XXX,XX |
| Min-Max | xxx.x - xxx.x | xxx.x - xxx.x | xxx.x - xxx.x |
| EQ-VAS | | | |
| N | XX | xx | XX |
| Mean (SD) | xxx.x (xxx.xx) | xxx.x (xxx.xx) | xxx.x (xxx.xx |
| Median | XXX,XX | xxx.xx | XXX.XX |
| Min-Max | xxx.x - xxx.x | xxx.x - xxx.x | xxx.x - xxx.x |
| SF-36 MCS | | | |
| N | XX | XX | XX |
| Mean (SD) | xxx.x (xxx.xx) | xxx.x (xxx.xx) | xxx.x (xxx.xx) |
| Median | xxx.xx | xxx.xx | xxx,xx |
| Min-Max | xxx.x - xxx.x | xxx.x - xxx.x | xxx.x - xxx.x |
| SF-36 PCS | | | |
| N | XX | xx | XX |
| Mean (SD) | xxx.x (xxx.xx) | xxx.x (xxx.xx) | xxx.x (xxx.xx) |
| Median | xxx.xx | xxx.xx | xxx.xx |
| Min-Max | xxx.x - xxx.x | xxx.x - xxx.x | xxx.x - xxx.x |

SETPOINT MEDICAL


May not be reproduced outside of SetPoint Medical without written permission from Document Control.

Number of prior b/ts DMARDs



#### Doc# CLP-004 Rev D, 15JUL2024

| | Treatment | Control | All |
|---|---|---|---|
| | (N=xxx) | (N=xxx) | (N=xxx) |
| N | xx | xx | xx |
| Mean (SD) | xxx.x (xxx.xx) | xxx.x (xxx.xx) | xxx.x (xxx.xx) |
| Median | xxx.xx | xxx.xx | xxx.xx |
| Min-Max | xxx.x - xxx.x | xxx.x - xxx.x | xxx.x - xxx.x |
| Number of prior b/ts DMARDs [1] | | | |
| 1 | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| 2 | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| 3 | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| 4 | | | |
| 5 | | | |
| 6 | | | |
| 7 | | | |
| 8 | | | |
| 9 | | | |
| 10+ | | | |
| Prior b/ts DMARDs [1] | | | |
| Anti-IL-1 agents | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Anti IL-6 agents | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Anti-TNF agents | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| B-cell depleting agents | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| JAKi | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| CTLA4-Ig | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |

Abbreviations: ACPA, anti-citrullinated protein antibodies; b/tsDMARD, biologic or targeted synthetic disease-modifying antirheumatic drug; CDAI, Clinical Disease Activity Index; CTLA4-Ig, cytotoxic T-lymphocyte-associated antigen-4 immunoglobulin; DAS, Disease Activity Score; HAQ-DI, Health Assessment Questionnaire Disability Index; hsCRP, high-sensitivity C-reactive protein; IL, interleukin; ITT, intent to treat; JAKi, Janus kinase inhibitor; RF, rheumatoid factor; SD, standard deviation; SJC, swollen joint count; TJC, tender joint count; TNF, tumor necrosis factor.

[1] Percentage calculated based on ITT population.

[2] Race selected based on all that applied.

Reference: Listing 16.x.x.x

SOURCE: xxxxx SAS 9.4 {program location} {run date/time}}


Doc# CLP-004 Rev D, 15JUL2024



Table 14.1.2.1 ACR20 Response (ITT Population)

| Variable | Treatment | Control |
|---|---|---|
| variable | (N=xxx) | (N=xxx) |
| ACR20 Response from baseline on the day of informed consent | | |
| Week 12 | | |
| N[1] | XX | XX |
| Yes | xx (xx.x%) | xx (xx.x%) |
| Difference [2] | XX.X% | |
| 95% CI for difference [2] | (xx.x, xx.x) | |
| p-value for difference [2] | 0.xxx | |
| ACR20 Response from Day 0* | | |
| Week 12 | | |
| N[1] | XX | XX |
| Yes | xx (xx.x%) | xx (xx.x%) |
| Difference [2] | XX.X% | |
| 95% CI for difference [2] | (xx.x, xx.x) | |
| p-value for difference [2] | 0.xxx | |

Abbreviations: ACR, American College of Rheumatology; CI, confidence interval; ITT, intent to treat.

Reference: Listing 16.x.x.x

SOURCE: xxxxx SAS 9.4 {program location} {run date/time}}


Percentage calculated based on ITT population.

<sup>[2]</sup> Difference in proportions and one-sided p-value based on the Cochran-Mantel-Haenszel test stratified by inadequate response or loss of response to JAKi and RA disease severity at Day 0 for Stage 1 subjects and RA disease severity at Day 0 and inadequate response or loss of response to ≥ 4 biological DMARDs with ≥ 2 mechanisms of action for Stage 2 subjects.

<sup>\*</sup>Day 0 post-Implant Procedure and before randomization and initiation of assigned treatment

Doc# CLP-004 Rev D, 15JUL2024



Table 14.1.2.1.0 ACR20 Response (PTE Population)

| Variable | Treatment | Control |
|---|---|---|
| variable | (N=xxx) | (N=xxx) |
| ACR20 Response from baseline on the day of informed consent | | |
| Week 12 | | |
| N[1] | XX | XX |
| Yes | xx (xx.x%) | xx (xx.x%) |
| Difference [2] | xx.x% | |
| 95% CI for difference [2] | (xx.x, xx.x) | |
| p-value for difference [2] | 0.xxx | |
| ACR20 Response from Day 0* | | |
| Week 12 | | |
| N[1] | XX | XX |
| Yes | xx (xx.x%) | xx (xx.x%) |
| Difference [2] | xx.x% | |
| 95% CI for difference [2] | (xx.x, xx.x) | |
| p-value for difference [2] | 0.xxx | |

Abbreviations: ACR, American College of Rheumatology; CI, confidence interval; ITT, intent to treat.

Reference: Listing 16.x.x.x

SOURCE: xxxxx SAS 9.4 {program location} {run date/time}}


Percentage calculated based on ITT population.

<sup>[2]</sup> Difference in proportions and one-sided p-value based on the Cochran-Mantel-Haenszel test stratified by inadequate response or loss of response to JAKi and RA disease severity at Day 0 for Stage 1 subjects and RA disease severity at Day 0 and inadequate response or loss of response to ≥ 4 biological DMARDs with ≥ 2 mechanisms of action for Stage 2 subjects.

<sup>\*</sup>Day 0 post-Implant Procedure and before randomization and initiation of assigned treatment



#### Table 14.1.2.1.1 Sensitivity Analysis of ACR20 Response: Rescue Treatment (ITT Population)

| Variable | Treatment | Control |
|---|---|---|
| уапавіе | (N=xxx) | (N=xxx) |
| ACR20 Response from baseline on the day of informed consent | | |
| Week 12 | | |
| N[1] | XX | XX |
| Yes | xx (xx.x%) | xx (xx.x%) |
| Difference [2] | xx.x% | |
| 95% CI for difference [2] | (xx.x, xx.x) | |
| p-value for difference [2] | 0.xxx | |
| ACR20 Response from Day 0 | | |
| Week 12 | | |
| N[1] | XX | XX |
| Yes | xx (xx.x%) | xx (xx.x%) |
| Difference [2] | xx.x% | |
| 95% CI for difference [2] | (xx.x, xx.x) | |
| p-value for difference [2] | 0.xxx | |

Abbreviations: ACR, American College of Rheumatology; ITT, intent to treat.

Reference: Listing 16.x.x.x

SOURCE: xxxxx SAS 9.4 {program location} {run date/time}}


Percentage calculated based on ITT Population.

<sup>[2]</sup> Difference in proportions and one-sided p-value based on the Cochran-Mantel-Haenszel test stratified by inadequate response or loss of response to JAKi and RA disease severity at Day 0 for Stage 1 subjects and RA disease severity at Day 0 and inadequate response or loss of response to ≥ 4 biological DMARDs with ≥ 2 mechanisms of action for Stage 2 subjects.

<sup>\*</sup>Day 0 post-Implant Procedure and before randomization and initiation of assigned treatment



#### Table 14.1.2.1.2 Sensitivity Analysis of ACR20 Response: Missing Data (ITT Population)

| Tipping Point Results | Treatment<br>(N=xxx) | Control<br>(N=xxx) | p-value |
|-----------------------|----------------------|--------------------|---------|
| ACR20 Non-responder | XX | xx | 0.xxx |
| ACR20 Responder | xx | xx | |

Abbreviations: ACR, American College of Rheumatology; ITT, intent to treat.

[1] Percentage calculated based on ITT population.

SOURCE: xxxxx SAS 9.4 {program location} {run date/time}}

Note to biostats: If more than 5% of primary efficacy data are missing, the table above is to be presented in addition to the multiple imputation approach of Berglund and Heeringa (2014) described in SAP Section 8.3.4.




#### Table 14.1.2.1.3 Sensitivity Analysis of ACR20 Response: Impact of COVID-19 (ITT Population)

| /ariable | Treatment | Control |
|---|---|---|
| | (N=xxx) | (N=xxx) |
| CR20 Response from baseline on the day of informed consent | | |
| No Covid-19 Diagnosis prior to Week 12 | | |
| N[1] | XX | XX |
| Yes | xx (xx.x%) | xx (xx.x%) |
| Difference [2] | xx.x% | |
| 95% CI for difference [2] | (xx.x, xx.x) | |
| p-value for difference [2] | 0.xxx | |
| Covid-19 Diagnosis prior to Week 12 | | |
| N[1] | XX | XX |
| Yes | xx (xx.x%) | xx (xx.x%) |
| Difference [2] | xx.x% | |
| 95% CI for difference [2] | (xx.x, xx.x) | |
| p-value for difference [2] | 0.xxx | |
| nteraction p-value [3] | 0.xxx | |

Abbreviations: ACR, American College of Rheumatology; ITT, intent to treat.

[3] Based on the Breslow Day test for homogeneity across subgroups.

SOURCE: xxxxx SAS 9.4 {program location} {run date/time}}


<sup>[1]</sup> Percentage calculated based on ITT Population.

<sup>[2]</sup> Difference in proportions and one-sided p-value based on the Cochran-Mantel-Haenszel test stratified by inadequate response or loss of response to JAKi and RA disease severity at Day 0 for Stage 1 subjects, and RA disease severity at Day 0 and inadequate response or loss of response to ≥ 4 biological DMARDs with ≥ 2 mechanisms of action for Stage 2 subjects.



Table 14.1.2.1.3.1 Descriptive Analysis of Diagnosis of COVID-19 (ITT Population)

| | All |
|--------------------------------------------------------|------------|
| | (N=xxx) |
| Diagnosed with Covid-19 post-procedure | |
| N[1] | xx |
| Yes | xx (xx.x%) |
| Received medication/treatment for Covid-19 | |
| N[1] | xx |
| Yes | xx (xx.x%) |
| Protocol Deviations associated with Covid-19 Diagnosis | |
| N[1] | xx |
| Yes | xx (xx.x%) |
| Adverse Events associated with Covid-19 Diagnosis | |
| N[1] | xx |
| Yes | xx (xx.x%) |

Abbreviations: ITT, intent to treat.

[1] Percentage calculated based on ITT population.

Reference: Listing 16.x.x.x

SOURCE: xxxxx SAS 9.4 {program location} {run date/time}}




#### Table 14.1.2.1.4 Subgroup Analysis of ACR20 Response: Age (ITT Population)

| Variable | Treatment (N=xxx) | Control<br>(N=xxx) |
|---|---|---|
| ACR20 Response from baseline on the day of informed consent | Ç. 1889 | ( |
| Age < 65 | | |
| Week 12 | | |
| N[1] | XX | XX |
| Yes | xx (xx.x%) | xx (xx.x%) |
| Difference [2] | xx.x% | |
| 95% CI for difference [2] | (xx.x, xx.x) | |
| p-value for difference [2] | 0.xxx | |
| $Age \ge 65$ | | |
| Week 12 | | |
| N[1] | XX | XX |
| Yes | xx (xx.x%) | xx (xx.x%) |
| Difference [2] | xx.x% | |
| 95% CI for difference [2] | (xx.x, xx.x) | |
| p-value for difference [2] | 0.xxx | |
| Interaction p-value [3] | 0.xxx | |

Abbreviations: ACR, American College of Rheumatology; ITT, intent to treat.

- [1] Percentage calculated based on ITT Population.
- [2] Difference in proportions and one-sided p-value based on the Cochran-Mantel-Haenszel test stratified by inadequate response or loss of response to JAKi and RA disease severity at Day 0 for Stage 1 subjects and RA disease severity at Day 0 and inadequate response or loss of response to ≥ 4 biological DMARDs with ≥ 2 mechanisms of action for Stage 2 subjects.
- [3] Based on the Breslow Day test for homogeneity across subgroups.

Reference: Listing 16.x.x.x

SOURCE: xxxxx SAS 9.4 {program location} {run date/time}}


Statistical Analysis Plan for Interim and Primary Analyses in SPM-020 (The RESET-RA Study) Doc# CLP-004 Rev D, 15JUL2024



Table 14.1.2.1.5 Subgroup Analysis of ACR20 Response: Gender (ITT Population)

Repeat Table 14.1.2.1.5 for Gender [Male vs. Female]

Table 14.1.2.1.6 Subgroup Analysis of ACR20 Response: Race (ITT Population)

Repeat Table 14.1.2.1.5 for Race [White vs. Non-White including Black or African American, American Indian or Alaska Native, Asian, Native Hawaiian or other Pacific Islander]

Table 14.1.2.1.7 Subgroup Analysis of ACR20 Response: RA Duration (ITT Population)

Repeat Table 14.1.2.1.5 for RA Duration [< 5 years vs.  $\ge 5$  to < 10 years vs.  $\ge 10$  years]

Table 14.1.2.1.8 Subgroup Analysis of ACR20 Response: Prior b/tsDMARDs (ITT Population)

Repeat Table 14.1.2.1.5 for Number of Prior b/tsDMARD [<4 vs. ≥ 4]

Add to abbreviations: DMARD, disease-modifying antirheumatic drug;

Table 14.1.2.1.9 Subgroup Analysis of ACR20 Response: Prior JAKi (ITT Population)

Repeat Table 14.1.2.1.5 for Prior JAKi [Yes vs. No]

Add to abbreviations: JAKi, Janus kinase inhibitor.


Statistical Analysis Plan for Interim and Primary Analyses in SPM-020 (The RESET-RA Study) Doc# CLP-004 Rev D, 15JUL2024



Table 14.1.2.1.10
Subgroup Analysis of ACR20 Response: RA Disease Activity at Screening (ITT Population)

Repeat Table 14.1.2.1.5 for RA Disease Activity at Screening [DAS28-CRP ≤ 5.1 vs DAS28-CRP > 5.1]

Add to abbreviations: DAS, Disease Activity Score.




#### Table 14.1.2.1.11 Subgroup Analysis of ACR20 Response: Moderate-to-severe RA at Day 0 (ITT Population)

| Variable | Treatment | Control |
|--------------------------------|--------------|------------|
| | (N=xxx) | (N=xxx) |
| Moderate-to-severe RA at Day 0 | | |
| < 4 TJC28 or < 4 SJC28 | | |
| Week 12 | | |
| N[1] | XX | XX |
| Yes | xx (xx.x%) | xx (xx.x%) |
| Difference [2] | xx.x% | |
| 95% CI for difference [2] | (xx.x, xx.x) | |
| p-value for difference [2] | 0.xxx | |
| ≥ 4 TJC28 and ≥ 4 SJC28 | | |
| Week 12 | | |
| N[1] | xx | XX |
| Yes | xx (xx.x%) | xx (xx.x%) |
| Difference [2] | xx.x% | |
| 95% CI for difference [2] | (xx.x, xx.x) | |
| p-value for difference [2] | 0.xxx | |
| Interaction p-value [3] | 0.xxx | |

Abbreviations: ACR, American College of Rheumatology; ITT, intent to treat.

- [1] Percentage calculated based on ITT Population.
- [2] Difference in proportions and one-sided p-value based on the Cochran-Mantel-Haenszel test stratified by inadequate response or loss of response to JAKi and RA disease severity at Day 0 for Stage 1 subjects and RA disease severity at Day 0 and inadequate response or loss of response to ≥ 4 biological DMARDs with ≥ 2 mechanisms of action for Stage 2 subjects.
- [3] Based on the Breslow Day test for homogeneity across subgroups.

Reference: Listing 16.x.x.x

SOURCE: xxxxx SAS 9.4 {program location} {run date/time}}




Table 14.1.2.2 Key Secondary Endpoints Adjusted for Multiplicity (ITT Population)

| Endpoint | Unadjusted p-value | Adjusted p-value [1] |
|---|---|---|
| ACR20 response at Week 12 from baseline at Day 0 | x.xxxx | x.xxxx |
| DAS28-CRP moderate/good EULAR response at Week 12 from baseline on the day of informed consent | x.xxxx | x.xxxx |
| DAS28-CRP response (MCID $\geq$ -1.2) at Week 12 from baseline on the day of informed consent | x.xxxx | x.xxxx |
| HAQ-DI response (MCID $\geq$ -0.22) at Week 12 from baseline on the day of informed consent | x.xxxx | x.xxxx |

Abbreviations: CRP, C-reactive protein; DAS, Disease Activity Score; EULAR, European League Against Rheumatism; HAQ-DI, Health Assessment Questionnaire Disability Index; ITT, intent to treat; MCID, minimal clinically important difference.

[1] Adjusted for multiplicity using Hochberg's Step-Up Method

Reference: Listing 16.x.x.x

SOURCE: xxxxx SAS 9.4 {program location} {run date/time}}




#### Table 14.1.2.2.1 Key Secondary Endpoints (PTE Population)

| Variable | Treatment (N=xxx) | Control<br>(N=xxx) |
|---|---|---|
| DAS28-CRP moderate/good EULAR response at Week 12 from Day 0 | (11 AAA) | (11 AAA) |
| Week 12 | | |
| N[1] | XX | xx |
| Yes | xx (xx.x%) | xx (xx.x%) |
| Difference [2] | xx.x% | |
| 95% CI for difference [2] | (xx.x%, xx.x%) | |
| p-value for difference [2] | 0.xxx | |
| DAS28-CRP response (MCID ≥ -1.2) at Week 12 | | |
| Week 12 | | |
| N[1] | XX | XX |
| Yes | xx (xx.x%) | xx (xx.x%) |
| Difference [2] | xx.x% | |
| 95% CI for difference [2] | (xx.x%, xx.x%) | |
| p-value for difference [2] | 0.xxx | |
| HAQ-DI response (MCID $\geq$ -0.22) at Week 12 | | |
| Week 12 | | |
| N[1] | XX | XX |
| Yes | xx (xx.x%) | xx (xx.x%) |
| Difference [2] | xx.x% | |
| 95% CI for difference [2] | (xx.x%, xx.x%) | |
| p-value for difference [2] | 0.xxx | |
| Mean HAQ-DI score change at Week 12 | | |
| Week 12 | | |
| N[1] | xx | xx |
| Yes | xx (xx.x%) | xx (xx.x%) |
| Difference [2] | xx.x | |
| 95% CI for difference [2] | (xx.x, xx.x) | |
| p-value for difference [2] | 0.xxx | |

Abbreviations: ACR, American College of Rheumatology; CRP, C-reactive protein; DAS, Disease Activity Score; EULAR, European League Against Rheumatism; HAQ-DI, Health Assessment Questionnaire Disability Index; ITT, intent to treat; MCID, minimal clinically important difference.




Doc# CLP-004 Rev D, 15JUL2024

| Variable | Treatment | Control |
|----------|-----------|---------|
| Variable | (N=xxx) | (N=xxx) |

<sup>[1]</sup> Percentage calculated based on ITT Population.

Reference: Listing 16.x.x.x

SOURCE: xxxxx SAS 9.4 {program location} {run date/time}}


<sup>[2]</sup> Difference in proportions and one-sided p-value based on the Cochran-Mantel-Haenszel test stratified by inadequate response or loss of response to JAKi and RA disease severity at Day 0 for Stage 1 subjects and RA disease severity at Day 0 and inadequate response or loss of response to ≥ 4 biological DMARDs with ≥ 2 mechanisms of action for Stage 2 subjects.



Table 14.1.2.2.2 Sensitivity Analysis of Key Secondary Endpoints: Timing of Baseline (ITT Population)

| Variable | Treatment (N=xxx) | Control<br>(N=xxx) |
|---|---|---|
| DAS28-CRP moderate/good EULAR response at Week 12 from Day 0 | ( | (cr state) |
| Week 12 | | |
| N[1] | XX | XX |
| Yes | xx (xx.x%) | xx (xx.x%) |
| Difference [2] | xx.x% | |
| 95% CI for difference [2] | (xx.x%, xx.x%) | |
| p-value for difference [2] | 0.xxx | |
| DAS28-CRP response (MCID ≥ -1.2) at Week 12 from Day 0 | | |
| Week 12 | | |
| N[1] | XX | XX |
| Yes | xx (xx.x%) | xx (xx.x%) |
| Difference [2] | xx.x% | |
| 95% CI for difference [2] | (xx.x%, xx.x%) | |
| p-value for difference [2] | 0.xxx | |
| HAQ-DI response (MCID ≥ -0.22) at Week 12 from Day 0 | | |
| Week 12 | | |
| N[1] | XX | XX |
| Yes | xx (xx.x%) | xx (xx.x%) |
| Difference [2] | xx.x% | |
| 95% CI for difference [2] | (xx.x%, xx.x%) | |
| p-value for difference [2] | 0.xxx | |
| Mean HAQ-DI score change at Week 12 from Day 0 | | |
| Week 12 | | |
| N[1] | XX | XX |
| Yes | xx (xx.x%) | xx (xx.x%) |
| Difference [2] | XX.X | |
| 95% CI for difference [2] | (xx.x, xx.x) | |
| p-value for difference [2] | 0.xxx | |
| p-value for difference [2] | 0.xxx | |




#### Doc# CLP-004 Rev D, 15JUL2024

| Variable | Treatment | Control |
|----------|-----------|---------|
| variable | (N=xxx) | (N=xxx) |

Abbreviations: ACR, American College of Rheumatology; CRP, C-reactive protein; DAS, Disease Activity Score; EULAR, European League Against Rheumatism; HAQ-DI, Health Assessment Questionnaire Disability Index; ITT, intent to treat; MCID, minimal clinically important difference.

[1] Percentage calculated based on ITT Population.

[2] Difference in proportions and one-sided p-value based on the Cochran-Mantel-Haenszel test stratified by inadequate response or loss of response to JAKi and RA disease severity at Day 0 for Stage 1 subjects and RA disease severity at Day 0 and inadequate response or loss of response to ≥ 4 biological DMARDs with ≥ 2 mechanisms of action for Stage 2 subjects.

Reference: Listing 16.x.x.x

SOURCE: xxxxx SAS 9.4 {program location} {run date/time}}




#### Table 14.1.2.2.3 Sensitivity Analysis of Key Secondary Endpoints: Rescue Treatments (ITT Population)

| (CTT Optimion | Treatment | Control |
|---|---|---|
| Variable Variable | (N=xxx) | (N=xxx) |
| CR20 response at Week 12 from Day 0 | * | , |
| Week 12 | | |
| N[1] | XX | XX |
| Yes | xx (xx.x%) | xx (xx.x%) |
| Difference [2] | xx.x% | |
| 95% CI for difference [2] | (xx.x%, xx.x%) | |
| p-value for difference [2] | 0.xxx | |
| DAS28-CRP moderate/good EULAR response at Week 12 from baseline on the day of infor | med consent | |
| Week 12 | | |
| N[1] | XX | XX |
| Yes | xx (xx.x%) | xx (xx.x%) |
| Difference [2] | xx.x% | |
| 95% CI for difference [2] | (xx.x%, xx.x%) | |
| p-value for difference [2] | 0.xxx | |
| DAS28-CRP response (MCID ≥ -1.2) at Week 12 from baseline on the day of informed of | consent | |
| Week 12 | | |
| N[1] | XX | XX |
| Yes | xx (xx.x%) | xx (xx.x%) |
| Difference [2] | xx.x% | |
| 95% CI for difference [2] | (xx.x%, xx.x%) | |
| p-value for difference [2] | 0.xxx | |
| IAQ-DI response (MCID ≥ -0.22) at Week 12 from baseline on the day of informed cons | sent | |
| Week 12 | | |
| N[1] | XX | XX |
| Yes | xx (xx.x%) | xx (xx.x%) |
| Difference [2] | xx.x% | |
| 95% CI for difference [2] | (xx.x%, xx.x%) | |
| p-value for difference [2] | 0.xxx | |




Doc# CLP-004 Rev D, 15JUL2024

Variable Treatment Control (N=xxx) (N=xxx)

Abbreviations: ACR, American College of Rheumatology; CRP, C-reactive protein; DAS, Disease Activity Score; EULAR, European League Against Rheumatism; HAQ-DI, Health Assessment Questionnaire Disability Index; ITT, intent to treat; MCID, minimal clinically important difference.

- [1] Percentage calculated based on ITT Population.
- [2] Difference in proportions and one-sided p-value based on the Cochran-Mantel-Haenszel test stratified by inadequate response or loss of response to JAKi and RA disease severity at Day 0 for Stage 1 subjects and RA disease severity at Day 0 and inadequate response or loss of response to ≥ 4 biological DMARDs with ≥ 2 mechanisms of action for Stage 2 subjects.

Reference: Listing 16.x.x.x

SOURCE: xxxxx SAS 9.4 {program location} {run date/time}}

Table 14.1.2.2.4 Sensitivity Analysis of Key Secondary Endpoints: Missing Values (ITT Population)

Insert 2 x 2 table with tipping point results

Note to biostats: If more than 5% of primary efficacy data are missing, the table above is to be presented in addition to the multiple imputation approach of Berglund and Heeringa (2014) described in SAP Section 8.3.4.




#### Table 14.1.2.2.5 Subgroup Analysis of Key Secondary Endpoints: Prior b/tsDMARDs (ITT Population)

| Variable | Treatment<br>(N=xxx) | Control<br>(N=xxx) |
|---|---|---|
| ACR20 response from Day 0 | (11-333) | (11-111) |
| < 4 Prior b/tsDMARD | | |
| Week 12 | | |
| N[1] | xx | XX |
| Yes | xx (xx.x%) | xx (xx.x%) |
| Difference [2] | xx.x% | |
| 95% CI for difference [2] | (xx.x, xx.x) | |
| p-value for difference [2] | 0.xxx | |
| ≥ 4 Prior b/tsDMARD | | |
| Week 12 | | |
| N[1] | xx | XX |
| Yes | xx (xx.x%) | xx (xx.x%) |
| Difference [2] | XX.X% | |
| 95% CI for difference [2] | (xx.x, xx.x) | |
| p-value for difference [2] | 0.xxx | |
| Interaction p-value [3] | 0.xxx | |
| Repeat for: | | |
| DAS28-CRP moderate/good EULAR response at Week 12 from baseline | | |
| DAS28-CRP response (MCID ≥ -1.2) at Week 12 from baseline | | |
| HAQ-DI response (MCID $\geq$ -0.22) at Week 12 from baseline | | |
| 117Q-D1 response (WCID = -0.22) at week 12 from baseline | | |

Abbreviations: ACR, American College of Rheumatology; ITT, intent to treat.

- [1] Percentage calculated based on ITT Population.
- [2] Difference in proportions and one-sided p-value based on the Cochran-Mantel-Haenszel test stratified by inadequate response or loss of response to JAKi and RA disease severity at Day 0 for Stage 1 subjects and RA disease severity at Day 0 and inadequate response or loss of response to ≥ 4 biological DMARDs with ≥ 2 mechanisms of action for Stage 2 subjects.




#### Doc# CLP-004 Rev D, 15JUL2024

| Vorighto | Treatment | Control |
|----------|-----------|---------|
| Variable | (N=xxx) | (N=xxx) |

[3] Based on the Breslow Day test for homogeneity across subgroups.

Reference: Listing 16.x.x.x

SOURCE: xxxxx SAS 9.4 {program location} {run date/time}}




Table 14.1.2.2.6 Subgroup Analysis of Key Secondary Endpoints: Prior JAKi (ITT Population)

Repeat Table 14.1.2.2.5 for Prior JAKi [Yes vs. No]

Table 14.1.2.2.7
Subgroup Analysis of Key Secondary Endpoints: RA Disease Activity at Screening (ITT Population)

Repeat Table 14.1.2.2.5 for RA Disease Activity at Screening [DAS28-CRP ≤ 5.1 vs DAS28-CRP > 5.1]

Table 14.1.2.2.8
Subgroup Analysis of Key Secondary Endpoints: Moderate-to-severe RA at Day 0
(ITT Population)

Repeat Table 14.1.2.2.5 for Moderate-to-severe RA at Day 0 [<4 TJC28 or <4 SJC28 vs. ≥4 TJC28 and ≥4 SJC28]




Table 14.1.2.3 ACR50/70 (ITT Population)

| Variable | Treatment | Control<br>(N=xxx) |
|----------------------------|--------------|--------------------|
| | (N=xxx) | |
| ACR50 Response | | |
| Week 12 | | |
| N[1] | XX | XX |
| Yes | xx (xx.x%) | xx (xx.x%) |
| Difference [2] | XX.X% | |
| 95% CI for difference [2] | (xx.x, xx.x) | |
| p-value for difference [2] | 0.xxx | |
| ACR70 Response | | |
| Week 12 | | |
| N[1] | xx | XX |
| Yes | xx (xx.x%) | xx (xx.x%) |
| Difference [2] | xx.x% | |
| 95% CI for difference [2] | (xx.x, xx.x) | |
| p-value for difference [2] | 0.xxx | |

Abbreviations: ACR, American College of Rheumatology; ITT, intent to treat.

Reference: Listing 16.x.x.x

SOURCE: xxxxx SAS 9.4 {program location} {run date/time}}


<sup>[1]</sup> Percentage calculated based on ITT Population.

<sup>[2]</sup> Difference in proportions and one-sided p-value based on the Cochran-Mantel-Haenszel test stratified by inadequate response or loss of response to JAKi and RA disease severity at Day 0 for Stage 1 subjects and RA disease severity at Day 0 and inadequate response or loss of response to ≥ 4 biological DMARDs with ≥ 2 mechanisms of action for Stage 2 subjects.



Table 14.1.2.4 TJC28 (ITT Population)

| Variable | Treatment | Control |
|----------------------------|----------------|----------------|
| | (N=xxx) | (N=xxx) |
| JC28 Score | | |
| Screening (baseline) | | |
| N[1] | xx (xx.x%) | xx (xx,x%) |
| Mean (SD) | xxx.x (xxx.xx) | xxx.x (xxx.xx) |
| Median | XXX,XX | XXX.XX |
| Min-Max | xxx.x - xxx.x | xxx.x - xxx.x |
| Day 0 | | |
| N[1] | xx (xx.x%) | xx (xx.x%) |
| Mean (SD) | xxx.x (xxx.xx) | xxx.x (xxx.xx) |
| Median | xxx.xx | xxx.xx |
| Min-Max | xxx.x - xxx.x | xxx.x - xxx.x |
| Change from baseline | | |
| N[1] | xx (xx.x%) | xx (xx.x%) |
| Mean (SD) | xxx.x (xxx.xx) | xxx.x (xxx.xx) |
| Median | xxx.xx | xxx.xx |
| Min-Max | xxx.x - xxx.x | xxx.x - xxx.x |
| 95% CI for difference [2] | (xx.x, xx.x) | |
| p-value for difference [2] | 0.xxx | |
| Week 4 | | |
| N[1] | xx (xx.x%) | xx (xx.x%) |
| Mean (SD) | xxx.x (xxx.xx) | xxx.x (xxx.xx) |
| Median | xxx.xx | xxx.xx |
| Min-Max | xxx.x - xxx.x | xxx.x - xxx.x |
| Change from baseline | | |
| N[1] | xx (xx.x%) | xx (xx.x%) |
| Mean (SD) | xxx.x (xxx.xx) | xxx.x (xxx.xx) |
| Median | xxx.xx | XXX.XX |
| Min-Max | xxx.x - xxx.x | xxx.x - xxx.x |


# SETPOINT MEDICAL

#### Doc# CLP-004 Rev D, 15JUL2024

| /ariable | Treatment<br>(N=xxx) | Control<br>(N=xxx) |
|----------------------------|----------------------|--------------------|
| 95% CI for difference [2] | (XX.X, XX.X) | (IN-XXX) |
| p-value for difference [2] | 0.xxx | |
| W-1.0 | | |
| Week 8 | (0/) | (0/) |
| N[1] | xx (xx.x%) | xx (xx.x%) |
| Mean (SD) | xxx.x (xxx.xx) | xxx.x (xxx.xx) |
| Median | XXX.XX | XXX.XX |
| Min-Max | xxx.x - xxx.x | xxx.x - xxx.x |
| Change from baseline | | |
| N[1] | xx (xx.x%) | xx (xx.x%) |
| Mean (SD) | xxx.x (xxx.xx) | xxx.x (xxx.xx) |
| Median | XXX.XX | xxx.xx |
| Min-Max | xxx.x - xxx.x | xxx.x - xxx.x |
| 95% CI for difference [2] | (xx.x, xx.x) | |
| p-value for difference [2] | 0.xxx | |
| Week 12 | | |
| N[1] | xx (xx.x%) | xx (xx.x%) |
| Mean (SD) | xxx.x (xxx.xx) | xxx.x (xxx.xx) |
| Median | XXX.XX | XXX.XX |
| Min-Max | xxx.x - xxx.x | xxx.x - xxx.x |
| Change from baseline | | |
| N[1] | xx (xx.x%) | xx (xx.x%) |
| Mean (SD) | xxx.x (xxx.xx) | xxx.x (xxx.xx) |
| Median | XXX.XX | XXX.XX |
| Min-Max | xxx.x - xxx.x | xxx.x - xxx.x |
| 95% CI for difference [2] | (xx.x, xx.x) | |
| p-value for difference [2] | 0.xxx | |
| p-value for unrecence [2] | Villa | |
| [C28 20% Response [1] | | |
| Week 12 | | |
| N[1] | XX | XX |
| Yes | xx (xx.x%) | xx (xx.x%) |
| Difference [2] | xx.x% | |




| Variable | Treatment (N=xxx) | Control<br>(N=xxx) |
|----------------------------|-------------------|--------------------|
| 95% CI for difference [2] | (xx.x, xx.x) | (IV-XXX) |
| p-value for difference [2] | 0.xxx | |
| TJC28 50% Response [1] | | |
| Week 12 | | |
| N[1] | XX | XX |
| Yes | xx (xx.x%) | xx (xx.x%) |
| Difference [2] | XX.X% | |
| 95% CI for difference [2] | (xx.x, xx.x) | |
| p-value for difference [2] | 0.xxx | |
| TJC28 70% Response [1] | | |
| Week 12 | | |
| N[1] | XX | XX |
| Yes | xx (xx.x%) | xx (xx.x%) |
| Difference [2] | XX.X% | |
| 95% CI for difference [2] | (xx.x, xx.x) | |
| p-value for difference [2] | 0.xxx | |

Abbreviations: TJC, tender joint count for 28 different joints; ITT, intent to treat.

Reference: Listing 16.x.x.x

SOURCE: xxxxx SAS 9.4 {program location} {run date/time}}


<sup>[1]</sup> Percentage calculated based on ITT Population.

<sup>[2]</sup> Difference in mean score change from baseline and one-sided p-value based on the Mixed-effect Model Repeated Measure model with PROC MIXED. Difference in proportions and one-sided p-value based on the Cochran-Mantel-Haenszel test. Stratification factors are inadequate response or loss of response to JAKi and RA disease severity at Day 0 For Stage 1 subjects and RA disease severity at Day 0 and inadequate response or loss of response to ≥ 4 biological DMARDs with ≥ 2 mechanisms of action for Stage 2 subjects.



Table 14.1.2.5 SJC28 (ITT Population)

| Variable | Treatment | Control |
|----------------------------|-----------------------------|----------------|
| SJC28 Score | (N=xxx) | (N=xxx) |
| Screening (baseline) | xx (xx.x%) | xx (xx.x%) |
| N [1]<br>Mean (SD) | XX (XX.X/6) XXX.X (XXX.XX) | xxx.x (xxx.xx) |
| Median (SD) | XXX.XX | XXX.X (XXX.XX) |
| Min-Max | XXX.X – XXX.X | xxx.x – xxx.x |
| Day 0 | | |
| N[1] | xx (xx.x%) | xx (xx,x%) |
| Mean (SD) | xxx.x (xxx.xx) | xxx.x (xxx.xx) |
| Median | XXX.XX | xxx.xx |
| Min-Max | xxx.x - xxx.x | xxx.x - xxx.x |
| Change from baseline | | |
| N[1] | xx (xx.x%) | xx (xx.x%) |
| Mean (SD) | xxx.x (xxx.xx) | xxx.x (xxx.xx) |
| Median | xxx.xx | xxx.xx |
| Min-Max | xxx.x - xxx.x | xxx.x - xxx.x |
| 95% CI for difference [2] | (xx.x, xx.x) | |
| p-value for difference [2] | 0.xxx | |
| Week 4 | | |
| N[1] | xx (xx.x%) | xx (xx.x%) |
| Mean (SD) | xxx.x (xxx.xx) | xxx.x (xxx.xx) |
| Median | xxx.xx | xxx.xx |
| Min-Max | xxx.x - xxx.x | xxx.x - xxx.x |
| Change from baseline | | |
| N[1] | xx (xx.x%) | xx (xx.x%) |
| Mean (SD) | xxx.x (xxx.xx) | xxx.x (xxx.xx) |


# SETPOINT MEDICAL

#### Doc# CLP-004 Rev D, 15JUL2024

| /ariable | Treatment | Control |
|----------------------------|-------------------|-------------------|
| Median | (N=xxx)<br>xxx.xx | (N=xxx)<br>xxx.xx |
| Min-Max | xxx.x - xxx.x | XXX.X – XXX.X |
| 95% CI for difference [2]f | (xx.x, xx.x) | AAA,A — AAA,A |
| p-value for difference [2] | 0.xxx | |
| Week 8 | | |
| N[1] | xx (xx.x%) | xx (xx.x%) |
| Mean (SD) | xxx.x (xxx.xx) | xxx.x (xxx.xx) |
| Median | xxx.xx | xxx.xx |
| Min-Max | xxx.x - xxx.x | xxx.x - xxx.x |
| Change from baseline | | |
| N[1] | xx (xx.x%) | xx (xx.x%) |
| Mean (SD) | xxx.x (xxx.xx) | xxx.x (xxx.xx) |
| Median | XXX.XX | XXX,XX |
| Min-Max | xxx.x - xxx.x | xxx.x - xxx.x |
| 95% CI for difference [2] | (xx.x, xx.x) | |
| p-value for difference [2] | 0.xxx | |
| Week 12 | | |
| N[1] | xx (xx.x%) | xx (xx.x%) |
| Mean (SD) | xxx.x (xxx.xx) | xxx,x (xxx,xx) |
| Median | XXX.XX | XXX,XX |
| Min-Max | xxx.x - xxx.x | xxx.x - xxx.x |
| Change from baseline | | |
| N[1] | xx (xx.x%) | xx (xx.x%) |
| Mean (SD) | xxx.x (xxx.xx) | xxx.x (xxx.xx) |
| Median | xxx.xx | xxx.xx |
| Min-Max | xxx.x - xxx.x | xxx.x - xxx.x |
| 95% CI for difference [2] | (xx.x, xx.x) | |
| p-value for difference [2] | 0.xxx | |
| JC28 20% Response [1] | | |
| Week 12 | | |
| N[1] | xx | XX |



| Variable | Treatment | Control |
|----------------------------|--------------|------------|
| variable | (N=xxx) | (N=xxx) |
| Yes | xx (xx.x%) | xx (xx.x%) |
| Difference [2] | xx.x% | |
| 95% CI for difference [2] | (xx.x, xx.x) | |
| p-value for difference [2] | 0.xxx | |
| SJC28 50% Response [1] | | |
| Week 12 | | |
| N[1] | XX | XX |
| Yes | xx (xx.x%) | xx (xx.x%) |
| Difference [2] | XX.X% | |
| 95% CI for difference [2] | (xx.x, xx.x) | |
| p-value for difference [2] | 0.xxx | |
| SJC28 70% Response [1] | | |
| Week 12 | | |
| N[1] | XX | XX |
| Yes | xx (xx.x%) | xx (xx.x%) |
| Difference [2] | XX.X% | |
| 95% CI for difference [2] | (xx.x, xx.x) | |
| p-value for difference [2] | 0.xxx | |

Abbreviations: SJC, swollen joint count for 28 different joints; ITT, intent to treat.

Reference: Listing 16.x.x.x

SOURCE: xxxxx SAS 9.4 {program location} {run date/time}}


<sup>[1]</sup> Percentage calculated based on ITT Population.

<sup>[2]</sup> Difference in mean score change from baseline and one-sided p-value based on the Mixed-effect Model Repeated Measure model with PROC MIXED. Difference in proportions and one-sided p-value based on the Cochran-Mantel-Haenszel test. Stratification factors are inadequate response or loss of response to JAKi and RA disease severity at Day 0 for Stage 1 subjects and RA disease severity at Day 0 and inadequate response or loss of response to ≥ 4 biological DMARDs with ≥ 2 mechanisms of action for Stage 2 subjects.



## Table 14.1.2.6 Subject's Assessment of Pain (ITT Population)

| Variable | Treatment<br>(N=xxx) | Control<br>(N=xxx) |
|---------------------------------|----------------------|--------------------|
| Subject's Pain Assessment (NRS) | (11-111) | (11-1111) |
| Screening (baseline) | | |
| N[1] | xx (xx.x%) | xx (xx.x%) |
| Mean (SD) | xxx.x (xxx.xx) | xxx.x (xxx.xx) |
| Median | xxx.xx | xxx.xx |
| Min-Max | xxx.x - xxx.x | xxx.x - xxx.x |
| Day 0 | | |
| N[1] | xx (xx.x%) | xx (xx.x%) |
| Mean (SD) | xxx.x (xxx.xx) | xxx.x (xxx.xx) |
| Median | xxx.xx | xxx.xx |
| Min-Max | xxx.x - xxx.x | xxx.x - xxx.x |
| Change from baseline | | |
| N[1] | xx (xx.x%) | xx (xx.x%) |
| Mean (SD) | xxx.x (xxx.xx) | xxx.x (xxx.xx) |
| Median | xxx.xx | xxx.xx |
| Min-Max | xxx.x - xxx.x | xxx.x - xxx.x |
| 95% CI for difference [2] | (xx.x, xx.x) | |
| p-value for difference [2] | 0.xxx | |
| Week 4 | | |
| N[1] | xx (xx.x%) | xx (xx.x%) |
| Mean (SD) | xxx.x (xxx.xx) | xxx.x (xxx.xx) |
| Median | xxx.xx | xxx.xx |
| Min-Max | xxx.x - xxx.x | xxx.x - xxx.x |
| Change from baseline | | |
| N[1] | xx (xx.x%) | xx (xx.x%) |
| Mean (SD) | xxx.x (xxx.xx) | xxx.x (xxx.xx) |
| Median | xxx.xx | xxx.xx |
| Min-Max | xxx.x - xxx.x | xxx.x - xxx.x |


## Doc# CLP-004 Rev D, 15JUL2024

| ariable | Treatment | Control |
|--------------------------------|-------------------------|----------------|
| 95% CI for difference [2] | (N=xxx)<br>(xx.x, xx.x) | (N=xxx) |
| p-value for difference [2] | 0.xxx | |
| p-value for difference [2] | V.AAA | |
| Week 8 | | |
| N[1] | xx (xx.x%) | xx (xx.x%) |
| Mean (SD) | xxx.x (xxx.xx) | xxx.x (xxx.xx) |
| Median | XXX,XX | XXX,XX |
| Min-Max | xxx.x - xxx.x | xxx.x - xxx.x |
| Change from baseline | | |
| N[1] | xx (xx.x%) | xx (xx.x%) |
| Mean (SD) | xxx.x (xxx.xx) | xxx.x (xxx.xx) |
| Median | xxx.xx | xxx.xx |
| Min-Max | xxx.x - xxx.x | xxx.x - xxx.x |
| 95% CI for difference [2] | (xx.x, xx.x) | |
| p-value for difference [2] | 0.xxx | |
| Week 12 | | |
| N[1] | xx (xx.x%) | xx (xx.x%) |
| Mean (SD) | xxx.x (xxx.xx) | xxx.x (xxx.xx |
| Median | XXX.XX | xxx.xx |
| Min-Max | xxx.x - xxx.x | xxx.x - xxx.x |
| Change from baseline | | |
| N[1] | xx (xx.x%) | xx (xx.x%) |
| Mean (SD) | xxx.x (xxx.xx) | xxx.x (xxx.xx |
| Median | XXX.XX | XXX,XX |
| Min-Max | xxx.x - xxx.x | xxx.x - xxx.x |
| 95% CI for difference [2] | (xx.x, xx.x) | |
| p-value for difference [2] | 0.xxx | |
| ıbject's Pain 20% Response [1] | | |
| Week 12 | | |
| N[1] | XX | xx |
| Yes | xx (xx.x%) | xx (xx.x%) |
| Difference [2] | xx.x% | |


## Statistical Analysis Plan for Interim and Primary Analyses in SPM-020 (The RESET-RA Study)



### Doc# CLP-004 Rev D, 15JUL2024

| Variable | Treatment (N=xxx) | Control<br>(N=xxx) |
|---------------------------------|-------------------|--------------------|
| 95% CI for difference [2] | (XX.X, XX.X) | (14-333) |
| p-value for difference [2] | 0.xxx | |
| Subject's Pain 50% Response [1] | | |
| Week 12 | | |
| N[1] | xx | XX |
| Yes | xx (xx.x%) | xx (xx.x%) |
| Difference [2] | XX.X% | |
| 95% CI for difference [2] | (xx.x, xx.x) | |
| p-value for difference [2] | 0.xxx | |
| Subject's Pain 70% Response [1] | | |
| Week 12 | | |
| N[1] | XX | XX |
| Yes | xx (xx.x%) | xx (xx.x%) |
| Difference [2] | xx.x% | |
| 95% CI for difference [2] | (xx.x, xx.x) | |
| p-value for difference [2] | 0.xxx | |

Abbreviations: NRS, Numerical Rating Scale; ITT, intent to treat.

- [1] Percentage calculated based on ITT Population.
- [2] Difference in mean score change from baseline and one-sided p-value based on the Mixed-effect Model Repeated Measure model with PROC MIXED. Difference in proportions and one-sided p-value based on the Cochran-Mantel-Haenszel test. Stratification factors are inadequate response or loss of response to JAKi and RA disease severity at Day 0 for Stage 1 subjects and RA disease severity at Day 0 and inadequate response or loss of response to ≥ 4 biological DMARDs with ≥ 2 mechanisms of action for Stage 2 subjects.

Reference: Listing 16.x.x.x

SOURCE: xxxxx SAS 9.4 {program location} {run date/time}}




Table 14.1.2.7 SGA (ITT Population)

| Variable | Treatment<br>(N=xxx) | Control<br>(N=xxx) |
|---|---|---|
| SGA Score | (, , | (51 11111) |
| Screening (baseline) | | |
| N[1] | xx (xx.x%) | xx (xx.x%) |
| Mean (SD) | xxx.x (xxx.xx) | xxx.x (xxx.xx) |
| Median | XXX.XX | xxx.xx |
| Min-Max | xxx.x - xxx.x | xxx.x - xxx.x |
| Day 0 | | |
| N[1] | xx (xx.x%) | xx (xx,x%) |
| Mean (SD) | xxx.x (xxx.xx) | xxx.x (xxx.xx) |
| Median | xxx.xx | XXX,XX |
| Min-Max | xxx.x - xxx.x | xxx.x - xxx.x |
| Change from baseline | | |
| N[1] | xx (xx.x%) | xx (xx.x%) |
| Mean (SD) | xxx.x (xxx.xx) | xxx.x (xxx.xx) |
| Median | XXX.XX | xxx,xx |
| Min-Max | xxx.x - xxx.x | xxx.x - xxx.x |
| 95% CI for difference [2] | (xx.x, xx.x) | |
| p-value for difference [2] | 0.xxx | |
| Week 4 | | |
| N[1] | xx (xx.x%) | xx (xx.x%) |
| Mean (SD) | xxx.x (xxx.xx) | xxx.x (xxx.xx) |
| Median | XXX.XX | XXX.XX |
| Min-Max | xxx.x - xxx.x | xxx.x - xxx.x |
| Change from baseline | | |
| N[1] | xx (xx.x%) | xx (xx.x%) |
| Mean (SD) | xxx.x (xxx.xx) | xxx.x (xxx.xx) |
| Median | xxx.xx | xxx.xx |
| Min-Max | xxx.x - xxx.x | xxx.x - xxx.x |


## Doc# CLP-004 Rev D, 15JUL2024

| ariable | Treatment<br>(N=xxx) | Control<br>(N=xxx) |
|----------------------------|----------------------|--------------------|
| 95% CI for difference [2] | (xx.x, xx.x) | (11 444) |
| p-value for difference [2] | 0.xxx | |
| Week 8 | | |
| N[1] | xx (xx.x%) | xx (xx.x%) |
| Mean (SD) | xxx.x (xxx.xx) | xxx.x (xxx.xx) |
| Median | XXX.XX | xxx,xx |
| Min-Max | xxx.x - xxx.x | xxx.x - xxx.x |
| Change from baseline | | |
| N[1] | xx (xx.x%) | xx (xx.x%) |
| Mean (SD) | xxx.x (xxx.xx) | xxx.x (xxx.xx) |
| Median | xxx.xx | XXX.XX |
| Min-Max | xxx.x - xxx.x | xxx.x - xxx.x |
| 95% CI for difference [2] | (xx.x, xx.x) | |
| p-value for difference [2] | 0.xxx | |
| Week 12 | | |
| N[1] | xx (xx.x%) | xx (xx.x%) |
| Mean (SD) | xxx.x (xxx.xx) | xxx.x (xxx.xx) |
| Median | XXX.XX | XXX,XX |
| Min-Max | xxx.x - xxx.x | xxx.x - xxx.x |
| Change from baseline | | |
| N[1] | xx (xx.x%) | xx (xx.x%) |
| Mean (SD) | xxx.x (xxx.xx) | xxx.x (xxx.xx) |
| Median | XXX.XX | XXX,XX |
| Min-Max | xxx.x - xxx.x | xxx.x - xxx.x |
| 95% CI for difference [2] | (xx.x, xx.x) | |
| p-value for difference [2] | 0.xxx | |
| A 20% Response [1] | | |
| Week 12 | | |
| N[1] | XX | XX |
| Yes | xx (xx.x%) | xx (xx.x%) |
| Difference [2] | xx.x% | |




| Variable | Treatment | Control |
|----------------------------|--------------|------------|
| variable | (N=xxx) | (N=xxx) |
| 95% CI for difference [2] | (xx.x, xx.x) | |
| p-value for difference [2] | 0.xxx | |
| SGA 50% Response [1] | | |
| Week 12 | | |
| N[1] | XX | xx |
| Yes | xx (xx.x%) | xx (xx.x%) |
| Difference [2] | xx.x% | |
| 95% CI for difference [2] | (xx.x, xx.x) | |
| p-value for difference [2] | 0.xxx | |
| GGA 70% Response [1] | | |
| Week 12 | | |
| N[1] | XX | XX |
| Yes | xx (xx.x%) | xx (xx.x%) |
| Difference [2] | xx.x% | |
| 95% CI for difference [2] | (xx.x, xx.x) | |
| p-value for difference [2] | 0.xxx | |

Abbreviations: SGA, subject's global assessment; ITT, intent to treat.

- [1] Percentage calculated based on ITT Population.
- [2] Difference in mean score change from baseline and one-sided p-value based on the Mixed-effect Model Repeated Measure model with PROC MIXED. Difference in proportions and one-sided p-value based on the Cochran-Mantel-Haenszel test. Stratification factors are inadequate response or loss of response to JAKi and RA disease severity at Day 0 for Stage 1 subjects and RA disease severity at Day 0 and inadequate response or loss of response to ≥ 4 biological DMARDs with ≥ 2 mechanisms of action for Stage 2 subjects.

Reference: Listing 16.x.x.x

SOURCE: xxxxx SAS 9.4 {program location} {run date/time}}




Table 14.1.2.8 EGA (ITT Population)

| Variable | Treatment<br>(N=xxx) | Control<br>(N=xxx) |
|----------------------------|----------------------|--------------------|
| EGA Score | (14-333) | (14-333) |
| Screening (baseline) | | |
| N[1] | xx (xx.x%) | xx (xx.x%) |
| Mean (SD) | xxx.x (xxx.xx) | xxx.x (xxx.xx) |
| Median | xxx.xx | XXX.XX |
| Min-Max | xxx.x - xxx.x | xxx.x - xxx.x |
| Day 0 | | |
| N[1] | xx (xx.x%) | xx (xx.x%) |
| Mean (SD) | xxx.x (xxx.xx) | xxx.x (xxx.xx) |
| Median | xxx.xx | xxx.xx |
| Min-Max | xxx.x - xxx.x | xxx.x - xxx.x |
| Change from baseline | | |
| N[1] | xx (xx.x%) | xx (xx.x%) |
| Mean (SD) | xxx.x (xxx.xx) | xxx.x (xxx.xx) |
| Median | xxx.xx | xxx.xx |
| Min-Max | xxx.x - xxx.x | xxx.x - xxx.x |
| 95% CI for difference [2] | (xx.x, xx.x) | |
| p-value for difference [2] | 0.xxx | |
| Week 4 | | |
| N[1] | xx (xx.x%) | xx (xx.x%) |
| Mean (SD) | xxx.x (xxx.xx) | xxx.x (xxx.xx) |
| Median | xxx.xx | xxx.xx |
| Min-Max | xxx.x - xxx.x | xxx.x - xxx.x |
| Change from baseline | | |
| N[1] | xx (xx.x%) | xx (xx.x%) |
| Mean (SD) | xxx.x (xxx.xx) | xxx.x (xxx.xx) |
| Median | xxx.xx | xxx.xx |
| Min-Max | xxx.x - xxx.x | xxx.x - xxx.x |


## Doc# CLP-004 Rev D, 15JUL2024

| Variable Variable | Treatment (N=xxx) | Control<br>(N=xxx) |
|----------------------------|-------------------|--------------------|
| 95% CI for difference [2] | (xx.x, xx.x) | (11 11111) |
| p-value for difference [2] | 0.xxx | |
| Week 8 | | |
| N[1] | xx (xx.x%) | xx (xx.x%) |
| Mean (SD) | xxx.x (xxx.xx) | xxx,x (xxx,xx) |
| Median | XXX.XX | XXX.XX |
| Min-Max | xxx.x - xxx.x | xxx.x - xxx.x |
| Change from baseline | | |
| N[1] | xx (xx.x%) | xx (xx,x%) |
| Mean (SD) | xxx.x (xxx.xx) | xxx.x (xxx.xx) |
| Median | xxx.xx | XXX,XX |
| Min-Max | xxx.x - xxx.x | xxx.x - xxx.x |
| 95% CI for difference [2] | (xx.x, xx.x) | |
| p-value for difference [2] | 0.xxx | |
| Week 12 | | |
| N[1] | xx (xx.x%) | xx (xx.x%) |
| Mean (SD) | xxx.x (xxx.xx) | xxx,x (xxx,xx) |
| Median | xxx.xx | XXX.XX |
| Min-Max | xxx.x - xxx.x | xxx.x - xxx.x |
| Change from baseline | | |
| N[1] | xx (xx.x%) | xx (xx.x%) |
| Mean (SD) | xxx.x (xxx.xx) | xxx.x (xxx.xx) |
| Median | XXX.XX | XXX,XX |
| Min-Max | xxx.x - xxx.x | xxx.x - xxx.x |
| 95% CI for difference [2] | (xx.x, xx.x) | |
| p-value for difference [2] | 0.xxx | |
| GA 20% Response [1] | | |
| Week 12 | | |
| N[1] | XX | XX |
| Yes | xx (xx.x%) | xx (xx.x%) |
| Difference [2] | xx.x% | |




| Variable | Treatment | Control |
|----------------------------|--------------|------------|
| V апавіе | (N=xxx) | (N=xxx) |
| 95% CI for difference [2] | (xx.x, xx.x) | |
| p-value for difference [2] | 0.xxx | |
| EGA 50% Response [1] | | |
| Week 12 | | |
| N[1] | XX | XX |
| Yes | xx (xx.x%) | xx (xx.x%) |
| Difference [2] | XX.X% | |
| 95% CI for difference [2] | (xx.x, xx.x) | |
| p-value for difference [2] | 0.xxx | |
| EGA 70% Response [1] | | |
| Week 12 | | |
| N[1] | XX | XX |
| Yes | xx (xx.x%) | xx (xx.x%) |
| Difference [2] | XX.X% | |
| 95% CI for difference [2] | (xx.x, xx.x) | |
| p-value for difference [2] | 0.xxx | |

Abbreviations: EGA, evaluator's global assessment; ITT, intent to treat.

Reference: Listing 16.x.x.x

SOURCE: xxxxx SAS 9.4 {program location} {run date/time}}


Percentage calculated based on ITT Population.

<sup>[2]</sup> Difference in mean score change from baseline and one-sided p-value based on the Mixed-effect Model Repeated Measure model with PROC MIXED. Difference in proportions and one-sided p-value based on the Cochran-Mantel-Haenszel test. Stratification factors are inadequate response or loss of response to JAKi and RA disease severity at Day 0 for Stage 1 subjects and RA disease severity at Day 0 and inadequate response or loss of response to ≥ 4 biological DMARDs with ≥ 2 mechanisms of action for Stage 2 subjects.



Table 14.1.2.9 hsCRP (ITT Population)

| Variable | Treatment | Control |
|----------------------------|----------------|----------------|
| | (N=xxx) | (N=xxx) |
| hsCRP (mg/L) | | |
| Screening (baseline) | | |
| N[1] | xx (xx.x%) | xx (xx.x%) |
| Mean (SD) | xxx.x (xxx.xx) | xxx.x (xxx.xx) |
| Median | XXX.XX | XXX.XX |
| Min-Max | xxx.x - xxx.x | xxx.x - xxx.x |
| Day 0 | | |
| N[1] | xx (xx.x%) | xx (xx.x%) |
| Mean (SD) | xxx.x (xxx.xx) | xxx.x (xxx.xx) |
| Median | xxx.xx | xxx.xx |
| Min-Max | xxx.x - xxx.x | xxx.x - xxx.x |
| Change from baseline | | |
| N[1] | xx (xx.x%) | xx (xx.x%) |
| Mean (SD) | xxx.x (xxx.xx) | xxx.x (xxx.xx) |
| Median | xxx.xx | xxx.xx |
| Min-Max | xxx.x - xxx.x | xxx.x - xxx.x |
| 95% CI for difference [2] | (xx.x, xx.x) | |
| p-value for difference [2] | 0.xxx | |
| Week 4 | | |
| N[1] | xx (xx.x%) | xx (xx.x%) |
| Mean (SD) | xxx.x (xxx.xx) | xxx.x (xxx.xx) |
| Median | xxx.xx | XXX.XX |
| Min-Max | xxx.x - xxx.x | xxx.x - xxx.x |
| Change from baseline | | |
| N[1] | xx (xx.x%) | xx (xx.x%) |
| Mean (SD) | xxx.x (xxx.xx) | xxx.x (xxx.xx) |
| Median | XXX.XX | XXX.XX |
| Min-Max | XXX.X — XXX.X | XXX.X – XXX.X |


## Doc# CLP-004 Rev D, 15JUL2024

| ariable | Treatment<br>(N=xxx) | Control<br>(N=xxx) |
|----------------------------|----------------------|--------------------|
| 95% CI for difference [2] | (xx.x, xx.x) | (IT AAA) |
| p-value for difference [2] | 0.xxx | |
| Week 8 | | |
| N[1] | xx (xx.x%) | xx (xx.x%) |
| Mean (SD) | xxx.x (xxx.xx) | xxx.x (xxx.xx) |
| Median | XXX.XX | xxx.xx |
| Min-Max | xxx.x - xxx.x | xxx.x - xxx.x |
| Change from baseline | | |
| N[1] | xx (xx.x%) | xx (xx.x%) |
| Mean (SD) | xxx.x (xxx.xx) | xxx.x (xxx.xx) |
| Median | xxx.xx | xxx,xx |
| Min-Max | xxx.x - xxx.x | xxx.x - xxx.x |
| 95% CI for difference [2] | (xx.x, xx.x) | |
| p-value for difference [2] | 0.xxx | |
| Week 12 | | |
| N[1] | xx (xx.x%) | xx (xx.x%) |
| Mean (SD) | xxx.x (xxx.xx) | xxx.x (xxx.xx) |
| Median | XXX.XX | xxx.xx |
| Min-Max | xxx.x - xxx.x | xxx.x - xxx.x |
| Change from baseline | | |
| N[1] | xx (xx.x%) | xx (xx.x%) |
| Mean (SD) | xxx.x (xxx.xx) | xxx.x (xxx.xx) |
| Median | XXX.XX | XXX,XX |
| Min-Max | xxx.x - xxx.x | xxx.x - xxx.x |
| 95% CI for difference [2] | (xx.x, xx.x) | |
| p-value for difference [2] | 0.xxx | |
| CRP 20% Response [1] | | |
| Week 12 | | |
| N[1] | xx | XX |
| Yes | xx (xx.x%) | xx (xx.x%) |
| Difference [2] | xx.x% | |




| Variable | Treatment | Control |
|-----------------------------------------------|--------------|------------|
| Vапавіе — | (N=xxx) | (N=xxx) |
| 95% CI for difference [2] | (xx.x, xx.x) | |
| p-value for difference [2] | 0.xxx | |
| hsCRP 50% Response [1] | | |
| Week 12 | | |
| N[1] | XX | XX |
| Yes | xx (xx.x%) | xx (xx.x%) |
| Difference [2] | xx.x% | |
| 95% CI for difference [2] | (xx.x, xx.x) | |
| p-value for difference [2] | 0.xxx | |
| hsCRP 70% Response [1] | | |
| Week 12 | | |
| N[1] | XX | XX |
| Yes | xx (xx.x%) | xx (xx.x%) |
| Difference [2] | XX.X% | |
| 95% CI for difference [2] | (xx.x, xx.x) | |
| p-value for difference [2] | 0.xxx | |

Abbreviations: hsCRP, high sensitivity C-reactive protein; ITT, intent to treat...

Reference: Listing 16.x.x.x

SOURCE: xxxxx SAS 9.4 {program location} {run date/time}}


<sup>[1]</sup> Percentage calculated based on ITT Population.

<sup>[2]</sup> Difference in mean score change from baseline and one-sided p-value based on the Mixed-effect Model Repeated Measure model with PROC MIXED. Difference in proportions and one-sided p-value based on the Cochran-Mantel-Haenszel test. Stratification factors are inadequate response or loss of response to JAKi and RA disease severity at Day 0 for Stage 1 subjects and RA disease severity at Day 0 and inadequate response or loss of response to ≥ 4 biological DMARDs with ≥ 2 mechanisms of action for Stage 2 subjects.



Table 14.1.2.10 HAQ-DI (ITT Population)

| Variable | Treatment | Control |
|----------------------------|----------------|----------------|
| | (N=xxx) | (N=xxx) |
| HAQ-DI Score | | |
| Screening (baseline) | | |
| N[1] | xx (xx.x%) | xx (xx.x%) |
| Mean (SD) | xxx.x (xxx.xx) | xxx.x (xxx.xx) |
| Median | XXX,XX | XXX,XX |
| Min-Max | xxx.x - xxx.x | xxx.x - xxx.x |
| Day 0 | | |
| N[1] | xx (xx.x%) | xx (xx.x%) |
| Mean (SD) | xxx.x (xxx.xx) | xxx.x (xxx.xx) |
| Median | xxx.xx | xxx.xx |
| Min-Max | xxx.x - xxx.x | xxx.x - xxx.x |
| Change from baseline | | |
| N[1] | xx (xx.x%) | xx (xx.x%) |
| Mean (SD) | xxx.x (xxx.xx) | xxx.x (xxx.xx) |
| Median | xxx.xx | xxx.xx |
| Min-Max | xxx.x - xxx.x | xxx.x - xxx.x |
| 95% CI for difference [2] | (xx.x, xx.x) | |
| p-value for difference [2] | 0.xxx | |
| Week 4 | | |
| N[1] | xx (xx.x%) | xx (xx.x%) |
| Mean (SD) | xxx.x (xxx.xx) | xxx.x (xxx.xx) |
| Median | xxx.xx | xxx.xx |
| Min-Max | xxx.x - xxx.x | xxx.x - xxx.x |
| Change from baseline | | |
| N[1] | xx (xx.x%) | xx (xx.x%) |
| Mean (SD) | xxx.x (xxx.xx) | xxx.x (xxx.xx) |
| Median | XXX.XX | XXX.XX |
| Min-Max | xxx.x – xxx.x | XXX.X – XXX.X |


## Doc# CLP-004 Rev D, 15JUL2024

| ariable | Treatment<br>(N=xxx) | Control<br>(N=xxx) |
|----------------------------|----------------------|--------------------|
| 95% CI for difference [2] | (xx.x, xx.x) | (II AAA) |
| p-value for difference [2] | 0.xxx | |
| Week 8 | | |
| N[1] | xx (xx.x%) | xx (xx.x%) |
| Mean (SD) | xxx.x (xxx.xx) | xxx.x (xxx.xx) |
| Median | XXX.XX | XXX,XX |
| Min-Max | xxx.x - xxx.x | xxx.x - xxx.x |
| Change from baseline | | |
| N[1] | xx (xx.x%) | xx (xx.x%) |
| Mean (SD) | xxx.x (xxx.xx) | xxx.x (xxx.xx) |
| Median | xxx.xx | xxx.xx |
| Min-Max | xxx.x - xxx.x | xxx.x - xxx.x |
| 95% CI for difference [2] | (xx.x, xx.x) | |
| p-value for difference [2] | 0.xxx | |
| Week 12 | | |
| N[1] | xx (xx.x%) | xx (xx.x%) |
| Mean (SD) | xxx.x (xxx.xx) | xxx.x (xxx.xx) |
| Median | XXX.XX | xxx.xx |
| Min-Max | xxx.x - xxx.x | xxx.x - xxx.x |
| Change from baseline | | |
| N[1] | xx (xx.x%) | xx (xx.x%) |
| Mean (SD) | xxx.x (xxx.xx) | xxx.x (xxx.xx) |
| Median | XXX.XX | XXX,XX |
| Min-Max | xxx.x - xxx.x | xxx.x - xxx.x |
| 95% CI for difference [2] | (xx.x, xx.x) | |
| p-value for difference [2] | 0.xxx | |
| Q-DI 20% Response [1] | | |
| Week 12 | | |
| N[1] | XX | XX |
| Yes | xx (xx.x%) | xx (xx.x%) |
| Difference [2] | xx.x% | |


## Doc# CLP-004 Rev D, 15JUL2024

| Variable | Treatment<br>(N=xxx) | Control<br>(N=xxx) |
|---|---|---|
| 95% CI for difference [2] | (xx.x, xx.x) | (*,) |
| p-value for difference [2] | 0.xxx | |
| HAQ-DI 50% Response [1] | | |
| Week 12 | | |
| N[1] | xx | XX |
| Yes | xx (xx.x%) | xx (xx.x%) |
| Difference [2] | xx.x% | |
| 95% CI for difference [2] | (xx.x, xx.x) | |
| p-value for difference [2] | 0.xxx | |
| HAQ-DI 70% Response [1] | | |
| Week 12 | | |
| N[1] | xx | XX |
| Yes | xx (xx.x%) | xx (xx.x%) |
| Difference [2] | xx.x% | |
| 95% CI for difference [2] | (xx.x, xx.x) | |
| p-value for difference [2] | 0.xxx | |
| HAQ-DI Mild Difficulties to Moderate Disability (score from 0 to < 1) [1]<br>Screening (baseline) | | |
| N[1] | xx | XX |
| Yes | xx (xx.x%) | xx (xx.x%) |
| Difference [2] | xx.x% | |
| Week 12 | | |
| N[1] | xx | xx |
| Yes | xx (xx.x%) | xx (xx.x%) |
| Difference [2] | xx.x% | |
| 95% CI for difference [2] | (xx.x, xx.x) | |
| p-value for difference [2] | 0.xxx | |
| HAQ-DI Moderate Disability (score from 1 to < 2) [1]<br>Screening (baseline) | | |
| N[1] | xx | xx |
| Yes | xx (xx.x%) | xx (xx.x%) |


### Doc# CLP-004 Rev D, 15JUL2024

| Variable | Treatment | Control |
|---|---|---|
| | (N=xxx) | (N=xxx) |
| Difference [2] | xx.x% | |
| Week 12 | | |
| N[1] | xx | XX |
| Yes | xx (xx.x%) | xx (xx,x%) |
| Difference [2] | xx.x% | |
| 95% CI for difference [2] | (xx.x, xx.x) | |
| p-value for difference [2] | 0.xxx | |
| HAQ-DI Subjects with Severe to Very Severe Disability (score from 2 to 3) [1] | | |
| Screening (baseline) | | |
| N[1] | XX | XX |
| Yes | xx (xx.x%) | xx (xx,x%) |
| Difference [2] | xx.x% | |
| Week 12 | | |
| N[1] | xx | XX |
| Yes | xx (xx.x%) | xx (xx.x%) |
| Difference [2] | xx.x% | |
| 95% CI for difference [2] | (xx.x, xx.x) | |
| p-value for difference [2] | 0.xxx | |
| HAQ-DI Response (MCID $\geq$ 0.22) [1] | | |
| Week 12 | | |
| N[1] | xx | XX |
| Yes | xx (xx.x%) | xx (xx,x%) |
| Difference [2] | xx.x% | |
| 95% CI for difference [2] | (xx.x, xx.x) | |
| p-value for difference [2] | 0.xxx | |

Abbreviations: HAQ-DI, Health Assessment Questionnaire Disability Index; ITT, intent to treat; MCID, Minimal clinically important difference.


<sup>[1]</sup> Percentage calculated based on ITT Population

<sup>[2]</sup> Difference in mean score change from baseline and one-sided p-value based on the Mixed-effect Model Repeated Measure model with PROC MIXED. Difference in proportions and one-sided p-value based on the Cochran-Mantel-Haenszel test. Stratification factors are inadequate response or loss of response to JAKi and RA disease severity at Day 0 for Stage 1 subjects and RA disease severity at Day 0 and inadequate response or loss of response to  $\geq$  4 biological DMARDs with  $\geq$  2 mechanisms of action for Stage 2 subjects.

Statistical Analysis Plan for Interim and Primary Analyses in SPM-020 (The RESET-RA Study)



## Doc# CLP-004 Rev D, 15JUL2024

Variable Treatment Control (N=xxx) (N=xxx)

Reference: Listing 16.x.x.x

SOURCE: xxxxx SAS 9.4 {program location} {run date/time}}




Table 14.1.2.11 DAS28-CRP (ITT Population)

| Variable | Treatment (N=xxx) | Control<br>(N=xxx) |
|----------------------------|-------------------|--------------------|
| DAS28-CRP Score | (11-333) | (11-222) |
| Screening (baseline) | | |
| N[1] | xx (xx.x%) | xx (xx.x%) |
| Mean (SD) | xxx.x (xxx.xx) | xxx.x (xxx.xx) |
| Median | xxx.xx | xxx.xx |
| Min-Max | xxx.x - xxx.x | xxx.x - xxx.x |
| Day 0 | | |
| N[1] | xx (xx.x%) | xx (xx.x%) |
| Mean (SD) | xxx.x (xxx.xx) | xxx.x (xxx.xx) |
| Median | xxx.xx | xxx.xx |
| Min-Max | xxx.x - xxx.x | xxx.x - xxx.x |
| Change from baseline | | |
| N[1] | xx (xx.x%) | xx (xx.x%) |
| Mean (SD) | xxx.x (xxx.xx) | xxx.x (xxx.xx) |
| Median | xxx.xx | xxx.xx |
| Min-Max | xxx.x - xxx.x | xxx.x - xxx.x |
| 95% CI for difference [2] | (xx.x, xx.x) | |
| p-value for difference [2] | 0.xxx | |
| Week 4 | | |
| N[1] | xx (xx.x%) | xx (xx.x%) |
| Mean (SD) | xxx.x (xxx.xx) | xxx.x (xxx.xx) |
| Median | xxx.xx | xxx.xx |
| Min-Max | xxx.x - xxx.x | xxx.x - xxx.x |
| Change from baseline | | |
| N[1] | xx (xx.x%) | xx (xx.x%) |
| Mean (SD) | xxx.x (xxx.xx) | xxx.x (xxx.xx) |
| Median | xxx.xx | xxx.xx |
| Min-Max | xxx.x - xxx.x | xxx.x - xxx.x |


## Doc# CLP-004 Rev D, 15JUL2024

| Variable | Treatment<br>(N=xxx) | Control<br>(N=xxx) |
|---|---|---|
| 95% CI for difference [2] | (xx.x, xx.x) | (1, 1111) |
| p-value for difference [2] | 0.xxx | |
| Week 8 | | |
| N[1] | xx (xx.x%) | xx (xx.x%) |
| Mean (SD) | xxx.x (xxx.xx) | xxx.x (xxx.xx) |
| Median | xxx.xx | xxx.xx |
| Min-Max | xxx.x - xxx.x | xxx.x - xxx.x |
| Change from baseline | | |
| N[1] | xx (xx.x%) | xx (xx.x%) |
| Mean (SD) | xxx.x (xxx.xx) | xxx.x (xxx.xx) |
| Median | XXX.XX | XXX,XX |
| Min-Max | xxx.x - xxx.x | xxx,x - xxx,x |
| 95% CI for difference [2] | (xx.x, xx.x) | |
| p-value for difference [2] | 0.xxx | |
| Week 12 | | |
| N[1] | xx (xx.x%) | xx (xx.x%) |
| Mean (SD) | xxx.x (xxx.xx) | xxx.x (xxx.xx) |
| Median | xxx.xx | XXX,XX |
| Min-Max | xxx.x - xxx.x | xxx.x - xxx.x |
| Change from baseline | | |
| N[1] | xx (xx.x%) | xx (xx.x%) |
| Mean (SD) | xxx.x (xxx.xx) | xxx.x (xxx.xx) |
| Median | XXX.XX | XXX.XX |
| Min-Max | xxx.x - xxx.x | xxx.x - xxx.x |
| 95% CI for difference [2] | (xx.x, xx.x) | |
| p-value for difference [2] | 0.xxx | |
| AS28-CRP MCID Response (score reduction from Baseline by 1.2) [1] | | |
| Week 12 | | |
| N[1] | xx | XX |
| Yes | xx (xx.x%) | xx (xx.x%) |
| Difference [2] | xx.x% | |


### Doc# CLP-004 Rev D, 15JUL2024

| Variable | Treatment<br>(N=xxx) | Control<br>(N=xxx) |
|---|---|---|
| 95% CI for difference [2] | (xx.x, xx.x) | (11 1111) |
| p-value for difference [2] | 0.xxx | |
| DAS28-CRP Low Disease Activity (score 2.6 to < 3.2) [1] | | |
| Week 12 | | |
| N[1] | | |
| Yes | xx (xx.x%) | xx (xx.x%) |
| Difference [2] | xx.x% | |
| 95% CI for difference [2] | (xx.x, xx.x) | |
| p-value for difference [2] | 0.xxx | |
| DAS28-CRP Remission (score 0 to < 2.6) [1] | | |
| Week 12 | | |
| N[1] | xx | XX |
| Yes | xx (xx.x%) | xx (xx.x%) |
| Difference [2] | xx.x% | |
| 95% CI for difference [2] | (xx.x, xx.x) | |
| p-value for difference [2] | 0.xxx | |
| DAS28-CRP EULAR Good Response [1][3] | | |
| Week 12 | | |
| N[1] | XX | XX |
| Yes | xx (xx.x%) | xx (xx.x%) |
| Difference [2] | xx.x% | |
| 95% CI for difference [2] | (xx.x, xx.x) | |
| p-value for difference [2] | 0.xxx | |
| DAS28-CRP EULAR Moderate Response [1][4] | | |
| Week 12 | | |
| N[1] | xx | XX |
| Yes | xx (xx.x%) | xx (xx.x%) |
| Difference [2] | xx.x% | |
| 95% CI for difference [2] | (xx.x, xx.x) | |
| p-value for difference [2] | 0.xxx | |

Abbreviations: CRP, C-reactive protein; DAS, Disease Activity Score; EULAR, European League Against Rheumatism; ITT, intent to treat.

[1] Percentage calculated based on ITT Population


Statistical Analysis Plan for Interim and Primary Analyses in SPM-020 (The RESET-RA Study)



Doc# CLP-004 Rev D, 15JUL2024

Variable Treatment Control (N=xxx) (N=xxx)

- [3] EULAR good treatment response if DAS28-CRP score reduced from baseline to a given timepoint by > 1.2 and is ≤ 3.2 at a given timepoint
- [4] EULAR moderate treatment response if DAS28-CRP score reduced from baseline to a given timepoint by > 0.6 to ≤ 1.2, and is ≤ 5.1 at a given timepoint; or DAS28-CRP score reduced from baseline to a given timepoint by > 1.2, and is > 3.2 at a given timepoint

Reference: Listing 16.x.x.x

SOURCE: xxxxx SAS 9.4 {program location} {run date/time}}


<sup>[2]</sup> Difference in mean score change from baseline and one-sided p-value based on the Mixed-effect Model Repeated Measure model with PROC MIXED. Difference in proportions and one-sided p-value based on the Cochran-Mantel-Haenszel test. Stratification factors are inadequate response or loss of response to JAKi and RA disease severity at Day 0 for Stage 1 subjects and RA disease severity at Day 0 and inadequate response or loss of response to  $\geq$  4 biological DMARDs with  $\geq$  2 mechanisms of action for Stage 2 subjects.



Table 14.1.2.12 CDAI (ITT Population)

| | Treatment | Control |
|----------------------------|----------------|----------------|
| CD LLC | (N=xxx) | (N=xxx) |
| CDAI Score | | |
| Screening (baseline) | | |
| N[1] | xx (xx.x%) | xx (xx.x%) |
| Mean (SD) | xxx.x (xxx.xx) | xxx.x (xxx.xx) |
| Median | XXX.XX | XXX,XX |
| Min-Max | xxx.x - xxx.x | xxx.x - xxx.x |
| Day 0 | | |
| N[1] | xx (xx.x%) | xx (xx.x%) |
| Mean (SD) | xxx.x (xxx.xx) | xxx.x (xxx.xx) |
| Median | xxx.xx | xxx.xx |
| Min-Max | xxx.x - xxx.x | xxx.x - xxx.x |
| Change from baseline | | |
| N[1] | xx (xx.x%) | xx (xx.x%) |
| Mean (SD) | xxx.x (xxx.xx) | xxx.x (xxx.xx) |
| Median | xxx.xx | xxx.xx |
| Min-Max | xxx.x - xxx.x | xxx.x - xxx.x |
| 95% CI for difference [2] | (xx.x, xx.x) | |
| p-value for difference [2] | 0.xxx | |
| Week 4 | | |
| N[1] | xx (xx.x%) | xx (xx.x%) |
| Mean (SD) | xxx.x (xxx.xx) | xxx.x (xxx.xx) |
| Median | xxx.xx | xxx.xx |
| Min-Max | xxx.x - xxx.x | xxx.x - xxx.x |
| Change from baseline | | |
| N[1] | xx (xx.x%) | xx (xx.x%) |
| Mean (SD) | xxx.x (xxx.xx) | xxx.x (xxx.xx) |
| Median | XXX.XX | XXX.XX |
| Min-Max | xxx.x – xxx.x | xxx.x - xxx.x |


## Doc# CLP-004 Rev D, 15JUL2024

| | Treatment | Control |
|---|---|---|
| 050/ CI for difference [2] | (N=xxx) | (N=xxx) |
| 95% CI for difference [2] | (xx.x, xx.x) | |
| p-value for difference [2] | 0.xxx | |
| Week 8 | | |
| N[1] | xx (xx.x%) | xx (xx.x%) |
| Mean (SD) | xxx.x (xxx.xx) | xxx.x (xxx.xx) |
| Median | XXX.XX | XXX,XX |
| Min-Max | xxx.x - xxx.x | xxx.x - xxx.x |
| Change from baseline | | |
| N[1] | xx (xx.x%) | xx (xx.x%) |
| Mean (SD) | xxx.x (xxx.xx) | xxx.x (xxx.xx) |
| Median | XXX.XX | xxx.xx |
| Min-Max | xxx.x - xxx.x | xxx.x - xxx.x |
| 95% CI for difference [2] | (xx.x, xx.x) | |
| p-value for difference [2] | 0.xxx | |
| Week 12 | | |
| N[1] | xx (xx.x%) | xx (xx.x%) |
| Mean (SD) | xxx.x (xxx.xx) | xxx.x (xxx.xx) |
| Median | xxx.xx | xxx.xx |
| Min-Max | xxx.x - xxx.x | xxx.x - xxx.x |
| Change from baseline | | |
| N[1] | xx (xx.x%) | xx (xx.x%) |
| Mean (SD) | xxx.x (xxx.xx) | xxx.x (xxx.xx) |
| Median | xxx.xx | xxx.xx |
| Min-Max | xxx.x - xxx.x | xxx.x - xxx.x |
| 95% CI for difference [2] | (xx.x, xx.x) | |
| p-value for difference [2] | 0.xxx | |
| OAI Low Disease Activity (Score >2.8 to ≤10) [1] | | |
| Screning (baseline) | | |
| N[1] | xx | xx |
| Yes | xx (xx.x%) | xx (xx.x%) |
| Difference [2] | xx.x% | AA (AAA/0) |
| | nact/V | |


### Doc# CLP-004 Rev D, 15JUL2024

| | Treatment | Control |
|---------------------------------------|--------------|------------|
| | (N=xxx) | (N=xxx) |
| 95% CI for difference | (xx.x, xx.x) | |
| p-value for difference [2] | 0.xxx | |
| Week 12 | | |
| N[1] | XX | XX |
| Yes | xx (xx.x%) | xx (xx.x%) |
| Difference [2] | xx.x% | |
| 95% CI for difference [2] | (xx.x, xx.x) | |
| p-value for difference [2] | 0.xxx | |
| CDAI Remission (Score 0 to ≤ 2.8) [1] | | |
| Screening (baseline) | | |
| N[1] | XX | XX |
| Yes | xx (xx.x%) | xx (xx.x%) |
| Difference [2] | xx.x% | |
| 95% CI for difference [2] | (xx.x, xx.x) | |
| p-value for difference [2] | 0.xxx | |
| Week 12 | | |
| N[1] | XX | XX |
| Yes | xx (xx.x%) | xx (xx,x%) |
| Difference [2] | xx.x% | |
| 95% CI for difference [2] | (xx.x, xx.x) | |
| p-value for difference [2] | 0.xxx | |
| CDAI Response (MCID) [1][3] | | |
| Week 12 | | |
| N[1] | xx | XX |
| Yes | xx (xx.x%) | xx (xx,x%) |
| Difference [2] | xx.x% | |
| 95% CI for difference [2] | (xx.x, xx.x) | |
| p-value for difference [2] | 0.xxx | |

Abbreviations: CDAI, Clinical Disease Activity Index; ITT, intent to treat; MCID, Minimal clinically important difference.


<sup>[1]</sup> Percentage calculated based on ITT Population.

<sup>[2]</sup> Difference in mean score change from baseline and one-sided p-value based on the Mixed-effect Model Repeated Measure model with PROC MIXED. Difference in proportions and one-sided p-value based on the Cochran-Mantel-Haenszel test. Stratification factors are inadequate response or loss of response to JAKi and RA disease

## Statistical Analysis Plan for Interim and Primary Analyses in SPM-020 (The RESET-RA Study)



Doc# CLP-004 Rev D, 15JUL2024

| associate at Day O for Stock 1 subjects and DA disease associate at Day O and inclosurate representation of representation A bio- | logical DMADDs with > 2 m | a salamiama af |
|---|---|---|
| | (N=xxx) | (N=xxx) |
| | Treatment | Control |

severity at Day 0 for Stage 1 subjects and RA disease severity at Day 0 and inadequate response or loss of response to ≥ 4 biological DMARDs with ≥ 2 mechanisms of action for Stage 2 subjects.

[3] MCID is -12 if starting in high disease (> 22), -6 if starting in moderate disease (10-22); and 1 if starting in low disease (< 10).CDAI ranges from 0 to 76 with higher values representing higher disease activity.

Reference: Listing 16.x.x.x

SOURCE: xxxxx SAS 9.4 {program location} {run date/time}}




Table 14.1.2.13 RAMRIS (ITT Population)

| Variable | Treatment<br>(N=xxx) | Control<br>(N=xxx) |
|---|---|---|
| RAMRIS Bone Erosion Score | (14-333) | (11-111) |
| Screening (baseline) | | |
| N[1] | xx (xx.x%) | xx (xx.x%) |
| Mean (SD) | xxx.x (xxx.xx) | xxx.x (xxx.xx) |
| Median | xxx.xx | xxx.xx |
| Min-Max | xxx.x - xxx.x | xxx.x - xxx.x |
| Week 12 | | |
| N[1] | xx (xx.x%) | xx (xx.x%) |
| Mean (SD) | xxx.x (xxx.xx) | xxx.x (xxx.xx) |
| Median | xxx.xx | xxx.xx |
| Min-Max | xxx.x - xxx.x | xxx.x - xxx.x |
| Change from baseline (SDC: x.xx) | | |
| N[1] | xx (xx.x%) | xx (xx.x%) |
| Mean (SD) | xxx.x (xxx.xx) | xxx.x (xxx.xx) |
| Median | xxx.xx | xxx.xx |
| Min-Max | xxx.x - xxx.x | xxx.x - xxx.x |
| 95% CI for difference [2] | (xx.x, xx.x) | |
| p-value for difference [2] | 0.xxx | |
| Progression rate from baseline (> 0.5) | | |
| N[1] | XX | XX |
| Yes | xx (xx.x%) | xx (xx.x%) |
| Difference [2] | xx.x% | |
| 95% CI for difference [2] | (xx.x, xx.x) | |
| p-value for difference [2] | 0.xxx | |
| RAMRIS Osteitis Score | | |
| Screening (baseline) | | |
| N[1] | xx (xx.x%) | xx (xx.x%) |
| Mean (SD) | xxx.x (xxx.xx) | xxx.x (xxx.xx) |


## Doc# CLP-004 Rev D, 15JUL2024

| Variable | Treatment<br>(N=xxx) | Control<br>(N=xxx) |
|----------------------------------|----------------------|--------------------|
| Median | xxx.xx | xxx.xx |
| Min-Max | xxx.x - xxx.x | xxx.x - xxx.x |
| Week 12 | | |
| N[1] | xx (xx.x%) | xx (xx.x%) |
| Mean (SD) | xxx.x (xxx.xx) | xxx.x (xxx.xx |
| Median | xxx.xx | xxx,xx |
| Min-Max | xxx.x - xxx.x | xxx.x - xxx.x |
| Change from baseline (SDC: x.xx) | | |
| N[1] | xx (xx.x%) | xx (xx.x%) |
| Mean (SD) | xxx.x (xxx.xx) | xxx.x (xxx.xx |
| Median | xxx.xx | xxx.xx |
| Min-Max | xxx.x - xxx.x | xxx.x - xxx.x |
| 95% CI for difference [2] | (xx.x, xx.x) | |
| p-value for difference [2] | 0.xxx | |
| RAMRIS Synovitis Score | | |
| Screening (baseline) | | |
| N[1] | xx (xx.x%) | xx (xx,x%) |
| Mean (SD) | xxx.x (xxx.xx) | xxx.x (xxx.xx |
| Median | XXX,XX | XXX.XX |
| Min-Max | xxx.x - xxx.x | xxx.x - xxx.x |
| Week 12 | | |
| N[1] | xx (xx.x%) | xx (xx.x%) |
| Mean (SD) | xxx.x (xxx.xx) | xxx,x (xxx,xx |
| Median | xxx.xx | XXX,XX |
| Min-Max | xxx.x - xxx.x | xxx.x - xxx.x |
| Change from baseline (SDC: x.xx) | | |
| N[1] | xx (xx.x%) | xx (xx.x%) |
| Mean (SD) | xxx.x (xxx.xx) | xxx.x (xxx.xx |
| Median | xxx.xx | xxx.xx |
| Min-Max | xxx.x - xxx.x | xxx.x - xxx.x |
| 95% CI for difference [2] | (xx.x, xx.x) | |




| Variable | Treatment | Control |
|----------------------------------|----------------|----------------|
| | (N=xxx) | (N=xxx) |
| p-value for difference [2] | 0.xxx | |
| RAMRIS CARLOS Score | | |
| Screening (baseline) | | |
| N[1] | xx (xx.x%) | xx (xx.x%) |
| Mean (SD) | xxx.x (xxx.xx) | xxx.x (xxx.xx) |
| Median | xxx.xx | XXX.XX |
| Min-Max | xxx.x - xxx.x | xxx.x - xxx.x |
| Week 12 | | |
| N[1] | xx (xx.x%) | xx (xx.x%) |
| Mean (SD) | xxx.x (xxx.xx) | xxx.x (xxx.xx) |
| Median | XXX.XX | XXX.XX |
| Min-Max | xxx.x - xxx.x | xxx.x - xxx.x |
| Change from baseline (SDC: x.xx) | | |
| N[1] | xx (xx.x%) | xx (xx.x%) |
| Mean (SD) | xxx.x (xxx.xx) | xxx.x (xxx.xx) |
| Median | xxx.xx | xxx.xx |
| Min-Max | xxx.x - xxx.x | xxx.x - xxx.x |
| 95% CI for difference [2] | (xx.x, xx.x) | |
| p-value for difference [2] | 0.xxx | |

Abbreviations: CARLOS, cartilage loss score; ITT, intent to treat; RAMRIS, Rheumatoid Arthritis MRI Scoring System; SDC, Smallest Detectable Change

Reference: Listing 16.x.x.x

SOURCE: xxxxx SAS 9.4 {program location} {run date/time}}


<sup>[1]</sup> Percentage calculated based on ITT Population.

<sup>[2]</sup> Difference in mean score change from baseline and one-sided p-value based on the Mixed-effect Model Repeated Measure model with PROC MIXED. Difference in proportions and one-sided p-value based on the Cochran-Mantel-Haenszel test. Stratification factors are inadequate response or loss of response to JAKi and RA disease severity at Day 0 for Stage 1 subjects and RA disease severity at Day 0 and inadequate response or loss of response to  $\geq$  4 biological DMARDs with  $\geq$  2 mechanisms of action for Stage 2 subjects.



Table 14.1.2.14 EQ-5D-5L (ITT Population)

| Variable | Treatment (N=xxx) | Control<br>(N=xxx) |
|----------------------------|-------------------|--------------------|
| EQ-5D-5L Index Score | (11 444) | (11 222) |
| Screening (baseline) | | |
| N[1] | xx (xx.x%) | xx (xx.x%) |
| Mean (SD) | xxx.x (xxx.xx) | xxx.x (xxx.xx) |
| Median | xxx.xx | xxx.xx |
| Min-Max | xxx.x - xxx.x | xxx.x-xxx.x |
| Day 0 | | |
| N[1] | xx (xx.x%) | xx (xx.x%) |
| Mean (SD) | xxx.x (xxx.xx) | xxx.x (xxx.xx) |
| Median | xxx.xx | xxx,xx |
| Min-Max | xxx.x - xxx.x | xxx.x-xxx.x |
| Change from baseline | | |
| N[1] | xx (xx.x%) | xx (xx.x%) |
| Mean (SD) | xxx.x (xxx.xx) | xxx.x (xxx.xx) |
| Median | xxx.xx | xxx,xx |
| Min-Max | xxx.x - xxx.x | xxx,x-xxx,x |
| Difference [2] | xx (xx.x%) | |
| 95% CI for difference [2] | (xx.x, xx.x) | |
| p-value for difference [2] | 0.xxx | |
| Week 4 | | |
| N[1] | xx (xx.x%) | xx (xx.x%) |
| Mean (SD) | xxx.x (xxx.xx) | xxx.x (xxx.xx) |
| Median | xxx.xx | xxx,xx |
| Min-Max | xxx.x - xxx.x | xxx.x-xxx.x |
| Change from baseline | | |
| N[1] | xx (xx.x%) | xx (xx.x%) |
| Mean (SD) | xxx.x (xxx.xx) | xxx.x (xxx.xx) |
| Median | xxx.xx | xxx.xx |


## Doc# CLP-004 Rev D, 15JUL2024

| ariable | Treatment | Control |
|-------------------------------|----------------|-----------------|
| | (N=xxx) | (N=xxx) |
| Min-Max | xxx.x - xxx.x | xxx.x - xxx.x |
| Difference [2] | xx (xx.x%) | |
| 95% CI for difference [2] | (xx.x, xx.x) | |
| p-value for difference [2] | 0.xxx | |
| Week 8 | | |
| N[1] | xx (xx.x%) | xx (xx.x%) |
| Mean (SD) | xxx.x (xxx.xx) | xxx.x (xxx.xx) |
| Median | xxx.xx | XXX.XX |
| Min-Max | xxx.x - xxx.x | xxx.x-xxx.x |
| Change from baseline | | |
| N[1] | xx (xx.x%) | xx (xx.x%) |
| Mean (SD) | xxx.x (xxx.xx) | xxx.x (xxx.xx) |
| Median | xxx.xx | xxx.xx |
| Min-Max | xxx.x - xxx.x | xxx.x-xxx.x |
| Difference [2] | xx (xx.x%) | |
| 95% CI for difference [2] | (xx.x, xx.x) | |
| p-value for difference [2] | 0.xxx | |
| Week 12 | | |
| N[1] | xx (xx.x%) | xx (xx.x%) |
| Mean (SD) | xxx.x (xxx.xx) | xxx.x (xxx.xx |
| Median | xxx.xx | xxx.xx |
| Min-Max | xxx.x - xxx.x | xxx, x - xxx, x |
| Change from baseline | | |
| N[1] | xx (xx.x%) | xx (xx.x%) |
| Mean (SD) | xxx.x (xxx.xx) | xxx.x (xxx.xx |
| Median | xxx.xx | xxx.xx |
| Min-Max | xxx.x - xxx.x | xxx.x-xxx.x |
| Difference [2] | xx (xx.x%) | |
| 95% CI for difference [2] | (xx.x, xx.x) | |
| p-value for difference [2] | 0.xxx | |
| -5D-5L Mobility Dimension [1] | | |


## Doc# CLP-004 Rev D, 15JUL2024

| Variable | Treatment | Control |
|---|---|---|
| | (N=xxx) | (N=xxx) |
| Screening (baseline) | | |
| Level 1 (No problem) | xx (xx.x%) | xx (xx.x%) |
| Level 2 (Slight problems) | xx (xx.x%) | xx (xx.x%) |
| Level 3 (Moderate problems) | xx (xx.x%) | xx (xx.x%) |
| Level 4 (Severe problems) | xx (xx.x%) | xx (xx.x%) |
| Level 5 (Extreme problems) | xx (xx.x%) | xx (xx.x%) |
| Repeat each level for. Day 0, Week 4, Week 8, and Week 12 | | |
| Repeat for other dimensions: | | |
| EQ-5D-5L Self-care | | |
| EQ-5D-5L Usual activities | | |
| EQ-5D-5L Pain/discomfort | | |
| EQ-5D-5L Anxiety/depression | | |
| EQ VAS | | |
| Screening (baseline) | | |
| N[1] | xx (xx.x%) | xx (xx.x%) |
| Mean (SD) | xxx.x (xxx.xx) | xxx.x (xxx.xx) |
| Median | xxx.xx | XXX.XX |
| Min-Max | xxx.x - xxx.x | xxx.x-xxx.x |
| Day 0 | | |
| N[1] | xx (xx.x%) | xx (xx.x%) |
| Mean (SD) | xxx.x (xxx.xx) | xxx.x (xxx.xx) |
| Median | XXX.XX | XXX.XX |
| Min-Max | xxx.x – xxx.x | xxx.x-xxx.x |
| Change from baseline | | |
| N[1] | xx (xx.x%) | xx (xx.x%) |
| Mean (SD) | xxx.x (xxx.xx) | xxx.x (xxx.xx) |
| Median | XXX.XX | XXX.XX |
| Min-Max | | XXX.XX<br>XXX.X – XXX.X |
| Difference [2] | xxx.x – xxx.x<br>xx (xx.x%) | $\lambda \lambda \lambda, \lambda - \lambda \lambda \lambda, \lambda$ |
| 95% CI for difference [2] | | |
| | (xx.x, xx.x) | |
| p-value for difference [2] | 0.xxx | |


## Doc# CLP-004 Rev D, 15JUL2024

| ariable | Treatment (N=xxx) | Control<br>(N=xxx) |
|----------------------------|-------------------|--------------------|
| Week 4 | | |
| N[1] | xx (xx.x%) | xx (xx.x%) |
| Mean (SD) | xxx.x (xxx.xx) | xxx.x (xxx.xx) |
| Median | xxx.xx | xxx.xx |
| Min-Max | xxx.x - xxx.x | xxx.x-xxx.x |
| Change from baseline | | |
| N[1] | xx (xx.x%) | xx (xx,x%) |
| Mean (SD) | xxx.x (xxx.xx) | xxx.x (xxx.xx) |
| Median | xxx.xx | xxx.xx |
| Min-Max | xxx.x - xxx.x | xxx.x - xxx.x |
| Difference [2] | xx (xx.x%) | |
| 95% CI for difference [2] | (xx.x, xx.x) | |
| p-value for difference [2] | 0.xxx | |
| Week 8 | | |
| N[1] | xx (xx.x%) | xx (xx.x%) |
| Mean (SD) | xxx.x (xxx.xx) | xxx.x (xxx.xx) |
| Median | xxx.xx | xxx.xx |
| Min-Max | xxx.x - xxx.x | xxx,x-xxx,x |
| Change from baseline | | |
| N[1] | xx (xx.x%) | xx (xx.x%) |
| Mean (SD) | xxx.x (xxx.xx) | xxx.x (xxx.xx) |
| Median | xxx.xx | xxx.xx |
| Min-Max | xxx.x - xxx.x | xxx.x - xxx.x |
| Difference [2] | xx (xx.x%) | |
| 95% CI for difference [2] | (xx.x, xx.x) | |
| p-value for difference [2] | 0.xxx | |
| Week 12 | | |
| N[1] | xx (xx.x%) | xx (xx.x%) |
| Mean (SD) | xxx.x (xxx.xx) | xxx.x (xxx.xx) |
| Median | XXX.XX | xxx.xx |
| Min-Max | xxx.x - xxx.x | xxx.x-xxx.x |


## Statistical Analysis Plan for Interim and Primary Analyses in SPM-020 (The RESET-RA Study)



### Doc# CLP-004 Rev D, 15JUL2024

| ariable | Treatment (N=xxx) | Control<br>(N=xxx) |
|----------------------------|-------------------|--------------------|
| Change from baseline | | |
| N[1] | xx (xx.x%) | xx (xx.x%) |
| Mean (SD) | xxx.x (xxx.xx) | xxx.x (xxx.xx) |
| Median | xxx.xx | XXX,XX |
| Min-Max | xxx.x - xxx.x | xxx.x-xxx.x |
| Difference [2] | xx (xx.x%) | |
| 95% CI for difference [2] | (xx.x, xx.x) | |
| p-value for difference [2] | 0.xxx | |

Abbreviations: EQ-5D-5L, EuroQol 5 domains 5 levels; ITT, intent to treat.

Reference: Listing 16.x.x.x

SOURCE: xxxxx SAS 9.4 {program location} {run date/time}}


<sup>[1]</sup> Percentage calculated based on ITT Population

<sup>[2]</sup> Difference in mean score change from baseline and one-sided p-value based on the Mixed-effect Model Repeated Measure model with PROC MIXED. Stratification factors are inadequate response or loss of response to JAKi and RA disease severity at Day 0 for Stage 1 subjects and RA disease severity at Day 0 and inadequate response or loss of response to ≥ 4 biological DMARDs with ≥ 2 mechanisms of action for Stage 2 subjects.



Table 14.1.2.15 SF-36 (ITT Population)

| Variable | Treatment | Control |
|----------------------------|----------------|----------------|
| | (N=xxx) | (N=xxx) |
| SF-36 MCS Score | | |
| Screening (baseline) | | |
| N[1] | xx (xx.x%) | xx (xx,x%) |
| Mean (SD) | xxx.x (xxx.xx) | xxx,x (xxx,xx) |
| Median | xxx.xx | xxx,xx |
| Min-Max | xxx.x - xxx.x | xxx.x - xxx.x |
| Day 0 | | |
| N[1] | xx (xx.x%) | xx (xx,x%) |
| Mean (SD) | xxx.x (xxx.xx) | xxx.x (xxx.xx) |
| Median | XXX.XX | XXX.XX |
| Min-Max | xxx.x - xxx.x | xxx.x - xxx.x |
| Change from baseline | | |
| N[1] | xx (xx.x%) | xx (xx.x%) |
| Mean (SD) | xxx.x (xxx.xx) | xxx.x (xxx.xx) |
| Median | xxx.xx | xxx.xx |
| Min-Max | xxx.x - xxx.x | xxx.x - xxx.x |
| 95% CI for difference [2] | (xx.x, xx.x) | |
| p-value for difference [2] | 0.xxx | |
| Week 4 | | |
| N[1] | xx (xx.x%) | xx (xx.x%) |
| Mean (SD) | xxx.x (xxx.xx) | xxx.x (xxx.xx) |
| Median | xxx.xx | xxx.xx |
| Min-Max | xxx.x - xxx.x | xxx.x - xxx.x |
| Change from baseline | | |
| N[1] | xx (xx.x%) | xx (xx.x%) |
| Mean (SD) | xxx.x (xxx.xx) | xxx.x (xxx.xx) |
| Median | xxx.xx | xxx.xx |
| Min-Max | xxx.x - xxx.x | xxx.x - xxx.x |


### Doc# CLP-004 Rev D, 15JUL2024

| Variable | Treatment (N=xxx) | Control<br>(N=xxx) |
|----------------------------|-------------------|--------------------|
| 95% CI for difference [2] | (xx.x, xx.x) | (11-111) |
| p-value for difference [2] | 0.xxx | |
| Week 8 | | |
| N[1] | xx (xx.x%) | xx (xx,x%) |
| Mean (SD) | xxx.x (xxx.xx) | xxx,x (xxx,xx) |
| Median | xxx.xx | XXX,XX |
| Min-Max | xxx.x - xxx.x | xxx.x - xxx.x |
| Change from baseline | | |
| N[1] | xx (xx.x%) | xx (xx.x%) |
| Mean (SD) | xxx.x (xxx.xx) | xxx.x (xxx.xx) |
| Median | xxx.xx | XXX,XX |
| Min-Max | xxx.x - xxx.x | xxx.x - xxx.x |
| 95% CI for difference [2] | (xx.x, xx.x) | |
| p-value for difference [2] | 0.xxx | |
| Week 12 | | |
| N[1] | xx (xx.x%) | xx (xx.x%) |
| Mean (SD) | xxx.x (xxx.xx) | xxx.x (xxx.xx) |
| Median | xxx.xx | xxx.xx |
| Min-Max | xxx.x - xxx.x | xxx.x - xxx.x |
| Change from baseline | | |
| N[1] | xx (xx.x%) | xx (xx.x%) |
| Mean (SD) | xxx.x (xxx.xx) | xxx.x (xxx.xx) |
| Median | xxx.xx | XXX.XX |
| Min-Max | xxx.x - xxx.x | xxx.x - xxx.x |
| 95% CI for difference [2] | (xx.x, xx.x) | |
| p-value for difference [2] | 0.xxx | |
| Repeat for: | | |
| SF-36 PCS Score | | |

Abbreviations: ITT, intent to treat; MCS, Mental Component Summary; PCS, Physical Component Summary; SF-36, Short Form Survey with 36 items.

[1] Percentage calculated based on ITT Population



Doc# CLP-004 Rev D, 15JUL2024

Variable Treatment Control (N=xxx) (N=xxx)

[2] Difference in mean score change from baseline and one-sided p-value based on the Mixed-effect Model Repeated Measure model with PROC MIXED. Stratification factors are inadequate response or loss of response to JAKi and RA disease severity at Day 0 for Stage 1 subjects and RA disease severity at Day 0 and inadequate response or loss of response to ≥ 4 biological DMARDs with ≥ 2 mechanisms of action for Stage 2 subjects.

Reference: Listing 16.x.x.x

SOURCE: xxxxx SAS 9.4 {program location} {run date/time}}


Doc# CLP-004 Rev D, 15JUL2024



### Table 14.1.2.16 Subject's Blinding Assessment (ITT Population)

| | | BI | | | | |
|---|---|---|---|---|---|---|
| Assignment | Treatment | Treatment | Control | Control | | |
| Assignment | Strongly Believe | Somewhat Believe | Somewhat Believe | Strongly Believe | Don't Know | (95% CI) |
| Week 4 | | | | | | |
| Treatment | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | 0.xx(0.xx, 0.xx) |
| Control | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | 0.xx(0.xx, 0.xx) |
| Week 12 | | | | | | |
| Treatment | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | 0.xx(0.xx, 0.xx) |
| Control | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | 0.xx(0.xx, 0.xx) |

Abbreviations: BI, Bang's blinding index; ITT, intent to treat.

Reference: Listing 16.x.x.x

SOURCE: xxxxx SAS 9.4 {program location} {run date/time}}

Table 14.1.2.16.1 Subject's Blinding Assessment (PTE Population)

Repeat Table 14.2.16 for PTE population


Doc# CLP-004 Rev D, 15JUL2024



### Table 14.1.2.17 Joint Evaluator's Blinding Assessment (ITT Population)

| | | BI | | | | |
|---|---|---|---|---|---|---|
| Assisanment | Treatment | Treatment | Control | Control | | _ |
| Assignment | Strongly Believe | Somewhat Believe | Somewhat Believe | Strongly Believe | Don't Know | (95% CI) |
| Week 4 | | | | | | |
| Treatment | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | 0.xx(0.xx, 0.xx) |
| Control | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | 0.xx(0.xx, 0.xx) |
| Week 12 | | | | | | |
| Treatment | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | 0.xx(0.xx, 0.xx) |
| Control | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | 0.xx(0.xx, 0.xx) |

Abbreviations: BI, Bang's blinding index; ITT, intent to treat.

Reference: Listing 16.x.x.x

SOURCE: xxxxx SAS 9.4 {program location} {run date/time}}

Table 14.1.2.17.1 Evaluator's Blinding Assessment (PTE Population)

Repeat Table 14.2.17 for PTE population






Table 14.1.2.18 Co-PI Rheumatologist's Blinding Assessment (ITT Population)

| | Co-PI Rheumatologist believes subject is in | | | | | |
|---|---|---|---|---|---|---|
| Assissment | Treatment | Treatment | Control | Control | | _ |
| Assignment | Strongly Believe | Somewhat Believe | Somewhat Believe | Strongly Believe | Don't Know | (95% CI) |
| Week 4 | | | | | | |
| Treatment | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | 0.xx(0.xx, 0.xx) |
| Control | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | 0.xx(0.xx, 0.xx) |
| Week 12 | | | | | | |
| Treatment | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | 0.xx(0.xx, 0.xx) |
| Control | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | 0.xx(0.xx, 0.xx) |

Abbreviations: BI, Bang's blinding index; ITT, intent to treat.

Reference: Listing 16.x.x.x

SOURCE: xxxxx SAS 9.4 {program location} {run date/time}}

Table 14.1.2.18.1 Co-PI Rheumatologist's Blinding Assessment (PTE Population)

Repeat Table 14.2.18 for PTE population


Doc# CLP-004 Rev D, 15JUL2024



### Table 14.1.2.19 Inflammatory Biomarkers (ITT Population)

| 'ariable | Treatment (N=xxx) | Control<br>(N=xxx) |
|----------------------|-------------------|--------------------|
| L-6 (pg/mL) | (11-111) | (14-222) |
| Screening (baseline) | | |
| N[1] | xx (xx.x%) | xx (xx.x%) |
| Mean (SD) | xxx.x (xxx.xx) | xxx.x (xxx.xx) |
| Median | xxx.xx | xxx.xx |
| Min-Max | xxx.x - xxx.x | xxx.x - xxx.x |
| Day 0 | | |
| N[1] | xx (xx.x%) | xx (xx.x%) |
| Mean (SD) | xxx.x (xxx.xx) | xxx.x (xxx.xx) |
| Median | xxx.xx | xxx.xx |
| Min-Max | xxx.x - xxx.x | xxx.x - xxx.x |
| Week 4 | | |
| N[1] | xx (xx.x%) | xx (xx.x%) |
| Mean (SD) | xxx.x (xxx.xx) | xxx.x (xxx.xx) |
| Median | XXX.XX | xxx.xx |
| Min-Max | xxx.x - xxx.x | xxx.x - xxx.x |
| Week 8 | | |
| N[1] | xx (xx.x%) | xx (xx.x%) |
| Mean (SD) | xxx.x (xxx.xx) | xxx.x (xxx.xx) |
| Median | XXX.XX | xxx.xx |
| Min-Max | xxx.x - xxx.x | xxx.x - xxx.x |
| Week 12 | | |
| N[1] | xx (xx.x%) | xx (xx.x%) |
| Mean (SD) | xxx.x (xxx.xx) | xxx.x (xxx.xx) |
| | xxx.xx | xxx.xx |
| Median | | xxx.x - xxx.x |




#### Doc# CLP-004 Rev D, 15JUL2024

| Variable | Treatment | Control |
|----------------------------|----------------|----------------|
| variable | (N=xxx) | (N=xxx) |
| N[1] | xx (xx.x%) | xx (xx,x%) |
| Mean (SD) | xxx.x (xxx.xx) | xxx.x (xxx.xx) |
| Median | XXX.XX | xxx.xx |
| Min-Max | xxx.x - xxx.x | xxx.x - xxx.x |
| Percent change | xx.x% | xx.x% |
| Relative difference [2] | xx.x% | |
| 95% CI for difference [2] | (xx.x%, xx.x%) | |
| p-value for difference [2] | 0.xxx | |

Repeat for: SAA (µg/mL) MMP-3 (pg/mL)

Abbreviations: IL, interleukin; ITT, intent to treat; MMP, matrix metalloproteinase; SAA, serum amyloid A.

[1] Percentage calculated based on ITT Population.

[2] Relative difference in mean score change from baseline and one-sided p-value based on the Mixed-effect Model Repeated Measure model with PROC MIXED. Stratification factors are inadequate response or loss of response to JAKi and RA disease severity at Day 0 for Stage 1 subjects and RA disease severity at Day 0 and inadequate response or loss of response to ≥ 4 biological DMARDs with ≥ 2 mechanisms of action for Stage 2 subjects.

Reference: Listing 16.x.x.x

SOURCE: xxxxx SAS 9.4 {program location} {run date/time}}


Doc# CLP-004 Rev D, 15JUL2024



# Table 14.1.2.20 RA Rescue Treatments and Follow-up Interventions (ITT Population)

| | Treatment | Control |
|---|---|---|
| | (N=xxx) | (N=xxx) |
| Received any post-procedure RA rescue treatment | | |
| Yes [1] | xxx (xx.x%) | xxx (xx.x%) |
| If yes, first noted at [2] | xxx (xx.x%) | xxx (xx.x%) |
| Post-Surgical Clearance | xxx (xx.x%) | xxx (xx.x%) |
| Day 0 | xxx (xx.x%) | xxx (xx.x%) |
| Titration 1 | xxx (xx.x%) | xxx (xx.x%) |
| Titration 2 | xxx (xx.x%) | xxx (xx.x%) |
| Titration 3 | xxx (xx.x%) | xxx (xx.x%) |
| Week 4 | xxx (xx.x%) | xxx (xx.x%) |
| Week 8 | xxx (xx.x%) | xxx (xx.x%) |
| Week 12 | xxx (xx.x%) | xxx (xx.x%) |
| Received csDMARD for RA (other than 1 at stable dose from Informed Consent to Week 12, as required per protocol) [1] | | |
| Yes [1] | xxx (xx.x%) | xxx (xx.x%) |
| If yes, first noted at [2] | xxx (xx.x%) | xxx (xx.x%) |
| Post-Surgical Clearance | xxx (xx.x%) | xxx (xx.x%) |
| Day 0 | xxx (xx.x%) | xxx (xx.x%) |
| Titration 1 | xxx (xx.x%) | xxx (xx.x%) |
| Titration 2 | xxx (xx.x%) | xxx (xx.x%) |
| Titration 3 | xxx (xx.x%) | xxx (xx.x%) |
| Week 4 | xxx (xx.x%) | xxx (xx.x%) |
| Week 8 | xxx (xx.x%) | xxx (xx.x%) |
| Week 12 | xxx (xx.x%) | xxx (xx.x%) |
| Received b/tsDMARDs for RA [1] | | |
| Yes [1] | xxx (xx.x%) | xxx (xx.x%) |
| If yes, first noted at [2] | xxx (xx.x%) | xxx (xx.x%) |
| Post-Surgical Clearance | xxx (xx.x%) | xxx (xx.x%) |
| Day 0 | xxx (xx.x%) | xxx (xx.x%) |
| Titration 1 | xxx (xx.x%) | xxx (xx.x%) |
| Titration 2 | xxx (xx.x%) | xxx (xx.x%) |
| THAUOH Z | XXX (XX.X70) | XXX (XX.X70) |




### Doc# CLP-004 Rev D, 15JUL2024

| | Treatment | Control |
|---|---|---|
| | (N=xxx) | (N=xxx) |
| Titration 3 | xxx (xx.x%) | xxx (xx.x%) |
| Week 4 | xxx (xx.x%) | xxx (xx.x%) |
| Week 8 | xxx (xx.x%) | xxx (xx,x%) |
| Week 12 | xxx (xx.x%) | xxx (xx.x%) |
| deceived corticosteroids (equivalent >10mg/day average dose prednisone) for RA [1] | | |
| Yes [1] | xxx (xx.x%) | xxx (xx.x%) |
| If yes, first noted at [2] | xxx (xx.x%) | xxx (xx.x%) |
| Post-Surgical Clearance | xxx (xx.x%) | xxx (xx.x%) |
| Baseline | xxx (xx.x%) | xxx (xx.x%) |
| Titration 1 | xxx (xx.x%) | xxx (xx.x%) |
| Titration 2 | xxx (xx.x%) | xxx (xx.x%) |
| Titration 3 | xxx (xx.x%) | xxx (xx.x%) |
| Week 4 | xxx (xx.x%) | xxx (xx.x%) |
| Week 8 | xxx (xx.x%) | xxx (xx.x%) |
| Week 12 | xxx (xx.x%) | xxx (xx.x%) |

Repeat for other RA rescue treatments as reported in CRFs

Abbreviations: b/tsDMARD, biologic or targeted synthetic disease-modifying anti-rheumatic drug.

- [1] Percentage calculated based on ITT Population.
- [2] Percent is calculated based on the start date noted on the Concomitant Medication log.

Reference: Listing 16.x.x.x

SOURCE: xxxxx SAS 9.4 {program location} {run date/time}}




Table 14.1.2.22 Implant Performance (ITT Population)

| Variable | Treatment | Control | All |
|---|---|---|---|
| Status of Study Implant at Study Exit [1] | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| Subjects with active implant | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| Subjects with deactivated/decommissioned implant | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| Subjects with explanted implant | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| Unknown | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| Other | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |

[1] Percentage calculated based on ITT Population.

Reference: Listing 16.x.x.x

SOURCE: xxxxx SAS 9.4 {program location} {run date/time}


Doc# CLP-004 Rev D, 15JUL2024



Table 14.1.3.1 Adverse Events (Safety Population)

| | Treatment | Control | All |
|---|---|---|---|
| Variable | (N=xxx) | (N=xxx) | (N=xxx) |
| | Events n (%) | Events n (%) | Events n (%) |
| Any AE | xx xx (xx.x%) | xx xx (xx.x%) | xx xx (xx.x%) |
| Not Related | xx xx (xx.x%) | xx xx (xx.x%) | xx xx (xx.x%) |
| Implant Procedure | xx xx (xx.x%) | xx xx (xx.x%) | xx xx (xx.x%) |
| Implant Device | xx xx (xx.x%) | xx xx (xx.x%) | xx xx (xx.x%) |
| Stimulation | xx xx (xx.x%) | xx xx (xx.x%) | xx xx (xx.x%) |
| Explant Procedure | xx xx (xx.x%) | xx xx (xx.x%) | xx xx (xx.x%) |
| Related [1] | | | |
| Implant Procedure | xx xx (xx.x%) | xx xx (xx.x%) | xx xx (xx.x%) |
| Implant Device | xx xx (xx.x%) | xx xx (xx.x%) | xx xx (xx.x%) |
| Stimulation | xx xx (xx.x%) | xx xx (xx.x%) | xx xx (xx.x%) |
| Explant Procedure | xx xx (xx.x%) | xx xx (xx.x%) | xx xx (xx.x%) |
| Indeterminate | | | |
| Implant Procedure | xx xx (xx.x%) | xx xx (xx.x%) | xx xx (xx.x%) |
| Implant Device | xx xx (xx.x%) | xx xx (xx.x%) | xx xx (xx.x%) |
| Stimulation | xx xx (xx.x%) | xx xx (xx.x%) | xx xx (xx.x%) |
| Explant Procedure | xx xx (xx.x%) | xx xx (xx.x%) | xx xx (xx.x%) |
| AE resulting in discontinuation | xx xx (xx.x%) | xx xx (xx.x%) | xx xx (xx.x%) |
| AE by maximum severity | | | |
| Mild | xx xx (xx.x%) | xx xx (xx.x%) | xx xx (xx.x%) |
| Moderate | xx xx (xx.x%) | xx xx (xx.x%) | xx xx (xx.x%) |
| Severe | xx xx (xx.x%) | xx xx (xx.x%) | xx xx (xx.x%) |
| Implant Procedure AE by maximum severity | | | |
| Mild | xx xx (xx.x%) | xx xx (xx.x%) | xx xx (xx.x%) |
| Moderate | xx xx (xx.x%) | xx xx (xx.x%) | xx xx (xx.x%) |


# SETPOINT MEDICAL

#### Doc# CLP-004 Rev D, 15JUL2024

| | Treatment | Control | All |
|---|---|---|---|
| Variable | (N=xxx) | (N=xxx) | (N=xxx) |
| | Events n (%) | Events n (%) | Events n (%) |
| Severe | xx xx (xx.x%) | xx xx (xx.x%) | xx xx (xx.x%) |
| Implant Device AE by maximum severity | | | |
| Mild | xx xx (xx.x%) | xx xx (xx.x%) | xx xx (xx.x%) |
| Moderate | xx xx (xx.x%) | xx xx (xx.x%) | xx xx (xx.x%) |
| Severe | xx xx (xx.x%) | xx xx (xx.x%) | xx xx (xx.x%) |
| Stimulation AE by maximum severity | | | |
| Mild | xx xx (xx.x%) | xx xx (xx.x%) | xx xx (xx.x%) |
| Moderate | xx xx (xx.x%) | xx xx (xx.x%) | xx xx (xx.x%) |
| Severe | xx xx (xx.x%) | xx xx (xx.x%) | xx xx (xx.x%) |
| Explant Procedure AE by maximum severity [1] | | | |
| Mild | xx xx (xx.x%) | xx xx (xx.x%) | xx xx (xx.x%) |
| Moderate | xx xx (xx.x%) | xx xx (xx.x%) | xx xx (xx.x%) |
| Severe | xx xx (xx.x%) | xx xx (xx.x%) | xx xx (xx.x%) |
| SAE [1] | xx xx (xx.x%) | xx xx (xx.x%) | xx xx (xx.x%) |
| Implant Procedure SAE | xx xx (xx.x%) | xx xx (xx.x%) | xx xx (xx.x%) |
| Implant Device SAE | xx xx (xx.x%) | xx xx (xx.x%) | xx xx (xx.x%) |
| Stimulation SAE | xx xx (xx.x%) | xx xx (xx.x%) | xx xx (xx.x%) |
| Energizer SAE | xx xx (xx.x%) | xx xx (xx.x%) | xx xx (xx.x%) |
| Explant Procedure SAE | xx xx (xx.x%) | xx xx (xx.x%) | xx xx (xx.x%) |

Abbreviations: AE, adverse event; RA, rheumatoid arthritis; SAE, serious adverse event.

Note: AEs coded using the MedDRA dictionary Version 21.0 or later. Given in the table are subject counts and percentages. At each level of summation, subjects are counted only once. Subjects experiencing AEs of more than one severity are summarized according to the maximum severity experienced over all episodes of an AE.

[1] AEs judged to be "Definitely related" or "Probably related" are reported as "Related".

Reference: Listing 16.x.x.x

SOURCE: xxxxx SAS 9.4 {program location} {run date/time}}


Doc# CLP-004 Rev D, 15JUL2024



Table 14.1.3.2

Adverse Events by SOC and Maximum Severity: All Events
Safety Population

| | | Treat<br>(N=) | | | | Contro<br>(N=xx | | | | A<br>(N=2 | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| SOC | Mild | Moderate | Severe | Total | Mild | Moderate | Severe | Total | Mild | Moderate | Severe | Total |
| Preferred Term | Events | Events | Events | Events | Events | Events | Events | Events | Events | Events | Events | Events |
| | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) |
| Prior to Implant Procedure | | | | | | | | | | | | |
| Any AE [1] | xx | xx | xx | xx | xx | xx | xx | xx | xx | xx | xx | xx |
| | x (xx%) | x (xx%) | x (xx%) | x (xx%) | x (xx%) | x (xx%) | x (xx%) | x (xx%) | x (xx%) | x (xx%) | x (xx%) | x (xx%) |
| SOC 1 [1] | xx | xx | xx | xx | xx | xx | xx | xx | xx | xx | xx | xx |
| | x (xx%) | x (xx%) | x (xx%) | x (xx%) | x (xx%) | x (xx%) | x (xx%) | x (xx%) | x (xx%) | x (xx%) | x (xx%) | x (xx%) |
| Preferred Term 1 | XX | XX | XX | XX | XX | XX | XX | XX | XX | XX | XX | XX |
| | x (xx%) | x (xx%) | x (xx%) | x (xx%) | x (xx%) | x (xx%) | x (xx%) | x (xx%) | x (xx%) | x (xx%) | x (xx%) | x (xx%) |
| Preferred Term 2 | XX | XX | XX | XX | XX | xx | xx | XX | xx | XX | XX | xx |
| | x (xx%) | x (xx%) | x (xx%) | x (xx%) | x (xx%) | x (xx%) | x (xx%) | x (xx%) | x (xx%) | x (xx%) | x (xx%) | x (xx%) |
| Preferred Term 3 | XX | XX | XX | XX | XX | xx | xx | XX | xx | XX | XX | xx |
| | x (xx%) | x (xx%) | x (xx%) | x (xx%) | x (xx%) | x (xx%) | x (xx%) | x (xx%) | x (xx%) | x (xx%) | x (xx%) | x (xx%) |
| Preferred Term 4 | XX | XX | xx | XX | XX | xx | xx | | xx | XX | xx | xx |
| | x (xx%) | x (xx%) | x (xx%) | x (xx%) | x (xx%) | x (xx%) | x (xx%) | x (xxxx%) | x (xx%) | x (xx%) | x (xx%) | x (xx%) |
| SOC 2 [1] | xx | xx | xx | xx | xx | xx | xx | xx | xx | xx | xx | xx |
| | x (xx%) | x (xx%) | x (xx%) | x (xx%) | x (xx%) | x (xx%) | x (xx%) | x (xx%) | x (xx%) | x (xx%) | x (xx%) | x (xx%) |
| Preferred Term 1 | XX | XX | XX | XX | XX | xx | xx | XX | xx | XX | xx | xx |
| | x (xx%) | x (xx%) | x (xx%) | x (xx%) | x (xx%) | x (xx%) | x (xx%) | x (xx%) | x (xx%) | x (xx%) | x (xx%) | x (xx%) |
| Preferred Term 2 | xx | xx | xx | xx | XX | xx | xx | xx | xx | xx | xx | xx |
| | x (xx%) | x (xx%) | x (xx%) | x (xx%) | x (xx%) | x (xx%) | x (xx%) | x (xx%) | x (xx%) | x (xx%) | x (xx%) | x (xx%) |
| Preferred Term 3 | xx | xx | xx | xx | XX | xx | xx | xx | XX | xx | XX | xx |
| | x (xx%) | x (xx%) | x (xx%) | x (xx%) | x (xx%) | x (xx%) | x (xx%) | x (xx%) | x (xx%) | x (xx%) | x (xx%) | x (xx%) |
| Preferred Term 4 | xx | xx | xx | xx | XX | xx | xx | xx | xx | xx | xx | xx |
| | x (xx%) | x (xx%) | x (xx%) | x (xx%) | x (xx%) | x (xx%) | x (xx%) | x (xx%) | x (xx%) | x (xx%) | x (xx%) | x (xx%) |






| | | Treat<br>(N=) | ment | | | Contro<br>(N=xx | | | | A (N=) | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| SOC | Mild | Moderate | Severe | Total | Mild | Moderate | Severe | Total | Mild | Moderate | Severe | Total |
| Preferred Term | Events | Events | Events | Events | Events | Events | Events | Events | Events | Events | Events | Events |
| Ticicirca Tellii | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) |
| Continue to report all | | ,, | 1 | 1 | | , , , , | 1 | | | | 1, -, | |
| reported events | | | | | | | | | | | | |
| At and Post-Implant | | | | | | | | | | | | |
| Procedure | | | | | | | | | | | | |
| Any AE [1] | xx | XX | XX | xx | xx | xx | xx | XX | XX | XX | XX | xx |
| | x (xx%) | x (xx%) | x (xx%) | x (xx%) | x (xx%) | x (xx%) | x (xx%) | x (xx%) | x (xx%) | x (xx%) | x (xx%) | x (xx%) |
| SOC 1 [1] | xx | xx | xx | xx | xx | xx | xx | xx | xx | xx | xx | xx |
| | x (xx%) | x (xx%) | x (xx%) | x (xx%) | x (xx%) | x (xx%) | x (xx%) | x (xx%) | x (xx%) | x (xx%) | x (xx%) | x (xx% |
| Preferred Term 1 | XX | XX | XX | XX | XX | XX | XX | XX | XX | XX | XX | XX |
| | x (xx%) | x (xx%) | x (xx%) | x (xx%) | x (xx%) | x (xx%) | x (xx%) | x (xx%) | x (xx%) | x (xx%) | x (xx%) | x (xx% |
| Preferred Term 2 | XX | XX | XX | XX | XX | xx | XX | XX | XX | XX | XX | XX |
| | x (xx%) | x (xx%) | x (xx%) | x (xx%) | x (xx%) | x (xx%) | x (xx%) | x (xx%) | x (xx%) | x (xx%) | x (xx%) | x (xx%) |
| Preferred Term 3 | XX | XX | XX | XX | XX | XX | XX | XX | XX | XX | XX | XX |
| | x (xx%) | x (xx%) | x (xx%) | x (xx%) | x (xx%) | x (xx%) | x (xx%) | x (xx%) | x (xx%) | x (xx%) | x (xx%) | x (xx% |
| Preferred Term 4 | XX | XX | XX | XX | XX | XX | XX | XX | XX | XX | XX | XX |
| | x (xx%) | x (xx%) | x (xx%) | x (xx%) | x (xx%) | x (xx%) | x (xx%) | x (xx%) | x (xx%) | x (xx%) | x (xx%) | x (xx%) |
| SOC 2 [1] | xx | xx | xx | xx | xx | xx | xx | xx | xx | xx | xx | xx |
| | x (xx%) | x (xx%) | x (xx%) | x (xx%) | x (xx%) | x (xx%) | x (xx%) | x (xx%) | x (xx%) | x (xx%) | x (xx%) | x (xx% |
| Preferred Term 1 | XX | XX | XX | XX | XX | xx | xx | xx | XX | XX | xx | XX |
| | x (xx%) | x (xx%) | x (xx%) | x (xx%) | x (xx%) | x (xx%) | x (xx%) | x (xx%) | x (xx%) | x (xx%) | x (xx%) | x (xx% |
| Preferred Term 2 | xx | xx | xx | xx | XX | xx | xx | xx | xx | XX | xx | XX |
| | x (xx%) | x (xx%) | x (xx%) | x (xx%) | x (xx%) | x (xx%) | x (xx%) | x (xx%) | x (xx%) | x (xx%) | x (xx%) | x (xx% |
| Preferred Term 3 | XX | XX | XX | XX | XX | xx | XX | xx | XX | XX | xx | XX |
| | x (xx%) | x (xx%) | x (xx%) | x (xx%) | x (xx%) | x (xx%) | x (xx%) | x (xx%) | x (xx%) | x (xx%) | x (xx%) | x (xx% |
| Preferred Term 4 | XX | XX | XX | XX | XX | XX | XX | XX | XX | XX | XX | XX |
| | x (xx%) | x (xx%) | x (xx%) | x (xx%) | x (xx%) | x (xx%) | x (xx%) | x (xx%) | x (xx%) | x (xx%) | x (xx%) | x (xx% |
| Continue to report all | | | | | | | | | | | | |
| reported events | | | | | | | | | | | | |


n (%)



n (%)

| | | Treatment | | | | Control | | | | All | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | (N=xxx) | | | | (N=xxx) | | | | (N=xxx) | | |
| SOC | Mild | Moderate | Severe | Total | Mild | Moderate | Severe | Total | Mild | Moderate | Severe | Total |
| Preferred Term | Events | Events | Events | Events | Events | Events | Events | Events | Events | Events | Events | Events |

Abbreviations: AE, adverse event; SOC, system organ class.

Note: AEs coded using the MedDRA dictionary Version 21.0 or later. Given in the table are subject counts and percentages. At each level of summation, subjects are counted only once. Subjects experiencing AEs of more than one severity are summarized according to the maximum severity experienced over all episodes of an AE.

n (%)

[1] Percentage calculated based on ITT Population.

Doc# CLP-004 Rev D, 15JUL2024

Reference: Listing 16.x.x.x

SOURCE: xxxxx SAS 9.4 {program location} {run date/time}}

CONFIDENTIAL 122 of 158 Doc# CLP-004 Rev D, 15JUL2024



Table 14.1.3.3 Implant Procedure-Related Adverse Events by SOC and Maximum Severity: All Events (Safety Population)

| | | Treat<br>(N=: | | | | Contro<br>(N=xx | | | | A<br>(N=) | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| SOC | Mild | Moderate | Severe | Total | Mild | Moderate | Severe | Total | Mild | Moderate | Severe | Total |
| Preferred Term | Events | Events | Events | Events | Events | Events | Events | Events | Events | Events | Events | Events |
| | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) |
| Subjects with any AE [1,2] | xx | xx | xx | xx | xx | xx | xx | xx | xx | xx | xx | xx |
| , , , | x (xx%) | x (xx%) | x (xx%) | x (xx%) | x (xx%) | x (xx%) | x (xx%) | x (xx%) | x (xx%) | x (xx%) | x (xx%) | x (xx%) |
| System Organ Class 1 [1,2] | xx | xx | xx | xx | xx | xx | xx | xx | xx | xx | xx | xx |
| | x (xx%) | x (xx%) | x (xx%) | x (xx%) | x (xx%) | x (xx%) | x (xx%) | x (xx%) | x (xx%) | x (xx%) | x (xx%) | x (xx%) |
| Preferred Term 1 | XX | XX | XX | XX | XX | XX | XX | XX | XX | XX | XX | XX |
| | x (xx%) | x (xx%) | x (xx%) | x (xx%) | x (xx%) | x (xx%) | x (xx%) | x (xx%) | x (xx%) | x (xx%) | x (xx%) | x (xx%) |
| Preferred Term 2 | XX | XX | XX | XX | XX | XX | XX | XX | XX | XX | XX | XX |
| | x (xx%) | x (xx%) | x (xx%) | x (xx%) | x (xx%) | x (xx%) | x (xx%) | x (xx%) | x (xx%) | x (xx%) | x (xx%) | x (xx%) |
| Preferred Term 3 | XX | XX | XX | XX | XX | XX | XX | XX | XX | XX | XX | XX |
| | x (xx%) | x (xx%) | x (xx%) | x (xx%) | x (xx%) | x (xx%) | x (xx%) | x (xx%) | x (xx%) | x (xx%) | x (xx%) | x (xx%) |
| Preferred Term 4 | XX | XX | XX | XX | XX | XX | XX | XX | XX | XX | XX | XX |
| | x (xx%) | x (xx%) | x (xx%) | x (xx%) | x (xx%) | x (xx%) | x (xx%) | x (xx%) | x (xx%) | x (xx%) | x (xx%) | x (xx%) |
| System Organ Class 2 [1,2] | xx | xx | xx | xx | xx | xx | xx | xx | xx | xx | xx | xx |
| | x (xx%) | x (xx%) | x (xx%) | x (xx%) | x (xx%) | x (xx%) | x (xx%) | x (xx%) | x (xx%) | x (xx%) | x (xx%) | x (xx%) |
| Preferred Term 1 | XX | XX | XX | XX | XX | XX | XX | XX | XX | XX | XX | XX |
| | x (xx%) | x (xx%) | x (xx%) | x (xx%) | x (xx%) | x (xx%) | x (xx%) | x (xx%) | x (xx%) | x (xx%) | x (xx%) | x (xx%) |
| Preferred Term 2 | XX | XX | XX | XX | XX | XX | XX | XX | XX | XX | XX | XX |
| | x (xx%) | x (xx%) | x (xx%) | x (xx%) | x (xx%) | x (xx%) | x (xx%) | x (xx%) | x (xx%) | x (xx%) | x (xx%) | x (xx%) |
| Preferred Term 3 | XX | XX | XX | XX | XX | XX | XX | XX | XX | XX | XX | XX |
| | x (xx%) | x (xx%) | x (xx%) | x (xx%) | x (xx%) | x (xx%) | x (xx%) | x (xx%) | x (xx%) | x (xx%) | x (xx%) | x (xx%) |
| Preferred Term 4 | XX | XX | XX | XX | XX | XX | XX | XX | XX | XX | XX | XX |
| | x (xx%) | x (xx%) | x (xx%) | x (xx%) | x (xx%) | x (xx%) | x (xx%) | x (xx%) | x (xx%) | x (xx%) | x (xx%) | x (xx%) |
| Continue to report all reported events | | | | | | | | | | | | |




Doc# CLP-004 Rev D, 15JUL2024

Abbreviations: AE, adverse event; SOC, system organ class.

Note: AEs coded using the MedDRA dictionary Version 21.0 or later. Given in the table are subject counts and percentages. At each level of summation, subjects are counted only once. Subjects experiencing AEs of more than one severity are summarized according to the maximum severity experienced over all episodes of an AE.

[1] Percentage calculated based on ITT Population.

[2] AEs judged to be "Definitely Related" or "Probably Related" "to Implant Procedure are reported.

Reference: Listing 16.x.x.x

SOURCE: xxxxx SAS 9.4 {program location} {run date/time}}




Table 14.1.3.4 Implant Device-Related Adverse Events by SOC and Maximum Severity: All Events (Safety Population)

Repeat Table 14.1.3.4 for implant device-related adverse events




Table 14.1.3.5 Stimulation-Related Adverse Events by SOC and Maximum Severity: All Events (Safety Population)

Repeat Table 14.1.3.4 for stimulation-related adverse events

Table 14.1.3.6
Explant Procedure-Related Adverse Events by SOC and Maximum Severity: All Events (Safety Population)

Repeat Table 14.1.3.4 for explant procedure-related adverse events

Table 14.1.3.7
Energizer-Related Adverse Events by SOC and Maximum Severity: All Events (Safety Population)

Repeat Table 14.1.3.4 for Energizer-related adverse events


Doc# CLP-004 Rev D, 15JUL2024



Table 14.1.3.8 Device Deficiency (Safety Population)

| Variable | Treatment<br>(N=xxx) | Control<br>(N=xxx) | All<br>(N=xxx) |
|---|---|---|---|
| | Events n (%) | Events n (%) | Events n (%) |
| Any study device deficiency [1] | xx xx (xx.x%) | xx xx (xx.x%) | xx xx (xx.x%) |
| Relationship of study device deficiency [1] | | | |
| MicroRegulator (Implant) | xx xx (xx.x%) | xx xx (xx.x%) | xx xx (xx.x%) |
| POD | xx xx (xx.x%) | xx xx (xx.x%) | xx xx (xx.x%) |
| Energizer | xx xx (xx.x%) | xx xx (xx.x%) | xx xx (xx.x%) |
| Stimulation | xx xx (xx.x%) | xx xx (xx.x%) | xx xx (xx.x%) |
| Prescription Pad | xx xx (xx.x%) | xx xx (xx.x%) | xx xx (xx.x%) |
| IFU/Labeling | xx xx (xx.x%) | xx xx (xx.x%) | xx xx (xx.x%) |
| Study device deficiency associated with AE [1] | xx xx (xx.x%) | xx xx (xx.x%) | xx xx (xx.x%) |
| Study device deficiency associated with SAE [1] | xx xx (xx.x%) | xx xx (xx.x%) | xx xx (xx.x%) |

Abbreviations: AE, adverse event; POD, Positioning Orientation Device; SAE, serious adverse event.

Note: Given in the table are subject counts and percentages. At each level of summation, subjects are counted only once. Subject experiencing several episodes of the same type of study device deficiency is counted once.

[1] Percentage calculated based on safety ITT population.

Reference: Listing 16.x.x.x

SOURCE: xxxxx SAS 9.4 {program location} {run date/time}}


Doc# CLP-004 Rev D, 15JUL2024



Table 14.1.3.9 Protocol Deviations (ITT Population)

| Treatment | Control | All |
|---|---|---|
| (N=xxx) | (N=xxx) | (N=xxx) |
| Events n (%) | Events n (%) | Events n (%) |
| xx xx (xx.x%) | xx xx (xx.x%) | xx xx (xx.x%) |
| | Events n (%) xx xx (xx.x%) | Events n (%) Events n (%) xx xx |

Abbreviations: AE, adverse event; SAE, serious adverse event.

Note: Given in the table are subject counts and percentages. At each level of summation, subjects are counted only once.

[1] Percentage calculated based on safety ITT population.

Reference: Listing 16.x.x.x

SOURCE: xxxxx SAS 9.4 {program location} {run date/time}}




### Appendix C: Listing Mockups

| Listing 16.1.1 | Eligibility and Treatment Assignment | 130 |
|---|---|---|
| Listing 16.1.2.1.1 | Subject Disposition | 131 |
| Listing 16.1.2.1.2 | Eligibility Not Met | 132 |
| Listing 16.1.2.2 | Protocol Deviations | 133 |
| Listing 16.1.2.3 | Analysis Populations | 134 |
| Listing 16.1.2.4 | Demographics and Baseline Characteristics | 135 |
| Listing 16.1.2.5.1 | Prior and Concomitant Medication | 138 |
| Listing 16.1.2.5.2 | Implant and Explant Procedure | 139 |
| Listing 16.1.2.5.3 | Stimulation Prescription (Part 1) | 140 |
| Listing 16.1.2.5.3 | Stimulation Prescription (Part 2) | 141 |
| Listing 16.1.2.6.1 | RA Disease Activity Assessments | 142 |
| Listing 16.1.2.6.2 | ACR20 Response from Baseline on the Day of Informed Consent | 143 |
| Listing 16.1.2.6.2.1 | ACR20 Response from Day 0 | 144 |
| Listing 16.1.2.6.2 | ACR50 Response | 145 |
| Listing 16.1.2.6.2 | ACR70 Response | 146 |
| Listing 16.1.2.6.5 | CDAI | 147 |
| Listing 16.1.2.6.6 | DAS28-CRP | 148 |
| Listing 16.1.2.6.7 | HAQ-DI | 149 |
| Listing 16.1.2.6.8 | RAMRIS | 150 |
| Listing 16.1.2.6.9 | EQ-5D-5L | 151 |
| Listing 16.1.2.6.10 | SF-36 | 152 |
| Listing 16.1.2.6.11 | Inflammatory Biomarkers | 153 |
| Listing 16.1.2.6.12 | Subject's Blinding Assessment | 154 |
| Listing 16.1.2.6.13 | Joint Evaluator's Blinding Assessment | 155 |
| Listing 16.1.2.6.14 | Co-PI Rheumatologist's Blinding Assessment | 156 |
| Listing 16.1.2.7 | Adverse Events | 157 |
| Listing 16.1.2.8 | Device Deficiencies | 158 |


SETPOINT MEDICAL

Doc# CLP-004 Rev D, 15JUL2024

### Listing 16.1.1 Eligibility and Treatment Assignment

| Subject ID | Enrolled | Randomized | Randomization Number | Randomization Date | Treatment Assignment |
|---|---|---|---|---|---|
| xx-xxxx | Yes | Yes | xx-xx | DD-MMM-YYYY | Treatment |
| xx-xxxx | Yes | Yes | xx-xx | DD-MMM-YYYY | Control |

SOURCE: xxxxx SAS 9.4 {program location} {run date/time}




Listing 16.1.2.1.1 Subject Disposition

| Treatment<br>Group | Subject ID | Subject ID Consent Date Implant Procedure Date | | Randomization<br>Date | Subject Status | Date of Exit | Reason for<br>Withdrawal | Implant Status at<br>Study Exit |
|---|---|---|---|---|---|---|---|---|
| | xx-xxxx | DD-MMM-YYYY | DD-MMM-YYYY | DD-MMM-YYYY | | | | |

<u>Programming note:</u> This listing will include all consented subjects including screen failures, all other listings should only include all enrolled subjects.

Subject Status: Consented, Screen Failure, Enrolled, Implanted, Randomized, Withdrawn, Completed Study

Reason for withdrawal: Subject decision to withdraw consent, Investigator decision or medical judgement, Lost to follow-up, Device malfunction, Adverse event, Subject no longer eligible, Death, Study terminated, Sponsor or IRB decision, Other

SOURCE: xxxxx SAS 9.4 {program location} {run date/time}




Listing 16.1.2.1.2 Eligibility Not Met

| | | | Inclusion | | Exclusion |
|---|---|---|---|---|---|
| Subject<br>ID | Date of Screening Visit<br>DD-MMM-YYYY | Met All? | Criteria Not Met | Met Any? | Criteria Met |
| xx-xxxx | DD-MMM-YYYY (-x) | Yes | | Yes | xx-xxxxxxxxxxxxxxxxxxxxxx |
| xx-xxxx | DD-MMM-YYYY (-x) | No | xx -xxxxxxxxxxxxxxxxx | No | |
| xx-xxxx | DD-MMM-YYYY (-x) | Yes | | No | |

SOURCE: xxxxx SAS 9.4 {program location} {run date/time}


Doc# CLP-004 Rev D, 15JUL2024



#### Listing 16.1.2.2 Protocol Deviations

| Treatmen<br>t Group | Subject<br>ID | Deviation<br>ID | Visit | Deviation<br>Date | Classification | Category | Reason | Associated with AE? | Associated with SAE? | Reported to IRB? | Description |
|---|---|---|---|---|---|---|---|---|---|---|---|
| Treatmen<br>t | xx-xxxx | | | | | | | | | | |
| Control | xx-xxxx | | | | | | | | | | |

SOURCE: xxxxx SAS 9.4 {program location} {run date/time}


Doc# CLP-004 Rev D, 15JUL2024



### Listing 16.1.2.3 Analysis Populations

| Treatment | | Popu | ulation | |
|---|---|---|---|---|
| Group | Subject ID | ITT [1] | PTE [2] | Reason for Exclusion from PTE |
| Treatment | xx-xxxx | Yes | Yes | |
| Treatment | xx-xxxx | No | Yes | |
| Control | xx-xxxx | No | Yes | xxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxx |

Abbreviations: ITT, intent to treat; PTE, per-treatment-evaluable; RA, rheumatoid arthritis.

SOURCE: xxxxx SAS 9.4 {program location} {run date/time}


<sup>[1]</sup> ITT population comprises all enrolled and randomized subjects in Stage 1 and 2

<sup>[2]</sup> PTE population comprises subjects from ITT population who have received the assigned treatment, have no major procedural protocol deviations, and for whom follow-up data are available

Doc# CLP-004 Rev D, 15JUL2024



### Listing 16.1.2.4 Demographics and Baseline Characteristics (Part 1)

| Treatment<br>Group | Subject<br>ID | Age<br>(year) | Gender | Ethnicity | Race | RA<br>Duration<br>(year) | BMI<br>(kg/m²) | RF | ACPA | hsCRP<br>(mg/L) | TJC28 | SJC28 |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Treatment | xx-xxxx | xx | F | Non-Hispanic | White | | | Negative | Positive | | | |
| Control | | xx | M | Hispanic | White | | | Positive | Negative | | | |

SOURCE: xxxxx SAS 9.4 {program location} {run date/time}




Listing 16.1.2.4 Demographics and Baseline Characteristics (Part 2)

| Treatment<br>Group | Subject ID | CDAI Score | DAS28-CRP<br>Score | HAQ-DI Score | Number of<br>Prior<br>b/tsDMARDs | Prior b/tsDMARDs | Prior Jaki (Y/N) | Ongoing<br>Medical<br>Condition |
|---|---|---|---|---|---|---|---|---|
| Treatment | xx-xxxx | | | | | | | |
| Control | | | | | | | | |

SOURCE: xxxxx SAS 9.4 {program location} {run date/time}




### Listing 16.1.2.5.1 Subjects Receiving Rescue Treatment Prior to Week 12 (ITT Population)

| Subject ID | CDAI at baseline | CDAI prior to start<br>of rescue | Type of rescue | Start date /<br>Stop date | Rescue type<br>ongoing in<br>OL/LTFU (Y/N) | Rescue start relative<br>to Day 0 (days) |
|---|---|---|---|---|---|---|
| xx-xxxx | Baseline: xx.x | Day 0: xx.x | | | | |


Doc# CLP-004 Rev D, 15JUL2024



### Listing 16.1.2.5.1 Prior and Concomitant Medication

| | | | Start | | Stop | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|
| | | ATC level | | Study | | Study | | | | |
| Treatment | Subject | Preferred Term/ | Date | Day | Date | Day | | Dosage | | |
| Group | ID | Medication | | | | | Primary Indication | (Unit) | Route | Frequency |

XX-XXXX

XX-XXXX

#### Programming Note:

- 1. If Ongoing is checked "Yes" list "Ongoing" under stop date column
- 2. Concatenate dose and unit for listing, if other unit exists then list it for units
- 3. Route, if Other Route is not blank, list it under "Route" column
- 4. Frequency, if Other Frequency is not blank, list it under 'Frequency' Column

SOURCE: xxxxx SAS 9.4 {program location} {run date/time}




### Listing 16.1.2.5.2 Implant and Explant Procedure

| Treatment<br>Group | Subject<br>ID | Procedure<br>Date | MicroRegulator<br>Serial# | Procedure<br>Start Time | Procedure<br>Stop<br>Time | Procedure type<br>(Implant/Explant) | Post-Op<br>Clearance<br>Date |
|---|---|---|---|---|---|---|---|
| | xx-xxxx | | | | | | |

XX-XXXX

SOURCE: xxxxx SAS 9.4 {program location} {run date/time}


Doc# CLP-004 Rev D, 15JUL2024



Listing 16.1.2.5.3 Stimulation Prescription (Part 1)

| Treatment | Subject | | Strength | | Dose Changed | | | |
|---|---|---|---|---|---|---|---|---|
| Group | ID | Visit | (uA) | Duration | Frequency | Schedule | at this Visit? | Dose Change Reason |
| | XX-XXXX | | | | | | | |
| | XX-XXXX | | | | | | | |




200, 221 00110, 2,10022021

Listing 16.1.2.5.3 Stimulation Prescription (Part 2)

| Treatment<br>Group | Subject<br>ID | Energizer App<br>Firmware | Energizer<br>Bluetooth<br>Firmware | Implant App<br>Firmware | Implant Impedance | MicroRegulator<br>Suspended?/<br>Reason |
|---|---|---|---|---|---|---|
| | xx-xxxx | | | | | |
| | xx-xxxx | | | | | |




Listing 16.1.2.6.1 RA Disease Activity Assessments

| Treatment<br>Group | Subject<br>ID | Visit | SJC28 | TJC28 | HAQ-DI<br>Score | Subject's<br>Pain | Subject's<br>Global<br>Assessment | Evaluator's<br>Global<br>Assessment | hsCRP<br>(mg/mL) |
|---|---|---|---|---|---|---|---|---|---|
| Treatment | xx-xxxx | Screening<br>Day 0<br>Week 4<br>Week 8<br>Week 12 | xx | xx | xxx | xxx | xx | xxx | xx |
| Control | xx-xxxx | | | | | | | | |

SOURCE: xxxxx SAS 9.4 {program location}


Doc# CLP-004 Rev D, 15JUL2024



Listing 16.1.2.6.2
ACR20 Response from Baseline on the Day of Informed Consent

| Treatment<br>Group | Subject<br>ID | Visit | ACR20<br>Response | SJC28 | TJC28 | HAQ-DI<br>Score | Subject's<br>Pain | Subject's<br>Global<br>Assessment | Evaluator's<br>Global<br>Assessment | hsCRP<br>(mg/mL) |
|---|---|---|---|---|---|---|---|---|---|---|
| Treatment | xx-xxxx | Day 0 | N | N | N | N | N | N | N | N |
| | | Week 4 | N | N | N | N | N | N | N | N |
| | | Week 8 | Y | N | N | N | N | N | N | N |
| | | Week 12 | Y | Y | Y | N | Y | Y | N | Y |
| Control | xx-xxxx | Day 0 | N | N | N | N | N | N | N | N |
| | | Week 4 | Y | N | N | N | N | N | N | N |
| | | Week 8<br>Week 12 | N | N | N | N | N | N | N | N |

Note: Response defined by at least 20% reduction from baseline on the day of informed consent in TJC28 and SJC28 and 3 our 5 outcomes, according to ACR definition.

SOURCE: xxxxx SAS 9.4 {program location} {run date/time}


Doc# CLP-004 Rev D, 15JUL2024



Listing 16.1.2.6.2.1 ACR20 Response from Day 0

| Treatment<br>Group | Subject<br>ID | Visit | ACR20<br>Response | SJC28 | TJC28 | HAQ-DI<br>Score | Subject's<br>Pain | Subject's<br>Global<br>Assessment | Evaluator's<br>Global<br>Assessment | hsCRP<br>(mg/mL) |
|---|---|---|---|---|---|---|---|---|---|---|
| Treatment | xx-xxxx | Week 4 | N | N | N | N | N | N | N | N |
| | | Week 8 | Y | N | N | N | N | N | N | N |
| | | Week 12 | Y | Y | Y | N | Y | Y | N | Y |
| Control | xx-xxxx | Week 4 | N | N | N | N | N | N | N | N |
| | | Week 8 | Y | N | N | N | N | N | N | N |
| | | Week 12 | Y | Y | Y | N | Y | Y | N | Y |

Note: Response defined by at least 20% reduction from Day 0 in TJC28 and SJC28 and 3 our 5 outcomes, according to ACR definition.

SOURCE: xxxxx SAS 9.4 {program location} {run date/time}

# Statistical Analysis Plan for Interim and Primary Analyses in SPM-020 (The RESET-RA Study)

Doc# CLP-004 Rev D, 15JUL2024



Listing 16.1.2.6.2 ACR50 Response

| Treatment<br>Group | Subject<br>ID | Visit | ACR50<br>Response | SJC28 | TJC28 | HAQ-DI<br>Score | Subject's<br>Pain | Subject's<br>Global<br>Assessment | Evaluator's<br>Global<br>Assessment | hsCRP<br>(mg/mL) |
|---|---|---|---|---|---|---|---|---|---|---|
| Treatment | xx-xxxx | Day 0 | N | N | N | N | N | N | N | N |
| | | Week 4 | Y | N | N | N | N | N | N | N |
| | | Week 8 | Y | Y | Y | N | Y | Y | N | Y |
| | | Week 12 | | | | | | | | |
| Control | xx-xxxx | Day 0 | N | N | N | N | N | N | N | N |
| | | Week 4 | Y | N | N | N | N | N | N | N |
| | | Week 8 | N | N | N | N | N | N | N | N |
| | | Week 12 | | | | | | | | |

Note: Response defined by at least 50% reduction from baseline on the day of informed consent in TJC28 and SJC28 and 3 our 5 outcomes, according to ACR definition.

SOURCE: xxxxx SAS 9.4 {program location} {run date/time}






Listing 16.1.2.6.2 ACR70 Response

| Treatment<br>Group | Subject<br>ID | Visit | ACR70<br>Response | SJC28 | TJC28 | HAQ-DI<br>Score | Subject's<br>Pain | Subject's<br>Global<br>Assessment | Evaluator's<br>Global<br>Assessment | hsCRP<br>(mg/mL) |
|---|---|---|---|---|---|---|---|---|---|---|
| Treatment | xx-xxxx | Day 0<br>Week 4<br>Week 8 | N<br>Y<br>Y | N<br>N<br>Y | N<br>N<br>Y | N<br>N<br>N | N<br>N<br>Y | N<br>N<br>Y | N<br>N<br>N | N<br>N<br>Y |
| Control | xx-xxxx | Week 12<br>Day 0 | N | N | N | N | N | N | N | N |
| | | Week 4<br>Week 8<br>Week 12 | Y<br>N | N<br>N | N<br>N | N<br>N | N<br>N | N<br>N | N<br>N | N<br>N |

Note: Response defined by at least 70% reduction from baseline on the day of informed consent in TJC28 and SJC28 and 3 our 5 outcomes, according to ACR definition.

SOURCE: xxxxx SAS 9.4 {program location} {run date/time}


Statistical Analysis Plan for Interim and Primary Analyses in SPM-020 (The RESET-RA Study)

Doc# CLP-004 Rev D, 15JUL2024



Listing 16.1.2.6.5 CDAI

| Treatment<br>Group | Subject<br>ID | Visit | CDAI Score | CDAI<br>LDA<br>(>2.8 to ≤ 10) | CDAI<br>Remission<br>(0 to ≤ 2.8) | CDAI<br>MCID Response |
|---|---|---|---|---|---|---|
| Treatment | xx-xxxx | Screening | XX.X | | | |
| | | Day 0 | | | | |
| | | Week 4 | | No | No | No |
| | | Week 8 | | Yes | No | Yes |
| | | Week 12 | | Yes | Yes | Yes |

SOURCE: xxxxx SAS 9.4 {program location} {run date/time}


# Statistical Analysis Plan for Interim and Primary Analyses in SPM-020 (The RESET-RA Study)

Doc# CLP-004 Rev D, 15JUL2024



Listing 16.1.2.6.6 DAS28-CRP

| Treatment<br>Group | Subject<br>ID | Visit | DAS28-CRP<br>Score | DAS28-CRP<br>LDA<br>(0.6 to < 3.2) | DAS28-CRP<br>Remission<br>(0 to < 2.6) | DAS28-CRP<br>MCID Response<br>(-1.2) | DAS28-CRP<br>Good/Moderate<br>EULAR<br>Response |
|---|---|---|---|---|---|---|---|
| Treatment | xx-xxxx | Screening | XX | _ | | | |
| | | Day 0 | xx | _ | | | |
| | | Week 4 | XX | No | No | No | |
| | | Week 8 | XX | Yes | No | Yes | Moderate |
| | | Week 12 | XX | Yes | Yes | Yes | Good |

SOURCE: xxxxx SAS 9.4 {program location} {run date/time}


Statistical Analysis Plan for Interim and Primary Analyses in SPM-020 (The RESET-RA Study) Doc# CLP-004 Rev D, 15JUL2024



Listing 16.1.2.6.7 HAQ-DI

| Treatment<br>Group | Subject<br>ID | Visit | HAQ-DI<br>Score | HAQ-DI<br>Response<br>(MCID -0.22) |
|---|---|---|---|---|
| Treatment | xx-xxxx | Screening | xx | |
| | | Day 0 | XX | No |
| | | Week 4 | XX | No |
| | | Week 8 | XX | Yes |
| | | Week 12 | xx | Yes |

SOURCE: xxxxx SAS 9.4 {program location} {run date/time}


Statistical Analysis Plan for Interim and Primary Analyses in SPM-020 (The RESET-RA Study)

Doc# CLP-004 Rev D, 15JUL2024



#### Listing 16.1.2.6.8 RAMRIS

| Treatment<br>Group | Subject<br>ID | Visit | Synovitis score | Osteitis score | Bone erosion<br>score | Progression?<br>(bone erosion<br>increase > 0.5) | CARLOS |
|---|---|---|---|---|---|---|---|
| Treatment | xx-xxxx | Screening<br>Week 12<br>Change from<br>baseline | | | | No | |

SOURCE: xxxxx SAS 9.4 {program location} {run date/time}


# Statistical Analysis Plan for Interim and Primary Analyses in SPM-020 (The RESET-RA Study) Doc# CLP-004 Rev D, 15JUL2024



Listing 16.1.2.6.9 EQ-5D-5L

| Treatment<br>Group | Subject<br>ID | Visit | Mobility | Self-Care | Usual<br>Activities | Pain/Discomfort | Anxiety/Depression | EQ-VAS | Index<br>value |
|---|---|---|---|---|---|---|---|---|---|
| Treatment | xx-xxxx | Screening<br>Day 0<br>Week 4<br>Week 8<br>Week 12 | x | x | x | x | х | xxx | xx |

SOURCE: xxxxx SAS 9.4 {program location} {run date/time}


# Statistical Analysis Plan for Interim and Primary Analyses in SPM-020 (The RESET-RA Study)



Doc# CLP-004 Rev D, 15JUL2024

Listing 16.1.2.6.10 SF-36

| Treatment<br>Group | Subject<br>ID | Visit | PCS score | MCS score |
|---|---|---|---|---|
| Treatment | xx-xxxx | Screening<br>Day 0<br>Week 4<br>Week 8<br>Week 12 | | |

SOURCE: xxxxx SAS 9.4 {program location} {run date/time}


Statistical Analysis Plan for Interim and Primary Analyses in SPM-020 (The RESET-RA Study)

Doc# CLP-004 Rev D, 15JUL2024



# Listing 16.1.2.6.11 Inflammatory Biomarkers

| Treatment<br>Group | Subject<br>ID | Visit | IL-6<br>(pg/mL) | IL-6<br>% Change | SAA<br>(µg/mL) | SAA<br>% Change | MMP-3<br>(pg/mL) | MMP-3<br>% Change |
|---|---|---|---|---|---|---|---|---|
| Treatment | xx-xxxx | Screening | | | | | | _ |
| | | Day 0<br>Week 4<br>Week 8<br>Week 12 | | | | | | - |

SOURCE: xxxxx SAS 9.4 {program location} {run date/time}


Statistical Analysis Plan for Interim and Primary Analyses in SPM-020 (The RESET-RA Study) Doc# CLP-004 Rev D, 15JUL2024



# Listing 16.1.2.6.12 Subject's Blinding Assessment

| Treatment<br>Group | Subject<br>ID | Visit Date<br>(Study Day) | Week 4 | Why? | Week 12 | Why? |
|---|---|---|---|---|---|---|
| xxx | xx-xxxx | | | | | |

SOURCE: xxxxx SAS 9.4 {program location} {run date/time}


Statistical Analysis Plan for Interim and Primary Analyses in SPM-020 (The RESET-RA Study) Doc# CLP-004 Rev D, 15JUL2024



### Listing 16.1.2.6.13 Joint Evaluator's Blinding Assessment

| Treatment<br>Group | Subject<br>ID | Visit Date<br>(Study Day) | Week 4 | Why? | Week 12 | Why? |
|---|---|---|---|---|---|---|
| xxx | xx-xxxx | | | | | |

SOURCE: xxxxx SAS 9.4 {program location} {run date/time}


Statistical Analysis Plan for Interim and Primary Analyses in SPM-020 (The RESET-RA Study)

SETPOINT MEDICAL

Doc# CLP-004 Rev D, 15JUL2024

## Listing 16.1.2.6.14 Co-PI Rheumatologist's Blinding Assessment

| Treatment<br>Group | Subject<br>ID | Visit Date<br>(Study Day) | Week 4 | Why? | Week 12 | Why? |
|---|---|---|---|---|---|---|
| xxx | xx-xxxx | | | | | |

SOURCE: xxxxx SAS 9.4 {program location} {run date/time}


# Statistical Analysis Plan for Interim and Primary Analyses in SPM-020 (The RESET-RA Study)

Doc# CLP-004 Rev D, 15JUL2024



#### Listing 16.1.2.7 Adverse Events

| Treatment<br>Group | Subject ID | System Organ<br>Class/<br>Preferred Term/<br>Adverse Event<br>Verbatim | Onset Date<br>(Day) | Resolution Date<br>(Day) | Severity | SAE? | Relationship | Treatment/<br>outcome |
|---|---|---|---|---|---|---|---|---|
| Treatment | xx-xxxx | xxxxxx/<br>xxxxxx/<br>xxxxxx/ | DD-MMM-YYYY<br>(xx) | DD-MMM-YYYY<br>(xx) | | | | xxxxxx/<br>xxxxxx |
| | | xxxxxx/<br>xxxxxx/<br>xxxxxx/ | | | | | | |
| Control | xx-xxxx | None | | | | | | |

Note: If a Subject has no AEs then "None" will be displayed. Adverse Events are coded in MedDRA.

Programming Note: If Ongoing is checked then list "Continuing" in the place for "Resolution Date (Day)".

SOURCE: xxxxx SAS 9.4 {program location} {run date/time}


Statistical Analysis Plan for Interim and Primary Analyses in SPM-020 (The RESET-RA Study) Doc# CLP-004 Rev D, 15JUL2024



Listing 16.1.2.8 Device Deficiencies

| Treatment<br>Group | Subject ID | Deficiency ID | Deficiency Date Deficiency Rela | Associated with AE? | Associated with SAE? | Description |
|---|---|---|---|---|---|---|
| Treatment | xx-xxxx | | | | | |
| Control | xx-xxxx | | | | | |

SOURCE: xxxxx SAS 9.4 {program location} {run date/time}




### STATISTICAL ANALYSIS PLAN

For Long-Term Safety and Exploratory Analyses

#### 1 TITLE PAGE

| Study Title | Vagus Nerve Stimulation Using the SetPoint System for Moderate-to-Severe<br>Rheumatoid Arthritis: The RESET-RA Study |
|---|---|
| Protocol Number | SPM-020 |
| ClinicalTrials.gov<br>Identifier | NCT04539964 |
| Investigational Device | The SetPoint System |
| Study Sponsor's Name<br>and Address | SetPoint Medical, Inc.<br>25101 Rye Canyon Loop<br>Valencia, CA 91355 |
| Biostatistics and Data<br>Analysis | SetPoint Medical, Inc. |

#### CONFIDENTIALITY STATEMENT

This document is the property of SetPoint Medical, Inc. The document is highly confidential and is to be used only in connection with matters authorized by a senior representative of SetPoint Medical, and no part of it is to be disclosed to a third party without prior written permission from SetPoint Medical.




### TABLE OF CONTENTS

| 1 | TITL | E PAGE | 1 |
|------|-------|-----------------------------------------------|----|
| 2 | LIST | OF ABBREVIATIONS | 5 |
| 3 | INTR | ODUCTION | 7 |
| | 3.1 | Study Objective | 7 |
| | 3.2 | Study Design | 7 |
| | 3.3 | Study Visits and Assessments During Extension | 7 |
| 4 | TYPE | E OF PLANNED ANALYSES | 7 |
| | 4.1 | DMC Analysis | 7 |
| | 4.2 | Exploratory Analysis | 8 |
| 5 | STAT | TISTICAL METHODS | 9 |
| | 5.1 | General Considerations for Data Analyses | 9 |
| | 5.2 | Analysis Populations | 10 |
| | 5.3 | Study Day Calculation | 10 |
| | 5.4 | Change from Baseline Calculation. | 10 |
| | 5.5 | Missing Data | 11 |
| | 5.6 | Data Assurance. | 11 |
| | 5.7 | Coding Dictionaries | 11 |
| 6 | EXPI | ORATORY EFFICACY ANALYSES | 11 |
| | 6.1 | General Considerations | 12 |
| | 6.2 | Clinical Variables | 13 |
| | 6.3 | Subgroup Analyses. | 17 |
| 7 | SAFE | TY EVALUATION | 18 |
| | 7.1 | AE and SAEs | 18 |
| | 7.2 | Protocol Deviations | 19 |
| | 7.3 | Device Deficiencies | 19 |
| 8 | STAT | TISTICAL CONSIDERATIONS RELATED TO COVID-19 | 19 |
| | 8.1 | Impact of COVID-19 on Study Integrity | 19 |
| | 8.2 | COVID-19 Analysis Considerations | 19 |
| 9 | REFE | ERENCES | 20 |
| 10 | APPE | ENDICES | 21 |
| APPE | ENDIX | A: SCHEDULE OF ASSESSMENTS | 21 |
| APPE | ENDIX | B: TABLE MOCKUPS | 22 |



| APPENDIX C: LISTING MOCKUPS | 106 |
|---------------------------------------------------------|-----|
| LIST OF TABLES | |
| Table 1: Data Access Matrix During Open-Label Extension | 8 |
| Table 2: Summary of Exploratory Efficacy Endpoints | 9 |
| Table 3: EULAR Response Criteria | 14 |






# **Revision History**

| Revision | Revision Date | Summary of Changes |
|---|---|---|
| A | 05MAY2021 | Document created |
| В | 29JAN2024 | <ul> <li>Updates made for consistency with current revision of CLP-001, Clinical Investigational Protocol SPM-020 (The RESET-RA Study) (p. 7)</li> <li>Updates made for consistency with current version of CLP-003, Data Monitoring Committee Charter for SPM-020 (The RESET-RA Study) (pp. 7-8)</li> <li>Added subgroup analyses for subjects receiving augmented therapy (pp. 9, 18, Appendix B pp. 17, 23, 29, 35, 74-77)</li> <li>Generalized language pertaining to software requirements for statistical analysis (p. 10)</li> <li>Change in nomenclature from Open-label PTE population to Treatment to Open Label (TOL), and crossover PTE population to Control to Open Label (TOL) for accuracy (p. 10, table and listing headers and footers throughout Appendices B &amp; C)</li> <li>Removed reference to collecting safety data once a subject is withdrawn from the study (p. 10)</li> <li>Rescue language and penalty as treatment failures is removed because additional RA treatment is allowed during open-label follow-up per protocol (p. 11)</li> <li>Added detail on missing analytes/retests (p. 11)</li> <li>Clarified missing data approaches (p. 12)</li> <li>Descriptions of ACR components removed as the section is duplicative with CLP-004; CLP-004 is referenced (p. 13)</li> <li>Added detail on methods for calculating and analyzing RAMRIS scores (p. 16)</li> <li>Removed information on calculation of SF-36 scores and replaced with reference to the same information which is found in the SF-36 User's Manual (p. 16)</li> <li>Clarified information on calculation of the EQ-5D-5L score (p. 17, Appendix B, pp. 63-67)</li> <li>Updated description of how AEs are categorized for consistency with study protocol (p. 18, Appendix B, p. 88)</li> <li>Added listing of subjects receiving augmented therapy (Appendix C, p. 6)</li> </ul> |
| C | 15JUL2024 | <ul> <li>Extended study duration by adding 6 visits as part of open-label,<br/>long-term follow-up after completion of Week 12 (pp. 7-8, 21)</li> </ul> |


Serial Number: c700c42a-b18e-4af7-8a24-9d2146ac6503 accessed by Melissa Evangelista (MEVANGELISTA) on Thu, 28 Aug 2025 18:20:31 GMT.



### 2 LIST OF ABBREVIATIONS

| Abbreviation | Expansion |
|--------------|--------------------------------------------------|
| ACR | American College of Rheumatology |
| AE | Adverse event |
| CARLOS | Cartilage Loss Score |
| CDAI | Clinical Disease Activity Index |
| CI | Confidence interval |
| СМО | Chief Medical Officer |
| COL | Control to Open Label |
| CRF | Case report form |
| DAS | Disease Activity Score |
| DMARD | Disease-modifying antirheumatic drug |
| DMC | Data monitoring committee |
| EDC | Electronic data capture |
| EGA | Evaluator's global assessment |
| EQ-5D-5L | EuroQol 5 domains 5 levels |
| EULAR | European League Against Rheumatism |
| HAQ-DI | Health Assessment Questionnaire Disability Index |
| hsCRP | High-sensitivity C-reactive protein |
| IL | Interleukin |
| IRB | Institutional Review Board |
| ITT | Intent to treat |
| JAKi | Janus kinase inhibitors |
| LDA | Low disease activity |
| LOCF | Last observation carried forward |
| MCID | Minimal clinically important difference |
| MedDRA | Medical Dictionary for Regulatory Activities |
| MRI | Magnetic resonance imaging |
| NRI | Non-responder imputation |
| NRS | Numerical rating scale |


# Statistical Analysis Plan for Long-Term Safety and Exploratory Analyses in SPM-020 (The RESET-RA Study)



# Doc# CLP-008 Rev C, 15JUL2024

| Abbreviation | Expansion |
|--------------|---------------------------------------------|
| ос | Observed case |
| PCS | Physical component summary |
| PD | Protocol deviation |
| PMA | Premarket Approval |
| PT | Preferred term |
| PTE | Per-treatment evaluable |
| RA | Rheumatoid arthritis |
| RAMRIS | Rheumatoid Arthritis MRI Scoring System |
| RF | Rheumatoid factor |
| SADE | Serious adverse device effect |
| SAE | Serious adverse event |
| SAP | Statistical analysis plan |
| SAS | Statistical Analysis Software |
| SD | Standard deviation |
| SF-36 | Short Form Survey with 36 items |
| SGA | Subject's global assessment |
| SJC28 | Swollen joint count for 28 different joints |
| SOC | System organ class |
| SOP | Standard operating procedure |
| TEAE | Treatment emergent adverse event |
| TJC28 | Tender joint count for 28 different joints |
| TOL | Treatment to Open Label |
| UADE | Unanticipated adverse device effect |
| USADE | Unanticipated serious adverse device effect |
| WHO | World Health Organization |




### 3 INTRODUCTION

This document outlines the statistical analysis plan (SAP) for the exploratory analysis during the open-label, long-term follow-up period in the RESET-RA study conducted by SetPoint Medical under protocol SPM-020 entitled "Vagus Nerve Stimulation Using the SetPoint System for Moderate to Severe Rheumatoid Arthritis: The RESET-RA Study." The SAP specifies the listings and tabular summaries for the exploratory data analyses to be performed using the data collected during the open-label, long-term follow-up.

Note: The primary, secondary and exploratory efficacy analyses of the randomized, shamcontrolled, double-blind data through Week 12 are detailed in a separate SAP (CLP-004).

### 3.1 Study Objective

The overall objective of this study is to evaluate the safety and efficacy of the SetPoint System for the treatment of adult patients with active, moderate-to-severe RA who have had an inadequate response or intolerance to biologic or targeted synthetic DMARDs.

The specific objective of the open-label follow-up with all subjects receiving active stimulation is to gather long-term safety and exploratory efficacy data.

# 3.2 Study Design

This is an operationally seamless, 2-stage, randomized, sham-controlled, double-blind, multicenter pivotal study enrolling up to 250 randomized subjects at up to 45 study centers across the U.S. After completing a 12-week follow-up for the primary efficacy endpoint, there is a one-way crossover of the control group and a 252-week follow-up of all subjects on active stimulation for long-term safety and exploratory efficacy data. The blinding to the original treatment assignment will be maintained until the last subject completes Week 12 assessments, and the study dataset for the primary analysis is locked.

## 3.3 Study Visits and Assessments During Extension

The open-label follow-up will begin after completion of assessments at Week 12 and a one-way crossover of the control group to active stimulation. Subjects receiving active stimulation will continue on active stimulation. Subjects will return for 3 device titration visits (Titration 4, 5 and 6 at Week 13, 14, 15, respectively), and 21 follow-up assessment visits every 12 weeks from Week 24 through Week 264 (end of study). See **Appendix A** for Schedule of Assessments.

#### 4 TYPE OF PLANNED ANALYSES

# 4.1 DMC Analysis

An independent Data Monitoring Committee (DMC) consisting of external, independent rheumatology, surgery and biostatistics experts will continue to provide ongoing monitoring of the safety, efficacy and overall study conduct. The DMC's role and responsibilities and the scope of




study oversight are detailed in the DMC Charter, which defines the DMC membership, meeting logistics, and meeting frequency.

During long-term extension, once the last study subject has been enrolled, the DMC will continue to meet once every 6 months and provide recommendations for continuing or stopping the study based on their ongoing review of cumulative safety data, including AEs, SAEs, device deficiencies, protocol deviations, and concomitant medications, as well as descriptive summaries of TJC28 and SJC28.

The DMC meetings will be performed in closed sessions until the study is unblinded. Data access is described in **Table 1** 

Table 1: Data Access Matrix During Open-Label Extension

| Department/Role | Blinded | Unblinded | Note |
|---|---|---|---|
| CEO | В | | Receiving DMC recommendations |
| Clinical<br>Operations <sup>1</sup> | В | | Not having access to randomization assignments or DMC Closed<br>Session reports to preserve blinding of everyone involved directly<br>or indirectly in the study conduct until locking the study dataset<br>for the primary efficacy analysis at Week 12 |
| Clinical Data<br>Management | В | | Consultants to sponsor responsible for managing EDC and IRT, generating data exports and not having access to randomization assignments until locking the study dataset for the primary efficacy analysis at Week 12 |
| Study<br>Biostatisticians | В | | Consultants to sponsor responsible for programming but not having access to randomization assignments until locking the study dataset for the primary efficacy analysis at Week12. |
| Independent<br>Biostatistician | | U | Non-voting statistician reporting to DMC responsible for receiving blinded data exports, accessing randomization assignments, conducting unblinded analyses and preparing outputs for review during DMC closed sessions |
| DMC | | U | DMC chairperson, biostatistician, and clinicians participating in closed meetings |

Abbreviations: B, blinded; CEO, Chief Executive Officer; DMC, data monitoring committee; EDC, electronic data capture; U, unblinded.

### 4.2 Exploratory Analysis

During the open-label follow-up, changes in exploratory efficacy endpoints at Week 24, 48, 96, 144 and 264 (end of study) will be evaluated in comparison to baseline and Day 0 for the treatment population and Week 12 for the crossover population using data for all subjects available at a given timepoint (**Table 2**). Refer to Section **5.2** for definitions of populations.


<sup>&</sup>lt;sup>1</sup>Clinical operations includes but is not limited to Chief Medical Officer, Vice President of Clinical Affairs, Managers of Clinical Affairs/Operations, Clinical Research Associates, Field Clinical Engineers.



Doc# CLP-008 Rev C, 15JUL2024

Table 2: Summary of Exploratory Efficacy Endpoints

| Endpoint | Display | TOL | COL | Subgroup |
|---|---|---|---|---|
| ACR20/50/70 response | T, L | Y | Y | Y[1] |
| DAS28-CRP moderate/good EULAR response | T, L | Y | Y | Y |
| DAS28-CRP response (MCID) | T, L | Y | Y | Y |
| HAQ-DI score change and response (MCID) | T, L | Y | Y | Y |
| ACR components (TJC28, SJC28, Subject Pain, SGA, HAQ-DI, EGA, hsCRP) 20/50/70response | T, L | Y | Y | |
| DAS28-CRP score change, LDA/remission | T, L | Y | Y | |
| CDAI score change, LDA/remission, response (MCID) | T, L | Y | Y | |
| RAMRIS (bone erosion, osteitis, synovitis, CARLOS)<br>score change, progression (bone erosion) at Week 24 | T, L | Y | Y | |
| EQ-5D-5L score change | T, L | Y | Y | |
| SF-36/PCS/MCS score change | T, L | Y | Y | |
| Percent change in inflammatory biomarkers at Week 24 | T, L | Y | Y | |
| Subject satisfaction at Week 24 | T, L | Y | Y | |

Abbreviations: ACR, American College of Rheumatology; CARLOS, cartilage loss score; CDAI, Clinical Disease Activity Index; COL, control to open label; CRP, C-reactive protein; DAS, Disease Activity Score; EGA, evaluator's global assessment; EQ-5d-5L, EuroQol 5 domains 5 levels; EULAR, European League Against Rheumatism; HAQ-DI, Health Assessment Questionnaire Disability Index; hsCRP, high sensitivity CRP; L, listings; LDA, low disease activity; RAMRIS, Rheumatoid Arthritis MRI Scoring System; SF-36, Short Form Survey with 36 items; SGA, subject's global assessment; T, tables; TJC, tender joint count; TOL, treatment to open label; SJC, swollen joint count; Y, yes.

[1] Subgroup analyses as defined in Section 6.3

Note: All score values are determined at all timepoints, unless stated otherwise. All response rates are determined based on change from baseline (i.e., on the day of informed consent for OL PTE population and Week 12 for CO PTE population) to a specified timepoint. Refer to Section **5.2** for definitions of populations Sections **6.2** for definition of response for specific endpoints.

#### 5 STATISTICAL METHODS

#### 5.1 General Considerations for Data Analyses

The exploratory analyses and safety evaluations are considered *a priori* analyses because they have been prespecified in the SAP prior to locking the database. All other analyses, if any, designed subsequent to locking the database will be considered *post-hoc* analyses, and their results will be considered exploratory. Any *post hoc* analyses will be clearly identified in the clinical study report.

Continuous data will be summarized in terms of the mean, SD, median, minimum, maximum and number of observations, unless otherwise stated. The minimum and maximum will be reported to the same number of decimal places as the raw data recorded in the database. The mean and median will be reported to 1 more decimal place than the raw data recorded in the database. The SD will be reported to 2 more decimal places than the raw data recorded in the database. In general, the maximum number of decimal places reported shall be 4 for any summary statistic.




Categorical data will be summarized in terms of the number of subjects providing data at the relevant time point, frequency counts and percentages. If not stated otherwise, percentages will be presented with one decimal place. Percentages will not be presented for zero counts. Percentages will be calculated using n as the denominator. 100% will be presented without decimal places.

95% Confidence intervals (CI) will be presented to 1 more decimal place than the raw data. Unless stated otherwise, a two-sided 95% confidence level will be calculated when confidence interval is presented.

Data from the protocol-specified visits (i.e., as reported in CRF) will be used in the summary tables (**Appendix B**) and data listings (**Appendix C**). All report outputs will be produced using a software package widely recognized as acceptable for analyzing clinical data in a secure and validated environment.

# 5.2 Analysis Populations

Analysis population defines the subjects to be included in an analysis. The exploratory analyses will be conducted on the Treatment to Open Label (TOL) and Control to Open Label (COL) populations. The safety analyses will be evaluated on the safety population. All analysis populations are defined below and the exploratory endpoints summarized in **Table 2**.

- Treatment to Open Label (TOL): The TOL population comprises treatment subjects from ITT population who received active stimulation through Week 12, completed Week 12 assessments, continued to receive active stimulation during open-label follow-up, and for whom follow-up data are available.
- Control to Open Label (COL): The COL population comprises Control subjects from ITT population who received non-active (sham) stimulation through Week 12, switched to active stimulation after completing Week 12 assessments, continued to receive active stimulation during open-label follow-up, and for whom follow-up data are available.
- Safety population. All enrolled subjects.

#### 5.3 Study Day Calculation

Study day is calculated relative to the date of Day 0 (randomization) and will appear in the listings where applicable. If the date of event is on or after Day 0, study day will be calculated as:

Study day = date of event – date of Day 0 (randomization)

### 5.4 Change from Baseline Calculation

Percent change from baseline to any time point will be calculated as follows:

[Value (Post-baseline) - Value (Baseline)] / Value (Baseline) x 100

A negative value reflects a decrease in a given parameter, while a positive relative difference reflects an increase in the parameter.


# SETPOINT MEDICAL

#### 5.5 Missing Data

For continuous endpoints, change from baseline will be set to missing at visits with missing values or where data were imputed to missing.

For binary endpoints, subjects with missing efficacy data or early withdrawals will be set to missing.

Additional rules for handling of missing data are detailed below:

- Missing efficacy data. Visits with missing data (due to a missed visit or missing component
  of a composite endpoint) will be set to missing.
- Early withdrawals. Visits following the early withdrawal will be set to missing.
- Missing baseline value. For efficacy endpoints, a missing value at baseline will not be imputed, and the endpoint will be set to missing for all visits.
- Missing analytes/ retests. If an analyte value is missing/ its concentration cannot be reliably
  determined (eg. sample was lost, damaged, etc.), a retest value will be used for that analyte. If
  an initial value is non-missing and reliable but the analyte was retested, the value that coincides
  with the date of clinical assessment will be used. If neither an initial and nor retest value are
  available, the analyte value will be set to missing.
- For missing dates, refer to Section 5.8 of CLP-004.

### 5.5.1 Multiple Assessments and Visits

If a variable (e.g., MRI, TJC, SJC) has been assessed multiple times at the same visit, only the last assessment will be used.

Only completed scheduled visits will be included in summary tables (**Appendix B**). Listings will include scheduled and unscheduled visits (**Appendix C**).

#### 5.6 Data Assurance

All tables, figures and data listings to be included in the report will be independently checked for consistency, integrity and in accordance with the study sponsor's SOPs.

### 5.7 Coding Dictionaries

AEs will be coded using the Medical Dictionary for Regulatory Activities (MedDRA, version 21.0 or later). Concomitant medications will be coded using the March 2019 or later version of the WHO Drug Global dictionary.

#### 6 EXPLORATORY EFFICACY ANALYSES




#### 6.1 General Considerations

For each follow-up time point, all dichotomous variables will be reported as responders / patients who have achieved that follow-up duration, percentage of responders, and 95% CI.

Values will be reported at each follow-up timepoint.

For continuous measures, mean, SD, median, minimum and maximum will be presented at each time point.

Time will be measured from initiation of stimulation. Therefore study participants originally randomized to stimulation will, for example, have Week 24 visits represented at 24 weeks of follow-up while study participants randomized to sham will have Week 24 visits represented as 12 weeks, since they will have been on stimulation on for 12 weeks at the Week 24 visit.

# 6.1.1 Missing endpoint data imputation

Below are the descriptions for the imputation methods that may be used throughout the efficacy analyses:

- Observed case (OC). Missing values remain missing. For the categorical composite endpoints, in the case that some components are missing, the composite endpoint assessment will be derived based on the non-missing components. If non-missing components are not sufficient to determine final composite endpoint, then the composite endpoint will be set as missing. For continuous composite endpoints, if any components are missing, the composite endpoints will be set as missing.
- Last observation carried forward (LOCF). Baseline and Day 0 measurements will not be carried forward to post-baseline. Only measurements post Day 0 will be LOCF for continuous and binary response measures. For the composite endpoints, the last non-missing, post-Day 0 observation will be carried forward to subsequent visits for each individual component first, and then the composite endpoints using individual components imputed by LOCF will be calculated as described above. If a subject does not have a non-missing observed record for a post-Day 0 visit, the last post-Day 0 record prior to the missed visit will be used. If the last non-missing observation prior to the missing visits cannot be determined due to multiple measurements occurring at the same time or the time not available within the same day, the worst outcome will be used for LOCF. If missing components still exist after LOCF, the composite endpoints will be calculated using the same rules as described in OC.
- Non-responder imputation (NRI). For all binary response measurements, starting from OC, all
  missing will be set as non-responders.

If subject only had baseline measurements, LOCF and OC analyses will not include this subject. But this subject will be treated as non-responder in NRI analyses.


# SETPOINT MEDICAL

# Doc# CLP-008 Rev C, 15JUL2024

Clinical Variables

For descriptions and definitions of ACR components (TJC28, SJC28, Subject's Pain Assessment, SGA, EGA, HAO-DI, hsCRP), refer to Section 8.2 of CLP-004.

#### 6.2.1 ACR20/50/70

A subject achieves ACR20/50/70 response when this subject experiences a  $\geq$  20%/50%/70%, respectively improvement from baseline to a given timepoint in TJC28, SJC28, and at least 3 of the following 5 items:

- Subject's pain assessment
- SGA

6.2

- EGA
- HAQ-DI
- hsCRP

For all visits, if any of the component scores are missing, then those scores will be considered as not having met the criteria for improvement. If 3 or more of the 5 remaining ACR measures are missing, ACR20/50/70 will each be considered missing.

For component scores with missing baseline values or a baseline value of 0, the percentage improvement cannot be calculated, and the component will be considered as not having met the criteria for improvement for all visits.

20/50/70 response for each component (TJC28, SJC28, Subject's Pain Assessment, SGA, HAQ-DI, EGA, hsCRP) corresponds to 20, 50 and 70% improvement from baseline to a given timepoint, respectively.

#### 6.2.2 DAS28-CRP

The Disease Activity Score (DAS) is a derived measurement of 4 components with differential weighting:

- TJC28
- SJC28
- hsCRP (mg/L)
- SGA

A total score ranges from 0 to 10 and is computed as follows:

DAS28-CRP = 0.56 \* sqrt(TJC28) + 0.28 \* sqrt(SJC28) + 0.36 \* ln(CRP+1) + 0.014 \* SGA + 0.96




Doc# CLP-008 Rev C, 15JUL2024

If one of the components is missing at an individual assessment point, the DAS28-CRP value for that assessment will be set to missing. An alternative imputation method for missing components may be applied as described in Section **6.1.1**.

The DAS28-CRP score corresponds to the current RA activity:

- 0 to < 2.6 Remission</li>
- 2.6 to < 3.2 Low disease activity (LDA)</li>
- 3.2 to ≤ 5.1 Moderate activity
- > 5.1 High activity

A DAS28-CRP score reduction by 1.2 represents the MCID.

# 6.2.3 DAS28-CRP Good/Moderate EULAR Response

DAS28-CRP good/moderate EULAR response is defined based on the combination of the current DAS28-CRP score and its improvement relative to baseline as illustrated in **Table 3**.

A subject is considered having a moderate treatment response if:

- DAS28-CRP score improvement from baseline to a given timepoint is > 0.6 and ≤ 1.2, and the DAS28-CRP score at that timepoint is ≤ 5.1; or
- DAS28-CRP score improvement from baseline to a given timepoint is > 1.2, and the DAS28-CRP score at that timepoint is > 3.2.

A subject is considered having a good treatment response if:

 DAS28-CRP score improvement from baseline to a given timepoint is > 1.2 and the DAS28-CRP score at that timepoint is ≤ 3.2.

Table 3: EULAR Response Criteria

| DAS28-CRP Score at | DAS28-CRP Score Decrease from Baseline Value to a Given Timepoint | | |
|---|---|---|---|
| a Given Timepoint | > 1.2 | > 0.6 to ≤ 1.2 | ≤ 0.6 |
| ≤3.2 | Good response | Moderate response | No response |
| $> 3.2 \text{ to} \le 5.1$ | Moderate response | Moderate response | No response |
| > 5.1 | Moderate response | No response | No response |

If the post-baseline DAS28-CRP score is missing, then the corresponding EULAR category will be missing.

Missing DAS28-CRP values will be set as missing.


#### Doc# CLP-008 Rev C, 15JUL2024



#### 6.2.4 CDAI

The Clinical Disease Activity Index (CDAI) is a composite score consisting of the sum of:

- SJC28
- TJC28
- SGA/10
- EGA/10

The CDAI score is calculated as follows and ranges from 0 to 76 with higher values representing higher disease activity:

$$CDAI = TJC28 + SJC28 + SGA + EGA$$

The CDAI score corresponds to the current RA activity:

- 0 to ≤ 2.8 Remission
- >2.8 to ≤ 10 Low disease activity (LDA)
- >10 to ≤ 22 Moderate activity
- > 22 High activity

The MCID varies depending on RA activity at baseline:

- -12 for high activity
- -6 for moderate activity
- 1 for low activity

If one of the components is missing at a given assessment point, no imputations will be done, and the CDAI value for that assessment will be set to missing. An alternative imputation method for missing components may be applied as described in Section **6.1.1**.

#### 6.2.5 RAMRIS

RAMRIS is the standardized system for RA MRI scoring of 4 different types of joint pathologies in the wrist and the hand. A total score for each pathology is generated by the summation of individual joint/bone scores as follows:

- Synovitis. 8 joints each scored on a scale from 0 = normal to 3 = severe, resulting in a total score from 0 to 24.
- Bone erosion. 25 bones each scored on a scale from 0 to 10, resulting in a total score from 0 to 250. An increase of > 0.5 from baseline to Week 12 will represent disease progression.
- Osteitis. 25 bones scored on a scale from 0 to 3, resulting in a total score from 0 to 75.




 CARLOS (cartilage loss). 25 joints each scored on a scale from 0 to 4, resulting in a total score from 0 to 100.

Subjects will undergo MRI at Week 24, and the MRI images will be scored by the same independent centralized blinded readers who scored baseline and Week 12 MRIs. Scores for each bone/joint will be calculated as the average of the score provided by each of the two readers. If a RAMRIS score from one of the readers is missing, then the RAMRIS score from the other reader will be used. If the score was missing for both readers at any given time point, the average score is considered missing. An imputation method for missing components may be applied as described in Section 6.1.1.

The smallest detectable change (SDC) will be calculated for each of the joint pathologies to assess whether a patient experienced a change beyond measurement error. The SDC is calculated as:

 $\pm 1.96 \text{ x SD}_{\Delta(\text{CHANGE SCORES})} / (\sqrt{2} \text{ x } \sqrt{k})$ 

where CHANGE SCORE = change in RAMRIS total score between two timepoints,  $SD_{\Delta(CHANGESCORES)}$  represents the standard deviation of difference in change scores between the two readers, and k= the number of readers (Bruynesteyn et al., 2005).

In addition, subgroup analyses will be performed for subjects with and without baseline joint damage that is predictive of future progression (Gandjbakhch et al, 2014).

#### 6.2.6 SF-36

Health-related quality of life will be assessed using the subject-completed Medical Outcomes Study Short-Form 36 (SF-36), which is a generic health survey that contains 36 questions covering eight domains of health. The SF-36 yields an 8-scale profile of functional health and well-being scores as well as physical and mental component health summary scores. The version 2, 4-week recall questionnaire will be used. Recoding, calculations and standardization will be done as recommended in the User's manual for the SF-36 (Mariush, 2011). Each of the 8 domain scores is the sum of some of the overall 36 item scores.

The initial domain scores are the sum of individual item scores:

- General Health
- Physical Functioning
- Role Physical
- Role Emotional
- Social Functioning
- Bodily Pain
- Vitality




#### Mental Health

Domain scores will only be calculated if less than half of the item scores are missing. An imputation method for missing components may be applied as described in Section 5.5.1.

# 6.2.7 EQ-5D-5L

A standardized instrument for measuring general health status within the following 5 dimensions:

- Mobility
- Self-care
- Usual activities
- Pain/discomfort
- Anxiety/depression

Each dimension is scored on 5-point scale as:

- 1 = No problems
- 2 = Slight problems
- 3 = Moderate problems
- 4 = Severe problems
- 5 = Extreme problems

General health status is scored on a VAS (0 = poor to 100 = the best). An imputation method for missing components may be applied as described in Section 5.5.1.

Reduction in the proportion of subjects with problems (moderate, severe or extreme) will represent improvement.

An EQ-5D summary index score can be derived by applying a formula that attaches weights, or index values, to each of the levels in each dimension. The index is calculated by deducting the appropriate weights from the value for full health (i.e., 1). Value sets are country specific and can be obtained from the EuroQol website (EuroQol Research Foundation, 2023).

# 6.3 Subgroup Analyses

Response rates for the key exploratory efficacy endpoints, as specified in **Table 2**, will be examined using the following subgroups:

- Number of prior biologic and targeted synthetic DMARDs (e.g., < 4 vs. ≥ 4)</li>
- Prior use of JAKi (Yes vs. No)
- RA activity at baseline (DAS28-CRP ≤ 5.1 vs. DAS28-CRP > 5.1)




- RA severity at imitation of stimulation (< 4 TJC28 or < 4 SJC28 vs. ≥ 4 TJC28 and ≥ 4 SJC28)</li>
- Augmented therapy (yes, no)

After completion of Week 12 assessments, additional treatment for RA may be provided at any time. The decision about the need, type and timing of treatment is left to the discretion of the Co-PI Rheumatologist and the subject. The initiation of these treatments with study treatment during open-label follow-up is considered "augmented therapy". Subjects combining stimulation with the following additions to RA therapy will fall into the augmented therapy subgroup for analysis of response rates for key exploratory efficacy endpoints at specific timepoints:

- Prednisone equivalent >10 mg/day. If average daily corticosteroid use exceeds 10 mg/day prednisone after a period (time from previous visit up to the day before the current visit), the subject is assigned to the augmented therapy subgroup for that visit.
- Corticosteroid injection. If subject received a corticosteroid injection within 30 days prior to
  a study visit, the subject is assigned to the augmented therapy subgroup for that visit.
- b/ts/csDMARD. Subjects who receive treatment with biologic, targeted synthetic, or additional
  conventional synthetic DMARD, or increased dose of background conventional synthetic
  DMARD will be assigned to the augmented therapy subgroup for all subsequent visits.

#### 7 SAFETY EVALUATION

#### 7.1 AE and SAEs

The incidence of AEs and SAEs in the safety population (see Section 5.2) will be tabulated through Week 264 (end of study). Each AE will be evaluated by clinical investigators in terms of seriousness, severity (i.e., mild, moderate, severe) and strength of relationship (i.e., not related, unlikely related, probably related, definitely related, indeterminate) to the implant procedure, explant procedure, implant device, stimulation and Energizer. Any AE that is determined by a participating investigator to be related (definitely related or probably related) to the implant procedure, explant procedure, implant device, stimulation or Energizer will be categorized as device related.

For all AE tables, a subject reporting the same adverse event more than once will be counted once when calculating the number and percentage of subjects with that particular event. If a subject reports the same AE more than once or has the same AE on multiple occasions, the maximum severity grade and relationship to the study implant and/or study drug will be presented.

The frequencies and percentages of treatment-emergent adverse events will be presented by MedDRA system organ class (SOC) and preferred term (PT). Complete subject listings of all AE will be provided. For each AE the following will be specified: start and stop dates, severity grade, MedDRA SOC and PT, relationship (unlikely related, probably related, definitely related or indeterminate) to the implant procedure, explant procedure, implant device, stimulation or Energizer, and, as well as action taken, outcome of the adverse event, and seriousness.




#### 7.2 Protocol Deviations

All protocol deviations will be tabulated with reasons for deviations reviewed by sponsor and reported in compliance with the study protocol, IRB requirements and sponsor's SOPs.

Summary tables with the number and percentage of subjects with protocol deviations will be provided by type of deviation (**Appendix B**). A by-subject listing of all protocol deviations will be provided (**Appendix C**).

#### 7.3 Device Deficiencies

All device deficiencies related to the identity, quality, durability, reliability, safety or performance of the study device, including device malfunctions, use errors, and inadequate labelling will be tabulated. Summary tables with the number and percentage of device deficiencies will be provided by type (**Appendix B**). A by-subject listing of all device malfunctions will be provided (**Appendix C**).

#### 8 STATISTICAL CONSIDERATIONS RELATED TO COVID-19

The statistical considerations detailed in this section are consistent with the FDA's guidance on the conduct of clinical trials during the COVID-19 pandemic and recommendations for the statistical analysis of the primary and key secondary endpoints to help ensure that the COVID-19-related changes to the RESET-RA study conduct will provide interpretable findings with correct statistical quantification of uncertainty.

# 8.1 Impact of COVID-19 on Study Integrity

Unavoidable protocol modifications may be required due to COVID-19 illness and/or COVID-19 control measures to protect subject safety and the to address its impact on the ability to collect data. The context and/or reasons for post-baseline events as they relate to COVID-19, such as discontinuation of treatment, withdrawal from the trial, use of alternative or rescue treatments, missed endpoint assessments, and the use of alternative endpoint assessment methods will be captured at the subject level. Information not specific to individual subjects, such as information on site closure (rheumatology or surgery) and its impact on disrupting administration of the investigational study device (i.e., implant procedure, device titration, device adjustments) will also be captured. This information at both the subject and site levels may be useful for incorporating into additional sensitivity analyses related to the impact of COVID-19.

### 8.2 COVID-19 Analysis Considerations

The impact of COVID-19 on the study integrity will be assessed and included into data summaries, including information on missing data, protocol deviations, subject discontinuation or interruption of the investigational treatment, subject withdrawal, and changes in endpoint assessments (e.g., virtual visit).

Extending the protocol-defined windows and using alternative remote methods for assessment of the exploratory efficacy endpoints may be warranted to address the impact of COVID-19. The data




from these late or modified assessments can be leveraged based on scientifically based rationale and clinical judgement.

The available data at baseline and post-baseline, including COVID-19-related information will be leveraged using the prespecified methods for handling missing data.

#### 9 REFERENCES

Bruynesteyn K, Boers M, Kostense P, van der Linden S, van der Heijde D. Deciding on progression of joint damage in paired films of individual patients: smallest detectable difference or change. Ann Rheum Dis. 2005;64:179-182.

EuroQol Research Foundation. EQ-5D-5L. Online Available: https://euroqol.org/eq-5d-instruments/eq-5d-5l-about/. 2023. Accessed: 16Oct2023

FDA Guidance for Industry on Statistical Considerations for Clinical Trials During the COVID-19 Public Health Emergency. June 2020.

FDA Guidance for Industry, Investigators, and Institutional Review Boards on Conduct of Clinical Trials of Medical Products During COVID-19 Public Health Emergency. 2020; updated September 21, 2020.

Gandjbakhch F, et al. Determining a magnetic resonance imaging inflammatory activity acceptable state without subsequent radiographic progression in rheumatoid arthritis: results from a followup MRI study of 254 patients in clinical remission or low disease activity. J Rheumatol. 2014 Feb;41(2):398-406.

Maruish, M.. (Ed.). User's manual for the SF-36v2 Health Survey (3rd ed.). Lincoln, RI: QualityMetric Incorporated. 2011.






#### 10 APPENDICES

# Appendix A: Schedule of Assessments

| Assessment | Titration 4<br>(91 ± 2d³) | Titration 5<br>(98 ± 2d <sup>2</sup> ) | <b>Titration 6</b> (105 ± 2d²) | Week 24<br>(168 ± 7d²) | Week 36 $(252 \pm 14d^2)$ | Week 48 $(336 \pm 14d^2)$ | Week 60 $(420 \pm 14d^2)$ | Week 72 $(504 \pm 14d^2)$ | Week 84 $(588 \pm 14d^2)$ | Week 96 $(672 \pm 14d^2)$ | Week 108 $(756 \pm 14d^2)$ | Week 120 $(840 \pm 14d^2)$ | Week 132 $(924 \pm 14d^2)$ | Week 144<br>(1,008 ± 14d²) | Week 156 $(1,092 \pm 144^2)$ | Week 168<br>(1,176 ± 14d²) | Week 180 $(1,260 \pm 1444^2)$ | Week 192<br>(1,344 ± 14d²) | Week 204 $(1,428 \pm 14d^2)$ | Week 216<br>(1,512 ± 14d²) | Week 228<br>(1,396 ± 14d²) | Week 240<br>(1,1680 ± 14¢) | Week 252<br>(1,764± 14d²) | Week 264<br>(1,848 ± 14d²)<br>(End of Study) |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Vital signs | | | | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X |
| Pregnancy test (childbearing female) | X | X | X | X | X | X | X | x | x | X | X | x | X | X | X | X | X | X | X | X | X | X | X | X |
| RA disease activity<br>assessments <sup>1</sup> | | | | x | X | X | X | X | X | x | X | X | x | X | X | X | X | X | X | x | X | X | X | X |
| SF-36 & EQ-5D-5L<br>questionnaires | | | | X | | X | | | | X | | | | X | | | | X | | | | | | |
| Satisfaction questionnaire | П | | | X | | | | | | | | | | | | | | | | | | | | |
| Blood collection (CBC) | | | | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X |
| Blood collection (biomarkers) | | | | X | | | | | | | | | | | | | | | | | | | | |
| Hand MRI | | | | X | | | | | | | | | | | | | | | | | | | | |
| 12-lead ECG | | | | X | | X | | | | X | | | | X | | | | X | | | | | | |
| Device check & dose titration | X <sup>3</sup> | X <sup>3</sup> | $X^3$ | | | | | | | | | | | | | | | | | | | | | |
| Device check & dose<br>adjustment if needed | | | | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X |
| Device deficiency reporting | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X |
| Adverse event reporting | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X |
| Concomitant medication | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X |

Abbreviations: CBC, complete blood count; d, day; EGA, evaluator's global assessment; HAQ-DI, Health Assessment Questionnaire Disability Index; hsCRP, high-sensitivity C-reactive protein; MRI, magnetic resonance imaging; RA, rheumatoid arthritis; SGA, subject's global assessment; SJC, swollen joint count.


<sup>1</sup> RA disease activity assessments include: HAQ-DI, SGA, subject's pain assessment, TJC28, SJC28, EGA, and hsCRP. Subjects must have  $\geq$  4TJC28 and  $\geq$  4SJC28 at consent to be eligible.

<sup>&</sup>lt;sup>2</sup>From Day 0 (randomization).

<sup>3</sup> Dose titration is not performed if subject and Co-PI Rheumatologist decide that subject should not receive active stimulation in open-label, long-term follow-up period.



# Appendix B: Table Mockups

| Table 14.8.1.1 | Subject Disposition | 24 |
|---|---|---|
| Table 14.8.1.2 | Demographic and Baseline Characteristics | 25 |
| Table 14.8.2.1 | ACR20/50/70 Response | 29 |
| Table 14.8.2.1.1 | Subgroup Analysis of ACR20 Response: Prior b/tsDMARDs | 33 |
| Table 14.8.2.1.1.1 | Subgroup Analysis of ACR50 Response: Prior b/tsDMARDs | 36 |
| Table 14.8.2.1.1.2 | Subgroup Analysis of ACR70 Response: Prior b/tsDMARDs | 36 |
| Table 14.8.2.1.2 | Subgroup Analysis of ACR20 Response: Prior JAKi | 36 |
| Table 14.8.2.1.2.1 | Subgroup Analysis of ACR50 Response: Prior JAKi | 36 |
| Table 14.8.2.1.2.2 | Subgroup Analysis of ACR70 Response: Prior JAKi | 36 |
| Table 14.8.2.1.3 | Subgroup Analysis of ACR20 Response: RA Activity at Baseline | 37 |
| Table 14.8.2.1.3.1 | Subgroup Analysis of ACR50 Response: RA Activity at Baseline | 37 |
| Table 14.8.2.1.3.2 | Subgroup Analysis of ACR70 Response: RA Activity at Baseline | 37 |
| Table 14.8.2.1.4 | Subgroup Analysis of ACR20 Response: RA Severity at Initiation of Stimulation | 37 |
| Table 14.8.2.1.4.1 | Subgroup Analysis of ACR50 Response: RA Severity at Initiation of Stimulation | 37 |
| Table 14.8.2.1.4.2 | Subgroup Analysis of ACR70 Response: RA Severity at Initiation of Stimulation | 38 |
| Table 14.8.2.1.5 | Subgroup Analysis of ACR20 Response: RA Augmented Therapy | 38 |
| Table 14.8.2.1.5.1 S | Subgroup Analysis of ACR50 Response: RA Augmented Therapy | 38 |
| Table 14.8.2.1.5.2 S | Subgroup Analysis of ACR70 Response: RA Augmented Therapy | 38 |
| Table 14.8.2.2 | DAS28-CRP Moderate/Good EULAR Response | 38 |
| Table 14.8.2.2.1 | Subgroup Analysis EULAR Response: Prior b/tsDMARDs | 40 |
| Table 14.8.2.2.2 | Subgroup Analysis of EULAR Response: Prior JAKi | 43 |
| Table 14.8.2.2.3 | Subgroup Analysis of EULAR Response: RA Activity at Baseline | 43 |
| Table 14.8.2.2.4 | Subgroup Analysis of EULAR Response: RA Severity at Initiation of Stimulation | 43 |
| Table 14.8.2.2.5 | Subgroup Analysis of EULAR Response: RA Augmented Therapy | |
| Table 14.8.2.3 | DAS28-CRP MCID Response | |
| Table 14.8.2.3.1 | Subgroup Analysis DAS28-CRP MCID Response: Prior b/tsDMARDs | |
| Table 14.8.2.3.2 | Subgroup Analysis of DAS28-CRP MCID Response: Prior JAKi | 49 |
| Table 14.8.2.3.3 | Subgroup Analysis of DAS28-CRP MCID Response: RA Activity at Baseline | 49 |
| Table 14.8.2.3.4 | Subgroup Analysis of DAS28-CRP MCID Response: RA Severity at<br>Initiation of Stimulation | 49 |
| Table 14.8.2.3.5 | Subgroup Analysis of DAS28-CRP MCID Response: Augmented Therap | |
| Table 14.8.2.4 | HAQ-DI MCID Response | - |
| Table 14.8.2.4.1 | Subgroup Analysis HAQ-DI MCID Response: Prior b/tsDMARDs | 52 |
| Table 14.8.2.4.2 | Subgroup Analysis of HAQ-DI MCID Response: Prior JAKi | 55 |
| Table 14.8.2.4.3 | Subgroup Analysis of HAQ-DI MCID Response: RA Disease Activity at | |
| | Baseline | 55 |



## Doc# CLP-008 Rev C, 15JUL2024

| Table 14.8.2.4.4 | Subgroup Analysis of HAQ-DI MCID Response: RA Severity at Initiatio of Stimulation | |
|---|---|---|
| Table 14.8.2.4.5 | Subgroup Analysis of HAQ-DI MCID Response: Augmented Therapy | |
| Table 14.8.2.5 | TJC28 | 56 |
| Table 14.8.2.6 | SJC28 | 62 |
| Table 14.8.2.7 | Subject's Assessment of Pain | 68 |
| Table 14.8.2.8 | SGA | 68 |
| Table 14.8.2.9 | EGA | 68 |
| Table 14.8.2.10 | hsCRP | 68 |
| Table 14.8.2.11 | DAS28-CRP | 69 |
| Table 14.8.2.12 | CDAI | 73 |
| Table 14.8.2.13 | RAMRIS | 77 |
| Table 14.8.2.14 | EQ-5D-5L | 80 |
| Table 14.8.2.15 | SF-36 | 84 |
| Table 14.8.2.16 | Subject Satisfaction | 86 |
| Table 14.8.2.17 | Inflammatory Biomarkers | 87 |
| Table 14.8.2.18 | RA Augmented Therapy | 89 |
| Table 14.8.2.20 | Implant Performance | 92 |
| Table 14.8.3.1 | Adverse Events | 93 |
| Table 14.8.3.2 | Adverse Events by SOC and Maximum Severity: All Events | 96 |
| Table 14.8.3.3 | Implant Procedure-Related AEs by SOC and Maximum Severity: All Events | 98 |
| Table 14.8.3.4 | Implant Device-Related AEs by SOC and Maximum Severity: All Events | s100 |
| Table 14.8.3.5 | Stimulation-Related AEs by SOC and Maximum Severity: All Events | 101 |
| Table 14.8.3.6 | Energizer-Related AEs by SOC and Maximum Severity: All Events | 102 |
| Table 14.8.3.7 Expl | ant Procedure-Related Adverse Events by SOC and Maximum Severity: A Events | |
| Table 14.8.3.8 Devi | ice Deficiency | 103 |
| Table 14.8.3.9 Prote | ocol Deviations | 104 |



Table 14.8.1.1 Subject Disposition

| | TOL [1] | COL [2] | Overall |
|---|---|---|---|
| Number of subjects: | | | |
| TOL [1] | xxx | | |
| COL [2] | | xxx | |
| Overall population | | | XXX |
| Withdrawn | xxx | XXX | XXX |
| Completed study through Week 192 | XXX | XXX | xxx |
| Primary reason for withdrawal [3]: | | | |
| Subject decision to withdraw consent | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| Investigator decision or medical judgement | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| Lost to follow-up | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| Device malfunction | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| Adverse event | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| Subject no longer eligible | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| Death | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| Study terminated | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| Sponsor or IRB decision | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| Other | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |

Abbreviations: COL, Control to Open Label; ITT, intent to treat; TOL, Treatment to Open Label

[3] Percentage calculated based on each analysis population (i.e., TOL, COL, Overall).

Reference: Listing 16.x.x.x

SOURCE: xxxxx SAS 9.4 {program location} {run date/time}

Serial Number: c700c42a-b18e-4af7-8a24-9d2146ac6503 accessed by Melissa Evangelista (MEVANGELISTA) on Thu, 28 Aug 2025 18:20:31 GMT.

<sup>[1]</sup> Treatment to Open Label (TOL): The TOL population comprises treatment subjects from ITT population who received active stimulation through Week 12, completed Week 12 assessments, continued to receive active stimulation during open-label follow-up, and for whom follow-up data are available.

<sup>[2]</sup> Control to Open Label (COL): The COL population comprises control subjects from ITT population who received non-active (sham) stimulation through Week 12, switched to active stimulation after completing Week 12 assessments, continued to receive active stimulation during open-label follow-up, and for whom follow-up data are available.



Table 14.8.1.2 Demographic and Baseline Characteristics

| N | | TOL [1] | COL[2] | Overall [3] |
|---|---|---|---|---|
| N | N | | xxx (xx.x%) | xxx (xx.x%) |
| Mean (SD) XX, X (XX,XX) XX,X (XX,XX) XX,X (XX,XX) Median XX,XX XX,XX XX,XX Min-Max XX,X (XX,XX) XXX XXX,XX Gender [3] SXX (XX,X%) XXX (XX,X%) XXX (XX,X%) Female XXX (XX,X%) XXX (XX,X%) XXX (XX,X%) Female XXX (XX,X%) XXX (XX,X%) XXX (XX,X%) Hispanic or Latino XXX (XX,X%) XXX (XX,X%) XXX (XX,X%) Not Hispanic or Latino XXX (XX,X%) XXX (XX,X%) XXX (XX,X%) Not disclosed XXX (XX,X%) XXX (XX,X%) XXX (XX,X%) Race [3][4] XXX XXX (XX,X%) XXX (XX,X%) XXX (XX,X%) Asian XXX (XX,X%) XXX (XX,X%) XXX (XX,X%) XXX (XX,X%) Black or African American XXX (XX,X%) XXX (XX,X%) XXX (XX,X%) XXX (XX,X%) Native Hawaiian or other Pacific Islander XXX (XX,X%) XXX (XX,X%) XXX (XX,X%) White XXX XXX XXX XXX N XX XXX | Age (years) | | | |
| Median XXXXX XXXXX XXXXX XXXXX XXXXXX XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | N | XXX | xxx | xxx |
| Min-Max xxx, xxx xxx xxxx xxx xxxx Gender [3] Male xxx (xxx%) xxx (xxx%) xxx (xxxx%) Female xxx (xxxx%) xxx (xxxx%) xxx (xxxx%) Ethnicity [3] Thispanic or Latino xxx (xxxx%) xxx (xxxx%) xxx (xxxx%) Not Hispanic or Latino xxx (xxxx%) xxx (xxxx%) xxx (xxxx%) xxx (xxxx%) Not disclosed xxx (xxxx%) xxx (xxxx%) xxx (xxxx%) xxx (xxxx%) Race [3][4] Xxx (xxxx%) xxx (xxxx%) xxx (xxxx%) xxx (xxxx%) Asian xxx (xxxx%) xxx (xxxx%) xxx (xxxx%) xxx (xxxx%) Black or African American xxx (xxxx%) xxx (xxxx%) xxx (xxxx%) xxx (xxxx%) Native Hawaiian or other Pacific Islander xxx (xxxx%) xxx (xxxx%) xxx (xxxx%) xxx (xxxx%) White xxx (xxxx%) xxx (xxxx%) xxx (xxxx%) xxx (xxxx%) Other xxx (xxxx%) xxx (xxxx%) xxx (xxxx%) xxx (xxxx%) N xxx (xxxxx) xxx (xxxxx) xxx (xxxxx) <td>Mean (SD)</td> <td>xx.x (xx.xx)</td> <td>xx.x (xx.xx)</td> <td>xx.x (xx.xx)</td> | Mean (SD) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) |
| Gender [3] Male | Median | xx.xx | xx.xx | xx.xx |
| Male Female xxx (xx.x%) xxx (xx.x%) xxx (xx.x%) Ethnicity [3] Thispanic or Latino xxx (xx.x%) xxx (xx.x%) xxx (xx.x%) Not Hispanic or Latino xxx (xx.x%) xxx (xx.x%) xxx (xx.x%) xxx (xx.x%) Not disclosed xxx (xx.x%) xxx (xx.x%) xxx (xx.x%) xxx (xx.x%) Race [3][4] Thispanic or Latino xxx (xx.x%) xxx (xx.x%) xxx (xx.x%) American Indian or A laska Native xxx (xx.x%) xxx (xx.x%) xxx (xx.x%) Asian xxx (xx.x%) xxx (xx.x%) xxx (xx.x%) Asian American xxx (xx.x%) xxx (xx.x%) xxx (xx.x%) Native Hawaiian or other Pacific Islander xxx (xx.x%) xxx (xx.x%) xxx (xx.x%) White xxx (xx.x%) xxx (xx.x%) xxx (xx.x%) Other xxx (xx.x%) xxx (xx.x%) xxx (xx.x%) XX xxx (xx.x%) xxx (xx.x%) xxx (xx.x%) XX xxx (xx.xx) xxx (xx.x%) xxx (xx.x%) XX xxx (xx.x%) xxx (xx.x%) xxx (xx.x%) <td>Min-Max</td> <td>xx.x - xx.x</td> <td>xx.x - xx.x</td> <td>xx.x - xx.x</td> | Min-Max | xx.x - xx.x | xx.x - xx.x | xx.x - xx.x |
| Female xxx (xx.x%) xxx (xx.x%) xxx (xx.x%) Ethnicity [3] | Gender [3] | | | |
| Ethnicity [3] Hispanic or Latino Not Hispanic or Latino Not disclosed Race [3][4] American Indian or Alaska Native Assian Stanta American Black or African American Native Hawaiian or other Pacific Islander White Other Stanta (SD) Not Marked (SD) N | Male | xxx (xx.x%) | xxx (xx.x%) | xxx (xx,x%) |
| Hispanic or Latino xxx (xx.x%) xxx (xx.x%) xxx (xx.x%) Not Hispanic or Latino xxx (xx.x%) xxx (xx.x%) xxx (xx.x%) Not disclosed xxx (xx.x%) xxx (xx.x%) xxx (xx.x%) Race [3][4] | Female | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| Not Hispanic or Latino xxx (xx.x%) xxx (xx.x%) xxx (xx.x%) Not disclosed xxx (xx.x%) xxx (xx.x%) xxx (xx.x%) Race [3][4] | Ethnicity [3] | | | |
| Not Hispanic or Latino xxx (xx.x%) xxx (xx.x%) xxx (xx.x%) Not disclosed xxx (xx.x%) xxx (xx.x%) xxx (xx.x%) Race [3][4] | Hispanic or Latino | xxx (xx.x%) | xxx (xx.x%) | xxx (xx,x%) |
| Race [3][4] XXX (XX.X%) XXX (XX.XX) | Not Hispanic or Latino | xxx (xx.x%) | | xxx (xx,x%) |
| American Indian or Alaska Native xxx (xx.x%) xxx (xx.x%) xxx (xx.x%) Asian xxx (xx.x%) xxx (xx.x%) xxx (xx.x%) Black or African American xxx (xx.x%) xxx (xx.x%) xxx (xx.x%) Native Hawaiian or other Pacific Islander xxx (xx.x%) xxx (xx.x%) xxx (xx.x%) White xxx (xx.x%) xxx (xx.x%) xxx (xx.x%) Other xxx (xx.x%) xxx (xx.x%) xxx (xx.x%) RA duration (years) [3] xxx xxx xxx xxx N xx xxx xxx xxx xxx Mean (SD) xx.x (xx.xx) xx.x (xx.xx) xx.x xx.x Min-Max xx xx.x xx.x xx.x xx.x BMI (kg/m²) xx xx xx xx xx N xx xx xx xx xx | Not disclosed | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| American Indian or Alaska Native xxx (xx.x%) xxx (xx.x%) xxx (xx.x%) Asian xxx (xx.x%) xxx (xx.x%) xxx (xx.x%) Black or African American xxx (xx.x%) xxx (xx.x%) xxx (xx.x%) Native Hawaiian or other Pacific Islander xxx (xx.x%) xxx (xx.x%) xxx (xx.x%) White xxx (xx.x%) xxx (xx.x%) xxx (xx.x%) Other xxx (xx.x%) xxx (xx.x%) xxx (xx.x%) RA duration (years) [3] xxx xxx xxx xxx N xx xxx xxx xxx xxx Mean (SD) xx.x (xx.xx) xx.x (xx.xx) xx.x xx.x Min-Max xx xx.x xx.x xx.x xx.x BMI (kg/m²) xx xx xx xx xx N xx xx xx xx xx | Race [3][4] | | | |
| Black or African American xxx (xx.x%) xxx (xx.x%) xxx (xx.x%) Native Hawaiian or other Pacific Islander xxx (xx.x%) xxx (xx.x%) xxx (xx.x%) White xxx (xx.x%) xxx (xx.x%) xxx (xx.x%) Other xxx (xx.x%) xxx (xx.x%) xxx (xx.x%) RA duration (years) [3] xxx xxx xxx xxx N xx xx.x (xx.xx) xxx xxx Mean (SD) xx.x (xx.xx) xx.x (xx.xx) xx.x (xx.xx) Median xx.x xx.x xx.x xx.x Min-Max xx.x - xx.x xx.x - xx.x xx.x - xx.x BMI (kg/m²) xx xx xx xx N xx xx xx xx Mean (SD) xxx.x (xxx.xx) xxx.x (xxx.xx) xxx.x (xxx.xx) | | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| Native Hawaiian or other Pacific Islander xxx (xx.x%) xxx (xx.x%) xxx (xx.x%) White xxx (xx.x%) xxx (xx.x%) xxx (xx.x%) Other xxx (xx.x%) xxx (xx.x%) xxx (xx.x%) RA duration (years) [3] xxx xxx xxx N xxx xxx xxx Mean (SD) xx.x (xx.xx) xx.x (xx.xx) xx.x (xx.xx) Median xx.xx xx.xx xx.xx Min-Max xx.x - xx.x xx.x - xx.x xx.x - xx.x BMI (kg/m²) xx xx xx xx N xx xx xx xx Mean (SD) xxx.x (xxx.xx) xxx.x (xxx.xx) xxx.x (xxx.xx) | Asian | xxx (xx.x%) | xxx (xx.x%) | xxx (xx,x%) |
| White Other xxx (xx.x%) xxx (xx.x%) xxx (xx.x%) xxx (xx.x%) xxx (xx.x%) RA duration (years) [3] xxx xxx xxx xxx xxx xxx xxx xxx xxx N | Black or African American | xxx (xx.x%) | xxx (xx.x%) | xxx (xx,x%) |
| Other xxx (xxx%) xxx (xxx%) xxx (xxx%) RA duration (years) [3] XXX XXX XXX N XXX XXX XXX Mean (SD) XX.X (XX.XX) XX.X (XX.XX) XX.X (XX.XX) Median XX.X (XXXX) XX.X (XXXXX) XX.X (XXX.XX) Min-Max XX XX.X - XX.X XX.X - XX.X BMI (kg/m²) XX XX XX N XX XX XX Mean (SD) XXX.X (XXX.XX) XXX.X (XXX.XX) XXX.X (XXX.XX) | Native Hawaiian or other Pacific Islander | xxx (xx.x%) | xxx (xx.x%) | xxx (xx,x%) |
| RA duration (years) [3] N xxx xxx xxx Mean (SD) xx.x (xx.xx) xx.x (xx.xx) xx.x (xx.xx) Median xx.xx xx.xx xx.xx Min-Max xx.x - xx.x xx.x - xx.x xx.x - xx.x BMI (kg/m²) xx xx xx N xx xx xx Mean (SD) xxx.x (xxx.xx) xxx.x (xxx.xx) xxx.x (xxx.xx) | White | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| N xxx xxx xxx Mean (SD) xx.x (xx.xx) xx.x (xx.xx) xx.x (xx.xx) Median xx.xx xx.xx xx.xx Min-Max xx.x - xx.x xx.x - xx.x xx.x - xx.x BMI (kg/m²) xx xx xx N xx xx xx Mean (SD) xxx.x (xxx.xx) xxx.x (xxx.xx) xxx.x (xxx.xx) | Other | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| Mean (SD) xx.x (xx.xx) xx.x (xx.xx) xx.x (xx.xx) Median xx.xx xx.xx xx.xx Min-Max xx.x - xx.x xx.x - xx.x xx.x - xx.x BMI (kg/m²) xx xx xx N xx xx xx Mean (SD) xxx.x (xxx.xx) xxx.x (xxx.xx) xxx.x (xxx.xx) | RA duration (years) [3] | | | |
| Median xx.xx xx.xx xx.xx Min-Max xx.x - xx.x xx.x - xx.x xx.x - xx.x BMI (kg/m²) xx xx xx N xx xx xx Mean (SD) xxx.x (xxx.xx) xxx.x (xxx.xx) xxx.x (xxx.xx) | N | xxx | xxx | XXX |
| Min-Max xx.x - xx.x xx.x - xx.x xx.x - xx.x BMI (kg/m²) xx xx xx N xx xx xx Mean (SD) xxx.x (xxx.xx) xxx.x (xxx.xx) xxx.x (xxx.xx) | Mean (SD) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) |
| BMI (kg/m²) N xx xx xx Mean (SD) xxx.x (xxx.xx) xxx.x (xxx.xx) | Median | xx.xx | XX.XX | xx.xx |
| N xx xx xx xx Mean (SD) xxx.x (xxx.xx) xx | Min-Max | xx.x - xx.x | xx.x - xx.x | xx.x - xx.x |
| N xx xx xx xx Mean (SD) xxx.x (xxx.xx) xx | BMI (kg/m²) | | | |
| | | xx | XX | xx |
| Median xxx.xx xxx.xx xxx.xx | Mean (SD) | xxx.x (xxx.xx) | xxx.x (xxx.xx) | xxx.x (xxx.xx) |
| | Median | xxx.xx | xxx.xx | xxx.xx |




## Doc# CLP-008 Rev C, 15JUL2024

| | TOL [1] | COL[2] | Overall [3] |
|---|---|---|---|
| Min-Max | xxx.x - xxx.x | xxx.x - xxx.x | xxx.x - xxx.x |
| F [3] | | | |
| Positive | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| CPA [3] | | | |
| Positive | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| erology for RF and/or ACPA [3] | | | |
| Positive | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| sCRP (mg/L) | | | |
| N | XX | XX | XX |
| Mean (SD) | xxx.x (xxx.xx) | xxx.x (xxx.xx) | xxx.x (xxx.xx) |
| Median | xxx.xx | xxx.xx | xxx,xx |
| Min-Max | xxx.x - xxx.x | xxx.x - xxx.x | xxx.x - xxx.x |
| JC28 | | | |
| N | XX | xx | XX |
| Mean (SD) | xxx.x (xxx.xx) | xxx.x (xxx.xx) | xxx.x (xxx.xx) |
| Median | xxx.xx | xxx.xx | XXX.XX |
| Min-Max | xxx.x - xxx.x | xxx.x - xxx.x | xxx.x - xxx.x |
| JC28 | | | |
| N | XX | xx | XX |
| Mean (SD) | xxx.x (xxx.xx) | xxx.x (xxx.xx) | xxx.x (xxx.xx) |
| Median | xxx.xx | xxx.xx | xxx,xx |
| Min-Max | xxx.x - xxx.x | xxx.x - xxx.x | xxx.x - xxx.x |
| DAI score | | | |
| N | xx | xx | XX |
| Mean (SD) | xxx.x (xxx.xx) | xxx.x (xxx.xx) | xxx.x (xxx.xx) |
| Median | xxx.xx | xxx.xx | xxx,xx |
| Min-Max | xxx.x - xxx.x | xxx.x - xxx.x | xxx.x - xxx.x |
| AS28-CRP score | | | |
| N | xx | xx | XX |
| Mean (SD) | xxx.x (xxx.xx) | xxx.x (xxx.xx) | xxx.x (xxx.xx) |



## Doc# CLP-008 Rev C, 15JUL2024

| | TOL [1] | COL[2] | Overall [3] |
|---|---|---|---|
| Median | xxx.xx | xxx.xx | XXX,XX |
| Min-Max | xxx.x - xxx.x | xxx.x - xxx.x | xxx.x - xxx.x |
| HAQ-DI score | | | |
| N | xx | xx | XX |
| Mean (SD) | xxx.x (xxx.xx) | xxx.x (xxx.xx) | xxx.x (xxx.xx) |
| Median | xxx.xx | xxx.xx | XXX.XX |
| Min-Max | xxx.x - xxx.x | xxx.x - xxx.x | xxx.x - xxx.x |
| EQ-5D-5L Index | | | |
| N | xx | XX | XX |
| Mean (SD) | xxx.x (xxx.xx) | xxx.x (xxx.xx) | xxx.x (xxx.xx) |
| Median | xxx.xx | xxx.xx | xxx.xx |
| Min-Max | xxx.x - xxx.x | xxx.x - xxx.x | xxx.x - xxx.x |
| EQ-VAS | | | |
| N | xx | XX | XX |
| Mean (SD) | xxx.x (xxx.xx) | xxx.x (xxx.xx) | xxx.x (xxx.xx) |
| Median | xxx.xx | xxx.xx | xxx.xx |
| Min-Max | xxx.x - xxx.x | xxx.x - xxx.x | xxx.x - xxx.x |
| SF-36 MCS | | | |
| N | xx | XX | XX |
| Mean (SD) | xxx.x (xxx.xx) | xxx.x (xxx.xx) | xxx.x (xxx.xx) |
| Median | xxx.xx | xxx.xx | xxx.xx |
| Min-Max | xxx.x - xxx.x | xxx.x - xxx.x | xxx.x - xxx.x |
| SF-36 PCS | | | |
| N | xx | xx | XX |
| Mean (SD) | xxx.x (xxx.xx) | xxx.x (xxx.xx) | xxx.x (xxx.xx) |
| Median | xxx.xx | xxx.xx | xxx.xx |
| Min-Max | xxx.x - xxx.x | xxx.x - xxx.x | xxx.x - xxx.x |
| Number of prior b/ts DMARDs | | | |
| N | xx | xx | XX |
| Mean (SD) | xxx.x (xxx.xx) | xxx.x (xxx.xx) | xxx.x (xxx.xx) |
| Median | xxx.xx | xxx.xx | xxx.xx |
| Min-Max | xxx.x - xxx.x | xxx.x - xxx.x | xxx.x - xxx.x |





| | TOL [1] | COL[2] | Overall [3] |
|---------------------------------|------------|------------|-------------|
| Number of prior b/ts DMARDs [3] | | | |
| 1 | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| 2 | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| 3 | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| 4 | | | |
| 5 | | | |
| 6 | | | |
| 7 | | | |
| 8 | | | |
| 9 | | | |
| 10+ | | | |
| Prior b/ts DMARDs [3] | | | |
| Anti-IL-1 agents | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Anti IL-6 agents | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Anti-TNF agents | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| B-cell depleting agents | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| JAKi | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| CTLA4-Ig | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |

Abbreviations: ACPA, anti-citrullinated protein antibodies; b/tsDMARD, biologic or targeted synthetic disease-modifying antirheumatic drug; CDAI, Clinical Disease Activity Index; COL, Control to Open Label; CTLA4-Ig, cytotoxic T-lymphocyte-associated antigen-4 immunoglobulin; DAS, Disease Activity Score; eGFR, estimated glomerular filtration rate; EQ-5D-5L Index, EuroQol-5D-5L Index; EQ-VAS, EuroQol Visual Analogue Scale; HAQ-DI, Health Assessment Questionnaire Disability Index; hsCRP, high-sensitivity C-reactive protein; IL, interleukin; ITT, intent to treat; JAKi, Janus Kinase inhibitor; OL, open label; PTE, per-treatment-evaluable; RF, rheumatoid factor; SD, standard deviation; SJC, swollen joint count; SF-36 MCS, Short Form 36 Mental Component Summary Score; SF-36 PCS, Short Form 36 Physical Component Score; TJC, tender joint count; TNF, tumor necrosis factor; TOL, Treatment to Open Label

- [1] Treatment to Open Label (TOL): The TOL population comprises treatment subjects from ITT population who received active stimulation through Week 12, completed Week 12 assessments, continued to receive active stimulation during open-label follow-up, and for whom follow-up data are available.
- [2] Control to Open Label (COL): The COL population comprises control subjects from ITT population who received non-active (sham) stimulation through Week 12, switched to active stimulation after completing Week 12 assessments, continued to receive active stimulation during open-label follow-up, and for whom follow-up data are available.
- [3] Percentage calculated based on each analysis population (i.e., TOL, COL, Overall).
- [4] Race selected based on all that applied.

Reference: Listing 16.x.x.x

SOURCE: xxxxx SAS 9.4 {program location} {run date/time}}

SETPOINT MEDICAL

Doc# CLP-008 Rev C, 15JUL2024

### Table 14.8.2.1 ACR20/50/70 Response

| Variable | TOL [1]<br>(N=xxx) | COL [2]<br>(N=xxx) |
|---|---|---|
| ACR20 response from baseline [4] | • | |
| Week 24 | | |
| N | xx | XX |
| Yes [3] | xx (xx.x%) | xx (xx.x%) |
| 95% CI | (xx.x, xx.x) | (xx.x, xx.x) |
| Repeat for: | | |
| Week 36 | | |
| Week 48 | | |
| Week 60 | | |
| Week 72 | | |
| Week 84 | | |
| Week 96 | | |
| Week 108 | | |
| Week 120 | | |
| Week 132 | | |
| Week 144 | | |
| Week 156 | | |
| Week 168 | | |
| Week 180 | | |
| Week 192 | | |
| ACR20 response from initiation of stimulation [5] | | |
| Week 24 | | |
| N | XX | XX |
| Yes [3] | xx (xx.x%) | xx (xx.x%) |
| 95% CI | (xx.x, xx.x) | (xx.x, xx.x) |
| Repeat for: | | |
| Week 36 | | |
| Week 48 | | |
| Week 60 | | |
| Week 72 | | |
| Week 84 | | |


# SETPOINT MEDICAL

## Doc# CLP-008 Rev C, 15JUL2024

| Variable | TOL [1]<br>(N=xxx) | COL [2]<br>(N=xxx) |
|---|---|---|
| Week 96 | (** *****) | (** ******) |
| Week 108 | | |
| Week 120 | | |
| Week 132 | | |
| Week 144 | | |
| Week 156 | | |
| Week 168 | | |
| Week 180 | | |
| Week 192 | | |
| ACR50 response from baseline [4] | | |
| Week 24 | | |
| N | XX | XX |
| Yes [3] | xx (xx.x%) | xx (xx.x%) |
| 95% CI | (xx.x, xx.x) | (xx.x, xx.x) |
| Repeat for: | | |
| Week 36 | | |
| Week 48 | | |
| Week 60 | | |
| Week 72 | | |
| Week 84 | | |
| Week 96 | | |
| Week 108 | | |
| Week 120 | | |
| Week 132 | | |
| Week 144 | | |
| Week 156 | | |
| Week 168 | | |
| Week 180 | | |
| Week 192 | | |
| ACR 50 response from initiation of stimulation [5] | | |
| Week 24 | | |
| N | xx | xx |
| Yes [3] | xx (xx.x%) | xx (xx.x%) |
| 95% CI | (xx.x, xx.x) | (xx.x, xx.x) |
| 7074 01 | (44.4, 44.4) | (1111, 1111) |




| Variable | TOL [1]<br>(N=xxx) | COL [2]<br>(N=xxx) |
|----------------------------------|--------------------|--------------------|
| Repeat for: | | |
| Week 36 | | |
| Week 48 | | |
| Week 60 | | |
| Week 72 | | |
| Week 84 | | |
| Week 96 | | |
| Week 108 | | |
| Week 120 | | |
| Week 132 | | |
| Week 144 | | |
| Week 156 | | |
| Week 168 | | |
| Week 180 | | |
| Week 192 | | |
| ACR70 Response from baseline [4] | | |
| Week 24 | | |
| N | XX | xx |
| Yes [3] | xx (xx.x%) | xx (xx.x%) |
| 95% CI | (xx.x, xx.x) | (xx.x, xx.x) |
| Repeat for: | | |
| Week 36 | | |
| Week 48 | | |
| Week 60 | | |
| Week 72 | | |
| Week 84 | | |
| Week 96 | | |
| Week 108 | | |
| Week 120 | | |
| Week 132 | | |
| Week 144 | | |
| Week 156 | | |
| Week 168 | | |
| Week 180 | | |




| Variable | TOL [1]<br>(N=xxx) | COL [2]<br>(N=xxx) |
|---|---|---|
| Week 192 | (iv and) | (11 720) |
| ACR70 response from initiation of stimulation [5] | | |
| Week 24 | | |
| N | XX | XX |
| Yes [3] | xx (xx.x%) | xx (xx,x%) |
| 95% CI | (xx.x, xx.x) | (xx.x, xx.x) |
| Repeat for: | | |
| Week 36 | | |
| Week 48 | | |
| Week 60 | | |
| Week 72 | | |
| Week 84 | | |
| Week 96 | | |
| Week 108 | | |
| Week 120 | | |
| Week 132 | | |
| Week 144 | | |
| Week 156 | | |
| Week 168 | | |
| Week 180 | | |
| Week 192 | | |

Abbreviations: ACR, American College of Rheumatology; CI, confidence interval; COL, Control to Open Label; TOL, Treatment to Open Label

- [1] Treatment to Open Label (TOL): The TOL population comprises treatment subjects from ITT population who received active stimulation through Week 12, completed Week 12 assessments, continued to receive active stimulation during open-label follow-up, and for whom follow-up data are available.
- [2] Control to Open Label (COL): The COL population comprises control subjects from ITT population who received non-active (sham) stimulation through Week 12, switched to active stimulation after completing Week 12 assessments, continued to receive active stimulation during open-label follow-up, and for whom follow-up data are available.
- [3] Percentage calculated based on each analysis population (i.e., TOL, COL)
- [4] Baseline on the day of informed consent for TOL and Week 12 for COL
- [5] Initiation of stimulation at Day 0 for TOL and Week 12 for COL

Reference: Listing 16.x.x.x

SOURCE: xxxxx SAS 9.4 {program location} {run date/time}}

Serial Number: c700c42a-b18e-4af7-8a24-9d2146ac6503 accessed by Melissa Evangelisfa (MEVANGELISTA) on Thu, 28 Aug 2025 18:20:31 GMT.


May not be reproduced outside of SetPoint Medical without written permission from Document Control.



Table 14.8.2.1.1 Subgroup Analysis of ACR20 Response: Prior b/tsDMARDs

| TOL [1] | COL [2] |
|-------------|--------------|
| (N=xxx) | (N=xxx) |
| XX | XX |
| x (xx.x%) | xx (xx.x%) |
| (x.x, xx.x) | (xx.x, xx.x) |
| XX | xx |
| x (xx.x%) | xx (xx.x%) |
| x.x, xx.x) | (xx.x, xx.x) |




| Variable | TOL [1]<br>(N=xxx) | COL [2]<br>(N=xxx) |
|---------------------|--------------------|--------------------|
| N | xx | xx |
| Yes [3] | xx (xx.x%) | xx (xx.x%) |
| 95% CI | (xx.x, xx.x) | (xx.x, xx.x) |
| Prior b/tsDMARD > 4 | | |
| Week 24 | | |
| N | xx | XX |
| Yes [3] | xx (xx.x%) | xx (xx.x%) |
| 95% CI | (xx.x, xx.x) | (xx.x, xx.x) |
| Repeat for: | | |
| Week 36 | | |
| Week 48 | | |
| Week 60 | | |
| Week 72 | | |
| Week 84 | | |
| Week 96 | | |
| Week 108 | | |
| Week 120 | | |
| Week 132 | | |
| Week 144 | | |
| Week 156 | | |
| Week 168 | | |
| Week 180 | | |
| Week 192 | | |

Abbreviations: ACR, American College of Rheumatology; CI, confidence interval; COL, Control to Open Label; TOL, Treatment to Open Label

- [1] Treatment to Open Label (TOL): The TOL population comprises treatment subjects from ITT population who received active stimulation through Week 12, completed Week 12 assessments, continued to receive active stimulation during open-label follow-up, and for whom follow-up data are available.
- [2] Control to Open Label (COL): The COL population comprises control subjects from ITT population who received non-active (sham) stimulation through Week 12, switched to active stimulation after completing Week 12 assessments, continued to receive active stimulation during open-label follow-up, and for whom follow-up data are available.
- [3] Percentage calculated based on each analysis population (i.e., TOL, COL)
- [4] Baseline on the day of informed consent for TOL and Week 12 for COL
- [5] Initiation of stimulation at Day 0 for TOL and Week 12 for COL


May not be reproduced outside of SetPoint Medical without written permission from Document Control.



Doc# CLP-008 Rev C, 15JUL2024

| Variable | TOL [1] | COL [2] |
|----------|---------|---------|
| Valiable | (N=xxx) | (N=xxx) |

Reference: Listing 16.x.x.x

SOURCE: xxxxx SAS 9.4 {program location} {run date/time}}


May not be reproduced outside of SetPoint Medical without written permission from Document Control.


Serial Number: c700c42a-b18e-4af7-8a24-9d2146ac6503 accessed by Melissa Evangelista (MEVANGELISTA) on Thu, 28 Aug 2025 18:20:31 GMT.



Table 14.8.2.1.1.1 Subgroup Analysis of ACR50 Response: Prior b/tsDMARDs

Repeat Table 14.8.2.1.1 for ACR50

Table 14.8.2.1.1.2 Subgroup Analysis of ACR70 Response: Prior b/tsDMARDs

Repeat Table 14.8.2.1.1 for ACR70

Table 14.8.2.1.2 Subgroup Analysis of ACR20 Response: Prior JAKi

Repeat Table 14.8.2.1.1 for Prior JAKi [Yes vs. No]

Add to abbreviations: JAKi, Janus kinase inhibitor.

Table 14.8.2.1.2.1 Subgroup Analysis of ACR50 Response: Prior JAKi

Repeat Table 14.8.2.1.1 for ACR50 and for Prior JAKi [Yes vs. No]

Table 14.8.2.1.2.2 Subgroup Analysis of ACR70 Response: Prior JAKi

Repeat Table 14.8.2.1.1 for ACR70 and for Prior JAKi [Yes vs. No]

Serial Number: c700c42a-b18e-4af7-8a24-9d2146ac6503 accessed by Melissa Evangelista (MEVANGELISTA) on Thu, 28 Aug 2025 18:20:31 GMT.



Table 14.8.2.1.3

Subgroup Analysis of ACR20 Response: RA Activity at Baseline

Repeat Table 14.8.2.1.1 for RA Disease Activity at Baseline [DAS28-CRP ≤ 5.1 vs DAS28-CRP > 5.1]

Add to abbreviations: DAS, Disease Activity Score.

Table 14.8.2.1.3.1

Subgroup Analysis of ACR50 Response: RA Activity at Baseline

Repeat Table 14.8.2.1.1 for ACR50 and RA Disease Activity at Baseline [DAS28-CRP ≤ 5.1 vs DAS28-CRP > 5.1]

Table 14.8.2.1.3.2

Subgroup Analysis of ACR70 Response: RA Activity at Baseline

Repeat Table 14.8.2.1.1 for ACR70 and for RA Disease Activity at Baseline [DAS28-CRP ≤ 5.1 vs DAS28-CRP > 5.1]

Table 14.8.2.1.4

Subgroup Analysis of ACR20 Response: RA Severity at Initiation of Stimulation

Repeat Table 14.8.2.1.1 for RA Severity at Initiation of Stimulation [<4 TJC28 or <4 SJC28 vs. ≥4 TJC28 and ≥4 SJC28]

Add to abbreviations: TJC, tender joint count; SJC, swollen joint count.

<u>Programming note</u>: For this analysis, remove the "from baseline" portion of the table.

Table 14.8.2.1.4.1

Subgroup Analysis of ACR50 Response: RA Severity at Initiation of Stimulation

Repeat Table 14.8.2.1.1 for ACR50 and for RA Severity at Initiation of Stimulation [<4 TJC28 or <4 SJC28 vs. ≥4 TJC28 and ≥4 SJC28]

Add to abbreviations: TJC, tender joint count; SJC, swollen joint count.




Programming note: For this analysis, remove the "from baseline" portion of the table.

Table 14.8.2.1.4.2

Subgroup Analysis of ACR70 Response: RA Severity at Initiation of Stimulation

Repeat Table 14.8.2.1.1 for ACR70 and for RA Severity at Initiation of Stimulation [<4 TJC28 or <4 SJC28 vs. ≥4 TJC28 and ≥4 SJC28]

Add to abbreviations: TJC, tender joint count; SJC, swollen joint count.

Programming note: For this analysis, remove the "from baseline" portion of the table.

Table 14.8.2.1.5

Subgroup Analysis of ACR20 Response: RA Augmented Therapy

Repeat Table 14.8.2.1.1 for ACR20 and RA Augmented Therapy [yes/no]

Table 14.8.2.1.5.1

Subgroup Analysis of ACR50 Response: RA Augmented Therapy

Repeat Table 14.8.2.1.1 for ACR50 and RA Augmented Therapy [yes/no]

Table 14.8.2.1.5.2

Subgroup Analysis of ACR70 Response: RA Augmented Therapy

Repeat Table 14.8.2.1.1 for ACR70 and RA Augmented Therapy [yes/no]

Table 14.8.2.2 DAS28-CRP Moderate/Good EULAR Response

| Variable | TOL [1] | COL [2] |
|----------|---------|---------|
| Variable | (N=xxx) | (N=xxx) |

DAS28-CRP moderate/good EULAR response from baseline [4]


# SETPOINT MEDICAL

## Doc# CLP-008 Rev C, 15JUL2024

| Variable | TOL [1]<br>(N=xxx) | COL [2]<br>(N=xxx) |
|---|---|---|
| Week 24 | ` ` ` | |
| N | xx | XX |
| Yes [3] | xx (xx.x%) | xx (xx.x%) |
| 95% CI | (xx.x%, xx.x%) | (xx.x%, xx.x%) |
| Repeat for: | | |
| Week 36 | | |
| Week 48 | | |
| Week 60 | | |
| Week 72 | | |
| Week 84 | | |
| Week 96 | | |
| Week 108 | | |
| Week 120 | | |
| Week 132 | | |
| Week 144 | | |
| Week 156 | | |
| Week 168 | | |
| Week 180 | | |
| Week 192 | | |
| DAS28-CRP moderate/good EULAR response from initiation of stimulation [5] | | |
| Week 24 | | |
| N | xx | xx |
| Yes [3] | xx (xx.x%) | xx (xx.x%) |
| 95% CI | (xx.x%, xx.x%) | (xx.x%, xx.x%) |
| Repeat for: | | |
| Week 36 | | |
| Week 48 | | |
| Week 60 | | |
| Week 72 | | |
| Week 84 | | |
| Week 96 | | |
| Week 108 | | |
| Week 120 | | |
| Week 132 | | |




Doc# CLP-008 Rev C, 15JUL2024

| Variable | TOL [1]<br>(N=xxx) | COL [2]<br>(N=xxx) |
|----------|--------------------|--------------------|
| Week 144 | | |
| Week 156 | | |
| Week 168 | | |
| Week 180 | | |
| Week 192 | | |

Abbreviations: CI, confidence interval; COL, Control to Open Label (COL): DAS, Disease Activity Score; EULAR, European League Against Rheumatism; hsCRP, High-sensitivity C-reactive protein; TOL, Treatment to Open Label (TOL)

- [1] Treatment to Open Label (TOL): The TOL population comprises treatment subjects from ITT population who received active stimulation through Week 12, completed Week 12 assessments, continued to receive active stimulation during open-label follow-up, and for whom follow-up data are available.
- [2] Control to Open Label (COL): The COL population comprises control subjects from ITT population who received non-active (sham) stimulation through Week 12, switched to active stimulation after completing Week 12 assessments, continued to receive active stimulation during open-label follow-up, and for whom follow-up data are available.
- [3] Percentage calculated based on each analysis population (i.e., TOL, COL)
- [4] Baseline on the day of informed consent for TOL and Week 12 for COL
- [5] Initiation of stimulation at Day 0 for TOL and Week 12 for COL

Reference: Listing 16.x.x.x

SOURCE: xxxxx SAS 9.4 {program location} {run date/time}}

#### Table 14.8.2.2.1 Subgroup Analysis EULAR Response: Prior b/tsDMARDs

| Variable | TOL [1]<br>(N=xxx) | COL [2]<br>(N=xxx) |
|---|---|---|
| DAS28-CRP moderate/severe EULAR response from baseline [4] | | |
| Prior b/tsDMARD < 4 Week 24 N Yes [3] 95% CI | xx<br>xx (xx.x%)<br>(xx.x, xx.x) | xx<br>xx (xx.x%)<br>(xx.x, xx.x) |
| Prior b/tsDMARD ≥ 4<br>Week 24 | | |




| Variable | TOL [1]<br>(N=xxx) | COL [2]<br>(N=xxx) |
|---|---|---|
| N | xx | xx |
| Yes [3] | xx (xx.x%) | xx (xx.x%) |
| 95% CI | (xx.x, xx.x) | (xx.x, xx.x) |
| Repeat for: | | |
| Week 36 | | |
| Week 48 | | |
| Week 60 | | |
| Week 72 | | |
| Week 84 | | |
| Week 96 | | |
| Week 108 | | |
| Week 120 | | |
| Week 132 | | |
| Week 144 | | |
| Week 156 | | |
| Week 168 | | |
| Week 180 | | |
| Week 192 | | |
| DAS28-CRP moderate/severe EULAR response from initiation of stimulation [5] Prior b/tsDMARD < 4 | | |
| Week 24 | | |
| N N | xx | xx |
| Yes [3] | xx (xx.x%) | xx (xx.x%) |
| 95% CI | (xx.x, xx.x) | (xx.x, xx.x) |
| 9370 C1 | (,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,, | (,,,,,,,,,,, |
| Harak A-DMADD S. A | | |
| Prior b/tsDMARD≥4 | | |
| Week 24 | | |
| Week 24<br>N | XX | XX |
| Week 24<br>N<br>Yes [3] | xx (xx.x%) | xx<br>xx (xx.x%) |
| Week 24<br>N | | |




Doc# CLP-008 Rev C, 15JUL2024

| /ariable | TOL [1]<br>(N=xxx) | COL [2]<br>(N=xxx) |
|----------|--------------------|--------------------|
| Week 36 | ( ) | ( |
| Week 48 | | |
| Week 60 | | |
| Week 72 | | |
| Week 84 | | |
| Week 96 | | |
| Week 108 | | |
| Week 120 | | |
| Week 132 | | |
| Week 144 | | |
| Week 156 | | |
| Week 168 | | |
| Week 180 | | |
| Week 192 | | |

Abbreviations: CI, confidence interval; COL, Control to Open Label; DAS, Disease Activity Score; EULAR, European League Against Rheumatism; hsCRP, High-sensitivity C-reactive protein; TOL, Treatment to Open Label

- [1] Treatment to Open Label (TOL): The TOL population comprises treatment subjects from ITT population who received active stimulation through Week 12, completed Week 12 assessments, continued to receive active stimulation during open-label follow-up, and for whom follow-up data are available.
- [2] Control to Open Label (COL): The COL population comprises control subjects from ITT population who received non-active (sham) stimulation through Week 12, switched to active stimulation after completing Week 12 assessments, continued to receive active stimulation during open-label follow-up, and for whom follow-up data are available.
- [3] Percentage calculated based on each analysis population (i.e., TOL, COL)
- [4] Baseline on the day of informed consent for TOL and Week 12 for COL
- [5] Initiation of stimulation at Day 0 for TOL and Week 12 for COL

Reference: Listing 16.x.x.x

SOURCE: xxxxx SAS 9.4 {program location} {run date/time}}



Table 14.8.2.2.2 Subgroup Analysis of EULAR Response: Prior JAKi

Repeat Table 14.8.2.2.1 for Prior JAKi [Yes vs. No]

Add to abbreviations: JAKi, Janus kinase inhibitor.

Table 14.8.2.2.3
Subgroup Analysis of EULAR Response: RA Activity at Baseline

Repeat Table 14.8.2.2.1 for RA Disease Activity at Baseline [DAS28-CRP ≤ 5.1 vs. DAS28-CRP > 5.1]

Add to abbreviations: DAS, Disease Activity Score.

Table 14.8.2.2.4
Subgroup Analysis of EULAR Response: RA Severity at Initiation of Stimulation

Repeat Table 14.8.2.2.1 for RA Severity at Initiation of Stimulation [<4 TJC28 or <4 SJC28 vs. ≥4 TJC28 and ≥4 SJC28]

Add to abbreviations: TJC, tender joint count; SJC, swollen joint count

Programming note: For this analysis, remove the "from baseline" portion of the table.

Table 14.8.2.2.5
Subgroup Analysis of EULAR Response: RA Augmented Therapy

Repeat Table 14.8.2.2.1 for RA Augmented Therapy [yes, no]



Table 14.8.2.3 DAS28-CRP MCID Response

| Variable | TOL [1]<br>(N=xxx) | COL[2]<br>(N=xxx) |
|---|---|---|
| DAS28-CRP response (MCID ≥ -1.2) from baseline [4] | (* : ::::/ | ( |
| Week 24 | | |
| N | xx | XX |
| Yes [3] | xx (xx.x%) | xx (xx.x%) |
| 95% CI | (xx.x%, xx.x%) | (xx.x%, xx.x% |
| Repeat for: | | |
| Week 36 | | |
| Week 48 | | |
| Week 60 | | |
| Week 72 | | |
| Week 84 | | |
| Week 96 | | |
| Week 108 | | |
| Week 120 | | |
| Week 132 | | |
| Week 144 | | |
| Week 156 | | |
| Week 168 | | |
| Week 180 | | |
| Week 192 | | |
| DAS28-CRP response (MCID ≥ -1.2) from initiation of stimulation [5] | | |
| Week 24 | | |
| N | XX | XX |
| Yes [3] | xx (xx.x%) | xx (xx.x%) |
| 95% CI | (xx.x%, xx.x%) | (xx.x%, xx.x% |
| Repeat for: | | |
| Week 36 | | |
| Week 48 | | |
| Week 60 | | |




Doc# CLP-008 Rev C, 15JUL2024

| Variable | TOL [1]<br>(N=xxx) | COL[2]<br>(N=xxx) |
|----------|--------------------|-------------------|
| Week 72 | (i, iiii) | (11 1111) |
| Week 84 | | |
| Week 96 | | |
| Week 108 | | |
| Week 120 | | |
| Week 132 | | |
| Week 144 | | |
| Week 156 | | |
| Week 168 | | |
| Week 180 | | |
| Week 192 | | |

Abbreviations: CI, confidence interval; COL, Control to Open Label; DAS, Disease Activity Score; CRP, C-reactive protein; MCID, minimal clinically important difference OL, TOL, Treatment to Open Label

- [1] Treatment to Open Label (TOL): The TOL population comprises treatment subjects from ITT population who received active stimulation through Week 12, completed Week 12 assessments, continued to receive active stimulation during open-label follow-up, and for whom follow-up data are available.
- [2] Control to Open Label (COL): The COL population comprises control subjects from ITT population who received non-active (sham) stimulation through Week 12, switched to active stimulation after completing Week 12 assessments, continued to receive active stimulation during open-label follow-up, and for whom follow-up data are available.
- [3] Percentage calculated based on each analysis population (i.e., TOL, COL)
- [4] Baseline on the day of informed consent for TOL and Week 12 for COL
- [5] Initiation of stimulation at Day 0 for TOL and Week 12 for COL

Reference: Listing 16.x.x.x

SOURCE: xxxxx SAS 9.4 {program location} {run date/time}}



### Table 14.8.2.3.1 Subgroup Analysis DAS28-CRP MCID Response: Prior b/tsDMARDs

| Variable | TOL [1]<br>(N=xxx) | COL [2]<br>(N=xxx) |
|---|---|---|
| DAS28-CRP response (MCID ≥ -1.2) from baseline [4] | (11 333) | (11 AAA) |
| Prior b/tsDMARD < 4 | | |
| Week 24 | | |
| N | XX | XX |
| Yes [3] | xx (xx.x%) | xx (xx.x%) |
| 95% CI | (xx.x, xx.x) | (xx.x, xx.x) |
| Prior b/tsDMARD ≥ 4 | | |
| Week 24 | | |
| N | XX | xx |
| Yes [3] | xx (xx.x%) | xx (xx.x%) |
| 95% CI | (xx.x, xx.x) | (xx.x, xx.x) |
| Repeat for: | | |
| Week 36 | | |
| Week 48 | | |
| Week 60 | | |
| Week 72 | | |
| Week 84 | | |
| Week 96 | | |
| Week 108 | | |
| Week 120 | | |
| Week 132 | | |
| Week 144 | | |
| Week 156 | | |
| Week 168 | | |
| Week 180 | | |
| Week 192 | | |
| DAS28-CRP Response (MCID ≥ -1.2) from initiation of stimulation [5] | | |
| Prior b/tsDMARD < 4 | | |




| Variable | TOL [1]<br>(N=xxx) | COL [2]<br>(N=xxx) |
|---------------------|--------------------|--------------------|
| Week 24 | , , | ì |
| N | XX | XX |
| Yes [3] | xx (xx.x%) | xx (xx.x%) |
| 95% CI | (xx.x, xx.x) | (xx.x, xx.x) |
| Prior b/tsDMARD ≥ 4 | | |
| Week 24 | | |
| N | XX | XX |
| Yes [3] | xx (xx.x%) | xx (xx.x%) |
| 95% CI | (xx.x, xx.x) | (xx.x, xx.x) |
| Repeat for: | | |
| Week 36 | | |
| Week 48 | | |
| Week 60 | | |
| Week 72 | | |
| Week 84 | | |
| Week 96 | | |
| Week 108 | | |
| Week 120 | | |
| Week 132 | | |
| Week 144 | | |
| Week 156 | | |
| Week 168 | | |
| Week 180 | | |
| Week 192 | | |

Abbreviations: CI, confidence interval; COL, Control to Open Label; DAS, Disease Activity Score; CRP, C-reactive protein; MCID, minimal clinically important difference; TOL, Treatment to Open Label

- [1] Treatment to Open Label (TOL): The TOL population comprises treatment subjects from ITT population who received active stimulation through Week 12, completed Week 12 assessments, continued to receive active stimulation during open-label follow-up, and for whom follow-up data are available.
- [2] Control to Open Label (COL): The COL population comprises control subjects from ITT population who received non-active (sham) stimulation through Week 12, switched to active stimulation after completing Week 12 assessments, continued to receive active stimulation during open-label follow-up, and for whom follow-up data are available.
- [3] Percentage calculated based on each analysis population (i.e., TOL, COL)
- [4] Baseline on the day of informed consent for TOL and Week 12 for COL




Doc# CLP-008 Rev C, 15JUL2024

| Variable | TOL [1]<br>(N=xxx) | COL [2]<br>(N=xxx) |
|---|---|---|
| [5] Initiation of stimulation at Day 0 for TOL and Week 12 for COL | | |

Reference: Listing 16.x.x.x

SOURCE: xxxxx SAS 9.4 {program location} {run date/time}}




Table 14.8.2.3.2 Subgroup Analysis of DAS28-CRP MCID Response: Prior JAKi

Repeat Table 14.8.2.3.1 for Prior JAKi [Yes vs. No]

Add to abbreviations: JAKi, Janus kinase inhibitor.

Table 14.8.2.3.3

Subgroup Analysis of DAS28-CRP MCID Response: RA Activity at Baseline

Repeat Table 14.8.2.3.1 for RA Activity at Baseline [DAS28-CRP ≤ 5.1 vs. DAS28-CRP > 5.1]

Add to abbreviations: DAS, Disease Activity Score.

Table 14.8.2.3.4

Subgroup Analysis of DAS28-CRP MCID Response: RA Severity at Initiation of Stimulation

Repeat Table 14.8.2.3.1 for RA Severity at Initiation of Stimulation [<4 TJC28 or <4 SJC28 vs. ≥4 TJC28 and ≥4 SJC28]

Add to abbreviations: TJC, tender joint count; SJC, swollen joint count

Programming note: For this analysis, remove the "from baseline" portion of the table.

Table 14.8.2.3.5

Subgroup Analysis of DAS28-CRP MCID Response: Augmented Therapy

Repeat Table 14.8.2.3.1 for RA Augmented Therapy [yes, no]





### Table 14.8.2.4 HAQ-DI MCID Response

| Variable | TOL [1]<br>(N=xxx) | COL [2]<br>(N=xxx) |
|---|---|---|
| HAQ-DI response (MCID ≥ -0.22) from baseline [4] | (11 1001) | (21 1414) |
| Week 24 | | |
| N | XX | xx |
| Yes [3] | xx (xx.x%) | xx (xx.x%) |
| 95% CI | (xx.x%, xx.x%) | (xx.x%, xx.x%) |
| Repeat for: | | |
| Week 36 | | |
| Week 48 | | |
| Week 60 | | |
| Week 72 | | |
| Week 84 | | |
| Week 96 | | |
| Week 108 | | |
| Week 120 | | |
| Week 132 | | |
| Week 144 | | |
| Week 156 | | |
| Week 168 | | |
| Week 180 | | |
| Week 192 | | |
| HAQ-DI response (MCID ≥ -0.22) from initiation of stimulation [5] | | |
| Week 24 | | |
| N | XX | XX |
| Yes [3] | xx (xx.x%) | xx (xx.x%) |
| 95% CI | (xx.x%, xx.x%) | (xx.x%, xx.x%) |
| Repeat for: | | |
| Week 36 | | |
| Week 48 | | |
| Week 60 | | |




Doc# CLP-008 Rev C, 15JUL2024

| Variable | TOL [1]<br>(N=xxx) | COL [2]<br>(N=xxx) |
|----------|--------------------|--------------------|
| Week 72 | | |
| Week 84 | | |
| Week 96 | | |
| Week 108 | | |
| Week 120 | | |
| Week 132 | | |
| Week 144 | | |
| Week 156 | | |
| Week 168 | | |
| Week 180 | | |
| Week 192 | | |

Abbreviations: CI, confidence interval; COL, Control to Open Label; HAQ-DI, Health Assessment Questionnaire Disability Index; MCID, minimal clinically important difference; TOL, Treatment to Open Label;

- [1] Treatment to Open Label (TOL): The TOL population comprises treatment subjects from ITT population who received active stimulation through Week 12, completed Week 12 assessments, continued to receive active stimulation during open-label follow-up, and for whom follow-up data are available.
- [2] Control to Open Label (COL): The COL population comprises control subjects from ITT population who received non-active (sham) stimulation through Week 12, switched to active stimulation after completing Week 12 assessments, continued to receive active stimulation during open-label follow-up, and for whom follow-up data are available.
- [3] Percentage calculated based on each analysis population (i.e., TOL, COL)
- [4] Baseline on the day of informed consent for TOL and Week 12 for COL
- [5] Initiation of stimulation at Day 0 for TOL and Week 12 for COL

Reference: Listing 16.x.x.x

SOURCE: xxxxx SAS 9.4 {program location} {run date/time}}




Table 14.8.2.4.1 Subgroup Analysis HAQ-DI MCID Response: Prior b/tsDMARDs

| Variable | TOL [1]<br>(N=xxx) | COL [2]<br>(N=xxx) |
|---|---|---|
| HAQ-DI response (MCID ≥ -0.22) from baseline [4] | , containing the same of the s | ( |
| Prior b/tsDMARD < 4 | | |
| Week 24 | | |
| N | xx | XX |
| Yes [3] | xx (xx.x%) | xx (xx,x%) |
| 95% CI | (xx.x, xx.x) | (xx.x, xx.x) |
| Prior b/tsDMARD ≥ 4 | | |
| Week 24 | | |
| N | xx | XX |
| Yes [3] | xx (xx.x%) | xx (xx.x%) |
| 95% CI | (xx.x, xx.x) | (xx.x, xx.x) |
| Repeat for: | | |
| Week 36 | | |
| Week 48 | | |
| Week 60 | | |
| Week 72 | | |
| Week 84 | | |
| Week 96 | | |
| Week 108 | | |
| Week 120 | | |
| Week 132 | | |
| Week 144 | | |
| Week 156 | | |
| Week 168 | | |
| Week 180 | | |
| Week 192 | | |

HAQ-DI response (MCID ≥ -0.22) from initiation of stimulation [5]



| Variable | TOL [1]<br>(N=xxx) | COL [2]<br>(N=xxx) |
|---|---|---|
| Prior b/tsDMARD < 4 | ( · | ( |
| Week 24 | | |
| N | xx | XX |
| Yes [3] | xx (xx.x%) | xx (xx.x%) |
| 95% CI | (xx.x, xx.x) | (xx.x, xx.x) |
| Prior b/tsDMARD ≥ 4 | | |
| Week 24 | | |
| N | xx | XX |
| Yes [3] | xx (xx.x%) | xx (xx.x%) |
| 95% CI | (xx.x, xx.x) | (xx.x, xx.x) |
| Repeat for: | | |
| Week 36 | | |
| Week 48 | | |
| Week 60 | | |
| Week 72 | | |
| Week 84 | | |
| Week 96 | | |
| Week 108 | | |
| Week 120 | | |
| Week 132 | | |
| Week 144 | | |
| Week 156 | | |
| Week 168 | | |
| Week 180 | | |
| Week 192 | | |

Abbreviations: CI, confidence interval; COL, Control to Open Label; HAQ-DI, Health Assessment Questionnaire Disability Index; MCID, minimal clinically important difference; TOL, Treatment to Open Label

- [1] Treatment to Open Label (TOL): The TOL population comprises treatment subjects from ITT population who received active stimulation through Week 12, completed Week 12 assessments, continued to receive active stimulation during open-label follow-up, and for whom follow-up data are available.
- [2] Control to Open Label (COL): The COL population comprises control subjects from ITT population who received non-active (sham) stimulation through Week 12, switched to active stimulation after completing Week 12 assessments, continued to receive active stimulation during open-label follow-up, and for whom follow-up data are available.
- [3] Percentage calculated based on each analysis population (i.e., TOL, COL)




Doc# CLP-008 Rev C, 15JUL2024

Variable TOL [1] COL [2] (N=xxx) (N=xxx)

[4] Baseline on the day of informed consent for TOL and Week 12 for COL

[5] Initiation of stimulation at Day 0 for TOL and Week 12 for COL

Reference: Listing 16.x.x.x

SOURCE: xxxxx SAS 9.4 {program location} {run date/time}}




Table 14.8.2.4.2 Subgroup Analysis of HAQ-DI MCID Response: Prior JAKi

Repeat Table 14.8.2.4.1 for Prior JAKi [Yes vs. No]

Add to abbreviations: JAKi, Janus kinase inhibitor.

Table 14.8.2.4.3
Subgroup Analysis of HAQ-DI MCID Response: RA Disease Activity at Baseline

Repeat Table 14.8.2.4.1 for RA Disease Activity at Baseline [DAS28-CRP ≤ 5.1 vs. DAS28-CRP > 5.1]

Add to abbreviations: DAS, Disease Activity Score.

Table 14.8.2.4.4
Subgroup Analysis of HAQ-DI MCID Response: RA Severity at Initiation of Stimulation

Repeat Table 14.8.2.4.1 for RA Severity at Initiation of Stimulation [<4 TJC28 or <4 SJC28 vs. ≥4 TJC28 and ≥4 SJC28]

Add to abbreviations: TJC, tender joint count; SJC, swollen joint count

Programming note: For this analysis, remove the "from baseline" portion of the table.

Table 14.8.2.4.5
Subgroup Analysis of HAQ-DI MCID Response: Augmented Therapy

Repeat Table 14.8.2.4.1 for RA Augmented Therapy [yes, no]



#### Table 14.8.2.5 TJC28

| Variable | TOL [1]<br>(N=xxx) | COL [2]<br>(N=xxx) |
|--------------------------|--------------------|--------------------|
| TJC28 Score | , | , , |
| Baseline [4] | | |
| N[3] | xx (xx.x%) | xx (xx,x%) |
| Mean (SD) | xxx.x (xxx.xx) | xxx.x (xxx.xx) |
| Median | xxx.xx | XXX,XX |
| Min-Max | xxx.x - xxx.x | xxx.x - xxx.x |
| Week 24 | | |
| N[3] | xx (xx.x%) | xx (xx.x%) |
| Mean (SD) | xxx.x (xxx.xx) | xxx.x (xxx.xx) |
| Median | xxx.xx | xxx.xx |
| Min-Max | xxx.x - xxx.x | xxx.x - xxx.x |
| Change from baseline [4] | | |
| N[3] | xx (xx.x%) | xx (xx.x%) |
| Mean (SD) | xxx.x (xxx.xx) | xxx.x (xxx.xx) |
| Median | xxx.xx | xxx.xx |
| Min-Max | xxx.x - xxx.x | xxx.x - xxx.x |
| 95% CI | (xx.x, xx.x) | (xx.x, xx.x) |
| Repeat for: | | |
| Week 36 | | |
| Week 48 | | |
| Week 60 | | |
| Week 72 | | |
| Week 84 | | |
| Week 96 | | |
| Week 108 | | |
| Week 120 | | |
| Week 132 | | |
| Week 144 | | |
| Week 156 | | |
| Week 168 | | |
| Week 180 | | |


## SETPOINT MEDICAL

## Doc# CLP-008 Rev C, 15JUL2024

| Variable | TOL [1]<br>(N=xxx) | COL [2]<br>(N=xxx) |
|---|---|---|
| Week 192 | (2. 1111) | ( |
| TJC28 20% response from baseline [4] | | |
| Week 24 | | |
| N | XX | XX |
| Yes [3] | xx (xx.x%) | xx (xx.x%) |
| 95% CI | (xx.x, xx.x) | (xx.x, xx.x) |
| Repeat for: | | |
| Week 36 | | |
| Week 48 | | |
| Week 60 | | |
| Week 72 | | |
| Week 84 | | |
| Week 96 | | |
| Week 108 | | |
| Week 120 | | |
| Week 132 | | |
| Week 144 | | |
| Week 156 | | |
| Week 168 | | |
| Week 180 | | |
| Week 192 | | |
| TJC28 50% response from baseline [4] | | |
| Week 24 | | |
| N | XX | XX |
| Yes [3] | xx (xx.x%) | xx (xx.x%) |
| 95% CI | (xx.x, xx.x) | (xx.x, xx.x) |
| Repeat for: | | |
| Week 36 | | |
| Week 48 | | |
| Week 60 | | |
| Week 72 | | |
| Week 84 | | |
| Week 96 | | |


# SETPOINT MEDICAL

## Doc# CLP-008 Rev C, 15JUL2024

| Variable | TOL [1]<br>(N=xxx) | COL [2]<br>(N=xxx) |
|---|---|---|
| Week 108 | (11 200) | (II AAA) |
| Week 120 | | |
| Week 132 | | |
| Week 144 | | |
| Week 156 | | |
| Week 168 | | |
| Week 180 | | |
| Week 192 | | |
| TJC28 70% response from baseline [4] | | |
| Week 24 | | |
| N | XX | XX |
| Yes [3] | xx (xx.x%) | xx (xx.x%) |
| 95% CI | (xx.x, xx.x) | (xx.x, xx.x) |
| Repeat for: | | |
| Week 36 | | |
| Week 48 | | |
| Week 60 | | |
| Week 72 | | |
| Week 84 | | |
| Week 96 | | |
| Week 108 | | |
| Week 120 | | |
| Week 132 | | |
| Week 144 | | |
| Week 156 | | |
| Week 168 | | |
| Week 180 | | |
| Week 192 | | |
| TJC28 change from initiation of stimulation | | |
| Day of Initiation of stimulation [5] | | |
| N[3] | xx (xx.x%) | xx (xx,x%) |
| Mean (SD) | xxx.x (xxx.xx) | xxx.x (xxx.xx) |
| Median | xxx.xx | xxx,xx |
| Min-Max | xxx.x - xxx.x | xxx.x - xxx.x |



| Variable | TOL [1]<br>(N=xxx) | COL [2]<br>(N=xxx) |
|---|---|---|
| Week 24 | | |
| Change from initiation of stimulation [5] | | |
| N[3] | xx (xx.x%) | xx (xx.x%) |
| Mean (SD) | xxx.x (xxx.xx) | xxx.x (xxx.xx) |
| Median | xxx.xx | xxx.xx |
| Min-Max | xxx.x - xxx.x | xxx.x - xxx.x |
| 95% CI | (xx.x, xx.x) | (xx.x, xx.x) |
| Repeat for: | | |
| Week 36 | | |
| Week 48 | | |
| Week 60 | | |
| Week 72 | | |
| Week 84 | | |
| Week 96 | | |
| Week 108 | | |
| Week 120 | | |
| Week 132 | | |
| Week 144 | | |
| Week 156 | | |
| Week 168 | | |
| Week 180 | | |
| Week 192 | | |
| TJC28 20% response from initiation of stimulation [5] | | |
| Week 24 | | |
| N | XX | XX |
| Yes [3] | xx (xx.x%) | xx (xx.x%) |
| 95% CI | (xx.x, xx.x) | (xx.x, xx.x) |
| Repeat for: | | |
| Week 36 | | |
| Week 48 | | |
| Week 60 | | |
| Week 72 | | |
| Week 84 | | |


## Doc# CLP-008 Rev C, 15JUL2024

| Variable Variable | TOL [1]<br>(N=xxx) | COL [2]<br>(N=xxx) |
|---|---|---|
| Week 96 | (** 1111) | (** ******) |
| Week 108 | | |
| Week 120 | | |
| Week 132 | | |
| Week 144 | | |
| Week 156 | | |
| Week 168 | | |
| Week 180 | | |
| Week 192 | | |
| GC28 50% response from initiation of stimulation [5] | | |
| Week 24 | | |
| N | XX | XX |
| Yes [3] | xx (xx.x%) | xx (xx.x%) |
| 95% CI | (xx.x, xx.x) | (xx.x, xx.x) |
| Repeat for: | | |
| Week 36 | | |
| Week 48 | | |
| Week 60 | | |
| Week 72 | | |
| Week 84 | | |
| Week 96 | | |
| Week 108 | | |
| Week 120 | | |
| Week 132 | | |
| Week 144 | | |
| Week 156 | | |
| Week 168 | | |
| Week 180 | | |
| Week 192 | | |
| GC28 70% response from initiation of stimulation [5] | | |
| Week 24 | | |
| N | xx | xx |
| Yes [3] | xx (xx.x%) | xx (xx.x%) |
| 95% CI | (xx.x, xx.x) | (11111111111111111111111111111111111111 |




| Variable | TOL [1]<br>(N=xxx) | COL [2]<br>(N=xxx) |
|-------------|--------------------|--------------------|
| Repeat for: | | |
| Week 36 | | |
| Week 48 | | |
| Week 60 | | |
| Week 72 | | |
| Week 84 | | |
| Week 96 | | |
| Week 108 | | |
| Week 120 | | |
| Week 132 | | |
| Week 144 | | |
| Week 156 | | |
| Week 168 | | |
| Week 180 | | |
| Week 192 | | |

Abbreviations: CI, confidence interval; COL, Control to Open Label; TJC, tender joint count; TOL, Treatment to Open Label

- [1] Treatment to Open Label (TOL): The TOL population comprises treatment subjects from ITT population who received active stimulation through Week 12, completed Week 12 assessments, continued to receive active stimulation during open-label follow-up, and for whom follow-up data are available.
- [2] Control to Open Label (COL): The COL population comprises control subjects from ITT population who received non-active (sham) stimulation through Week 12, switched to active stimulation after completing Week 12 assessments, continued to receive active stimulation during open-label follow-up, and for whom follow-up data are available.
- [3] Percentage calculated based on each analysis population (i.e., TOL, COL)
- [4] Baseline on the day of informed consent for TOL and Week 12 for COL
- [5] Initiation of stimulation at Day 0 for TOL and Week 12 for COL

Reference: Listing 16.x.x.x

SOURCE: xxxxx SAS 9.4 {program location} {run date/time}}

Serial Number: c700c42a-b18e-4af7-8a24-9d2146ac6503 accessed by Melissa Evangelista (MEVANGELISTA) on Thu, 28 Aug 2025 18:20:31 GMT.




Table 14.8.2.6 SJC28

| Variable | TOL [1]<br>(N=xxx) | COL [2]<br>(N=xxx) |
|--------------------------|--------------------|--------------------|
| SJC28 Score | • | |
| Baseline [4] | | |
| N[3] | xx (xx.x%) | xx (xx.x%) |
| Mean (SD) | xxx.x (xxx.xx) | xxx.x (xxx.xx) |
| Median | xxx.xx | XXX.XX |
| Min-Max | xxx.x - xxx.x | xxx.x - xxx.x |
| Week 24 | | |
| N[3] | xx (xx.x%) | xx (xx.x%) |
| Mean (SD) | xxx.x (xxx.xx) | xxx.x (xxx.xx) |
| Median | xxx.xx | xxx.xx |
| Min-Max | xxx.x - xxx.x | xxx.x - xxx.x |
| Change from baseline [4] | | |
| N[3] | xx (xx.x%) | xx (xx.x%) |
| Mean (SD) | xxx.x (xxx.xx) | xxx.x (xxx.xx) |
| Median | xxx.xx | xxx.xx |
| Min-Max | xxx.x - xxx.x | xxx.x - xxx.x |
| 95% CI | (xx.x, xx.x) | (xx.x, xx.x) |
| Repeat for: | | |
| Week 36 | | |
| Week 48 | | |
| Week 60 | | |
| Week 72 | | |
| Week 84 | | |
| Week 96 | | |
| Week 108 | | |
| Week 120 | | |
| Week 132 | | |
| Week 144 | | |
| Week 156 | | |
| Week 168 | | |
| Week 180 | | |


## Doc# CLP-008 Rev C, 15JUL2024

| Variable | TOL [1]<br>(N=xxx) | COL [2]<br>(N=xxx) |
|---|---|---|
| Week 192 | , , | |
| SJC28 20% response from baseline [4] | | |
| Week 24 | | |
| N | XX | XX |
| Yes [3] | xx (xx.x%) | xx (xx.x%) |
| 95% CI | (xx.x, xx.x) | (xx.x, xx.x) |
| Repeat for: | | |
| Week 36 | | |
| Week 48 | | |
| Week 60 | | |
| Week 72 | | |
| Week 84 | | |
| Week 96 | | |
| Week 108 | | |
| Week 120 | | |
| Week 132 | | |
| Week 144 | | |
| Week 156 | | |
| Week 168 | | |
| Week 180 | | |
| Week 192 | | |
| SJC28 50% response from baseline [4] | | |
| Week 24 | | |
| N | XX | XX |
| Yes [3] | xx (xx.x%) | xx (xx,x%) |
| 95% CI | (xx.x, xx.x) | (xx.x, xx.x) |
| Repeat for: | | |
| Week 36 | | |
| Week 48 | | |
| Week 60 | | |
| Week 72 | | |
| Week 84 | | |
| Week 96 | | |


## Doc# CLP-008 Rev C, 15JUL2024

| Variable | TOL [1]<br>(N=xxx) | COL [2]<br>(N=xxx) |
|---|---|---|
| Week 108 | (TV AMA) | (11 1221) |
| Week 120 | | |
| Week 132 | | |
| Week 144 | | |
| Week 156 | | |
| Week 168 | | |
| Week 180 | | |
| Week 192 | | |
| SJC28 70% response from baseline [4] | | |
| Week 24 | | |
| N | XX | XX |
| Yes [3] | xx (xx.x%) | xx (xx.x%) |
| 95% CI | (xx.x, xx.x) | (xx.x, xx.x) |
| Repeat for: | | |
| Week 36 | | |
| Week 48 | | |
| Week 60 | | |
| Week 72 | | |
| Week 84 | | |
| Week 96 | | |
| Week 108 | | |
| Week 120 | | |
| Week 132 | | |
| Week 144 | | |
| Week 156 | | |
| Week 168 | | |
| Week 180 | | |
| Week 192 | | |
| SJC28 change from initiation of stimulation | | |
| Day of Initiation of stimulation [5] | | |
| N[3] | xx (xx.x%) | xx (xx.x%) |
| Mean (SD) | xxx.x (xxx.xx) | xxx.x (xxx.xx) |
| Median | xxx.xx | xxx.xx |
| Min-Max | xxx.x - xxx.x | xxx.x - xxx.x |




| Variable | TOL [1]<br>(N=xxx) | COL [2]<br>(N=xxx) |
|---|---|---|
| Week 24 | | |
| Change from initiation of stimulation [5] | | |
| N[3] | xx (xx.x%) | xx (xx.x%) |
| Mean (SD) | xxx.x (xxx.xx) | xxx.x (xxx.xx) |
| Median | xxx.xx | xxx.xx |
| Min-Max | xxx.x - xxx.x | xxx.x - xxx.x |
| 95% CI | (xx.x, xx.x) | (xx.x, xx.x) |
| Repeat for: | | |
| Week 36 | | |
| Week 48 | | |
| Week 60 | | |
| Week 72 | | |
| Week 84 | | |
| Week 96 | | |
| Week 108 | | |
| Week 120 | | |
| Week 132 | | |
| Week 144 | | |
| Week 156 | | |
| Week 168 | | |
| Week 180 | | |
| Week 192 | | |
| SJC28 20% response from initiation of stimulation [5] | | |
| Week 24 | | |
| N | XX | XX |
| Yes [3] | xx (xx.x%) | xx (xx.x%) |
| 95% CI | (xx.x, xx.x) | (xx.x, xx.x) |
| Repeat for: | | |
| Week 36 | | |
| Week 48 | | |
| Week 60 | | |
| Week 72 | | |
| Week 84 | | |


## Doc# CLP-008 Rev C, 15JUL2024

| Variable | TOL [1]<br>(N=xxx) | COL [2]<br>(N=xxx) |
|---|---|---|
| Week 96 | (ii aay | (11 7000) |
| Week 108 | | |
| Week 120 | | |
| Week 132 | | |
| Week 144 | | |
| Week 156 | | |
| Week 168 | | |
| Week 180 | | |
| Week 192 | | |
| SJC28 50% response from initiation of stimulation [5] | | |
| Week 24 | | |
| N | XX | XX |
| Yes [3] | xx (xx.x%) | xx (xx.x%) |
| 95% CI | (xx.x, xx.x) | (xx.x, xx.x) |
| tepeat for: | | |
| Week 36 | | |
| Week 48 | | |
| Week 60 | | |
| Week 72 | | |
| Week 84 | | |
| Week 96 | | |
| Week 108 | | |
| Week 120 | | |
| Week 132 | | |
| Week 144 | | |
| Week 156 | | |
| Week 168 | | |
| Week 180 | | |
| Week 192 | | |
| JC28 70% response from initiation of stimulation [5] | | |
| Week 24 | | |
| N | XX | xx |
| Yes [3] | xx (xx.x%) | xx (xx.x%) |
| 95% CI | (xx.x, xx.x) | (xx.x, xx.x) |




| Variable | TOL [1]<br>(N=xxx) | COL [2]<br>(N=xxx) |
|-------------|--------------------|--------------------|
| Repeat for: | | |
| Week 36 | | |
| Week 48 | | |
| Week 60 | | |
| Week 72 | | |
| Week 84 | | |
| Week 96 | | |
| Week 108 | | |
| Week 120 | | |
| Week 132 | | |
| Week 144 | | |
| Week 156 | | |
| Week 168 | | |
| Week 180 | | |
| Week 192 | | |

Abbreviations: CI, confidence interval; COL, Control to Open Label; SJC, swollen joint count; TOL, Treatment to Open Label

- [1] Treatment to Open Label (TOL): The TOL population comprises treatment subjects from ITT population who received active stimulation through Week 12, completed Week 12 assessments, continued to receive active stimulation during open-label follow-up, and for whom follow-up data are available.
- [2] Control to Open Label (COL): The COL population comprises control subjects from ITT population who received non-active (sham) stimulation through Week 12, switched to active stimulation after completing Week 12 assessments, continued to receive active stimulation during open-label follow-up, and for whom follow-up data are available.
- [3] Percentage calculated based on each analysis population (i.e., TOL, COL)
- [4] Baseline on the day of informed consent for TOL and Week 12 for COL
- [5] Initiation of stimulation at Day 0 for TOL and Week 12 for COL

Reference: Listing 16.x.x.x

SOURCE: xxxxx SAS 9.4 {program location} {run date/time}}


#### Statistical Analysis Plan for Long-Term Safety and Exploratory Analyses in SPM-020 (The RESET-RA Study) Doc# CLP-008 Rev C, 15JUL2024



#### Table 14.8.2.7 Subject's Assessment of Pain

Repeat 14.8.2.6 for Subject's Pain Assessment

Note to Programmer: Remove SJC from footnote.

Table 14.8.2.8 SGA

Repeat 14.8.2.6 for SGA

Note to Programmer: Remove SJC from footnote and add SGA, subject's global assessment.

Table 14.8.2.9 EGA

Repeat 14.8.2.6 for EGA

Note to Programmer: Remove SJC from footnote and add EGA, evaluator's global assessment.

Table 14.8.2.10 hsCRP

Repeat 14.8.2.6 for hsCRP (mg/mL)

Note to Programmer: Remove SJC from footnote and add hsCRP, high sensitivity C-reactive protein.



#### Table 14.8.2.11 DAS28-CRP

| Variable | TOL [1]<br>(N=xxx) | COL [2]<br>(N=xxx) |
|--------------------------|--------------------|--------------------|
| DAS28-CRP Score | (N-XXX) | (IV-XXX) |
| Baseline [4] | | |
| N [3] | xx (xx.x%) | xx (xx.x%) |
| Mean (SD) | xxx.x (xxx.xx) | xxx.x (xxx.xx) |
| Median | XXX.XX | XXX.XX |
| Min-Max | XXX.X – XXX.X | XXX.X – XXX.X |
| THE THE | and and | aaa,a aaa,a |
| Week 24 | | |
| N[3] | xx (xx.x%) | xx (xx.x%) |
| Mean (SD) | xxx.x (xxx.xx) | xxx.x (xxx.xx) |
| Median | xxx.xx | xxx.xx |
| Min-Max | xxx.x - xxx.x | xxx.x - xxx.x |
| Change from baseline [4] | | |
| N[3] | xx (xx.x%) | xx (xx.x%) |
| Mean (SD) | xxx.x (xxx.xx) | xxx.x (xxx.xx) |
| Median | XXX.XX | XXX,XX |
| Min-Max | xxx.x - xxx.x | xxx.x - xxx.x |
| 95% CI | (xx.x, xx.x) | (xx.x, xx.x) |
| Repeat for: | | |
| Week 36 | | |
| Week 48 | | |
| Week 60 | | |
| Week 72 | | |
| Week 84 | | |
| Week 96 | | |
| Week 108 | | |
| Week 120 | | |
| Week 132 | | |
| Week 144 | | |
| Week 156 | | |
| Week 168 | | |


## Doc# CLP-008 Rev C, 15JUL2024

| Variable | TOL [1]<br>(N=xxx) | COL [2]<br>(N=xxx) |
|---|---|---|
| Week 180 | \ | , |
| Week 192 | | |
| DAS28-CRP low disease activity (score 2.6 to < 3.2) | | |
| Week 24 | | |
| N | XX | XX |
| Yes [3] | xx (xx.x%) | xx (xx.x%) |
| 95% CI | (xx.x, xx.x) | (xx.x, xx.x) |
| Repeat for: | | |
| Week 36 | | |
| Week 48 | | |
| Week 60 | | |
| Week 72 | | |
| Week 84 | | |
| Week 96 | | |
| Week 108 | | |
| Week 120 | | |
| Week 132 | | |
| Week 144 | | |
| Week 156 | | |
| Week 168 | | |
| Week 180 | | |
| Week 192 | | |
| DAS28-CRP remission (score 0 to < 2.6) | | |
| Week 24 | | |
| N | XX | XX |
| Yes [3] | xx (xx.x%) | xx (xx.x%) |
| 95% CI | (xx.x, xx.x) | (xx.x, xx.x) |
| Repeat for: | | |
| Week 36 | | |
| Week 48 | | |
| Week 60 | | |
| Week 72 | | |
| Week 84 | | |




| Variable | TOL [1]<br>(N=xxx) | COL [2]<br>(N=xxx) |
|---|---|---|
| Week 96 | , , | |
| Week 108 | | |
| Week 120 | | |
| Week 132 | | |
| Week 144 | | |
| Week 156 | | |
| Week 168 | | |
| Week 180 | | |
| Week 192 | | |
| DAS28-CRP score change from initiation of stimulation [5] | | |
| Day of initiation of stimulation [5] | | |
| N[3] | xx (xx.x%) | xx (xx.x%) |
| Mean (SD) | xxx.x (xxx.xx) | xxx.x (xxx.xx) |
| Median | xxx.xx | xxx.xx |
| Min-Max | xxx.x - xxx.x | xxx.x - xxx.x |
| Week 24 | | |
| Change from initiation of stimulation [5] | | |
| N[3] | xx (xx.x%) | xx (xx.x%) |
| Mean (SD) | xxx.x (xxx.xx) | xxx.x (xxx.xx) |
| Median | xxx.xx | xxx.xx |
| Min-Max | xxx.x - xxx.x | xxx.x - xxx.x |
| 95% CI | (xx.x, xx.x) | (xx.x, xx.x) |
| Repeat for: | | |
| Week 36 | | |
| Week 48 | | |
| Week 60 | | |
| Week 72 | | |
| Week 84 | | |
| Week 96 | | |
| Week 108 | | |
| Week 120 | | |
| Week 132 | | |
| Week 144 | | |
| Week 156 | | |


Statistical Analysis Plan for Long-Term Safety and Exploratory Analyses in SPM-020 (The RESET-RA Study)



Doc# CLP-008 Rev C, 15JUL2024

| Variable | TOL [1] | COL [2] |
|----------|---------|---------|
| | (N=xxx) | (N=xxx) |
| Week 168 | | |
| Week 180 | | |
| Week 192 | | |

Abbreviations: CI, confidence interval; COL, Control to Open Label; CRP, C-reactive protein; DAS, Disease Activity Score; TOL, Treatment to Open Label;

- [1] Treatment to Open Label (TOL): The TOL population comprises treatment subjects from ITT population who received active stimulation through Week 12, completed Week 12 assessments, continued to receive active stimulation during open-label follow-up, and for whom follow-up data are available.
- [2] Control to Open Label (COL): The COL population comprises control subjects from ITT population who received non-active (sham) stimulation through Week 12, switched to active stimulation after completing Week 12 assessments, continued to receive active stimulation during open-label follow-up, and for whom follow-up data are available.
- [3] Percentage calculated based on each analysis population (i.e., TOL, COL)
- [4] Baseline on the day of informed consent for TOL and Week 12 for COL
- [5] Initiation of stimulation at Day 0 for TOL and Week 12 for COL

Reference: Listing 16.x.x.x

SOURCE: xxxxx SAS 9.4 {program location} {run date/time}}




#### Table 14.8.2.12 CDAI

| Variable | TOL [1]<br>(N=xxx) | COL [2]<br>(N=xxx) |
|--------------------------|--------------------|--------------------|
| CDAI score | (11 202) | (ii aaa) |
| Baseline [4] | | |
| N [3] | xx (xx.x%) | xx (xx.x%) |
| Mean (SD) | xxx.x (xxx.xx) | xxx.x (xxx.xx) |
| Median | xxx.xx | XXX,XX |
| Min-Max | xxx.x - xxx.x | xxx.x - xxx.x |
| Week 24 | | |
| N [3] | xx (xx.x%) | xx (xx.x%) |
| Mean (SD) | xxx.x (xxx.xx) | xxx.x (xxx.xx) |
| Median | xxx.xx | xxx.xx |
| Min-Max | xxx.x - xxx.x | xxx.x - xxx.x |
| Change from baseline [4] | | |
| N [3] | xx (xx.x%) | xx (xx.x%) |
| Mean (SD) | xxx.x (xxx.xx) | xxx.x (xxx.xx) |
| Median | xxx.xx | xxx,xx |
| Min-Max | xxx.x - xxx.x | xxx.x - xxx.x |
| 95% CI | (xx.x, xx.x) | (xx.x, xx.x) |
| Repeat for: | | |
| Week 36 | | |
| Week 48 | | |
| Week 60 | | |
| Week 72 | | |
| Week 84 | | |
| Week 96 | | |
| Week 108 | | |
| Week 120 | | |
| Week 132 | | |
| Week 144 | | |
| Week 156 | | |
| Week 168 | | |




| Variable | TOL [1]<br>(N=xxx) | COL [2]<br>(N=xxx) |
|---|---|---|
| Week 180 | (11 000) | (IV AAA) |
| Week 192 | | |
| CDAI low disease activity (score $\geq$ 2.8 to $\leq$ 10) | | |
| Week 24 | | |
| N | XX | xx |
| Yes [3] | xx (xx.x%) | xx (xx.x%) |
| 95% CI | (xx.x, xx.x) | (xx.x, xx.x |
| Repeat for: | | |
| Week 36 | | |
| Week 48 | | |
| Week 60 | | |
| Week 72 | | |
| Week 84 | | |
| Week 96 | | |
| Week 108 | | |
| Week 120 | | |
| Week 132 | | |
| Week 144 | | |
| Week 156 | | |
| Week 168 | | |
| Week 180 | | |
| Week 192 | | |
| CDAI remission (score 0 to $\leq 2.8$ ) | | |
| Week 24 | | |
| N | XX | XX |
| Yes [3] | xx (xx.x%) | xx (xx.x% |
| 95% CI | (xx.x, xx.x) | (xx.x, xx.x |
| Repeat for: | | |
| Week 36 | | |
| Week 48 | | |
| Week 60 | | |
| Week 72 | | |
| Week 84 | | |




| Variable | TOL [1]<br>(N=xxx) | COL [2]<br>(N=xxx) |
|---|---|---|
| Week 96 | ( · | ( |
| Week 108 | | |
| Week 120 | | |
| Week 132 | | |
| Week 144 | | |
| Week 156 | | |
| Week 168 | | |
| Week 180 | | |
| Week 192 | | |
| CDAI score change from initiation of stimulation [5] | | |
| Day of initiation of stimulation [5] | | |
| N [3] | xx (xx.x%) | xx (xx.x%) |
| Mean (SD) | xxx.x (xxx.xx) | xxx.x (xxx.xx) |
| Median | xxx.xx | xxx.xx |
| Min-Max | xxx.x - xxx.x | xxx.x - xxx.x |
| Week 24 | | |
| Change from initiation of stimulation [5] | | |
| N [3] | xx (xx.x%) | xx (xx.x%) |
| Mean (SD) | xxx.x (xxx.xx) | xxx.x (xxx.xx) |
| Median | xxx.xx | xxx.xx |
| Min-Max | xxx.x - xxx.x | xxx.x - xxx.x |
| 95% CI | (xx.x, xx.x) | (xx.x, xx.x) |
| Repeat for: | | |
| Week 36 | | |
| Week 48 | | |
| Week 60 | | |
| Week 72 | | |
| Week 84 | | |
| Week 96 | | |
| Week 108 | | |
| Week 120 | | |
| Week 132 | | |
| Week 144 | | |
| Week 156 | | |


## Doc# CLP-008 Rev C, 15JUL2024

| Variable | | TOL [1]<br>(N=xxx) | COL [2]<br>(N=xxx) |
|---|---|---|---|
| Week 168 | - | (11 222) | (11 444) |
| Week 180 | | | |
| Week 192 | | | |
| DAI response (MCID) from baselin | ne [4] | | |
| Week 24 | | | |
| N | | xx | XX |
| Yes [3] | | xx (xx.x%) | xx (xx.x%) |
| 95% CI | | (xx.x%, xx.x%) | (xx.x%, xx.x%) |
| Repeat for: | | | |
| Week 36 | | | |
| Week 48 | | | |
| Week 60 | | | |
| Week 72 | | | |
| Week 84 | | | |
| Week 96 | | | |
| Week 108 | | | |
| Week 120 | | | |
| Week 132 | | | |
| Week 144 | | | |
| Week 156 | | | |
| Week 168 | | | |
| Week 180 | | | |
| Week 192 | | | |
| DAI response (MCID) from initiati | ion of stimulation [5] | | |
| Week 24 | | | |
| N | | XX | XX |
| Yes [3] | | xx (xx.x%) | xx (xx.x%) |
| 95% CI | | (xx.x%, xx.x%) | (xx.x%, xx.x%) |
| Repeat for: | | | |
| Week 36 | | | |
| Week 48 | | | |
| Week 60 | | | |
| Week 72 | | | |




| Variable | TOL [1]<br>(N=xxx) | COL [2]<br>(N=xxx) |
|----------|--------------------|--------------------|
| Week 84 | (11 202) | (III ALA) |
| Week 96 | | |
| Week 108 | | |
| Week 120 | | |
| Week 132 | | |
| Week 144 | | |
| Week 156 | | |
| Week 168 | | |
| Week 180 | | |
| Week 192 | | |

Abbreviations: CDAI, Clinical Disease Activity Index; CI, confidence interval; COL, Contol to Open Label; TOL, Treatment to Open Label

- [1] Treatment to Open Label (TOL): The TOL population comprises treatment subjects from ITT population who received active stimulation through Week 12, completed Week 12 assessments, continued to receive active stimulation during open-label follow-up, and for whom follow-up data are available.
- [2] Control to Open Label (COL): The COL population comprises control subjects from ITT population who received non-active (sham) stimulation through Week 12, switched to active stimulation after completing Week 12 assessments, continued to receive active stimulation during open-label follow-up, and for whom follow-up data are available.
- [3] Percentage calculated based on each analysis population (i.e., TOL, COL)
- [4] Baseline on the day of informed consent for TOL and Week 12 for COL
- [5] Initiation of stimulation at Day 0 for TOL and Week 12 for COL

Reference: Listing 16.x.x.x

SOURCE: xxxxx SAS 9.4 {program location} {run date/time}}

Table 14.8.2.13 RAMRIS

| Variable | TOL [1] | COL [2] |
|---------------------------|----------------|----------------|
| | (N=xxx) | (N=xxx) |
| RAMRIS bone erosion score | | |
| Baseline [4] | | |
| N[3] | xx (xx.x%) | xx (xx.x%) |
| Mean (SD) | xxx.x (xxx.xx) | xxx.x (xxx.xx) |
| Median | XXX.XX | XXX,XX |
| Min-Max | xxx.x - xxx.x | xxx.x - xxx.x |


## Doc# CLP-008 Rev C, 15JUL2024

| Variable | TOL [1]<br>(N=xxx) | COL [2]<br>(N=xxx) |
|---|---|---|
| Week 24 | | |
| N[3] | xx (xx.x%) | xx (xx.x%) |
| Mean (SD) | xxx.x (xxx.xx) | xxx.x (xxx.xx) |
| Median | xxx.xx | xxx.xx |
| Min-Max | xxx.x - xxx.x | xxx.x - xxx.x |
| Change from baseline [4] (SDC: x.xx) | | |
| N[3] | xx (xx.x%) | xx (xx.x%) |
| Mean (SD) | xxx.x (xxx.xx) | xxx.x (xxx.xx) |
| Median | xxx.xx | xxx.xx |
| Min-Max | xxx.x - xxx.x | xxx.x - xxx.x |
| 95% CI | (xx.x, xx.x) | (xx.x, xx.x) |
| Progression rate from baseline (> 0.5) | | |
| N[3] | xx (xx.x%) | xx (xx.x%) |
| Mean (SD) | xxx.x (xxx.xx) | xxx.x (xxx.xx) |
| Median | xxx.xx | XXX,XX |
| Min-Max | xxx.x - xxx.x | xxx.x - xxx.x |
| AMRIS osteitis score | | |
| Baseline [4] | | |
| N[3] | xx (xx.x%) | xx (xx.x%) |
| Mean (SD) | xxx.x (xxx.xx) | xxx.x (xxx.xx) |
| Median | xxx.xx | XXX,XX |
| Min-Max | xxx.x - xxx.x | xxx.x - xxx.x |
| Week 24 | | |
| N[3] | xx (xx.x%) | xx (xx.x%) |
| Mean (SD) | xxx.x (xxx.xx) | xxx.x (xxx.xx) |
| Median | xxx.xx | xxx.xx |
| Min-Max | xxx.x - xxx.x | xxx.x - xxx.x |
| Change from baseline [4] (SDC: x.xx) | | |
| N[3] | xx (xx.x%) | xx (xx.x%) |
| Mean (SD) | xxx.x (xxx.xx) | xxx.x (xxx.xx) |
| Median | xxx.xx | xxx.xx |



| Variable | TOL [1]<br>(N=xxx) | COL [2]<br>(N=xxx) |
|---|---|---|
| Min-Max | xxx.x - xxx.x | xxx.x - xxx.x |
| 95% CI | (xx.x, xx.x) | (xx.x, xx.x) |
| RAMRIS CARLOS score | | |
| Baseline [4] | | |
| N[3] | xx (xx.x%) | xx (xx.x%) |
| Mean (SD) | xxx.x (xxx.xx) | xxx.x (xxx.xx) |
| Median | xxx.xx | XXX,XX |
| Min-Max | xxx.x - xxx.x | xxx.x - xxx.x |
| Week 24 | | |
| N[3] | xx (xx.x%) | xx (xx.x%) |
| Mean (SD) | xxx.x (xxx.xx) | xxx.x (xxx.xx) |
| Median | xxx.xx | XXX,XX |
| Min-Max | xxx.x - xxx.x | xxx.x - xxx.x |
| Change from baseline [4] (SDC: x.xx) | | |
| N[3] | xx (xx.x%) | xx (xx.x%) |
| Mean (SD) | xxx.x (xxx.xx) | xxx.x (xxx.xx) |
| Median | xxx.xx | xxx.xx |
| Min-Max | xxx.x - xxx.x | xxx.x - xxx.x |
| 95% CI | (xx.x, xx.x) | (xx.x, xx.x) |

Abbreviations: CARLOS, cartilage loss score; CI, confidence interval; COL, Control to Open Label; RAMRIS, Rheumatoid Arthritis MRI Scoring System; SDC, Smallest Detectable Change; TOL, Treatment to Open Label

- [1] Treatment to Open Label (TOL): The TOL population comprises treatment subjects from ITT population who received active stimulation through Week 12, completed Week 12 assessments, continued to receive active stimulation during open-label follow-up, and for whom follow-up data are available.
- [2] Control to Open Label (COL): The COL population comprises control subjects from ITT population who received non-active (sham) stimulation through Week 12, switched to active stimulation after completing Week 12 assessments, continued to receive active stimulation during open-label follow-up, and for whom follow-up data are available.
- [3] Percentage calculated based on each analysis population (i.e., TOL, COL)
- [4] Baseline on the day of informed consent for TOL and Week 12 for COL
- [5] Initiation of stimulation at Day 0 for TOL and Week 12 for COL

Reference: Listing 16.x.x.x

SOURCE: xxxxx SAS 9.4 {program location} {run date/time}}



Table 14.8.2.14 EQ-5D-5L

| Variable | TOL [1] | COL[2] |
|----------------------------|----------------|----------------|
| | (N=xxx) | (N=xxx) |
| Q-5D-5L Index score | | |
| Baseline [4] | | |
| N[3] | xx (xx.x%) | xx (xx.x%) |
| Mean (SD) | xxx.x (xxx.xx) | xxx.x (xxx.xx) |
| Median | xxx.xx | XXX,XX |
| Min-Max | xxx.x - xxx.x | xxx.x - xxx.x |
| Week 24 | | |
| N[3] | xx (xx.x%) | xx (xx.x%) |
| Mean (SD) | xxx.x (xxx.xx) | xxx.x (xxx.xx |
| Median | xxx.xx | xxx.xx |
| Min-Max | xxx.x - xxx.x | xxx.x - xxx.x |
| Change from baseline [4] | | |
| N[3] | xx (xx.x%) | xx (xx.x%) |
| Mean (SD) | xxx.x (xxx.xx) | xxx,x (xxx,xx |
| Median | xxx.xx | xxx.xx |
| Min-Max | xxx.x - xxx.x | xxx.x - xxx.x |
| 95% CI | (xx.x, xx.x) | (xx.x, xx.x) |
| Repeat for: | | |
| Week 48 | | |
| Week 96 | | |
| Week 144 | | |
| Week 192 | | |
| Q-5D-5L Mobility Dimension | | |
| Baseline [4] | | |
| Level 1 (No problem) | xx (xx.x%) | xx (xx.x%) |
| Level 2 (Slight problems) | xx (xx.x%) | xx (xx.x%) |
| Level 3 (Moderate problem) | xx (xx.x%) | xx (xx.x%) |
| Level 4 (Severe problems) | xx (xx.x%) | xx (xx.x%) |
| Level 5 (Extreme problems) | xx (xx.x%) | xx (xx.x%) |


## Doc# CLP-008 Rev C, 15JUL2024

| Variable | TOL [1]<br>(N=xxx) | COL[2]<br>(N=xxx) |
|---|---|---|
| | (IN-XXX) | (IN-XXX) |
| Initiation of stimulation [5] | | |
| Level 1 (No problem) | xx (xx.x%) | xx (xx.x%) |
| Level 2 (Slight problems) | xx (xx.x%) | xx (xx.x%) |
| Level 3 (Moderate problems) | xx (xx.x%) | xx (xx,x%) |
| Level 4 (Severe problems) | xx (xx.x%) | xx (xx,x%) |
| Level 5 (Extreme problems) | xx (xx.x%) | xx (xx.x%) |
| Week 24 | | |
| Level 1 (No problem) | xx (xx.x%) | xx (xx.x%) |
| Level 2 (Slight problems) | xx (xx.x%) | xx (xx.x%) |
| Level 3 (Moderate problems) | xx (xx.x%) | xx (xx.x%) |
| Level 4 (Severe problems) | xx (xx.x%) | xx (xx.x%) |
| Level 5 (Extreme problems) | xx (xx.x%) | xx (xx,x%) |
| Repeat for: | | |
| Week 48 | | |
| Week 96 | | |
| Week 144 | | |
| Week 192 | | |
| Repeat for other dimensions: | | |
| EQ-5D-5L Self-care | | |
| EQ-5D-5L Usual activities | | |
| EQ-5D-5L Pain/discomfort | | |
| EQ-5D-5L Anxiety/depression | | |
| EQ-5D-5L Index score | | |
| Initiation of stimulation [5] | | |
| N[3] | xx (xx.x%) | xx (xx.x%) |
| Mean (SD) | xxx.x (xxx.xx) | xxx.x (xxx.xx) |
| Median | xxx.xx | xxx.xx |
| Min-Max | xxx.x - xxx.x | xxx.x - xxx.x |
| Week 24 | | |
| Change from initiation of stimulation [5] | | |
| N[3] | xx (xx.x%) | xx (xx.x%) |
| | ( | ( |


## Doc# CLP-008 Rev C, 15JUL2024

| Variable | TOL [1]<br>(N=xxx) | COL[2]<br>(N=xxx) |
|--------------------------|--------------------|-------------------|
| Mean (SD) | xxx.x (xxx.xx) | xxx.x (xxx.xx) |
| Median | xxx.xx | xxx.xx |
| Min-Max | xxx.x - xxx.x | xxx.x - xxx.x |
| 95% CI | (xx.x, xx.x) | (xx.x, xx.x) |
| Repeat for: | | |
| Week 48 | | |
| Week 96 | | |
| Week 144 | | |
| Week 192 | | |
| EQ-5D-5L VAS score | | |
| Baseline [4] | | |
| N[3] | xx (xx.x%) | xx (xx.x%) |
| Mean (SD) | xxx.x (xxx.xx) | xxx.x (xxx.xx) |
| Median | XXX.XX | XXX.XX |
| Min-Max | xxx.x - xxx.x | xxx.x - xxx.x |
| Week 24 | | |
| N[3] | xx (xx.x%) | xx (xx.x%) |
| Mean (SD) | xxx.x (xxx.xx) | xxx.x (xxx.xx) |
| Median | XXX.XX | XXX.XX |
| Min-Max | xxx.x - xxx.x | xxx.x - xxx.x |
| Change from baseline [4] | | |
| N[3] | xx (xx.x%) | xx (xx.x%) |
| Mean (SD) | xxx.x (xxx.xx) | xxx.x (xxx.xx) |
| Median | xxx.xx | XXX,XX |
| Min-Max | xxx.x - xxx.x | xxx.x - xxx.x |
| 95% CI | (xx.x, xx.x) | (xx.x, xx.x) |
| Repeat for: | | |
| Week 48 | | |
| Week 96 | | |
| Week 144 | | |
| Week 192 | | |



| ariable | TOL [1]<br>(N=xxx) | COL[2]<br>(N=xxx) |
|---|---|---|
| Q-5D-5L VAS score | ` , | |
| Initiation of stimulation [5] | | |
| N[3] | xx (xx.x%) | xx (xx.x%) |
| Mean (SD) | xxx.x (xxx.xx) | xxx.x (xxx.xx) |
| Median | xxx.xx | xxx.xx |
| Min-Max | xxx.x - xxx.x | xxx.x - xxx.x |
| Week 24 | | |
| Change from initiation of stimulation [5] | | |
| N[3] | xx (xx.x%) | xx (xx.x%) |
| Mean (SD) | xxx.x (xxx.xx) | xxx.x (xxx.xx) |
| Median | XXX.XX | XXX,XX |
| Min-Max | xxx.x - xxx.x | xxx.x - xxx.x |
| 95% CI | (xx.x, xx.x) | (xx.x, xx.x) |
| Repeat for: | | |
| Week 48 | | |
| Week 96 | | |
| Week 144 | | |
| Week 192 | | |

Abbreviations: CI, confidence interval; COL, Control to Open Label; EQ-5d-5L, EuroQol 5 domains 5 levels; OL, open label; TOL, Treamtent to Open Label

- [1] Treatment to Open Label (TOL): The TOL population comprises treatment subjects from ITT population who received active stimulation through Week 12, completed Week 12 assessments, continued to receive active stimulation during open-label follow-up, and for whom follow-up data are available.
- [2] Control to Open Label (COL): The COL population comprises control subjects from ITT population who received non-active (sham) stimulation through Week 12, switched to active stimulation after completing Week 12 assessments, continued to receive active stimulation during open-label follow-up, and for whom follow-up data are available.
- [3] Percentage calculated based on each analysis population (i.e., TOL, COL)
- [4] Baseline on the day of informed consent for TOL and Week 12 for COL
- [5] Initiation of stimulation at Day 0 for TOL and Week 12 for COL

Reference: Listing 16.x.x.x

SOURCE: xxxxx SAS 9.4 {program location} {run date/time}}



Table 14.8.2.15 SF-36

| Variable | TOL [1] | COL [2] |
|-------------------------------|-----------------|----------------|
| 77.44.400 | (N=xxx) | (N=xxx) |
| SF-36 MCS score | | |
| Baseline [4] | | |
| N[3] | xx (xx.x%) | xx (xx.x%) |
| Mean (SD) | xxx.x (xxx.xx) | xxx.x (xxx.xx) |
| Median | XXX.XX | XXX,XX |
| Min-Max | xxx, x - xxx, x | xxx.x - xxx.x |
| Week 24 | | |
| N[3] | xx (xx.x%) | xx (xx.x%) |
| Mean (SD) | xxx.x (xxx.xx) | xxx.x (xxx.xx) |
| Median | xxx.xx | xxx.xx |
| Min-Max | xxx.x - xxx.x | xxx.x - xxx.x |
| Change from baseline [4] | | |
| N[3] | xx (xx.x%) | xx (xx.x%) |
| Mean (SD) | xxx.x (xxx.xx) | xxx.x (xxx.xx) |
| Median | xxx.xx | xxx.xx |
| Min-Max | xxx.x - xxx.x | xxx.x - xxx.x |
| 95% CI | (xx.x, xx.x) | (xx.x, xx.x) |
| Repeat for: | | |
| Week 48 | | |
| Week 96 | | |
| Week 144 | | |
| Week 192 | | |
| Repeat for: | | |
| SF-36 PCS score | | |
| F-36 MCS score | | |
| Initiation of stimulation [5] | | |
| N[3] | xx (xx.x%) | xx (xx.x%) |
| Mean (SD) | xxx.x (xxx.xx) | xxx.x (xxx.xx) |
| Mean (SD) | AAA,A (AAA,AA) | AAA.A (AAA.AA) |




| /ariable | TOL [1]<br>(N=xxx) | COL [2]<br>(N=xxx) |
|---|---|---|
| Median | xxx.xx | xxx.xx |
| Min-Max | xxx.x - xxx.x | xxx.x - xxx.x |
| Week 24 | | |
| Change from initiation of stimulation [5] | | |
| N[3] | xx (xx.x%) | xx (xx.x%) |
| Mean (SD) | xxx.x (xxx.xx) | xxx.x (xxx.xx) |
| Median | xxx.xx | xxx.xx |
| Min-Max | xxx.x - xxx.x | xxx.x - xxx.x |
| 95% CI | (xx.x, xx.x) | (xx.x, xx.x) |
| Repeat for: | | |
| Week 48 | | |
| Week 96 | | |
| Week 144 | | |
| Week 192 | | |
| Repeat for: | | |
| SF-36 PCS score | | |

Abbreviations: CI, confidence interval; COL Control to Open Label; MCS, Mental Component Summary; PCS, Physical Component Summary; SF-36, Short Form Survey with 36 items; TOL, Treatment to Open Label

- [1] Treatment to Open Label (TOL): The TOL population comprises treatment subjects from ITT population who received active stimulation through Week 12, completed Week 12 assessments, continued to receive active stimulation during open-label follow-up, and for whom follow-up data are available.
- [2] Control to Open Label (COL): The COL population comprises control subjects from ITT population who received non-active (sham) stimulation through Week 12, switched to active stimulation after completing Week 12 assessments, continued to receive active stimulation during open-label follow-up, and for whom follow-up data are available.
- [3] Percentage calculated based on each analysis population (i.e., TOL, COL)
- [4] Baseline on the day of informed consent for TOL and Week 12 for COL
- [5] Initiation of stimulation at Day 0 for TOL and Week 12 for COL

Reference: Listing 16.x.x.x

SOURCE: xxxxx SAS 9.4 {program location} {run date/time}}



Table 14.8.2.16 Subject Satisfaction

| Variable | TOL [1] | COL [2] |
|---|---|---|
| | (N=xxx) | (N=xxx) |
| How satisfied are you with the SetPoint System for treatment of RA? | | |
| Week 24 | | |
| N[3] | xx (xx.x%) | xx (xx.x%) |
| Very satisfied | xx (xx.x%) | xx (xx.x%) |
| Satisfied | xx (xx.x%) | xx (xx.x%) |
| Neither satisfied nor dissatisfied | xx (xx.x%) | xx (xx.x%) |
| Somewhat dissatisfied | xx (xx.x%) | xx (xx.x%) |
| Very dissatisfied | xx (xx.x%) | xx (xx.x%) |
| Would you recommend the SetPoint System to a family member or a friend? | | |
| Week 24 | | |
| N[3] | xx (xx.x%) | xx (xx.x%) |
| Yes | xx (xx.x%) | xx (xx.x%) |
| No | xx (xx.x%) | xx (xx.x%) |

Abbreviations: COL, Control to Open Label; TOL, Treatment to Open Label

- [1] Treatment to Open Label (TOL): The TOL population comprises treatment subjects from ITT population who received active stimulation through Week 12, completed Week 12 assessments, continued to receive active stimulation during open-label follow-up, and for whom follow-up data are available.
- [2] Control to Open Label (COL): The COL population comprises control subjects from ITT population who received non-active (sham) stimulation through Week 12, switched to active stimulation after completing Week 12 assessments, continued to receive active stimulation during open-label follow-up, and for whom follow-up data are available.
- [3] Percentage calculated based on each analysis population (i.e., TOL, COL)

Reference: Listing 16.x.x.x

SOURCE: xxxxx SAS 9.4 {program location} {run date/time}}



#### Table 14.8.2.17 Inflammatory Biomarkers

| Variable | TOL [1]<br>(N=xxx) | COL [2]<br>(N=xxx) |
|---|---|---|
| IL-6 (pg/mL) | ( | (5.1.1.1.) |
| Baseline [4] | | |
| N[3] | xx (xx.x%) | xx (xx.x%) |
| Mean (SD) | xxx.x (xxx.xx) | xxx.x (xxx.xx) |
| Median | xxx.xx | XXX,XX |
| Min-Max | xxx.x - xxx.x | xxx.x - xxx.x |
| Week 24 | | |
| N[3] | xx (xx.x%) | xx (xx.x%) |
| Mean (SD) | xxx.x (xxx.xx) | xxx.x (xxx.xx) |
| Median | xxx.xx | xxx.xx |
| Min-Max | xxx.x - xxx.x | xxx.x - xxx.x |
| Change from baseline [4] | | |
| N[3] | xx (xx.x%) | xx (xx.x%) |
| Mean (SD) | xxx.x (xxx.xx) | xxx.x (xxx.xx) |
| Median | xxx.xx | XXX,XX |
| Min-Max | xxx.x - xxx.x | xxx.x - xxx.x |
| 95% CI | (xx.x, xx.x) | (xx.x, xx.x) |
| Repeat for: | | |
| SAA (μg/mL) | | |
| MMP-3 (pg/mL) | | |
| IL-6 (pg/mL) | | |
| Initiation of stimulation [5] | | |
| N[3] | xx (xx.x%) | xx (xx.x%) |
| Mean (SD) | xxx.x (xxx.xx) | xxx.x (xxx.xx) |
| Median | XXX.XX | XXX.XX |
| Min-Max | xxx.x - xxx.x | xxx.x - xxx.x |
| Week 24 | | |
| Change from initiation of stimulation [5] | | |
| N[3] | xx (xx.x%) | xx (xx.x%) |




| Variable | TOL [1]<br>(N=xxx) | COL [2]<br>(N=xxx) |
|---|---|---|
| Mean (SD) | xxx.x (xxx.xx) | xxx.x (xxx.xx) |
| Median | XXX.XX | XXX.XX |
| Min-Max | xxx.x - xxx.x | xxx.x - xxx.x |
| 95% CI | (xx.x, xx.x) | (xx.x, xx.x) |
| Repeat for:<br>SAA (µg/mL)<br>MMP-3 (pg/mL) | | |

Abbreviations: COL, Control to Open Label; IL, interleukin; MMP, matrix metalloproteinase; SAA, serum amyloid A; TOL, Treatment to Open Label

- [1] Treatment to Open Label (TOL): The TOL population comprises treatment subjects from ITT population who received active stimulation through Week 12, completed Week 12 assessments, continued to receive active stimulation during open-label follow-up, and for whom follow-up data are available.
- [2] Control to Open Label (COL): The COL population comprises control subjects from ITT population who received non-active (sham) stimulation through Week 12, switched to active stimulation after completing Week 12 assessments, continued to receive active stimulation during open-label follow-up, and for whom follow-up data are available.
- [3] Percentage calculated based on each analysis population (i.e., TOL, COL)
- [4] Baseline on the day of informed consent for TOL and Week 12 for COL
- [5] Initiation of stimulation at Day 0 for TOL and Week 12 for COL

Reference: Listing 16.x.x.x

SOURCE: xxxxx SAS 9.4 {program location} {run date/time}}

Serial Number: c700c42a-b18e-4af7-8a24-9d2146ac6503 accessed by Melissa Evangelista (MEVANGELISTA) on Thu, 28 Aug 2025 18:20:31 GMT.




Table 14.8.2.18 RA Augmented Therapy

| Variable | TOL [1] | COL [2] |
|-----------------------------------|-------------|------------|
| | (N=xxx) | (N=xxx) |
| Received any RA augmented therapy | | |
| Yes [3] | xxx (xx.x%) | xxx (xx.x% |
| If yes, first noted at [4] | xxx (xx.x%) | xxx (xx.x% |
| Titration 4 | xxx (xx.x%) | xxx (xx.x% |
| Titration 5 | xxx (xx.x%) | xxx (xx.x% |
| Titration 6 | xxx (xx.x%) | xxx (xx.x% |
| Week 24 | xxx (xx.x%) | xxx (xx.x% |
| Week 36 | xxx (xx.x%) | xxx (xx.x% |
| Week 48 | xxx (xx.x%) | xxx (xx.x% |
| Week 60 | xxx (xx.x%) | xxx (xx.x% |
| Week 72 | xxx (xx.x%) | xxx (xx.x% |
| Week 84 | xxx (xx.x%) | xxx (xx.x% |
| Week 96 | xxx (xx.x%) | xxx (xx.x% |
| Week 108 | xxx (xx.x%) | xxx (xx.x% |
| Week 120 | xxx (xx.x%) | xxx (xx.x% |
| Week 132 | xxx (xx.x%) | xxx (xx.x% |
| Week 144 | xxx (xx.x%) | xxx (xx.x% |
| Week 156 | xxx (xx.x%) | xxx (xx.x% |
| Week 168 | xxx (xx.x%) | xxx (xx.x% |
| Week 180 | xxx (xx.x%) | xxx (xx.x% |
| Week 192 | xxx (xx.x%) | xxx (xx.x% |
| Received csDMARD for RA | | |
| Yes [3] | xxx (xx.x%) | xxx (xx.x% |
| If yes, first noted at [4] | · · · | |
| Titration 4 | xxx (xx.x%) | xxx (xx.x% |
| Titration 5 | xxx (xx.x%) | xxx (xx.x% |
| Titration 6 | xxx (xx.x%) | xxx (xx.x% |
| Week 24 | xxx (xx.x%) | xxx (xx.x% |
| Week 36 | xxx (xx.x%) | xxx (xx.x% |
| Week 48 | xxx (xx.x%) | xxx (xx.x% |
| Week 60 | xxx (xx.x%) | xxx (xx.x% |
| Week 72 | xxx (xx.x%) | xxx (xx.x% |

## Doc# CLP-008 Rev C, 15JUL2024

| Variable | TOL [1] | COL [2] |
|---|---|---|
| | (N=xxx) | (N=xxx) |
| Week 84 | xxx (xx.x%) | xxx (xx.x%) |
| Week 96 | xxx (xx.x%) | xxx (xx.x%) |
| Week 108 | xxx (xx.x%) | xxx (xx.x%) |
| Week 120 | xxx (xx.x%) | xxx (xx.x%) |
| Week 132 | xxx (xx.x%) | xxx (xx.x%) |
| Week 144 | xxx (xx.x%) | xxx (xx.x%) |
| Week 156 | xxx (xx.x%) | xxx (xx.x%) |
| Week 168 | xxx (xx.x%) | xxx (xx.x%) |
| Week 180 | xxx (xx.x%) | xxx (xx,x%) |
| Week 192 | xxx (xx.x%) | xxx (xx.x%) |
| Received b/tsDMARDs for RA [1] | | |
| Yes [3] | xxx (xx.x%) | xxx (xx.x%) |
| If yes, first noted at [4] | | |
| Titration 4 | xxx (xx.x%) | xxx (xx.x%) |
| Titration 5 | xxx (xx.x%) | xxx (xx.x%) |
| Titration 6 | xxx (xx.x%) | xxx (xx.x%) |
| Week 24 | xxx (xx.x%) | xxx (xx.x%) |
| Week 36 | xxx (xx.x%) | xxx (xx.x%) |
| Week 48 | xxx (xx.x%) | xxx (xx.x%) |
| Week 60 | xxx (xx.x%) | xxx (xx.x%) |
| Week 72 | xxx (xx.x%) | xxx (xx.x%) |
| Week 84 | xxx (xx.x%) | xxx (xx.x%) |
| Week 96 | xxx (xx.x%) | xxx (xx.x%) |
| Week 108 | xxx (xx.x%) | xxx (xx.x%) |
| Week 120 | xxx (xx.x%) | xxx (xx.x%) |
| Week 132 | xxx (xx.x%) | xxx (xx.x%) |
| Week 144 | xxx (xx.x%) | xxx (xx.x%) |
| Week 156 | xxx (xx.x%) | xxx (xx.x%) |
| Week 168 | xxx (xx.x%) | xxx (xx.x%) |
| Week 180 | xxx (xx.x%) | xxx (xx.x%) |
| Week 192 | xxx (xx.x%) | xxx (xx.x%) |
| Received corticosteroids (equivalent >10mg/day mean dose prednisone) for RA | | |
| Yes [3] | xxx (xx.x%) | xxx (xx.x%) |
| If yes, first noted at [4] | ,, | |
| Titration 4 | xxx (xx.x%) | xxx (xx.x%) |

## Statistical Analysis Plan for Long-Term Safety and Exploratory Analyses in SPM-020 (The RESET-RA Study)



Doc# CLP-008 Rev C, 15JUL2024

| Variable | TOL [1] | COL [2] |
|-------------|-------------|-------------|
| | (N=xxx) | (N=xxx) |
| Titration 5 | xxx (xx.x%) | xxx (xx.x%) |
| Titration 6 | xxx (xx.x%) | xxx (xx.x%) |
| Week 24 | xxx (xx.x%) | xxx (xx.x%) |
| Week 36 | xxx (xx.x%) | xxx (xx.x%) |
| Week 48 | xxx (xx.x%) | xxx (xx.x%) |
| Week 60 | xxx (xx.x%) | xxx (xx.x%) |
| Week 72 | xxx (xx.x%) | xxx (xx.x%) |
| Week 84 | xxx (xx.x%) | xxx (xx.x%) |
| Week 96 | xxx (xx.x%) | xxx (xx.x%) |
| Week 108 | xxx (xx.x%) | xxx (xx.x%) |
| Week 120 | xxx (xx.x%) | xxx (xx.x%) |
| Week 132 | xxx (xx.x%) | xxx (xx.x%) |
| Week 144 | xxx (xx.x%) | xxx (xx.x%) |
| Week 156 | xxx (xx.x%) | xxx (xx.x%) |
| Week 168 | xxx (xx.x%) | xxx (xx.x%) |
| Week 180 | xxx (xx.x%) | xxx (xx.x%) |
| Week 192 | xxx (xx.x%) | xxx (xx.x%) |

Repeat for other RA augmented therapy as reported in CRFs

Abbreviations: COL, Control to Open Label; cs/b/tsDMARD, conventional synthetic, biologic or targeted synthetic disease-modifying anti-rheumatic drug; TOL, Treament to Open Label

- [1] Treatment to Open Label (TOL): The TOL population comprises treatment subjects from ITT population who received active stimulation through Week 12, completed Week 12 assessments, continued to receive active stimulation during open-label follow-up, and for whom follow-up data are available.
- [2] Control to Open Label (COL): The COL population comprises control subjects from ITT population who received non-active (sham) stimulation through Week 12, switched to active stimulation after completing Week 12 assessments, continued to receive active stimulation during open-label follow-up, and for whom follow-up data are available.
- [3] Percentage calculated based on each analysis population (i.e., TOL, COL)
- [4] Percentage calculated based on the start date noted on the Concomitant Medication log

Reference: Listing 16.x.x.x

SOURCE: xxxxx SAS 9.4 {program location} {run date/time}}



Table 14.8.2.20 Implant Performance

| Variable | TOL [1] | COL [2] | Overall |
|---|---|---|---|
| Status of study implant at study exit [3] | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| Subjects with active implant | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| Subjects with suspended implant | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| Subjects with explanted implant | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| Unknown | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| Other | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |

Abbreviations: COL, Control to Open Label; TOL, Treatment to Open Label

- Treatment to Open Label (TOL): The TOL population comprises treatment subjects from ITT population who received active stimulation through Week
   completed Week 12 assessments, continued to receive active stimulation during open-label follow-up, and for whom follow-up data are available.
- [2] Control to Open Label (COL): The COL population comprises control subjects from ITT population who received non-active (sham) stimulation through Week 12, switched to active stimulation after completing Week 12 assessments, continued to receive active stimulation during open-label follow-up, and for whom follow-up data are available.
- [3] Percentage calculated based on each analysis population (i.e., TOL, COL, Overall)

Reference: Listing 16.x.x.x

SOURCE: xxxxx SAS 9.4 {program location} {run date/time}

Serial Number: c700c42a-b18e-4af7-8a24-9d2146ac6503 accessed by Melissa Evangelista (MEVANGELISTA) on Thu, 28 Aug 2025 18:20:31 GMT.



Table 14.8.3.1 Adverse Events

| Variable | TOL [1]<br>(N=xxx) | COL [2]<br>(N=xxx) | Safety Population [3]<br>(N=xxx) |
|---|---|---|---|
| | Events n (%) | Events n (%) | Events n (%) |
| Any AE [4] | xx xx (xx.x%) | xx xx (xx.x%) | xx xx (xx.x%) |
| Not Related [4] | xx xx (xx.x%) | xx xx (xx.x%) | xx xx (xx.x%) |
| Implant Procedure | xx xx (xx.x%) | xx xx (xx.x%) | xx xx (xx.x%) |
| Implant Device | xx xx (xx.x%) | xx xx (xx.x%) | xx xx (xx.x%) |
| Stimulation | xx xx (xx.x%) | xx xx (xx.x%) | xx xx (xx.x%) |
| Explant Procedure | xx xx (xx.x%) | xx xx (xx.x%) | xx xx (xx.x%) |
| Related [4][5] | | | |
| Implant Procedure | xx xx (xx.x%) | xx xx (xx.x%) | xx xx (xx.x%) |
| Implant Device | xx xx (xx.x%) | xx xx (xx.x%) | xx xx (xx.x%) |
| Stimulation | xx xx (xx.x%) | xx xx (xx.x%) | xx xx (xx.x%) |
| Explant Procedure | xx xx (xx.x%) | xx xx (xx.x%) | xx xx (xx.x%) |
| Indeterminate [4] | | | |
| Implant Procedure | xx xx (xx.x%) | xx xx (xx.x%) | xx xx (xx.x%) |
| Implant Device | xx xx (xx.x%) | xx xx (xx.x%) | xx xx (xx.x%) |
| Stimulation | xx xx (xx.x%) | xx xx (xx.x%) | xx xx (xx.x%) |
| Explant Procedure | xx xx (xx.x%) | xx xx (xx.x%) | xx xx (xx.x%) |
| AE resulting in discontinuation [4] | xx xx (xx.x%) | xx xx (xx.x%) | xx xx (xx.x%) |
| AE by maximum severity [4] | | | |
| Mild | xx xx (xx.x%) | xx xx (xx.x%) | xx xx (xx.x%) |
| Moderate | xx xx (xx.x%) | xx xx (xx.x%) | xx xx (xx.x%) |
| Severe | xx xx (xx.x%) | xx xx (xx.x%) | xx xx (xx.x%) |
| Implant Procedure related AE by maximum | | | |
| severity [4][5] | | | |
| Mild | xx xx (xx.x%) | xx xx (xx.x%) | xx xx (xx.x%) |
| Moderate | xx xx (xx.x%) | xx xx (xx.x%) | xx xx (xx.x%) |
| Severe | xx xx (xx.x%) | xx xx (xx.x%) | xx xx (xx.x%) |

## Statistical Analysis Plan for Long-Term Safety and Exploratory Analyses in SPM-020 (The RESET-RA Study)



#### Doc# CLP-008 Rev C, 15JUL2024

| Variable | TOL [1]<br>(N=xxx) | COL [2]<br>(N=xxx) | Safety Population [3]<br>(N=xxx) |
|---|---|---|---|
| | Events n (%) | Events n (%) | Events n (%) |
| Implant Device AE by maximum severity | | | |
| [4][5] | | | |
| Mild | xx xx (xx.x%) | xx xx (xx.x%) | xx xx (xx.x%) |
| Moderate | xx xx (xx.x%) | xx xx (xx.x%) | xx xx (xx.x%) |
| Severe | xx xx (xx.x%) | xx xx (xx.x%) | xx xx (xx.x%) |
| Stimulation related AE by maximum severity | | | |
| [4][5] | | | |
| Mild | xx xx (xx.x%) | xx xx (xx.x%) | xx xx (xx.x%) |
| Moderate | xx xx (xx.x%) | xx xx (xx.x%) | xx xx (xx.x%) |
| Severe | xx xx (xx.x%) | xx xx (xx.x%) | xx xx (xx.x%) |
| Energizer related AE by maximum severity | | | |
| [4][5] | | | |
| Mild | xx xx (xx.x%) | xx xx (xx.x%) | xx xx (xx.x%) |
| Moderate | xx xx (xx.x%) | xx xx (xx.x%) | xx xx (xx.x%) |
| Severe | xx xx (xx.x%) | xx xx (xx.x%) | xx xx (xx.x%) |
| Explant Procedure related AE by maximum | | | |
| severity [4][5] | | | |
| Mild | xx xx (xx.x%) | xx xx (xx.x%) | xx xx (xx.x%) |
| Moderate | xx xx (xx.x%) | xx xx (xx.x%) | xx xx (xx.x%) |
| Severe | xx xx (xx.x%) | xx xx (xx.x%) | xx xx (xx.x%) |
| SAE [4][5] | xx xx (xx.x%) | xx xx (xx.x%) | xx xx (xx.x%) |
| Implant Procedure SAE | xx xx (xx.x%) | xx xx (xx.x%) | xx xx (xx.x%) |
| Implant Device SAE | xx xx (xx.x%) | xx xx (xx.x%) | xx xx (xx.x%) |
| Stimulation SAE | xx xx (xx.x%) | xx xx (xx.x%) | xx xx (xx.x%) |
| Energixer SAE | xx xx (xx.x%) | xx xx (xx.x%) | xx xx (xx.x%) |
| Explant Procedure SAE | xx xx (xx.x%) | xx xx (xx.x%) | xx xx (xx.x%) |

Abbreviations: AE, adverse event; COL, Control to Open Label; SAE, serious adverse event; TOL, Treatment to Open Label
Note: AEs coded using the MedDRA dictionary Version 21.0 or later. Given in the table are subject counts and percentages. At each level of summation, subjects are counted only once. Subjects experiencing AEs of more than one severity are summarized according to the maximum severity experienced over all episodes of an AE



Doc# CLP-008 Rev C, 15JUL2024

| | TOL [1] | COL [2] | Safety Population [3] |
|----------|--------------|--------------|-----------------------|
| Variable | (N=xxx) | (N=xxx) | (N=xxx) |
| | Events n (%) | Events n (%) | Events n (%) |

- Treatment to Open Label (TOL): The TOL population comprises treatment subjects from ITT population who received active stimulation through Week
   completed Week 12 assessments, continued to receive active stimulation during open-label follow-up, and for whom follow-up data are available.
- [2] Control to Open Label (COL): The COL population comprises control subjects from ITT population who received non-active (sham) stimulation through Week 12, switched to active stimulation after completing Week 12 assessments, continued to receive active stimulation during open-label follow-up, and for whom follow-up data are available.
- [3] Safety population comprises all enrolled subjects.
- [4] Percentage calculated based on each analysis population (i.e., TOL, CL, Safety).
- [5] AEs judged to be "Definitely related" or "Probably related" are reported as "Related".

Reference: Listing 16.x.x.x

SOURCE: xxxxx SAS 9.4 {program location} {run date/time}}




Table 14.8.3.2

Adverse Events by SOC and Maximum Severity: All Events

| | TOL [1]<br>(N=xxx) | | | | | COL [2]<br>(N=xxx) | | | | Safety Population [3]<br>(N=xxx) | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| SOC | Mild | Moderate | Severe | Total | Mild | Moderate | Severe | Total | Mild | Moderate | Severe | Total |
| Preferred Term | Events | Events | Events | Events | Events | Events | Events | Events | Events | Events | Events | Events |
| | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) |
| Any AE [4] | xx | XX | xx | xx | xx | xx | xx | xx | xx | xx | xx | xx |
| , , , | x (xx%) | x (xx%) | x (xx%) | x (xx%) | x (xx%) | x (xx%) | x (xx%) | x (xx%) | x (xx%) | x (xx%) | x (xx%) | x (xx%) |
| SOC 1 [4] | xx | xx | xx | xx | xx | xx | xx | xx | xx | xx | xx | xx |
| | x (xx%) | x (xx%) | x (xx%) | x (xx%) | x (xx%) | x (xx%) | x (xx%) | x (xx%) | x (xx%) | x (xx%) | x (xx%) | x (xx%) |
| Preferred Term 1 | XX | XX | XX | XX | XX | XX | XX | XX | XX | XX | XX | XX |
| | x (xx%) | x (xx%) | x (xx%) | x (xx%) | x (xx%) | x (xx%) | x (xx%) | x (xx%) | x (xx%) | x (xx%) | x (xx%) | x (xx%) |
| Preferred Term 2 | XX | XX | XX | XX | XX | XX | XX | XX | XX | XX | XX | XX |
| | x (xx%) | x (xx%) | x (xx%) | x (xx%) | x (xx%) | x (xx%) | x (xx%) | x (xx%) | x (xx%) | x (xx%) | x (xx%) | x (xx%) |
| Preferred Term 3 | XX | XX | XX | XX | XX | XX | XX | XX | XX | XX | XX | XX |
| | x (xx%) | x (xx%) | x (xx%) | x (xx%) | x (xx%) | x (xx%) | x (xx%) | x (xx%) | x (xx%) | x (xx%) | x (xx%) | x (xx%) |
| Preferred Term 4 | XX | XX | XX | XX | XX | XX | XX | XX | XX | XX | XX | XX |
| | x (xx%) | x (xx%) | x (xx%) | x (xx%) | x (xx%) | x (xx%) | x (xx%) | x (xx%) | x (xx%) | x (xx%) | x (xx%) | x (xx%) |
| SOC 2 [4] | xx | XX | xx | xx | xx | xx | xx | xx | xx | xx | xx | XX |
| | x (xx%) | x (xx%) | x (xx%) | x (xx%) | x (xx%) | x (xx%) | x (xx%) | x (xx%) | x (xx%) | x (xx%) | x (xx%) | x (xx%) |
| Preferred Term 1 | XX | XX | XX | XX | XX | XX | XX | XX | XX | XX | XX | XX |
| | x (xx%) | x (xx%) | x (xx%) | x (xx%) | x (xx%) | x (xx%) | x (xx%) | x (xx%) | x (xx%) | x (xx%) | x (xx%) | x (xx% |
| Preferred Term 2 | XX | XX | XX | XX | XX | XX | XX | XX | XX | XX | XX | XX |
| | x (xx%) | x (xx%) | x (xx%) | x (xx%) | x (xx%) | x (xx%) | x (xx%) | x (xx%) | x (xx%) | x (xx%) | x (xx%) | x (xx% |
| Preferred Term 3 | XX | XX | XX | XX | XX | XX | XX | XX | XX | XX | XX | XX |
| | x (xx%) | x (xx%) | x (xx%) | x (xx%) | x (xx%) | x (xx%) | x (xx%) | x (xx%) | x (xx%) | x (xx%) | x (xx%) | x (xx%) |
| Preferred Term 4 | XX | XX | XX | XX | XX | XX | XX | XX | XX | XX | XX | XX |
| | x (xx%) | x (xx%) | x (xx%) | x (xx%) | x (xx%) | x (xx%) | x (xx%) | x (xx%) | x (xx%) | x (xx%) | x (xx%) | x (xx%) |

Continue ...

Abbreviations: AE, adverse event; COL, Control to Open Label; SOC, system organ class; TOL, Treatment to Open Label

Note: AEs coded using the MedDRA dictionary Version 21.0 or later. Given in the table are subject counts and percentages. At each level of summation, subjects are counted only once. Subjects experiencing AEs of more than one severity are summarized according to the maximum severity experienced over all episodes of an AE.



Doc# CLP-008 Rev C, 15JUL2024

- [1] Treatment to Open Label (TOL): The TOL population comprises treatment subjects from ITT population who received active stimulation through Week 12, completed Week 12 assessments, continued to receive active stimulation during open-label follow-up, and for whom follow-up data are available.
- [2] Control to Open Label (COL): The COL population comprises control subjects from ITT population who received non-active (sham) stimulation through Week 12, switched to active stimulation after completing Week 12 assessments, continued to receive active stimulation during open-label follow-up, and for whom follow-up data are available.
- [3] Safety population comprises all enrolled subjects.
- [4] Percentage calculated based on each analysis population (i.e., TOL, CL, Safety).

Reference: Listing 16.x.x.x

SOURCE: xxxxx SAS 9.4 {program location} {run date/time}}




Table 14.8.3.3
Implant Procedure-Related AEs by SOC and Maximum Severity: All Events

| | TOL [1]<br>(N=xxx) | | | | | COL [<br>(N=xx | | | Safety Population [3]<br>(N=xxx) | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| SOC | Mild | Moderate | Severe | Total | Mild | Moderate | Severe | Total | Mild | Moderate | Severe | Total |
| Preferred Term | Events | Events | Events | Events | Events | Events | Events | Events | Events | Events | Events | Events |
| | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) |
| Any AE [4][5] | xx | xx | xx | xx | xx | xx | xx | xx | xx | xx | xx | xx |
| 2 6363 | x (xx%) | x (xx%) | x (xx%) | x (xx%) | x (xx%) | x (xx%) | x (xx%) | x (xx%) | x (xx%) | x (xx%) | x (xx%) | x (xx%) |
| SOC 1 [4][5] | xx | xx | xx | xx | xx | xx | xx | xx | xx | xx | xx | xx |
| | x (xx%) | x (xx%) | x (xx%) | x (xx%) | x (xx%) | x (xx%) | x (xx%) | x (xx%) | x (xx%) | x (xx%) | x (xx%) | x (xx%) |
| Preferred Term 1 | XX | XX | XX | XX | XX | XX | XX | XX | XX | XX | XX | XX |
| | x (xx%) | x (xx%) | x (xx%) | x (xx%) | x (xx%) | x (xx%) | x (xx%) | x (xx%) | x (xx%) | x (xx%) | x (xx%) | x (xx%) |
| Preferred Term 2 | XX | XX | XX | XX | XX | XX | XX | XX | XX | XX | XX | XX |
| | x (xx%) | x (xx%) | x (xx%) | x (xx%) | x (xx%) | x (xx%) | x (xx%) | x (xx%) | x (xx%) | x (xx%) | x (xx%) | x (xx%) |
| Preferred Term 3 | XX | XX | XX | XX | XX | XX | XX | XX | XX | XX | XX | XX |
| | x (xx%) | x (xx%) | x (xx%) | x (xx%) | x (xx%) | x (xx%) | x (xx%) | x (xx%) | x (xx%) | x (xx%) | x (xx%) | x (xx%) |
| Preferred Term 4 | XX | XX | XX | XX | XX | XX | XX | XX | XX | XX | XX | XX |
| | x (xx%) | x (xx%) | x (xx%) | x (xx%) | x (xx%) | x (xx%) | x (xx%) | x (xx%) | x (xx%) | x (xx%) | x (xx%) | x (xx%) |
| SOC 2 [4][5] | xx | xx | xx | xx | xx | xx | xx | xx | xx | xx | xx | xx |
| | x (xx%) | x (xx%) | x (xx%) | x (xx%) | x (xx%) | x (xx%) | x (xx%) | x (xx%) | x (xx%) | x (xx%) | x (xx%) | x (xx%) |
| Preferred Term 1 | XX | XX | XX | XX | XX | XX | XX | XX | XX | XX | XX | XX |
| | x (xx%) | x (xx%) | x (xx%) | x (xx%) | x (xx%) | x (xx%) | x (xx%) | x (xx%) | x (xx%) | x (xx%) | x (xx%) | x (xx%) |
| Preferred Term 2 | XX | XX | XX | XX | XX | XX | XX | XX | XX | XX | XX | XX |
| | x (xx%) | x (xx%) | x (xx%) | x (xx%) | x (xx%) | x (xx%) | x (xx%) | x (xx%) | x (xx%) | x (xx%) | x (xx%) | x (xx% |
| Preferred Term 3 | xx | xx | xx | xx | xx | xx | xx | xx | xx | xx | xx | xx |
| | x (xx%) | x (xx%) | x (xx%) | x (xx%) | x (xx%) | x (xx%) | x (xx%) | x (xx%) | x (xx%) | x (xx%) | x (xx%) | x (xx% |
| Preferred Term 4 | xx | xx | xx | XX | xx | xx | XX | XX | XX | xx | XX | xx |
| | x (xx%) | x (xx%) | x (xx%) | x (xx%) | x (xx%) | x (xx%) | x (xx%) | x (xx%) | x (xx%) | x (xx%) | x (xx%) | x (xx%) |

#### Continue ...

Abbreviations: AE, adverse event; COL, Control to Open Label, SOC, system organ class; TOL, Treatment to Open Label

Note: AEs coded using the MedDRA dictionary Version 21.0 or later. Given in the table are subject counts and percentages. At each level of summation, subjects are counted only once. Subjects experiencing AEs of more than one severity are summarized according to the maximum severity experienced over all episodes of an AE.

Doc# CLP-008 Rev C, 15JUL2024



- [1] Treatment to Open Label (TOL): The TOL population comprises treatment subjects from ITT population who received active stimulation through Week 12, completed Week 12 assessments, continued to receive active stimulation during open-label follow-up, and for whom follow-up data are available.
- [2] Control to Open Label (COL): The COL population comprises control subjects from ITT population who received non-active (sham) stimulation through Week 12, switched to active stimulation after completing Week 12 assessments, continued to receive active stimulation during open-label follow-up, and for whom follow-up data are available.
- [3] Safety population comprises all enrolled subjects.
- [4] Percentage calculated based on each analysis population (i.e., TOL, CL, Safety).
- [5] AEs judged to be "Definitely related" or "Probably related" are reported as "Related".

Reference: Listing 16.x.x.x

SOURCE: xxxxx SAS 9.4 {program location} {run date/time}}




Table 14.8.3.4
Implant Device-Related AEs by SOC and Maximum Severity: All Events

Repeat Table 14.8.3.3 for implant device-related adverse events


Serial Number: c700c42a-b18e-4af7-8a24-9d2146ac6503 accessed by Melissa Evangelista (MEVANGELISTA) on Thu, 28 Aug 2025 18:20:31 GMT.

May not be reproduced outside of SetPoint Medical without written permission from Document Control.



Table 14.8.3.5 Stimulation-Related AEs by SOC and Maximum Severity: All Events

Repeat Table 14.8.3.3 for stimulation-related adverse events




Table 14.8.3.6 Energizer-Related AEs by SOC and Maximum Severity: All Events

Repeat Table 14.8.3.3 for Energizer-related adverse events

Table 14.8.3.7
Explant Procedure-Related Adverse Events by SOC and Maximum Severity: All Events

Repeat Table 14.8.3.3 for explant procedure-related adverse events


May not be reproduced outside of SetPoint Medical without written permission from Document Control.


Serial Number: c700c42a-b18e-4af7-8a24-9d2146ac6503 accessed by Melissa Evangelista (MEVANGELISTA) on Thu, 28 Aug 2025 18:20:31 GMT.

Doc# CLP-008 Rev C, 15JUL2024



Table 14.8.3.8 Device Deficiency

| Variable | TOL [1]<br>(N=xxx) | COL [2]<br>(N=xxx) | Safety Population [3]<br>(N=xxx) |
|---|---|---|---|
| | Events n (%) | Events n (%) | Events n (%) |
| Any study device deficiency [4] | xx xx (xx.x%) | xx xx (xx.x%) | xx xx (xx.x%) |
| Relationship of study device deficiency [4] | xx xx (xx.x%) | xx xx (xx.x%) | xx xx (xx.x%) |
| MicroRegulator (Implant) | xx xx (xx.x%) | xx xx (xx.x%) | xx xx (xx.x%) |
| POD | xx xx (xx.x%) | xx xx (xx.x%) | xx xx (xx.x%) |
| Energizer | xx xx (xx.x%) | xx xx (xx.x%) | xx xx (xx.x%) |
| Stimulation | xx xx (xx.x%) | xx xx (xx.x%) | xx xx (xx.x%) |
| Prescription Pad | xx xx (xx.x%) | xx xx (xx.x%) | xx xx (xx.x%) |
| IFU/Labeling | xx xx (xx.x%) | xx xx (xx.x%) | xx xx (xx.x%) |
| Study device deficiency associated with AE [4] | xx xx (xx.x%) | xx xx (xx.x%) | xx xx (xx.x%) |
| Study device deficiency associated with SAE [4] | xx xx (xx.x%) | xx xx (xx.x%) | xx xx (xx.x%) |

Abbreviations: AE, adverse event; COL, Control to Open Label; POD, Positioning Orientation Device; SAE, serious adverse event; SOC, system organ class; TOL, Treatment to Open Label

Note: Given in the table are subject counts and percentages. At each level of summation, subjects are counted only once. Subject experiencing several episodes of the same type of study device deficiency is counted once.

- [1] Treatment to Open Label (TOL): The TOL population comprises treatment subjects from ITT population who received active stimulation through Week 12, completed Week 12 assessments, continued to receive active stimulation during open-label follow-up, and for whom follow-up data are available.
- [2] Control to Open Label (COL): The COL population comprises control subjects from ITT population who received non-active (sham) stimulation through Week 12, switched to active stimulation after completing Week 12 assessments, continued to receive active stimulation during open-label follow-up, and for whom follow-up data are available.
- [3] Safety population comprises all enrolled subjects.
- [4] Percentage calculated based on each analysis population (i.e., TOL, CL, Safety).

Reference: Listing 16.x.x.x

SOURCE: xxxxx SAS 9.4 {program location} {run date/time}}



Table 14.8.3.9 Protocol Deviations

| Variable | OL PTE [1]<br>(N=xxx) | CO PTE [2]<br>(N=xxx) | Safety Population [3] (N=xxx) |
|---|---|---|---|
| Any protocol deviation [4] | Events n (%)<br>xx xx (xx.x%) | Events n (%)<br>xx xx (xx.x%) | Events n (%)<br>xx xx (xx.x%) |
| (f | | | |
| Minor protocol deviations [4] | xx xx (xx.x%) | xx xx (xx.x%) | xx xx (xx.x%) |
| Improper documentation of consent | xx xx (xx.x%) | xx xx (xx.x%) | xx xx (xx.x%) |
| Visit or assessment not done | xx xx (xx.x%) | xx xx (xx.x%) | xx xx (xx.x%) |
| Visit or assessment completed out of window | xx xx (xx.x%) | xx xx (xx.x%) | xx xx (xx.x%) |
| AE not reported within required schedule | xx xx (xx.x%) | xx xx (xx,x%) | xx xx (xx.x%) |
| Received medication not allowed per protocol | xx xx (xx.x%) | xx xx (xx.x%) | xx xx (xx.x%) |
| Subject or study staff unblinded | xx xx (xx.x%) | xx xx (xx.x%) | xx xx (xx.x%) |
| Other, specify | xx xx (xx.x%) | xx xx (xx.x%) | xx xx (xx.x%) |
| Protocol deviations due to COVID-19 [4] | xx xx (xx.x%) | xx xx (xx.x%) | xx xx (xx.x%) |
| Visit or assessment not done | xx xx (xx.x%) | xx xx (xx.x%) | xx xx (xx.x%) |
| Visit or assessment completed out of window | xx xx (xx.x%) | xx xx (xx.x%) | xx xx (xx.x%) |
| Visit or assessment completed not per protocol | xx xx (xx.x%) | xx xx (xx.x%) | xx xx (xx.x%) |
| Protocol deviations associated with AE [4] | xx xx (xx.x%) | xx xx (xx.x%) | xx xx (xx.x%) |
| Protocol deviations associated with SAE [4] | xx xx (xx.x%) | xx xx (xx.x%) | xx xx (xx.x%) |

Abbreviations: AE, adverse event; COL, Control to Open Label; SAE, serious adverse event; TOL, Treatment to Open Label Note: Given in the table are subject counts and percentages. At each level of summation, subjects are counted only once.

- [3] Safety population comprises all enrolled subjects.
- [4] Percentage calculated based on each analysis population (i.e., TOL, CL, Safety).

Reference: Listing 16.x.x.x

<sup>[1]</sup> Treatment to Open Label (TOL): The TOL population comprises treatment subjects from ITT population who received active stimulation through Week 12, completed Week 12 assessments, continued to receive active stimulation during open-label follow-up, and for whom follow-up data are available.

<sup>[2]</sup> Control to Open Label (COL): The COL population comprises control subjects from ITT population who received non-active (sham) stimulation through Week 12, switched to active stimulation after completing Week 12 assessments, continued to receive active stimulation during open-label follow-up, and for whom follow-up data are available.



Doc# CLP-008 Rev C, 15JUL2024

| | OL PTE [1] | CO PTE [2] | Safety Population [3] |
|---|---|---|---|
| Variable | (N=xxx) | (N=xxx) | (N=xxx) |
| | Events n (%) | Events n (%) | Events n (%) |
| SOURCE: xxxxx SAS 9.4 {program location} | {run date/time}} | | |




## Appendix C: Listing Mockups

| Listing 16.8.2.1 | Subject Disposition | 107 |
|---|---|---|
| Listing 16.8.2.2 | Protocol Deviations | 108 |
| Listing 16.8.2.3 | Analysis Populations | 109 |
| Listing 16.8.2.4 | Concomitant Medication | 110 |
| Listing 16.8.2.5 Su | bjects Receiving Augmented Treatment After Week 12 | 111 |
| Listing 16.8.2.6.1 | Explant Procedure | 112 |
| Listing 16.8.2.6.2 | Stimulation Prescription (Part 1) | 113 |
| Listing 16.8.2.6.2 | Stimulation Prescription (Part 2) | 114 |
| Listing 16.8.2.7.1 | RA Disease Activity Assessments | 115 |
| Listing 16.8.2.7.2 | ACR20 Response from Baseline | 116 |
| Listing 16.8.2.7.2.1 | ACR20 Response from Initiation of Stimulation | 118 |
| Listing 16.8.2.7.3 | ACR50 Response from Baseline | 120 |
| Listing 16.8.2.7.3.1 | ACR50 Response from Initiation of Stimulation | 122 |
| Listing 16.8.2.7.4 | ACR70 Response from Baseline | 124 |
| Listing 16.8.2.7.4.1 | ACR70 Response from Initiation of Stimulation | 126 |
| Listing 16.8.2.7.5 | CDAI | 128 |
| Listing 16.8.2.7.6 | DAS28-CRP | 130 |
| Listing 16.8.2.7.7 | HAQ-DI | 132 |
| Listing 16.8.2.7.8 | RAMRIS | 134 |
| Listing 16.8.2.7.9 | EQ-5D-5L | 135 |
| Listing 16.8.2.7.10 | SF-36 | 136 |
| Listing 16.8.2.7.11 | Subject Satisfaction | 137 |
| Listing 16.8.2.7.12 | Inflammatory Biomarkers | 138 |
| Listing 16.8.2.8 | Adverse Events | 140 |
| Listing 16.8.2.9Dev | vice Deficiencies | 141 |



Listing 16.8.2.1 Subject Disposition

| Analysis<br>Populati<br>on | Subject<br>ID | Consent Date | Implant<br>Procedure<br>Date | Day 0 Date | Week 12<br>Date | Subject<br>Status | Date of Exit | Reason for<br>Withdrawal | Implant<br>Status at<br>Study Exit |
|---|---|---|---|---|---|---|---|---|---|
| TOL | xx-xxxx | DD-MMM-<br>YYYY | DD-MMM-<br>YYYY | DD-MMM-<br>YYYY | | | | | |
| COL | xx-xxxx | DD-MMM-<br>YYYY | DD-MMM-<br>YYYY | DD-MMM-<br>YYYY | | | | | |

#### Programming notes:

This listing will include all subjects from Control to Open Label (COL) and Treatment to Open Label (TOL) populations for whom follow-up data are available.

Subject Status: Withdrawn, Completed Study.

Reason for withdrawal: Subject decision to withdraw consent, Investigator decision or medical judgement, Lost to follow-up, Device malfunction, Adverse event, Subject no longer eligible, Death, Study terminated, Sponsor or IRB decision, Other

SOURCE: xxxxx SAS 9.4 {program location} {run date/time}



#### Listing 16.8.2.2 Protocol Deviations

| Analysis<br>Populati<br>on | Subject<br>ID | Deviation<br>ID | Visit | Deviation<br>Date | Classification | Category | Reason | Associated with AE? | Associated with SAE? | Reported to IRB? | Description |
|---|---|---|---|---|---|---|---|---|---|---|---|
| | xx-xxxx | | | | | | | | | | |
| | xx-xxxx | | | | | | | | | | |

SOURCE: xxxxx SAS 9.4 {program location} {run date/time}




Listing 16.8.2.3 Analysis Populations

| | Popu | ılation |
|------------|---------|---------|
| Subject ID | TOL [1] | COL [2] |
| xx-xxxx | Yes | No |
| xx-xxxx | No | Yes |
| xx-xxxx | No | Yes |

Abbreviations: COL, Control to Open Label; ITT, intent to treat; TOL, Treatment to Open Label

SOURCE: xxxxx SAS 9.4 {program location} {run date/time}

Serial Number: c700c42a-b18e-4af7-8a24-9d2146ac6503 accessed by Melissa Evangelista (MEVANGELISTA) on Thu, 28 Aug 2025 18:20:31 GMT.


<sup>[1]</sup> Treatment to Open Label (TOL): The TOL population comprises treatment subjects from ITT population who received active stimulation through Week 12, completed Week 12 assessments, continued to receive active stimulation during open-label follow-up, and for whom follow-up data are available.

<sup>[2]</sup> Control to Open Label (COL): The COL population comprises control subjects from ITT population who received non-active (sham) stimulation through Week 12, switched to active stimulation after completing Week 12 assessments, continued to receive active stimulation during open-label follow-up, and for whom follow-up data are available.



#### Listing 16.8.2.4 Concomitant Medication

| | | ATC level | Sta | art | St | ор | | | | |
|---|---|---|---|---|---|---|---|---|---|---|
| Analysis | Subject | Preferred Term/ | | Study | | Study | | Dosage | | |
| Population | ID | Medication | Date | Day | Date | Day | Primary Indication | (Unit) | Route | Frequency |
| OL PTE | XX-XXXX | | | | | | | | | |
| COPTE | XX-XXXX | | | | | | | | | |

#### Programming notes:

- . This listing will include all subjects from OL PTE and CO PTE populations for whom follow-up data are available.
- · If Ongoing is checked "Yes" list "Ongoing" under stop date column
- · Concatenate dose and unit for listing, if other unit exists then list it for units
- Route, if Other Route is not blank, list it under "Route" column
- · Frequency, if Other Frequency is not blank, list it under 'Frequency" Column

SOURCE: xxxxx SAS 9.4 {program location} {run date/time}



# Listing 16.8.2.5 Subjects Receiving Augmented Treatment After Week 12




Listing 16.8.2.6.1 Explant Procedure

| Population<br>Analysis | Subject<br>ID | Explant Procedure Date | MicroRegulator<br>Serial# | MicroRegulator<br>Explanted? | Post-Op Clearance<br>Date | Any AEs? |
|---|---|---|---|---|---|---|
| TOL | | | | | | |
| | XX-XXXX | | | | | |
| COL | | | | | | |
| | XX-XXXX | | | | | |

SOURCE: xxxxx SAS 9.4 {program location} {run date/time}

May not be reproduced outside of SetPoint Medical without written permission from Document Control.


Serial Number: c700c42a-b18e-4af7-8a24-9d2146ac6503 accessed by Melissa Evangelista (MEVANGELISTA) on Thu, 28 Aug 2025 18:20:31 GMT.



#### Listing 16.8.2.6.2 Stimulation Prescription (Part 1)

| Analysis<br>Populati<br>on | Subject<br>ID | Visit | Strength<br>(uA) | Duration | Frequency | Schedule | Dose<br>Changed at<br>this Visit? | Dose Change Reason |
|---|---|---|---|---|---|---|---|---|
| TOL | | | | | | | | |
| | XX-XXXX | | | | | | | |
| | xx-xxxx | | | | | | | |
| | AA AAAA | | | | | | | |
| COL | | | | | | | | |
| | XX-XXXX | | | | | | | |
| | xx-xxxx | | | | | | | |

SOURCE: xxxxx SAS 9.4 {program location} {run date/time}


May not be reproduced outside of SetPoint Medical without written permission from Document Control.




Listing 16.8.2.6.2 Stimulation Prescription (Part 2)

| Analysis<br>Population | Subject<br>ID | Energizer<br>Battery Charge | Energizer App<br>Firmware | Energizer<br>Bluetooth<br>Firmware | Implant App<br>Firmware | Implant<br>Impedance | MicroRegulator<br>Suspended?/Reason |
|---|---|---|---|---|---|---|---|
| OL | ID | Battery Charge | rimiware | rimiware | rimiware | impedance | |
| OL | xx-xxxx | | | | | | |
| | xx-xxxx | | | | | | |
| OL | | | | | | | |
| | xx-xxxx | | | | | | |
| | xx-xxxx | | | | | | |




#### Listing 16.8.2.7.1 RA Disease Activity Assessments

| Analysis<br>Population | Subject<br>ID | Visit | SJC28<br>Score | TJC28<br>Score | HAQ-DI<br>Score | Subject's<br>Pain Score | SGA<br>Score | EGA Score | hsCRP<br>(mg/mL) |
|---|---|---|---|---|---|---|---|---|---|
| TOL | | | | | | | | | |
| | XX-XXXX | | | | | | | | |
| | | Screening | XX | XX | XXX | XXX | XX | XXX | XX |
| | | Day 0 | | | | | | | |
| | | Week 12 | | | | | | | |
| | | Week 24 | | | | | | | |
| | | Week 36 | | | | | | | |
| | | Week 48 | | | | | | | |
| | | Week 60 | | | | | | | |
| | | Week 72 | | | | | | | |
| | | Week 84 | | | | | | | |
| | | Week 96 | | | | | | | |
| | | Week 108 | | | | | | | |
| | | Week 120 | | | | | | | |
| | | Week 132 | | | | | | | |
| | | Week 144 | | | | | | | |
| | | Week 156 | | | | | | | |
| | | Week 168 | | | | | | | |
| | | Week 180 | | | | | | | |
| | | Week 192 | | | | | | | |
| COL | | | | | | | | | |


Serial Number: c700c42a-b18e-4af7-8a24-9d2146ac6503 accessed by Melissa Evangelista (MEVANGELISTA) on Thu, 28 Aug 2025 18:20:31 GMT.



Listing 16.8.2.7.2 ACR20 Response from Baseline

| | | | | | | Redu | ced by at least | 20%? | | |
|---|---|---|---|---|---|---|---|---|---|---|
| Analysis<br>Population | Subject<br>ID | Visit | ACR20<br>Response | SJC28 | TJC28 | HAQ-DI | Subject's<br>Pain | SGA | EGA | hsCRP |
| TOL | | W1- 24 | N | N | NI | N | N | N | N | N |
| | XX-XXXX | Week 24 | N | N | N | N | N | N | N | N |
| | | Week 36 | N | N | N | N | N | N | N | N |
| | | Week 48 | Y | N | N | N | N | N | N | N |
| | | Week 60 | Y | Y | Y | N | Y | Y | N | Y |
| | | Week 72 | N | N | N | N | N | N | N | N |
| | | Week 84 | Y | N | N | N | N | N | N | N |
| | | Week 96 | | | | | | | | |
| | | Week 108 | | | | | | | | |
| | | Week 120 | | | | | | | | |
| | | Week 132 | | | | | | | | |
| | | Week 144 | | | | | | | | |
| | | Week 156 | | | | | | | | |
| | | Week 168 | | | | | | | | |
| | | Week 180 | | | | | | | | |
| | | Week 192 | | | | | | | | |
| COL | | | | | | | | | | |
| | xx-xxxx | Week 24 | N | N | N | N | N | N | N | N |
| | | Week 36 | N | N | N | N | N | N | N | N |
| | | Week 48 | Y | N | N | N | N | N | N | N |
| | | Week 60 | Y | Y | Y | N | Y | Y | N | Y |
| | | Week 72 | N | N | N | N | N | N | N | N |
| | | Week 84 | Y | N | N | N | N | N | N | N |
| | | Week 96 | | | | | | | | |
| | | Week 108 | | | | | | | | |
| | | Week 120 | | | | | | | | |
| | | Week 132 | | | | | | | | |
| | | Week 144 | | | | | | | | |
| | | Week 156 | | | | | | | | |
| | | Week 168 | 2 | | | | | | | |




Doc# CLP-008 Rev C, 15JUL2024

| | | | | Reduced by at least 20%? | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|
| Analysis<br>Population | Subject<br>ID | Visit | ACR20<br>Response | SJC28 | TJC28 | HAQ-DI | Subject's<br>Pain | SGA | EGA | hsCRP |
| | | Week 192 | - | | | | | | | |

Note: Response defined by at least 70% reduction from baseline (i.e., on the day of informed consent for TOL and Week 12 for COL) in TJC28 and SJC28 and 3 our 5 outcomes, according to ACR definition.

SOURCE: xxxxx SAS 9.4 {program location} {run date/time}


May not be reproduced outside of SetPoint Medical without written permission from Document Control.

Serial Number: c700c42a-b18e-4af7-8a24-9d2146ac6503 accessed by Melissa Evangelista (MEVANGELISTA) on Thu, 28 Aug 2025 18:20:31 GMT.



Listing 16.8.2.7.2.1
ACR20 Response from Initiation of Stimulation

| | | | | | | Redu | iced by at least | 20%? | | |
|---|---|---|---|---|---|---|---|---|---|---|
| Analysis | Subject | | ACR20 | | | | Subject's | | | |
| Population | IĎ | Visit | Response | SJC28 | TJC28 | HAQ-DI | Pain | SGA | EGA | hsCR1 |
| TOL | | | • | | | | | | | |
| | xx-xxxx | Week 24 | N | N | N | N | N | N | N | N |
| | | Week 36 | N | N | N | N | N | N | N | N |
| | | Week 48 | Y | N | N | N | N | N | N | N |
| | | Week 60 | Y | Y | Y | N | Y | Y | N | Y |
| | | Week 72 | N | N | N | N | N | N | N | N |
| | | Week 84 | Y | N | N | N | N | N | N | N |
| | | Week 96 | | | | | | | | |
| | | Week 108 | | | | | | | | |
| | | Week 120 | | | | | | | | |
| | | Week 132 | | | | | | | | |
| | | Week 144 | | | | | | | | |
| | | Week 156 | | | | | | | | |
| | | Week 168 | | | | | | | | |
| | | Week 180 | | | | | | | | |
| | | Week 192 | | | | | | | | |
| COL | | | | | | | | | | |
| | XX-XXXX | Week 24 | N | N | N | N | N | N | N | N |
| | | Week 36 | N | N | N | N | N | N | N | N |
| | | Week 48 | Y | N | N | N | N | N | N | N |
| | | Week 60 | Y | Y | Y | N | Y | Y | N | Y |
| | | Week 72 | N | N | N | N | N | N | N | N |
| | | Week 84 | Y | N | N | N | N | N | N | N |
| | | Week 96 | | | | | | | | |
| | | Week 108 | | | | | | | | |
| | | Week 120 | | | | | | | | |
| | | Week 132 | | | | | | | | |
| | | Week 144 | | | | | | | | |
| | | Week 156 | | | | | | | | |
| | | Week 168 | | | | | | | | |
| | | Week 180 | | | | | | | | |
| | | Week 192 | | | | | | | | |



Doc# CLP-008 Rev C, 15JUL2024

| | | | | | Reduced by at least 20%? |
|---|---|---|---|---|---|
| Analysis | Subject | | ACR20 | Subject's | |
| Population | ID | Visit | Response | SJC28 TJC28 HAQ-DI Pain SGA EGA hsCRP | |

Note: Response defined by at least 20% reduction from initiation of stimulation (i.e., Day 0 for subjects in TOL, and Week 12 for subjects in COL) in TJC28 and SJC28 and 3 our 5 outcomes, according to ACR definition.

#### Note to programmer:

Subjects from both TOL and COL populations are listed here.

SOURCE: xxxxx SAS 9.4 {program location} {run date/time}




#### Listing 16.8.2.7.3 ACR 50 Response from Baseline

| | | | | | | Redu | aced by at least: | 50%? | | |
|---|---|---|---|---|---|---|---|---|---|---|
| Analysis<br>Population | Subject<br>ID | Visit | ACR50<br>Response | SJC28 | TJC28 | HAQ-DI | Subject's<br>Pain | SGA | EGA | hsCRP |
| TOL | 110 | VISIT | Response | 33020 | 13020 | naq-bi | Taili | SUA | EUA | IISCKI |
| TOL | xx-xxxx | Week 24 | N | N | N | N | N | N | N | N |
| | AA ACAA | Week 36 | N | N | N | N | N | N | N | N |
| | | Week 48 | Y | N | N | N | N | N | N | N |
| | | Week 60 | Y | Y | Y | N | Y | Y | N | Y |
| | | Week 72 | N | N | N | N | N | N | N | N |
| | | Week 84 | Y | N | N | N | N | N | N | N |
| | | Week 96 | - | | | | | | | |
| | | Week 108 | | | | | | | | |
| | | Week 120 | | | | | | | | |
| | | Week 132 | | | | | | | | |
| | | Week 144 | | | | | | | | |
| | | Week 156 | | | | | | | | |
| | | Week 168 | | | | | | | | |
| | | Week 180 | | | | | | | | |
| | | Week 192 | | | | | | | | |
| COL | | | | | | | | | | |
| COL | xx-xxxx | Week 24 | N | N | N | N | N | N | N | N |
| | AA-AAAA | Week 36 | N | N | N | N | N | N | N | N |
| | | Week 48 | Y | N | N | N | N | N | N | N |
| | | Week 60 | Y | Y | Y | N | Y | Y | N | Y |
| | | Week 72 | N | N | N | N | N | N | N | N |
| | | Week 84 | Y | N | N | N | N | N | N | N |
| | | Week 96 | • | | - 1 | | | | | - 1 |
| | | Week 108 | | | | | | | | |
| | | Week 120 | | | | | | | | |
| | | Week 132 | | | | | | | | |
| | | Week 144 | | | | | | | | |
| | | Week 144<br>Week 156<br>Week 168 | | | | | | | | |




Doc# CLP-008 Rev C, 15JUL2024

| | | _ | Reduced by at least 50%? | | | | | | |
|---|---|---|---|---|---|---|---|---|---|
| | bject | ACR50 | axa** | | **** | Subject's | | na. | |
| ulation | ID Visit | Response | SJC28 | TJC28 | HAQ-DI | Pain | SGA | EGA | hsCRP |
| | Week 18<br>Week 19 | 80 | | | | | | | |

Note: Response defined by at least 70% reduction from baseline (i.e., on the day of informed consent for TOL and Week 12 for COL) in TJC28 and SJC28 and 3 our 5 outcomes, according to ACR definition.

SOURCE: xxxxx SAS 9.4 {program location} {run date/time}




Listing 16.8.2.7.3.1
ACR 50 Response from Initiation of Stimulation

| | | | | | | Redu | iced by at least: | 50%? | | |
|---|---|---|---|---|---|---|---|---|---|---|
| Analysis<br>Population | Subject<br>ID | Visit | ACR50<br>Response | SJC28 | TJC28 | HAQ-DI | Subject's<br>Pain | SGA | EGA | hsCRF |
| TOL | | | | | | | | | | |
| | XX-XXXX | Week 24 | N | N | N | N | N | N | N | N |
| | | Week 36 | N | N | N | N | N | N | N | N |
| | | Week 48 | Y | N | N | N | N | N | N | N |
| | | Week 60 | Y | Y | Y | N | Y | Y | N | Y |
| | | Week 72 | N | N | N | N | N | N | N | N |
| | | Week 84 | Y | N | N | N | N | N | N | N |
| | | Week 96 | | | | | | | | |
| | | Week 108 | | | | | | | | |
| | | Week 120 | | | | | | | | |
| | | Week 132 | | | | | | | | |
| | | Week 144 | | | | | | | | |
| | | Week 156 | | | | | | | | |
| | | Week 168 | | | | | | | | |
| | | Week 180 | | | | | | | | |
| | | Week 192 | | | | | | | | |
| COL | | | | | | | | | | |
| | XX-XXXX | Week 24 | N | N | N | N | N | N | N | N |
| | | Week 36 | N | N | N | N | N | N | N | N |
| | | Week 48 | Y | N | N | N | N | N | N | N |
| | | Week 60 | Y | Y | Y | N | Y | Y | N | Y |
| | | Week 72 | N | N | N | N | N | N | N | N |
| | | Week 84 | Y | N | N | N | N | N | N | N |
| | | Week 96 | | | | | | | | |
| | | Week 108 | | | | | | | | |
| | | Week 120 | | | | | | | | |
| | | Week 132 | | | | | | | | |
| | | Week 144 | | | | | | | | |
| | | Week 156 | | | | | | | | |
| | | Week 168 | | | | | | | | |
| | | Week 180 | | | | | | | | |
| | | Week 192 | | | | | | | | |



Doc# CLP-008 Rev C, 15JUL2024

| | | | | | Reduced by at least 50%? |
|---|---|---|---|---|---|
| Analysis | Subject | | ACR50 | Subject's | |
| Population | IĎ | Visit | Response | SJC28 TJC28 HAQ-DI Pain SGA EGA hsCRP | |

Note: Response defined by at least 50% reduction from initiation of stimulation (i.e., Day 0 for subjects in TOL, and Week 12 for subjects in COL) in TJC28 and SJC28 and 3 our 5 outcomes, according to ACR definition.

SOURCE: xxxxx SAS 9.4 {program location} {run date/time}




Listing 16.8.2.7.4 ACR70 Response from Baseline

| | | | | | | Redu | ced by at least | 70%? | | |
|---|---|---|---|---|---|---|---|---|---|---|
| Analysis | Subject | | ACR70 | | | | Subject's | | | |
| Population | ID | Visit | Response | SJC28 | TJC28 | HAQ-DI | Pain | SGA | EGA | hsCR |
| TOL | | | | | | | | | | |
| | XX-XXXX | Week 24 | N | N | N | N | N | N | N | N |
| | | Week 36 | N | N | N | N | N | N | N | N |
| | | Week 48 | Y | N | N | N | N | N | N | N |
| | | Week 60 | Y | Y | Y | N | Y | Y | N | Y |
| | | Week 72 | N | N | N | N | N | N | N | N |
| | | Week 84 | Y | N | N | N | N | N | N | N |
| | | Week 96 | | | | | | | | |
| | | Week 108 | | | | | | | | |
| | | Week 120 | | | | | | | | |
| | | Week 132<br>Week 144 | | | | | | | | |
| | | Week 156 | | | | | | | | |
| | | Week 168 | | | | | | | | |
| | | Week 180 | | | | | | | | |
| | | Week 192 | | | | | | | | |
| | | WCCK 192 | | | | | | | | |
| COL | | | | | | | | | | |
| | XX-XXXX | Week 24 | N | N | N | N | N | N | N | N |
| | | Week 36 | N | N | N | N | N | N | N | N |
| | | Week 48 | Y | N | N | N | N | N | N | N |
| | | Week 60 | Y | Y | Y | N | Y | Y | N | Y |
| | | Week 72 | N | N | N | N | N | N | N | N |
| | | Week 84 | Y | N | N | N | N | N | N | N |
| | | Week 96 | | | | | | | | |
| | | Week 108 | | | | | | | | |
| | | Week 120 | | | | | | | | |
| | | Week 132 | | | | | | | | |
| | | Week 144 | | | | | | | | |
| | | Week 156<br>Week 168 | | | | | | | | |




Doc# CLP-008 Rev C, 15JUL2024

| | | | | | | Redu | iced by at least | 70%? | | |
|---|---|---|---|---|---|---|---|---|---|---|
| Analysis | Subject | | ACR70 | | | | Subject's | | | |
| Population | ID | Visit | Response | SJC28 | TJC28 | HAQ-DI | Pain | SGA | EGA | hsCRP |
| | | Week 180 | - | | | | | | | |
| | | Week 192 | | | | | | | | |

Note: Response defined by at least 70% reduction from baseline (i.e., on the day of informed consent for TOL and Week 12 for COL) in TJC28 and SJC28 and 3 our 5 outcomes, according to ACR definition.

SOURCE: xxxxx SAS 9.4 {program location} {run date/time}




Listing 16.8.2.7.4.1
ACR 70 Response from Initiation of Stimulation

| | | | | | | Redu | iced by at least | 70%? | | |
|---|---|---|---|---|---|---|---|---|---|---|
| Analysis<br>Population | Subject<br>ID | Visit | ACR70<br>Response | SJC28 | TJC28 | HAQ-DI | Subject's<br>Pain | SGA | EGA | hsCRF |
| TOL | | | | | | | | | | |
| | XX-XXXX | Week 24 | N | N | N | N | N | N | N | N |
| | | Week 36 | N | N | N | N | N | N | N | N |
| | | Week 48 | Y | N | N | N | N | N | N | N |
| | | Week 60 | Y | Y | Y | N | Y | Y | N | Y |
| | | Week 72 | N | N | N | N | N | N | N | N |
| | | Week 84 | Y | N | N | N | N | N | N | N |
| | | Week 96 | | | | | | | | |
| | | Week 108 | | | | | | | | |
| | | Week 120 | | | | | | | | |
| | | Week 132 | | | | | | | | |
| | | Week 144 | | | | | | | | |
| | | Week 156 | | | | | | | | |
| | | Week 168 | | | | | | | | |
| | | Week 180 | | | | | | | | |
| | | Week 192 | | | | | | | | |
| COL | | | | | | | | | | |
| | XX-XXXX | Week 24 | N | N | N | N | N | N | N | N |
| | | Week 36 | N | N | N | N | N | N | N | N |
| | | Week 48 | Y | N | N | N | N | N | N | N |
| | | Week 60 | Y | Y | Y | N | Y | Y | N | Y |
| | | Week 72 | N | N | N | N | N | N | N | N |
| | | Week 84 | Y | N | N | N | N | N | N | N |
| | | Week 96 | | | | | | | | |
| | | Week 108 | | | | | | | | |
| | | Week 120 | | | | | | | | |
| | | Week 132 | | | | | | | | |
| | | Week 144 | | | | | | | | |
| | | Week 156 | | | | | | | | |
| | | Week 168 | | | | | | | | |
| | | Week 180 | | | | | | | | |
| | | Week 192 | | | | | | | | |



Doc# CLP-008 Rev C, 15JUL2024

| | | | _ | | | Redu | ced by at least | t 70%? | | |
|---|---|---|---|---|---|---|---|---|---|---|
| Analysis | Subject | | ACR70 | | | | Subject's | | | |
| Population | ID | Visit | Response | SJC28 | TJC28 | HAQ-DI | Pain | SGA | EGA | hsCRP |

Note: Response defined by at least 70% reduction from initiation of stimulation (i.e., Day 0 for subjects in TOL, and Week 12 for subjects in COL) in TJC28 and SJC28 and 3 our 5 outcomes, according to ACR definition.

#### Note to programmer:

Subjects from both TOL and COL populations are listed here.

SOURCE: xxxxx SAS 9.4 {program location} {run date/time}




Doc# CLP-008 Rev C, 15JUL2024

Listing 16.8.2.7.5 CDAI

| Population<br>Analysis | Subject<br>ID | Visit | CDAI Score | LDA (>2.8 to $\leq$ 10) | Remission $(0 \text{ to } \le 2.8)$ | MCID from<br>Baseline | MCID from<br>Initiation of<br>Stimulation |
|---|---|---|---|---|---|---|---|
| TOL | | | | | | | |
| | XX-XXXX | Baseline | XX,X | N | N | _ | - |
| | | Day 0 | XX.X | N | N | N | - |
| | | Week 12 | XX,X | N | N | N | N |
| | | Week 24 | | Y | N | Y | Y |
| | | Week 36 | | Y | Y | Y | Y |
| | | Week 48 | | | | | |
| | | Week 60 | | | | | |
| | | Week 72 | | | | | |
| | | Week 84 | | | | | |
| | | Week 96 | | | | | |
| | | Week 108 | | | | | |
| | | Week 120 | | | | | |
| | | Week 132 | | | | | |
| | | Week 144 | | | | | |
| | | Week 156 | | | | | |
| | | Week 168 | | | | | |
| | | Week 180 | | | | | |
| | | Week 192 | | | | | |
| COL | | | | | | | |
| | xx-xxxx | Week 12 | XX.X | N | N | _ | _ |
| | | Week 24 | | Y | N | Y | Y |
| | | Week 36 | | Y | Y | Y | Y |
| | | Week 48 | | | | | |
| | | Week 60 | | | | | |
| | | Week 72 | | | | | |
| | | Week 84 | | | | | |
| | | Week 96 | | | | | |
| | | Week 108 | | | | | |
| | | Week 120 | | | | | |
| | | Week 132 | | | | | |
| | | Week 144 | | | | | |
| | | Week 156 | | | | | |




#### Doc# CLP-008 Rev C, 15JUL2024

| Population<br>Analysis | Subject<br>ID | Visit | CDAI Score | LDA<br>(>2.8 to ≤10) | Remission $(0 \text{ to } \le 2.8)$ | MCID from<br>Baseline | MCID from<br>Initiation of<br>Stimulation |
|---|---|---|---|---|---|---|---|
| | | Week 168<br>Week 180<br>Week 192 | | | | | |

Note: The MCID varies depending on RA disease activity at baseline (i.e., on the day of informed consent for TOL and at Week 12 for COL) or initiation of stimulation (TOL, COL): -12 for high activity (CDAI > 22), -6 for moderate activity (>10 to  $\leq$  22), or 1 if low disease activity (>2.8 to  $\leq$  10).

Note to programmer: Baseline on the day of informed consent for TOL and at Week 12 for COL.

SOURCE: xxxxx SAS 9.4 {program location} {run date/time}


Serial Number: c700c42a-b18e-4af7-8a24-9d2146ac6503 accessed by Melissa Evangelista (MEVANGELISTA) on Thu, 28 Aug 2025 18:20:31 GMT.



Listing 16.8.2.7.6 DAS28-CRP

| Population<br>Analysis | Subject<br>ID | Visit | DAS28-CRP<br>Score | LDA<br>(0.6 to < 3.2) | Remission<br>(0 to < 2.6) | MCID from<br>Baseline<br>(-1.2) | MCID from<br>Initiation of<br>Stimulation<br>(-1.2) | DAS28-CRP<br>Good/Moderat<br>e EULAR<br>Response |
|---|---|---|---|---|---|---|---|---|
| TOL | | | | | | | | |
| | XX-XXXX | Baseline | XX | N | N | | _ | |
| | | Day 0 | XX | N | N | N | _ | N |
| | | Week 12 | XX | Y | N | Y | Y | Moderate |
| | | Week 24 | XX | Y | Y | Y | Y | Good |
| | | Week 36 | | | | | | |
| | | Week 48 | | | | | | |
| | | Week 60 | | | | | | |
| | | Week 72 | | | | | | |
| | | Week 84 | | | | | | |
| | | Week 96 | | | | | | |
| | | Week 108 | | | | | | |
| | | Week 120 | | | | | | |
| | | Week 132 | | | | | | |
| | | Week 144 | | | | | | |
| | | Week 156 | | | | | | |
| | | Week 168 | | | | | | |
| | | Week 180 | | | | | | |
| | | Week 192 | | | | | | |
| COL | | | | | | | | |
| | XX-XXXX | Week 12 | XX | N | N | | _ | |
| | | Week 24 | XX | N | N | N | Y | N |
| | | Week 36 | XX | Y | N | Y | Y | Moderate |
| | | Week 48 | XX | Y | Y | Y | Y | Good |
| | | Week 60 | | | | | | |
| | | Week 72 | | | | | | |
| | | Week 84 | | | | | | |
| | | Week 96 | | | | | | |
| | | Week 108 | | | | | | |
| | | Week 120 | | | | | | |
| | | Week 132 | | | | | | |
| | | Week 144 | | | | | | |




Week 156

Week 168

Week 180

Week 192

Note to programmer: Baseline on the day of informed consent for TOL and at Week 12 for COL.

SOURCE: xxxxx SAS 9.4 {program location} {run date/time}

Serial Number: c700c42a-b18e-4af7-8a24-9d2146ac6503 accessed by Melissa Evangelista (MEVANGELISTA) on Thu, 28 Aug 2025 18:20:31 GMT.

Doc# CLP-008 Rev C, 15JUL2024



#### Listing 16.8.2.7.7 HAQ-DI

| Population<br>Analysis | Subject<br>ID | Visit | HAQ-DI Score | MCID from Baseline<br>(-0.22) | MCID from Initiation of<br>Stimulation |
|---|---|---|---|---|---|
| TOL | 113 | * 1510 | III Q DI Score | (0.22) | Stillulation |
| | xx-xxxx | Baseline | XX | | |
| | | Day 0 | XX | N | |
| | | Week 12 | XX | N | N |
| | | Week 24 | XX | Y | Y |
| | | Week 36 | XX | Y | Y |
| | | Week 48 | | | |
| | | Week 60 | | | |
| | | Week 72 | | | |
| | | Week 84 | | | |
| | | Week 96 | | | |
| | | Week 108 | | | |
| | | Week 120 | | | |
| | | Week 132 | | | |
| | | Week 144 | | | |
| | | Week 156 | | | |
| | | Week 168 | | | |
| | | Week 180 | | | |
| | | Week 192 | | | |
| COL | | | | | |
| | XX-XXXX | Week 12 | XX | | |
| | | Week 24 | XX | N | N |
| | | Week 36 | XX | Y | Y |
| | | Week 48 | XX | Y | Y |
| | | Week 60 | | | |
| | | Week 72 | | | |
| | | Week 84 | | | |
| | | Week 96 | | | |
| | | Week 108 | | | |
| | | Week 120 | | | |
| | | Week 132 | | | |
| | | Week 144<br>Week 156 | | | |




Doc# CLP-008 Rev C, 15JUL2024

| Population<br>Analysis | Subject<br>ID | Visit | HAQ-DI Score | MCID from Baseline<br>(-0.22) | MCID from Initiation of<br>Stimulation |
|---|---|---|---|---|---|
| | | Week 168 | | | |
| | | Week 180 | | | |
| | | Week 192 | | | |

Note to programmer: Baseline on the day of informed consent for TOL and at Week 12 for COL

SOURCE: xxxxx SAS 9.4 {program location} {run date/time}


May not be reproduced outside of SetPoint Medical without written permission from Document Control.


Serial Number: c700c42a-b18e-4af7-8a24-9d2146ac6503 accessed by Melissa Evangelista (MEVANGELISTA) on Thu, 28 Aug 2025 18:20:31 GMT.



#### Listing 16.8.2.7.8 RAMRIS

| Population<br>Analysis | Subject<br>ID | Visit | Synovitis<br>Score | Osteitis<br>score | Bone<br>Erosion<br>score | Progression?<br>(Bone Erosion<br>Increase > 0.5) | CARLOS |
|---|---|---|---|---|---|---|---|
| TOL | xx-xxxx | Baseline (Screening)<br>Week 24<br>% Change from baseline | xx | xx | xx | -<br>-<br>N | xx |
| COL | xx-xxxx | Baseline (Week 12)<br>Week 24<br>Change from baseline | | | | | |

Note to programmer: Baseline during Screening for TOL and at Week 12 for COL

SOURCE: xxxxx SAS 9.4 {program location} {run date/time}

Serial Number: c700c42a-b18e-4af7-8a24-9d2146ac6503 accessed by Melissa Evangelista (MEVANGELISTA) on Thu, 28 Aug 2025 18:20:31 GMT.



#### Listing 16.8.2.7.9 EQ-5D-5L

| Population<br>Analysis | Subject<br>ID | Visit | Mobility | Self-Care | Usual<br>Activities | Pain/Discomfort | Anxiety/Depression | EQ-VAS | Index<br>value |
|---|---|---|---|---|---|---|---|---|---|
| TOL | | W. 1 24 | | | | | | | |
| | XX-XXXX | Week 24<br>Week 48<br>Week 96<br>Week 144 | х | х | х | х | х | XXX | XX |
| COL | | | | | | | | | |
| | XX-XXXX | Week 24<br>Week 48<br>Week 96<br>Week 144<br>Week 192 | х | х | x | х | х | xxx | xx |

SOURCE: xxxxx SAS 9.4 {program location} {run date/time}


May not be reproduced outside of SetPoint Medical without written permission from Document Control.




Listing 16.8.2.7.10 SF-36

| Population<br>Analysis | Subject<br>ID | Visit | PCS score | MCS score |
|------------------------|---------------|----------|-----------|-----------|
| TOL | | | | |
| | xx-xxxx | Week 24 | | |
| | | Week 48 | | |
| | | Week 96 | | |
| | | Week 144 | | |
| COL | | | | |
| | xx-xxxx | Week 24 | | |
| | | Week 48 | | |
| | | Week 96 | | |
| | | Week 144 | | |
| | | Week 192 | | |

SOURCE: xxxxx SAS 9.4 {program location} {run date/time}


May not be reproduced outside of SetPoint Medical without written permission from Document Control.




Listing 16.8.2.7.11 Subject Satisfaction

| Population<br>Analysis | Subject<br>ID | Visit SelPoint System for Insalment | | Would you recommend<br>it to a family member<br>or a friend? | Comment |
|---|---|---|---|---|---|
| TOL | | | | | |
| | xx-xxxx | Week 24 | Very satisfied | Yes | |
| | xx-xxxx | Week 24 | Satisfied | Yes | |
| | XX-XXXX | Week 24 | Neither satisfied nor dissatisfied | No | |
| | xx-xxxx | Week 24 | Somewhat dissatisfied | No | |
| | XX-XXXX | Week 24 | Very dissatisfied | No | |
| COL | | | | | |
| | xx-xxxx | Week 24 | Very satisfied | Yes | |
| | xx-xxxx | Week 24 | Satisfied | Yes | |
| | xx-xxxx | Week 24 | Neither satisfied nor dissatisfied | No | |
| | xx-xxxx | Week 24 | Somewhat dissatisfied | No | |
| | xx-xxxx | Week 24 | Very dissatisfied | No | |

SOURCE: xxxxx SAS 9.4 {program location} {run date/time}




Doc# CLP-008 Rev C, 15JUL2024

### Listing 16.8.2.7.12 Inflammatory Biomarkers

| Population<br>Analysis | Subject<br>ID | Visit | IL-6<br>(pg/mL) | IL-6<br>% Change | SAA<br>(µg/mL) | SAA<br>% Change | MMP-3<br>(pg/mL) | MMP-3<br>% Change |
|---|---|---|---|---|---|---|---|---|
| TOL | | | | | | | | |
| | xx-xxxx | Baseline | | _ | | | | |
| | | Day 0 | | | | | | |
| | | Week 12 | | | | | | |
| | | Week 24 | | | | | | |
| | | Week 36 | | | | | | |
| | | Week 48 | | | | | | |
| | | Week 60 | | | | | | |
| | | Week 72 | | | | | | |
| | | Week 84 | | | | | | |
| | | Week 96 | | | | | | |
| | | Week 108 | | | | | | |
| | | Week 120 | | | | | | |
| | | Week 132 | | | | | | |
| | | Week 144 | | | | | | |
| | | Week 156 | | | | | | |
| | | Week 168 | | | | | | |
| | | Week 180 | | | | | | |
| | | Week 192 | | | | | | |
| COL | | | | | | | | |
| | xx-xxxx | Week 12 | | _ | | | | |
| | | Week 24 | | | | | | |
| | | Week 36 | | | | | | |
| | | Week 48 | | | | | | |
| | | Week 60 | | | | | | |
| | | Week 72 | | | | | | |
| | | Week 84 | | | | | | |
| | | Week 96 | | | | | | |
| | | Week 108 | | | | | | |
| | | Week 120 | | | | | | |
| | | Week 132 | | | | | | |
| | | Week 144 | | | | | | |




Doc# CLP-008 Rev C, 15JUL2024

Week 156 Week 168 Week 180 Week 192

Note to programmer: Percent change from baseline (i.e., Screening for TOL and at Week 12 for COL).

SOURCE: xxxxx SAS 9.4 {program location} {run date/time}


May not be reproduced outside of SetPoint Medical without written permission from Document Control.


Serial Number: c700c42a-b18e-4af7-8a24-9d2146ac6503 accessed by Melissa Evangelista (MEVANGELISTA) on Thu, 28 Aug 2025 18:20:31 GMT.



Listing 16.8.2.8 Adverse Events

| Analysis<br>Population | Subject ID | System Organ<br>Class/<br>Preferred Term/<br>Adverse Event<br>Verbatim | Onset Date<br>(Day) | Resolution Date<br>(Day) | 5 | Severity | SAE? | Relationship | Treatment/<br>outcome |
|---|---|---|---|---|---|---|---|---|---|
| TOL | | | | | | | · | | |
| | xx-xxxx | xxxxxx/<br>xxxxxx/<br>xxxxxx/ | DD-MMM-YYYY<br>(xx) | DD-MMM-YYYY<br>(xx) | | | | | xxxxxx/<br>xxxxxx |
| | | xxxxxx/<br>xxxxxx/<br>xxxxxx/ | | | | | | | |
| COL | xx-xxxx | None | | | | | | | |

Note: If a Subject has no AEs then "None" will be displayed. Adverse Events are coded in MedDRA V21.0 or later.

Note to programmer: If Ongoing is checked then list "Continuing" in the place for "Resolution Date (Day)".

SOURCE: xxxxx SAS 9.4 {program location} {run date/time}



#### Listing 16.8.2.9 Device Deficiencies

| Analysis<br>Population | Subject ID | Deficiency ID | Deficiency<br>Date | Deficiency<br>Related To | Associated with AE? | Associated with SAE? | Description |
|---|---|---|---|---|---|---|---|
| TOL | | | | | | | |
| | xx-xxxx | | | | | | |
| ~~* | | | | | | | |
| COL | | | | | | | |
| | XX-XXXX | | | | | | |

SOURCE: xxxxx SAS 9.4 {program location} {run date/time}

May not be reproduced outside of SetPoint Medical without written permission from Document Control.
